## **Cover Page for Statistical Analysis Plan**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT03175120 |
| Sponsor trial ID: | NN9068-4166 |
| Official title of study: | A trial comparing the efficacy and safety of insulin degludec/liraglutide and insulin degludec in combination with metformin in Chinese subjects with type 2 diabetes mellitus inadequately controlled with basal insulin therapy and metformin $\pm$ one other OAD. DUAL <sup>TM</sup> II China |
| Document date: | 23 January 2020 |

Redacted statistical analysis plan Includes redaction of personal identifiable information only.

IDegLira Trial ID: NN9068-4166 Clinical Trial Report Appendix 16.1.9


Date: Version: Status:

23 January 2020 Novo Nordisk Final

#### 16.1.9 Documentation of statistical methods

### List of contents

| Statistical analysis plan | Link |
|---------------------------|------|
| Statistical documentation | Link |

Statistical Analysis Plan Trial ID:NN9068-4166 UTN:U1111-1154-6732 EudraCT No.:


Date: Version: Status: Page:

12 July 2019 | Novo Nordisk Final 1 of 19

#### Statistical Analysis Plan

**Trial ID: NN9068-4166** 

A trial comparing the efficacy and safety of insulin degludec/liraglutide and insulin degludec in combination with metformin in Chinese subjects with type 2 diabetes mellitus inadequately controlled with basal insulin therapy and metformin  $\pm$  one other OAD

Author:




Date: Version: Status: Page:

12 July 2019 | **Novo Nordisk**2.0
Final

### **Table of contents**

| | | | | | Page |
|---|---|---|---|---|---|
| Ta | ble of co | ontents | ••••• | | 2 |
| Lis | t of abb | reviation | s | | 3 |
| 1 | | | | | |
| | 1.1<br>1.2 | | | l analysis plan | |
| 2 | Statist | ical consi | derations | | 4 |
| | 2.1 | | | on | |
| | 2.2 | - | | sets | |
| | 2.3 | | | | |
| | | 2.3.1 | | analysis | |
| | 2.4 | Seconda | | | |
| | | 2.4.1 | | ory secondary endpoints | |
| | | 2.4.2 | | e secondary endpoints | |
| | | | 2.4.2.1 | | |
| | | | 2.4.2.2 | J 1 | |
| 3 | Chang | ges to the | statistical an | alyses planned in the protocol | 18 |
| 4 | Refere | ences | | | 19 |

Statistical Analysis Plan Trial ID:NN9068-4166 UTN:U1111-1154-6732 EudraCT No.:


Date: Version: Status: Page:

12 July 2019 | Novo Nordisk 2.0

Final


#### List of abbreviations

ADA American Diabetes Association

AE adverse event

ANCOVA analysis of covariance

BG blood glucose **BMI** body mass index CAS completer analysis set CTR clinical trial report **ECG** electrocardiogram **EOT** End of treatment ET End of treatment **FAS** full analysis set

**FDA** U.S. Food and Drug Administration

**FPG** fasting plasma glucose  $HbA_{1c}$ glycosylated haemoglobin **HDL** high density lipoprotein НОМА-В homeostatic model assessment IDegLira insulin degludec/liraglutide

insulin degludec **IDeg** ITT intention-to-treat

LDL low density lipoprotein lower limit of quantification LLOQ **LOCF** Last Observation Carried Forward

SAE serious adverse event SAP statistical analysis plan SAS safety analysis set SD standard deviation

**SMPG** self-measured plasma glucose

type 2 diabetes mellitus T2DM

**TEAEs** treatment emergent adverse events

**UNR** upper normal range UTN Universal Trial Number **VLDL** very low density lipoprotein

| EudraCT No.: Status: Final F | Statistical Analysis Plan<br>Trial ID:NN9068-4166<br>UTN:U1111-1154-6732<br>EudraCT No: | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 2.0<br>Final | Novo Nordisk |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

#### 1 Introduction

#### 1.1 Trial information

This is a 26 week, randomised, parallel two-arm, double-blind, multi-centre, treat-to-target (TTT) trial in Chinese subjects with T2DM inadequately controlled with basal insulin therapy and metformin  $\pm$  one other OAD:  $\alpha$ -glucosidase inhibitors (AGI), sulphonylureas (SU), glinides or thiazolidinediones (TZD). The trial is comparing efficacy and safety of insulin degludec/liraglutide (IDegLira) versus insulin degludec (IDeg) both in combination with Metformin. For further details please see the protocol.

#### 1.2 Scope of the statistical analysis plan

This Statistical Analysis Plan (SAP) is based on final Protocol version 5.0 (06-Dec-2016).

The scope of this SAP is to add one sensitivity analysis for change from baseline in  $HbA_{1c}$  after 26 weeks of treatment and several sensitivity analyses for confirmatory secondary endpoints, and performed other minor changes. For further details on the changes see section  $\underline{3}$ .

#### 2 Statistical considerations

Novo Nordisk will analyse and report data from all sites together.

All analyses of efficacy and safety endpoints will be based on the full analysis set (FAS). The analysis of the primary endpoint and the confirmatory secondary endpoint, change from baseline in body weight after 26 weeks of treatment, will be repeated on the per-protocol (PP) analysis set and the completer analysis set (CAS) for sensitivity purposes. All efficacy endpoints will be summarised using the FAS and safety endpoints will be summarised using the safety analysis set (SAS).

The impact of protocol deviations and outliers may be investigated further in sensitivity analyses if deemed relevant.

Unless otherwise specified, all continuous measurements will be summarised descriptively at each visit by treatment using observed data. After 26 weeks of treatment, descriptive statistics will be presented based both on observed and last observation carried forward (LOCF) imputed data. Endpoints that are analysed untransformed and endpoints that are not formally analysed are summarised by the arithmetic mean, standard deviation (SD), median, and minimum and maximum value. Endpoints that are analysed log-transformed are summarised by the geometric mean and coefficient of variation (CV).

| Statistical Analysis Plan | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: | Page: | 5 of 19 | |

For measurements over time, mean values will be plotted to explore the trajectory over time. LOCF imputed data will be used as the basis for plotting data, if not otherwise specified. For endpoints that are analysed log-transformed, the geometric mean values will be plotted.

A standard analysis of covariance (ANCOVA) model will be applied for the continuous primary and secondary endpoints. The model includes treatment and previous antidiabetic treatment (basal insulin and metformin or basal insulin, metformin and other OAD(s)) as fixed factors and the corresponding baseline value as a covariate. In the following, this model will be referred to as the standard ANCOVA model.

Presentation of results from a statistical analysis will include the estimated mean treatment effects (Least Square Means [LSMeans]) for absolute values and change from baseline. In addition, estimated mean treatment difference (or ratio) will be presented together with the two-sided 95% confidence interval and corresponding two-sided p-value.

#### Handling of missing data

The expected percentage of missing data is around 15%. In accordance with industry guidance<sup>1</sup>, endpoints will be assessed at frequent visits and also on subjects who withdraw prematurely. This will facilitate an analysis in accordance with ITT principles. Also, the combined information on frequent outcomes and information on reason for drop-out is assumed to account for the missing data anticipated.

If an assessment has been made both at screening (visit 1) and randomisation (visit 2), and if not otherwise specified, the value from the randomisation visit will be used as the baseline value. If the value measured at the randomisation visit is missing and the assessment also has been made at screening, then the screening value will be used as the baseline value.

Missing values (including intermittent missing values) will be imputed using the LOCF method. Subjects without data after randomisation will be included by carrying forward their baseline value. LOCF has been a standard approach in diabetes trials for many years and was used as the primary analysis in both IDegLira and IDeg phase 3a trials. LOCF is considered to be an appropriate method in the context of TTT trials, where subjects after withdrawal typically continue their therapy using commercially available insulin. In previous TTT trials with IDegLira and IDeg, LOCF has generally provided similar results to alternative methods applied to handle missing data, such as repeated measures models and completer analyses. In this trial, similar sensitivity analyses will be made to examine the robustness of the LOCF method. The LOCF approach will also be used to impute missing values in CAS.

#### 2.1 Sample size calculation

The primary objective of this trial is to confirm superiority of IDegLira vs. IDeg in controlling glycaemia in Chinese subjects with T2DM after 26 weeks of treatment. This is done by comparing

| Statistical Analysis Plan | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: | Page: | 6 of 19 | |

the difference in change from baseline in  $HbA_{1c}$  after 26 weeks of treatment to a superiority margin of 0.0% for IDegLira vs. IDeg.

Superiority in the primary endpoint for IDegLira versus IDeg will be considered confirmed if the upper bound of the two-sided 95% confidence interval for the estimated mean treatment difference in change from baseline in  $HbA_{1c}$  (for IDegLira - IDeg) is strictly below 0% or equivalently if the p-value for the two-sided test of

$$H_0$$
 D=0 against  $H_A$  D $\neq 0$ ,

is less than 5% and D<0, where D is the estimated treatment difference. This is equivalent to using a one-sided test of size 2.5%, which means that the type 1 error rate is controlled at 2.5% (1-sided).

The sample size is determined using a t-statistic under the assumption of a two-sided test of size 5%, a mean difference in treatment of - 0.4%, and a standard deviation of SD=1.2%. It is also assumed that 15% of the randomised subjects will be excluded from the PP analysis set. Superiority will be investigated for both the FAS and the PP analysis set in line with the Committee for Proprietary Medicinal Products (CPMP) Points to Consider<sup>2</sup>. The above assumptions are based on experience from the phase 3a development programmes for IDegLira and IDeg. From these assumptions and based on a 2:1 randomisation the sample size is set to 300 subjects in the IDegLira arm and 150 subjects in the IDeg arm; in total 450 subjects will be randomised. This will ensure a power of 91.4% for confirming the primary objective in the full analysis set. Reducing the mean difference to -0.35% yields a power of 83%.

#### 2.2 Definition of analysis sets

The following analysis sets are defined in accordance with the ICH-E9 guidance<sup>3</sup>.

- Full Analysis Set (FAS): includes all randomised subjects. In exceptional cases, subjects may be eliminated from the full analysis set. In such cases the elimination will be justified and documented. The statistical evaluation of the FAS will follow the intention-to-treat (ITT) principle and subjects will contribute to the evaluation "as randomised".
- **Per-Protocol (PP) analysis set:** includes all subjects in the FAS who fulfils the following criteria:
  - o Have not violated any inclusion criteria
  - o Have not fulfilled any exclusion criteria
  - Have a non-missing HbA<sub>1c</sub> at screening or randomisation
  - o Have at least one non-missing HbA<sub>1c</sub> after 12 weeks of exposure
  - o Have at least 12 weeks of exposure

Subjects will contribute to the evaluation "as treated".

| Statistical Analysis Plan | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: | Page: | 7 of 19 | |

- Safety Analysis Set (SAS): includes all subjects receiving at least one dose of the
  investigational product or comparator. Subjects in the safety set will contribute to the evaluation
  "as treated".
- Completer Analysis Set (CAS): includes all randomised subjects who have completed the trial. Subjects in the completer analysis set will contribute to the evaluation "as randomised".

Randomised subjects who are lost to follow up and where no exposure information of the investigational product or comparators is available after randomisation will be handled as unexposed.

Before data are released for statistical analysis, a review of all data will take place to identify protocol deviations that could potentially affect the results. Any decision to exclude any subject or observation from the statistical analysis is the joint responsibility of the members of the study group. The subjects or observations to be excluded, and the reasons for their exclusion must be documented and signed by those responsible before database lock. The subjects and observations excluded from analysis sets, and the reason for this, will be described in the clinical trial report.

#### 2.3 Primary endpoint

The primary endpoint is defined as change from baseline in HbA<sub>1c</sub> after 26 weeks of treatment.

The change from baseline in  $HbA_{1c}$  after 26 weeks of treatment will be analysed using an ANCOVA model with treatment, previous antidiabetic treatment (basal insulin and metformin or basal insulin, metformin and other OAD(s)) as fixed effects and baseline  $HbA_{1c}$  as covariate. Missing values after 26 weeks of treatment will be imputed LOCF using  $HbA_{1c}$  values at and after baseline.

Superiority of IDegLira vs. IDeg will be considered as confirmed if the 95% confidence interval for the mean treatment difference for change from baseline in  $HbA_{1c}$  lies entirely below 0.0%; equivalent to a one-sided test with significance level of 2.5%. Conclusion of superiority will be based on FAS. Analysis based on the PP analysis set will be regarded as sensitivity analysis.

#### 2.3.1 Sensitivity analysis

The primary efficacy analysis will be repeated on the PP analysis set and the CAS as sensitivity analysis. Furthermore, sensitivity analysis will be performed on FAS using the mixed model for repeated measurement (MMRM) to evaluate the sensitivity of using LOCF. All  $HbA_{1c}$  values available post baseline at scheduled measurement times will be analysed in a linear mixed normal model using an unstructured residual covariance matrix for  $HbA_{1c}$  measurements within the same subject. The model will include treatment, visit and previous antidiabetic treatment as fixed factors and baseline  $HbA_{1c}$  as a covariate. Interactions between visit and all factors and the covariate are also included in the model.

| Statistical Analysis Plan | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: | Page: | 8 of 19 | |

The result will be compared to the result of the ANCOVA method using LOCF for imputation of missing data. Any marked difference between the MMRM and ANCOVA LOCF approach regarding the estimated treatment difference will be commented upon in the CTR.

Further, a pattern mixture model approach, mimicking an intention-to-treat scenario will be applied. The imputation in the IDegLira arm will be based on IDeg values. It will be done as follows:

- In the first step intermittent missing values are imputed using a Markov Chain Monte Carlo method, in order to obtain a monotone missing data pattern. This imputation is done for each treatment group separately and 1000 copies of the dataset will be generated.
- In the second step, for each of the 1000 copies of the dataset, an analysis of variance model with previous anti-diabetic treatment as fixed factors, and baseline HbA1c as covariates is fitted to the change in HbA1c from baseline to 4 weeks (V10) for the IDeg group only. The estimated parameters, and their variances, from this model are used to impute missing values at 4 weeks for subjects in IDeg and IDegLira treatment groups, based on previous anti-diabetic treatment and HbA1c at baseline.
- In the third step, for each of the 1000 copies of the dataset, missing HbA1c values at 8 weeks (V15) are imputed in the same way as for 4 weeks. Now the imputations are based on an analysis of variance model with the same factors and the HbA1c values at baseline and 4 weeks as covariates, fitted to the IDeg group.
- This stepwise procedure is then repeated sequentially over the available planned visits, adding one visit in each step until the last planned visit at 26 weeks (V33).
- For each of the complete data sets, the change from baseline to 26 weeks is analysed using an analysis of variance model with treatment and previous anti-diabetic treatment as fixed factors and baseline HbA1c value as a covariate.

The estimates and standard deviations for data sets are pooled to one estimate and associated standard deviation using Rubin's rule<sup>4</sup>. From these pooled estimates the confidence interval for the treatment differences and the associated p-value are calculated.

#### 2.4 Secondary endpoints

#### 2.4.1 Confirmatory secondary endpoints

The following two confirmatory endpoints will be tested for superiority of IDegLira vs. IDeg:

- Change from baseline in body weight after 26 weeks of treatment
- Number of treatment emergent severe or BG confirmed hypoglycaemic episodes during 26 weeks of treatment

| Statistical Analysis Plan | | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|---|
| Trial ID:NN9068-4166 | CONFIDENTIAL | Version: | 2.0 | I |
| UTN:U1111-1154-6732 | CONFIDENTIAL | Status: | Final | 1 |
| FudraCT No · | | Page. | 9 of 19 | I |

The tests for superiority of the confirmatory secondary endpoints will be based on the FAS and will only be carried out if superiority of IDegLira vs. IDeg with regards to the primary endpoint is confirmed.

In order to control the overall type I error on a 2-sided 5% level with regards to the secondary endpoints, a hierarchical testing procedure will be used. If superiority is confirmed with respect to change from baseline in body weight after 26 weeks of treatment the number of treatment emergent severe or BG confirmed hypoglycaemic episodes during 26 weeks of treatment will be tested for superiority.

Superiority for change from baseline in body weight will be considered confirmed if the upper bound of the two-sided 95% confidence interval for the estimated mean treatment difference (IDegLira minus IDeg) is strictly below zero or equivalently if the p-value for the one-sided test of

$$H_0 D \ge 0.0$$
 against  $H_A D < 0.0$ ,

is less than 2.5%, where D is the treatment difference.

The change from baseline in body weight after 26 weeks of treatment will be analysed using an ANCOVA model with treatment and previous antidiabetic treatment (basal insulin and metformin or basal insulin, metformin and other OAD(s)) as fixed effect and baseline weight as covariate.

The similar sensitivity analyses as specified for the primary endpoint (ANCOVA on the PP analysis set and CAS, MMRM and the pattern mixture model) will be performed.

Superiority for hypoglycaemic episodes will be considered confirmed if the upper bound of the two-sided 95% confidence interval for the estimated mean treatment ratio (IDegLira vs. IDeg) is strictly below one or equivalently if the p-value for the one-sided test of

$$H_0$$
 RR $\geq$ 1.0 against  $H_A$  RR $\leq$ 1.0,

is less than 2.5%, where RR is the treatment rate ratio.

The number of treatment emergent severe or BG confirmed hypoglycaemic episodes during 26 weeks of treatment will be analysed using a negative binominal regression model with a log-link function and the logarithm of the time period in which a hypoglycaemic episode is considered treatment emergent as offset. The model will include treatment and previous antidiabetic treatment as fixed factors.

As a sensitivity analysis, for withdrawn subjects, the number of episodes in the missing period (time of withdrawal to planned treatment emergent period [max of 27 weeks and longest treatment emergent time observed in the trial]) will be imputed using a multiple imputation technique<sup>5</sup>, and

| Statistical Analysis Plan | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: | Page: | 10 of 19 | |

assuming that all subjects have an event rate in the period before and after withdrawal corresponding to the event rate in the comparator group (IDeg). This will be done as follows:

- As a first step, a Bayes negative binomial model with the same fixed factors used in the original
  confirmatory analysis model is fitted to the event rate data to obtain the posterior distribution of
  model parameters.
- In the second step, based on the estimated parameters for comparator (IDeg) in this model, the number of events in the missing period is imputed for all withdrawn subjects. I.e. pre and post withdrawal event rates in the conditional distribution used for imputation are as for comparator (IDeg). Multiple copies (1000 copies) of a complete data set are generated by sampling from the estimated distribution.
- In the third step, for each of the complete data sets, the number of events is analysed using a negative binomial model including the same fixed factors used in the original model.
- In the fourth step, the estimates and standard deviations for the 1000 data sets are pooled to one estimate and associated standard deviation using Rubin's rule<sup>4</sup>. From these pooled estimates the confidence interval for the treatment ratio and the associated p-value are calculated.

#### 2.4.2 Supportive secondary endpoints

#### 2.4.2.1 Efficacy endpoints

#### Insulin dose after 26 weeks of treatment

The actual daily insulin dose after 26 weeks of treatment will be analysed using an ANCOVA model including treatment and previous antidiabetic treatment as fixed factors and baseline  $HbA_{1c}$  value and insulin dose at screening as covariates.

#### Responder for HbA<sub>1c</sub> after 26 weeks of treatment

Two dichotomous endpoints (responder/non-responder) will be defined based on whether a subject has met a specific target level after 26 weeks of treatment:

- ADA HbA<sub>1c</sub> target (HbA<sub>1c</sub> < 7.0%)
- International Diabetes Federation (IDF)  $HbA_{1c}$  target ( $HbA_{1c} \le 6.5\%$ )

Analysis of each of the two responder endpoints will be based on a logistic regression model with treatment and previous antidiabetic treatment as fixed factors and baseline HbA<sub>1c</sub> value as a covariate.

| Statistical Analysis Plan | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: | Page: | 11 of 19 | |

#### HbA<sub>1c</sub> responder endpoints without weight gain

Responder for  $HbA_{1c}$  without weight gain after 26 weeks of treatment will be defined as  $HbA_{1c} < 7.0\%$  or  $\le 6.5\%$  at end of treatment and change from baseline in body weight below or equal to zero. Analysis of each of the two responder endpoints will be based on a logistic regression model with treatment and previous antidiabetic treatment as fixed factors and baseline  $HbA_{1c}$  and body weight values as covariates.

#### HbA<sub>1c</sub> responder endpoints without hypoglycaemic episodes

Responder for  $HbA_{1c}$  without hypoglycaemic episodes after 26 weeks of treatment will be defined as  $HbA_{1c} < 7.0\%$  or  $\le 6.5\%$  at end of treatment and without severe or BG confirmed episodes during the last 12 weeks of treatment. Analysis of each of the two responder endpoints will be based on a logistic regression model with treatment and previous antidiabetic treatment as fixed factors and baseline  $HbA_{1c}$  values as a covariate.

#### HbA<sub>1c</sub> responder endpoints without hypoglycaemic episodes and weight gain

Responder for  $HbA_{1c}$  without hypoglycaemic episodes and weight gain after 26 weeks of treatment will be defined as  $HbA_{1c} < 7.0\%$  or  $\le 6.5\%$  at end of treatment, without severe or BG confirmed episodes during the last 12 weeks of treatment, and change from baseline in body weight below or equal to zero. Analysis of each of the two responder endpoints will be based on a logistic regression model with treatment and previous antidiabetic treatment as fixed factors and baseline  $HbA_{1c}$  and body weight values as covariates.

#### Fasting plasma glucose (FPG)

Change from baseline in FPG after 26 weeks of treatment will be analysed using the standard ANCOVA model.

#### Waist circumference

Change from baseline in waist circumference after 26 weeks of treatment will be analysed using the standard ANCOVA model.

#### Beta-cell function (fasting insulin, fasting C-peptide, fasting glucagon, and HOMA-β)

In addition to fasting insulin, fasting C-peptide, and fasting glucagon, one derived parameter will be calculated; Beta-cell function (HOMA- $\beta$ ). The calculation of the HOMA endpoint will be done as follows:

• Beta-cell function (%) =  $20 \cdot \text{fasting insulin} [\mu \text{U/mL}]/(\text{FPG[mmol/L]}-3.5)$ 

These endpoints after 26 weeks of treatment will be analysed separately using the standard ANCOVA model. In these statistical analyses the endpoint will be log-transformed and so will the baseline covariate.

Statistical Analysis Plan
Trial ID:NN9068-4166
UTN:U1111-1154-6732
EudraCT No.:

Date:
12 July 2019
Version:
2.0
Status:
Final
Page:

#### Fasting lipid profile

Cholesterol, low density lipoprotein cholesterol (LDL cholesterol), high density lipoprotein cholesterol (HDL cholesterol), very low density lipoprotein cholesterol (VLDL cholesterol), triglycerides, and free fatty acids after 26 weeks of treatment will be analysed separately using the standard ANCOVA model. In these statistical analyses the endpoint will be log-transformed and so will the baseline covariate.

#### Self-measured plasma glucose (SMPG) 9-point profile

Three endpoints from the 9 point SMPG profile will be defined:

- 9-point profile
- Mean of the 9-point profile, defined as the area under the profile (calculated using the trapezoidal method) divided by the measurement time
- Post-prandial PG increments (from before meal to 90 min after for breakfast, lunch and dinner). The mean increment over all meals will be derived as the mean of all available meal increments

A linear mixed effect model will be fitted to the 9-point SMPG profile data. The model will include treatment, previous antidiabetic treatment, time, the interaction between treatment and time and the interaction between previous antidiabetic treatment and time as fixed factors and subject as random effect, where measurements within subjects will be assumed correlated with a compound symmetry covariance matrix. From the model mean profile by treatment and relevant treatment differences will be estimated and explored.

Change from baseline after 26 weeks of treatment in mean of the 9-point profile and post-prandial increment endpoints will be analysed separately using the standard ANCOVA model.

#### 2.4.2.2 Safety endpoints

#### Adverse events

AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) coding.

A TEAE is defined as an event that has onset date on or after the first day of exposure to randomised treatment and no later than seven days after the last day of randomised treatment. If the event has onset date before the first day of exposure on randomised treatment and increases in severity during the treatment period and until 7 days after the last drug date, then this event should also be considered as a TEAE. Major adverse cardiovascular events (MACEs, defined as all cardiovascular deaths, non-fatal myocardial infarctions and non-fatal strokes) are considered treatment-emergent until 30 calendar days after the last dose of trial product.

| Statistical Analysis Plan | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: | Page: | 13 of 19 | |

TEAEs are summarised descriptively, whereas non-TEAEs are presented in listings. TEAE data will be displayed in terms of the number of subjects with at least one event (N), the percentage of subjects with at least one event (%), the number of events (E) and the event rate per 100 years of exposure (R).

Summaries of TEAEs and of serious TEAEs will be presented as an overview including all AEs, AEs by seriousness, AEs by severity, AEs by relation to treatment, technical complaint AEs and AEs by outcome (including deaths).

Furthermore summary tables based on system organ class and preferred terms are made for:

- All TEAEs
- TEAEs leading to withdrawal
- Serious TEAEs
- Possibly or probably related TEAEs
- Severe, moderate and mild TEAEs
- TEAEs reported by safety areas of interest
- TEAEs with preferred term that are experienced by at least 5% of the subjects in any treatment arm or by at least 5% of all subjects

A listing for non-treatment emergent adverse events with onset date before the first day of exposure to randomised treatment will be presented. A listing will also be presented for non-treatment emergent adverse events collected after the treatment emergent period according to the definition of TEAE.

#### Classification of Hypoglycaemia

**Treatment emergent:** hypoglycaemic episodes will be defined as treatment emergent if the onset of the episode occurs on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.

**Nocturnal hypoglycaemic episodes:** are episodes with time of onset between 00:01 and 05.59 both inclusive.

Hypoglycaemic episodes are classified according to the Novo Nordisk classification of hypoglycaemia (see <u>Figure 1</u>) and the ADA classification of hypoglycaemia (see <u>Figure 2</u>).

#### Novo Nordisk classification of hypoglycaemia

In normal physiology, symptoms of hypoglycaemia occur below a plasma glucose level of 3.1 mmol/L. Therefore, Novo Nordisk has included hypoglycaemia with plasma glucose levels below this cut-off point in the definition of BG confirmed hypoglycaemia.

| Statistical Analysis Plan | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: | Page: | 14 of 19 | |

Novo Nordisk uses the following classification (see <u>Figure 1</u>) in addition to the ADA classification (see <u>Figure 2</u>)

- Severe or BG confirmed symptomatic hypoglycaemia: An episode that is severe according to the ADA classification<sup>7</sup> or BG confirmed by a plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia.
- Severe or BG confirmed hypoglycaemia: An episode that is severe according to the ADA classification<sup>7</sup> or BG confirmed by a plasma glucose value <3.1 mmol/L with or without symptoms consistent with hypoglycaemia.



Note: Glucose measurements are performed with capillary blood calibrated to plasma equivalent glucose values

BG: blood glucose PG: plasma glucose SMPG: Self-measured plasma glucose

Figure 1 Novo Nordisk classification of hypoglycaemia

#### ADA classification of hypoglycaemia<sup>7</sup>

- Severe hypoglycaemia: An episode requiring assistance of another person to actively administer
  carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not
  be available during an event, but neurological recovery following the return of plasma glucose
  to normal is considered sufficient evidence that the event was induced by a low plasma glucose
  concentration.
- Asymptomatic hypoglycaemia: An episode not accompanied by typical symptoms of hypoglycaemia, but with a measured plasma glucose concentration ≤ 3.9 mmol/L.
- Documented symptomatic hypoglycaemia: An episode during which typical symptoms of hypoglycaemia are accompanied by a measured plasma glucose concentration ≤ 3.9 mmol/L.
- Pseudo-hypoglycaemia: An episode during which the person with diabetes reports any of the typical symptoms of hypoglycaemia with a measured plasma glucose concentration > 3.9 mmol/L but approaching that level.

| Statistical Analysis Plan | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: | Page: | 15 of 19 | |

• Probable symptomatic hypoglycaemia: An episode during which symptoms of hypoglycaemia are not accompanied by a plasma glucose determination but that was presumably caused by a plasma glucose concentration ≤ 3.9 mmol/L.



Note: Glucose measurements are performed with capillary blood calibrated to plasma equivalent glucose values

PG: plasma glucose SMPG: Self-measured plasma glucose

Figure 2 ADA classification of hypoglycaemia

Data on treatment emergent hypoglycaemic episodes are presented in terms of the number of subjects with at least one event (N), the percentage of subjects with at least one event (%), the number of events (E) and the event rate per 100 years (R).

Separate summaries are made for severe or BG confirmed hypoglycaemic episodes, severe or BG confirmed symptomatic hypoglycaemic episodes, nocturnal severe or BG confirmed hypoglycaemic episodes, nocturnal severe or BG confirmed symptomatic hypoglycaemic episodes and the ADA classification of hypoglycaemia.

The number of hypoglycaemic episodes during 26 weeks of treatment will be analysed separately for each endpoint using a negative binominal regression model with a log-link function and the logarithm of the time period in which a hypoglycaemic episode is considered treatment emergent as offset. The model will include treatment and previous antidiabetic treatment as fixed factor.

| Statistical Analysis Plan | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: | Page: | 16 of 19 | |

#### Pulse

Change from baseline in pulse after 26 weeks of treatment will be analysed using the standard ANCOVA model.

#### Systolic and diastolic blood pressure

Change from baseline in systolic and diastolic blood pressure after 26 weeks of treatment will be analysed using the standard ANCOVA model.

#### Clinical evaluations (physical examination, fundoscopy or fundus photography and ECG)

Eye examination (dilated fundoscopy/fundus photography) and ECG findings will be summarised descriptively, including:

- Summaries
- The change from baseline after 26 weeks of treatment

Any findings in the physical examination evaluation at screening will be presented as listings. Any clinically significant deterioration of a pre-existing condition after the screening visit, as well as any new clinically significant findings will be recorded as adverse events.

#### **Laboratory assessments**

All laboratory parameters will be summarised descriptively. The following tables will be presented based on both observed and LOCF imputed data:

- Shift tables from baseline to after 26 weeks of treatment
- Proportion of subjects with measurements outside reference range by treatment and week.

Laboratory values will be presented graphically as box plots by treatment and week.

For each laboratory parameter, individual values outside the reference ranges (abnormal values) will be listed.

For lipase and amylase the following rule will apply in the evaluation of the result:

• If the amylase or lipase baseline (at screening) value is > 3xUNR the information were recorded as medical history for that subject.

#### Calcitonin

The purpose of the calcitonin analysis is to evaluate longitudinal changes in calcitonin, with main focus on subjects who develop persistently high levels of calcitonin during the trial.

| Statistical Analysis Plan | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: | Page: | 17 of 19 | |

Calcitonin will be displayed in terms of the number of subjects (N), the percentage of subjects (%) and the event rate per 100 years of exposure (R). The following criteria are defined for tabulations:

• Persistent (all post baseline measurements)

```
From < UNR to persistently \geq UNR
From < UNR to persistently \geq 1.5 UNR
From < UNR to persistently \geq 20 ng/L
From < UNR to persistently \geq 50 ng/L
From < 20 ng/L to persistently \geq 20 ng/L
From < 50 ng/L to persistently \geq 50 ng/L
```

• Incidental (at least one post baseline measurements)

```
From < UNR to \ge UNR
From < UNR to \ge 1.5 UNR
From < UNR to \ge 20 ng/L
From < UNR to \ge 50 ng/L
From < 20 ng/L to \ge 20 ng/L
From < 50 ng/L to \ge 50 ng/L
```

The distribution of all calcitonin measurements across treatment groups and time will be shown with box plots and corresponding cumulative plots for actual levels of calcitonin and change from baseline. The plots will be presented by treatment group at EOT using LOCF imputed values and within treatment group by week. Plots will be done by each gender, separately.

Summaries tables of calcitonin continuous measurements, will include number and percentage of observations < and  $\ge$  LLOQ, minimum, Q25, median, Q75 and maximum. Summaries will be presented for all subjects and by gender.

Longitudinal changes for subjects with calcitonin levels  $\geq 20$  ng/L will be plotted (longitudinal plots). The plots will be done by treatment and gender. They will be done for subjects in the persistent and incidental categories, separately.

A listing of subjects with at least one post baseline value  $\geq 20$  ng/l will be done. The listing will include age, gender, calcitonin measurements over time and AE history (including preferred term, onset and stop dates).

#### Urinalysis

Categorical urinalysis parameters will be summarised descriptively by:

- Shift from baseline to EOT (using the number of subjects in the different categories)
- Subjects with at least one post baseline measurement outside reference range will be listed

| Statistical Analysis Plan | Date: | 12 July 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: | Page: | 18 of 19 | |

#### Insulin and GLP-1 antibodies

Insulin antibodies (IDeg specific, cross-reacting to human insulin and total) will be summarised with arithmetic mean, standard deviation (SD), median, and minimum and maximum value by treatment and treatment week, and their mean over time will be plotted. Correlations will be explored graphically as follows. Insulin antibodies (IDeg specific, cross-reacting to human insulin and total) will be plotted against HbA<sub>1c</sub> after 26 weeks, HbA<sub>1c</sub> change from baseline after 26 weeks, and dose after 26 weeks. Change from baseline to FU1 in insulin antibodies (IDeg specific, cross-reacting to human insulin and total) will be plotted against HbA<sub>1c</sub> after 26 weeks, HbA<sub>1c</sub> change from baseline after 26 weeks, and dose after 26 weeks.

GLP-1 antibodies (liraglutide specific, cross-reacting to native GLP-1, liraglutide *in vitro* neutralising and *in vitro* neutralising to native GLP-1) will be summarised by number of subjects (N) and percentage of subjects (%) with positive and negative samples.

Antibody measurements will be listed by subject and visit together with associated age, sex, BMI, HbA<sub>1c</sub> and dose

### 3 Changes to the statistical analyses planned in the protocol

- Additional sensitivity analysis added to use pattern mixture model to evaluate the sensitivity of using LOCF for primary endpoint HbA<sub>1c</sub>
- Sensitivity analyses for confirmatory secondary endpoints have been added.
- One minor change regarding the analysis model to the supportive secondary endpoint of 9-point self-measured plasma glucose has been made

| Statistical Analysis Plan |
|---------------------------|
| Trial ID:NN9068-4166 |
| UTN:U1111-1154-6732 |
| EudraCT No.: |


Date: Version: Status: Page:

12 July 2019 | Novo Nordisk Final 19 of 19

#### References 4

<sup>&</sup>lt;sup>1</sup> U.S. Department of Health and Human Services, Food and Drug Administration. Guidance for Industry, Diabetes Mellitus: Developing Drugs and Therapeutic Biologics for Treatment and Prevention, Draft Guidance. 2008.

<sup>&</sup>lt;sup>2</sup> European Medicines Agency. Comitee for Proprietary Medical Products (CPMP): Points to consider on switching between superiority and non-inferiority (CPMP/EWP/482/99). EMEA 2000. 2000.

<sup>&</sup>lt;sup>3</sup> International Conference on Harmonisation. ICH Harmonised Tripartite Guideline E9. Statistical Principles for Clinical Trials. 5 Feb 1998.

<sup>&</sup>lt;sup>4</sup> Little RJA, Rubin D.B. Statistical analysis with missing data. New York: John Wiley & Sons, 1987.

<sup>&</sup>lt;sup>5</sup> Keene ONea. Missing data sensitivity analysis for recurrent event data using controlled imputation. Pharm Stat 2014; 13:258-264.

<sup>&</sup>lt;sup>6</sup> Schwartz NS, Clutter WE, Shah SD, Cryer PE. Glycemic thresholds for activation of glucose counterregulatory systems are higher than the threshold for symptoms. J Clin Invest. 1987;79(3):777-81.

<sup>&</sup>lt;sup>7</sup> Seaguist ER, Anderson J, Childs B, Cryer P, Dagogo-Jack S, Fish L, et al. Hypoglycemia and diabetes: a report of a workgroup of the American Diabetes Association and the Endocrine Society. Diabetes Care. 2013;36(5):1384-95.

| NN9068<br>NN9068-4166 | <del>CONFIDENTIAL</del> | Date:<br>Version: | 22 . |
|---|---|---|---|
| Clinical Trial Report<br>Statistical document | | Status:<br>Page: | |

January 2020 | Novo Nordisk 1.0 Final 1 of 334

## **Table of contents**

| | Page |
|---|---|
| 1: Actual daily total insulin dose after 26 weeks of treatment – supportive statistical analysis – full analysis set - appendix | 4 |
| 2: HbA1c after 26 weeks of treatment – change from baseline – confirmatory statistical analysis – full analysis set - appendix | 7 |
| 3: HbA1c after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – PP analysis set - appendix | 17 |
| 4: HbA1c after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – completer analysis set - appendix | 27 |
| 5: HbA1c after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – MMRM – full analysis set - appendix | |
| 5: HbA1c after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – conditional multiple imputation – full analysis set - appendix | 57 |
| 7: Responder for HbA1c treatment target – supportive statistical analysis – full analysis set | 67 |
| 8: Responder for HbA1c treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes – supportive statistical analysis – full analysis set | 71 |
| 9: Responder for HbA1c treatment target without weight gain – supportive statistical analysis – full analysis set | 75 |
| 10: Responder for HbA1c treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes and weight gain – supportive statistical analysis – full analysis set | 81 |
| 11: Body weight after 26 weeks of treatment – change from baseline – confirmatory statistical analysis – full analysis set - appendix | 87 |
| 12: Body weight after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – PP analysis set - appendix | 97 |
| 13: Body weight after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – completer analysis set - appendix | 107 |
| 14: Body weight after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – MMRM – full analysis set - appendix | 117 |
| 15: Body weight after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – conditional multiple imputation – full analysis set - appendix | 137 |
| 16: Waist circumference after 26 weeks of treatment – change from baseline – supportive statistical analysis – full analysis set - appendix | 147 |
| 17: Fasting plasma glucose after 26 weeks of treatment – change from baseline – supportive statistical analysis – full analysis set - appendix | |
| 18: 9-point self-measured plasma glucose profile after 26 weeks of treatment – supportive statistical analysis – full analysis set | |
| 19: Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment – change from haseline – supportive statistical analysis – full analysis set - appendix | 204 |

| NN9068<br>NN9068-4166<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 22 January 2020<br>1.0<br>Final<br>2 of 334 | Novo Nordisk |
|---|---|---|---|---|
| | ortive statistical analysis – full a | nalysis set - append | dix | 214 |
| 21: Fasting insulin after 26 weeks appendix | s of treatment – supportive statis | • | • | 254 |
| 22: Fasting C-peptide after 26 we appendix | eks of treatment – supportive sta | • | - | 257 |
| 23: Fasting glucagon after 26 wee appendix | eks of treatment – supportive sta | • | • | 263 |
| 24: HOMA-B after 26 weeks of tr | 11 | 2 | , ,,, | x266 |
| 11 | | | | 269 |
| 26: LDL cholesterol after 26 weed appendix | ks of treatment – supportive stat | • | • | 275 |
| 27: VLDL cholesterol after 26 we appendix | eeks of treatment – supportive st | - | • | 281 |
| 28: Triglycerides after 26 weeks of appendix | of treatment – supportive statistic | • | • | 287 |
| 29: Total cholesterol after 26 wee appendix | ks of treatment – supportive stat | | | 293 |
| 30: Free fatty acid after 26 weeks appendix | of treatment – supportive statist | | | 299 |
| 31: Hypoglycaemic episodes – tre | eatment emergent – confirmator | y statistical analysi | s – full analysis se | et305 |
| 32: Hypoglycaemic episodes – tro<br>imputation – full analysis set | eatment emergent – statistical se | | • | 307 |
| 33: Hypoglycaemic episodes – tro | | | | |
| 34: Nocturnal hypoglycaemic epi analysis set | sodes – treatment emergent – su | | • | 313 |
| 35: Pulse after 26 weeks of treatmanalysis set - appendix | nent – change from baseline – su | * * | • | 320 |
| 36: Systolic blood pressure after 2 | | from baseline – suj | pportive statistical | 1 |
| 37: Diastolic blood pressure after | | from baseline – su | apportive statistica | ıl |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 3 of 334 | |

#### **Statistical documentation**

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 4 of 334 | |

# 1: Actual daily total insulin dose after 26 weeks of treatment – supportive statistical analysis – full analysis set - appendix

Parameter Code=TOTDDAC

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 450

Number of Observations

Number of Observations Read 453 Number of Observations Used 450 Number of Observations Not Used 3

Covariance Parameter Estimates

Cov Parm Estimate
Residual 109.52

Fit Statistics

-2 Res Log Likelihood 3384.2
AIC (Smaller is Better) 3386.2
AICC (Smaller is Better) 3386.2
BIC (Smaller is Better) 3390.3

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept 7.9327 4.2569 1.86 trtpn -3.3593 1.0472 -3.21 trtpn 2 Ω BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD -1.0335 0.9944 PREAD 445 -1.04 PREAD 0.4191 0.08246 5.08 INSSCR 445

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 5 of 334 | |

Actual daily total insulin dose after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

Parameter Code=TOTDDAC

The Mixed Procedure

#### Solution for Fixed Effects

| Solution for Fixed Effects | | | | | | |
|---|---|---|---|---|---|---|
| Effect<br>HBA1CBL | Pre Trial anti-Diabetic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Estimate | Standard<br>Error<br>0.4169 | DF<br>445 | t Value |
| | Solution for Fixed Effect | S | | | | |
| | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial anti-Diabetic treatment | 01 (N) | Pr > t | Alpha | | |
| Intercept<br>trtpn<br>trtpn | | 1 2 | 0.0631<br>0.0014 | 0.05<br>0.05 | | |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | ۷ | 0.2992 | 0.05 | | |
| INSSCR<br>HBA1CBL | DAGAD INCODIN + METICAMIN + ONE OTHER OAD | | <.0001<br><.0001 | 0.05<br>0.05 | | |
| | Solution for Fixed Effec | cts | | | | |
| | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial anti-Diabetic treatment | 01 (N) | Lower | Upper | | |
| Intercept<br>trtpn<br>trtpn | | 1 2 | -0.4334<br>-5.4174 | 16.2989<br>-1.3013 | | |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | -2.9879 | 0.9209 | | |
| INSSCR<br>HBA1CBL | BAGAL INCOLIN METFORMIN ONE OTHER OND | | 0.2571<br>1.3742 | 0.5812<br>3.0130 | | |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 1 | 445 | 10.29 | 0.0014 |
| PREAD | 1 | 445 | 1.08 | 0.2992 |
| INSSCR | 1 | 445 | 25.83 | <.0001 |
| HBA1CBL | 1 | 445 | 27.68 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | WORK.ADATA2 | 34.2145 | 0.6057 | 445 | 56.49 | <.0001 | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | 37.5739 | 0.8529 | 445 | 44.05 | <.0001 | 0.05 |

| | | | CONI | FIDENTIAL | Vers<br>Stati | Date: 22 Version: Status: Page: | | anuary 202<br>1<br>Fin<br>6 of 33 | .0<br>al |
|---|---|---|---|---|---|---|---|---|---|
| | Actual daily total insulin dose after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix | | | | | | | | |
| Paramet | er Code=TOT | 'DDAC | | | | | | | |
| The Mix | The Mixed Procedure | | | | | | | | |
| Least Squares Means Estimates | | | | | | | | | |
| Effect | Label | | Lower | Upper Exp | onentiated | Exponent | iated<br>Lower | Exponent | ciated<br>Upper |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | | | .4049<br>.2501 | 7.231E14<br>2.08E16 | | 99E14<br>92E15 | | 378E15<br>L12E17 |
| | | | Least Squ | ares Means | Estimate | | | | |
| Effect | Label | | | Margins | Estima | Stand<br>ate Er | lard | DF t | Value |
| trtpn | Treatment | contrast, | IDegLira - IDeg | WORK.ADAT | A2 -3.35 | 593 1.0 | 472 | 445 | -3.21 |
| | Least Squares Means Estimate | | | | | | | | |
| Effect | Label | | | Pr > t | Alpha | Lower | Upper | Exponent | ciated |
| trtpn | Treatment | contrast, | IDegLira - IDeg | 0.0014 | 0.05 - | -5.4174 - | 1.3013 | 0 . | .03476 |

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.004439 0.2722

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 7 of 334 | |

# 2: HbA1c after 26 weeks of treatment – change from baseline – confirmatory statistical analysis – full analysis set - appendix

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values TRTPN 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.7569

Fit Statistics

-2 Res Log Likelihood 1171.1 AIC (Smaller is Better) 1173.1 AICC (Smaller is Better) 1173.1 BIC (Smaller is Better) 1177.2

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept 4.8895 0.3187 449 TRTPN -0.9186 0.08674 TRTPN 2 0 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD -0.2401 PREAD 0.08191 449 -2.93 PREAD 0.3580 0.03449 BASE 449 10.38

| NN9068 | | Date: | 22 January 2020 Novo Nordis | sk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 8 of 334 | |

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=C64849B

| The Mixe | ed Procedure | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Solution for | Fixed Effec | cts | | | | |
| Intercep<br>TRTPN<br>TRTPN<br>PREAD<br>PREAD | BASAL INSULIN + | METFORMIN | 1<br>2 | Pr > t <.0001 <.0001 0.0036 | 0.0 | )5<br>)5<br>)5 | | |
| BASE | | | | | <.0001 | 0.0 | )5 | |
| Solution for Fixed Effects | | | | | | | | |
| Effect | Pre Trial anti-D | liabetic treatm | nent | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | . Uŗ | pper | |
| Intercep<br>TRTPN<br>TRTPN | pt | 1 2 | 4.2631<br>-1.0891 | | 5159<br>7481 | | | |
| PREAD BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | | -0.4010 | -0.07 | 7910 | |
| BASE | DAGAH INGULIN | METI OTHIN 1 OF | VE OTHER OA | | 0.2902 | 0.4 | 1258 | |
| | Type 3 Tests of Fix | ed Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value F | ?r > F | | | | | |
| TRTPN<br>PREAD<br>BASE | 1 449<br>1 449<br>1 449 | 8.59 ( | <.0001<br>0.0036<br><.0001 | | | | | |
| | | Least | Squares Mea | ans Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| TRTPN<br>TRTPN | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | | 449<br>449 | 140.98<br>112.65 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least So | quares Means | s Estimates | | | | |
| Effect | Label | Lower | Upper I | Exponentiated | | entiated<br>Lower | | ted<br>per |
| TRTPN<br>TRTPN | LSMeans, IDegLira<br>LSMeans, IDeg | 6.9601<br>7.8379 | 7.1569<br>8.1162 | 1162.68<br>2913.40 | | 1053.72<br>2534.89 | 1282<br>3348 | |
| | | Least S | Squares Mean | ns Estimate | | | | |
| Effect | Label | | Margins | s Estima | | ndard<br>Error | DF t Va | lue |

TRTPN Treatment contrast, IDegLira - IDeg WORK.ADATA2 -0.9186 0.08674 449 -10.59

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 9 of 334 | |

 $\label{thm:hbalc} \mbox{HbAlc after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix$ 

Parameter Code=C64849B

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated TRTPN Treatment contrast, IDegLira - IDeg <.0001 0.05 -1.0891 -0.7481 0.3991

Least Squares Means Estimate

Effect Label Exponentiated Lower Upper TRTPN Treatment contrast, IDegLira - IDeg 0.3365 Exponentiated O.4733

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

HbAlc after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

TRTPN 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453
Number of Observations Used 453
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate Residual 90.4255

Fit Statistics

-2 Res Log Likelihood 3323.4
AIC (Smaller is Better) 3325.4
AICC (Smaller is Better) 3325.4
BIC (Smaller is Better) 3329.5

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 38.3549 2.7080 449 14.16 Intercept -10.0402 0.9481 TRTPN 1 -10.59 449 TRTPN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -2.6239 0.8952 449 -2.93 PREAD 0.3580 BASE 0.03449 449 10.38

#### NN9068 22 January 2020 | Novo Nordisk Date: NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=HBA1CONV

| The Mixe | ed Procedu | re | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Solution for | Fixed Effec | ts | | | | |
| Effect<br>Intercep<br>TRTPN | | ial anti-D | iabetic treat | ment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t<br><.0003<br><.0003 | 1 0.0 | )5 | |
| TRTPN<br>PREAD<br>PREAD | | INSULIN + 1 | METFORMIN<br>METFORMIN + C | ONE OTHER OAD | 2 | 0.003 | | | |
| BASE | DIIGIIL | INCOLIN . | indii Oidiiii | AND OTHER ONE | , | <.0000 | 1 0.0 | )5 | |
| | | | Solution fo | r Fixed Effe | ects | | | | |
| T. F. C. C. T. | Duo III n | ial anti D | iabetic treat | | Planned<br>Treatment<br>for<br>Period | Lava | | | |
| | | Idi dilli-D | iabetic treat | ment | 01 (N) | Lowe | | oper | |
| Intercept<br>TRTPN<br>TRTPN | | | | | 1 2 | 33.0330 | | | |
| PREAD<br>PREAD | | INSULIN + 1<br>INSULIN + 1 | METFORMIN<br>METFORMIN + C | NE OTHER OAD | ) | -4.3832 | 2 -0.8 | 3645 | |
| BASE | | | | | | 0.290 | 2 0.4 | 1258 | |
| | Type 3 Te | sts of Fix | ed Effects | | | | | | |
| Effect | Num<br>DF | | F Value | Pr > F | | | | | |
| TRTPN<br>PREAD<br>BASE | 1<br>1<br>1 | 449 | 8.59 | <.0001<br>0.0036<br><.0001 | | | | | |
| | | | Least | : Squares Mea | ıns Estimates | | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| TRTPN<br>TRTPN | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADATA2<br>WORK.ADATA2 | 53.6492<br>63.6894 | 0.5473<br>0.7740 | 449<br>449 | 98.03<br>82.29 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least S | Squares Means | Estimates | | | | |
| Effect | Label | | Lower | Upper E | Exponentiated | | entiated<br>Lower | - | ted<br>per |
| TRTPN<br>TRTPN | LSMeans,<br>LSMeans, | | | 54.7247<br>65.2106 | 1.993E23<br>4.571E27 | | 6.799E22<br>9.985E26 | 5.843<br>2.092 | |
| | | | Least | Squares Mean | s Estimate | | | | |
| Effect | Label | | | Margins | Estima | | andard<br>Error | DF t Va | lue |

TRTPN Treatment contrast, IDegLira - IDeg WORK.ADATA2 -10.0402 0.9481 449 -10.59

| NN9068 | | Date: | 22 January 2020 Novo Nordisk |
|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final |
| Statistical document | | Page: | 12 of 334 |

 $\label{thm:hbalc} \mbox{HbAlc after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix$ 

Parameter Code=HBA1CONV

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated TRTPN Treatment contrast, IDegLira - IDeg <.0001 0.05 -11.9034 -8.1770 0.000044

Least Squares Means Estimate

Exponentiated Lower Upper TRTPN Treatment contrast, IDegLira - IDeg 6.767E-6 0.000281


HbAlc after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

TRTPN 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453
Number of Observations Used 453
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.7569

Fit Statistics

-2 Res Log Likelihood 1171.1 AIC (Smaller is Better) 1173.1 AICC (Smaller is Better) 1173.1 BIC (Smaller is Better) 1177.2

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 4.8895 449 0.3187 15.34 Intercept -0.9186 0.08674 TRTPN -10.59 449 TRTPN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.2401 0.08191 449 -2.93 PREAD -0.6420 BASE 0.03449 449 -18.61


 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=C64849B

The Mixed Procedure

#### Solution for Fixed Effects

| Solution for Fixed Effects | | | | | | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| | | | | 1 2 | <.0001<br><.0001 | 0.05<br>0.05 | |
| PREAD | BASAL INS | | | 2 | 0.0036 | 0.05 | |
| PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD BASE | | | | | <.0001 | 0.05 | |
| | Solution for Fixed Effects | | | | | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>TRTPN<br>TRTPN | | | | | 1 2 | 4.2631<br>-1.0891 | 5.5159<br>-0.7481 |
| PREAD<br>PREAD | | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | -0.4010 | -0.07910 |
| BASE | DASAL INS | OLIN T I | MEIFORMIN T | ONE OTHER OAD | | -0.7098 | -0.5742 |
| Ту | pe 3 Tests | of Fixe | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| TRTPN<br>PREAD<br>BASE | 1<br>1<br>1 | 449<br>449<br>449 | 112.15<br>8.59<br>346.39 | <.0001<br>0.0036<br><.0001 | | | |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| TRTPN<br>TRTPN | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.05007<br>0.07082 | 449<br>449 | -37.64<br>-13.64 | <.0001<br><.0001 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| TRTPN<br>TRTPN | Change from baseline, IDegLira<br>Change from baseline, IDeg | | -1.9827<br>-1.1049 | -1.7859<br>-0.8266 | | | |


HbAlc after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

TRTPN 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453
Number of Observations Used 453
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 90.4255

Fit Statistics

-2 Res Log Likelihood 3323.4
AIC (Smaller is Better) 3325.4
AICC (Smaller is Better) 3325.4
BIC (Smaller is Better) 3329.5

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 38.3549 2.7080 449 14.16 Intercept -10.0402 TRTPN 0.9481 -10.59 449 TRTPN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -2.6239 0.8952 449 -2.93 PREAD -0.6420 BASE 0.03449 449 -18.61
#### NN9068 Date: 22 January 2020 | Novo Nordisk NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 16 of 334 Statistical document Page:

HbAlc after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=HBA1CONV

The Mixed Procedure

| Solution for Fixed Effects | | | | | | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-Di | abetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>TRTPN<br>TRTPN | | | | | 1 2 | <.0001<br><.0001 | 0.05<br>0.05 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | ۷ | 0.0036 | 0.05 |
| BASE BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | | <.0001 | 0.05 | |
| | Solution for Fixed Effects | | | | | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-Di | abetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>TRTPN<br>TRTPN | | | | | 1 2 | 33.0330<br>-11.9034 | 43.6767<br>-8.1770 |
| PREAD<br>PREAD | BASAL INS | | | ONE OTHER OAD | _ | -4.3832 | -0.8645 |
| BASE | DASAL INS | OLIN I P | EIFORMIN ( | ONE OTHER OAD | | -0.7098 | -0.5742 |
| Т | pe 3 Tests | of Fixe | d Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| TRTPN<br>PREAD<br>BASE | 1<br>1<br>1 | 449<br>449<br>449 | 112.15<br>8.59<br>346.39 | <.0001<br>0.0036<br><.0001 | | | |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| TRTPN<br>TRTPN | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.5473<br>0.7740 | 449<br>449 | -37.64<br>-13.64 | <.0001<br><.0001 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| TRTPN<br>TRTPN | Change from baseline, IDegLira<br>Change from baseline, IDeg | | 21.6714 | -19.5204<br>-9.0345 | | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 17 of 334 | |

### 3: HbA1c after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – PP analysis set - appendix

Parameter Code=C64849B

Levels

The Mixed Procedure

Class

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

trtan 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Values

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 431

Number of Observations

Number of Observations Read 431 Number of Observations Used 431 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.7326

Fit Statistics

-2 Res Log Likelihood 1100.6
AIC (Smaller is Better) 1102.6
AICC (Smaller is Better) 1102.6
BIC (Smaller is Better) 1106.6

Solution for Fixed Effects

Actual Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept 4.9698 0.3237 15.35 trtan -0.9065 0.08773 427 -10.33 trtan 2 Λ BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD -0.2699 PREAD 0.08260 427 -3.27 PREAD 0.3456 0.03506 9.86 BASE 427

#### NN9068 22 January 2020 | Novo Nordisk Date: NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

 $\label{thm:balc} \mbox{HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix$ 

Parameter Code=C64849B

| The Mixe | ed Procedure | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Solution for | Fixed Effec | ts | | | | |
| Effect<br>Intercer<br>trtan<br>trtan<br>PREAD<br>PREAD | BASAL INSULIN + | METFORMIN | | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t<br><.000<br><.000<br>0.001 | 1 0. | 05<br>05 | |
| BASE | | | | | <.000 | 1 0. | 05 | |
| | | Solution for | Fixed Effe | cts | | | | |
| Effect | Pre Trial anti-I | Diabetic treatm | nent | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lowe | r Uj | pper | |
| Intercep<br>trtan | pt | | | 1 | 4.333<br>-1.079 | | 6061<br>7341 | |
| trtan<br>PREAD | PREAD BASAL INSULIN + METFORMIN | | | 2 | -0.432 | 2 -0. | 1075 | |
| PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD BASE | | | | 0.276 | 7 0. | 4145 | | |
| | Type 3 Tests of Fix | ed Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value F | r > F | | | | | |
| trtan<br>PREAD<br>BASE | 1 427<br>1 427<br>1 427 | 10.67 | 3.0001<br>0.0012<br>3.0001 | | | | | |
| | | Least | Squares Mea | ns Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtan<br>trtan | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.05035<br>0.07183 | 427<br>427 | 139.64<br>110.50 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least So | quares Means | Estimates | | | | |
| Effect | Label | Lower | Upper E | xponentiated | | entiated<br>Lower | Exponentia<br>Up | ted<br>per |
| trtan<br>trtan | | 6.9318<br>7.7961 | 7.1298<br>8.0785 | 1130.93<br>2799.86 | | 1024.37<br>2431.19 | 1248<br>3224 | |
| | | Least S | Squares Mean | s Estimate | | | | |
| Effect | Label | | Margins | Estim | | andard<br>Error | DF t Va | lue |

trtan Treatment contrast, IDegLira - IDeg WORK.ADATA2

427 -10.33

-0.9065 0.08773

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
5tatus:
Final
Page:

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=C64849B

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtan Treatment contrast, IDegLira - IDeg <.0001 0.05 -1.0790 -0.7341 0.4039

Least Squares Means Estimate

Exponentiated Lower Upper trtan Treatment contrast, IDegLira - IDeg 0.3399 0.4799


HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtan 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 431

Number of Observations

Number of Observations Read 431
Number of Observations Used 431
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 87.5168

Fit Statistics

-2 Res Log Likelihood 3147.7 AIC (Smaller is Better) 3149.7 AICC (Smaller is Better) 3149.7 BIC (Smaller is Better) 3153.8

Solution for Fixed Effects

Actual

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 38.9418 2.7492 427 14.16 Intercept -9.9084 0.9589 1 -10.33 427 trtan trtan BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -2.9498 427 -3.27 PREAD 0.3456 BASE 0.03506 427 9.86

# NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

 $\label{thm:balc} \mbox{HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix$ 

Parameter Code=HBA1CONV

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial anti-D: | abetic treatmen | n† | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | а | |
|---|---|---|---|---|---|---|---|---|
| | | abetic treatmen | .10 | 01 (11) | | - | | |
| Intercep<br>trtan | t | | | 1 | <.0001<br><.0001 | 0.0 | | |
| trtan<br>PREAD | BASAL INSULIN + N | METFORMIN | | 2 | 0.0012 | 0.0 | 5 | |
| PREAD<br>BASE | BASAL INSULIN + N | METFORMIN + ONE | OTHER OAD | | <.0001 | 0.0 | 5 | |
| | | Solution for H | Fixed Effec | ts | | | | |
| | | | | Actual<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial anti-Di | abetic treatmen | nt | 01 (N) | Lower | Up | per | |
| Intercep<br>trtan<br>trtan | t | | | 1 2 | 33.5380<br>-11.7931 | 44.3<br>-8.0 | | |
| PREAD<br>PREAD | BASAL INSULIN + N | | OMITED OND | _ | -4.7244 | -1.1 | 752 | |
| BASE | | | | | 0.2767 | 0.4 | 145 | |
| | Type 3 Tests of Fixe | ed Effects | | | | | | |
| | Num Den | | | | | | | |
| Effect | DF DF | F Value Pr | > F | | | | | |
| trtan<br>PREAD<br>BASE | 1 427<br>1 427<br>1 427 | 10.67 0.0 | 0001<br>0012<br>0001 | | | | | |
| | | Least So | quares Mean | s Estimates | | | | |
| | | | - | Standard | | | | |
| Effect | Label | Margins | Estimate | Error | DF t | Value | Pr > t | Alpha |
| | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 53.3466<br>63.2550 | 0.5503<br>0.7851 | 427<br>427 | 96.94<br>80.57 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least Squa | ares Means | Estimates | | | | |
| Effect | Label | Lower | Upper Ex | ponentiated | | tiated<br>Lower | | ted<br>per |
| | LSMeans, IDegLira<br>LSMeans, IDeg | | 4.4283<br>4.7982 | 1.473E23<br>2.96E27 | | 993E22<br>325E26 | 4.344<br>1.385 | |
| | | Least Squ | uares Means | Estimate | | | | |
| | | | | | Stan | ıdard | | |
| Effect | Label | | Margins | Estim | ate E | rror | DF t Va | lue |

trtan Treatment contrast, IDegLira - IDeg WORK.ADATA2 -9.9084 0.9589 427 -10.33

NN9068 Date: 22 January 2020 Novo Nordisk
NN9068-4166 Version: 1.0
Clinical Trial Report Status: Final
Statistical document 

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=HBA1CONV

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtan Treatment contrast, IDegLira - IDeg <.0001 0.05 -11.7931 -8.0237 0.000050

Least Squares Means Estimate

Exponentiated Lower Upper trtan Treatment contrast, IDegLira - IDeg 7.557E-6 0.000328


HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtan 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 431

Number of Observations

Number of Observations Read 431 Number of Observations Used 431 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.7326

Fit Statistics

-2 Res Log Likelihood 1100.6 AIC (Smaller is Better) 1102.6 AICC (Smaller is Better) 1102.6 BIC (Smaller is Better) 1106.6

Solution for Fixed Effects

Actual Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 4.9698 0.3237 427 15.35 Intercept -0.9065 0.08773 -10.33 427 trtan trtan BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.2699 0.08260 427 -3.27 PREAD -0.6544 BASE 0.03506 427 -18.66

#### NN9068 Date: 22 January 2020 | Novo Nordisk NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 24 of 334 Statistical document Page:

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=C64849B

The Mixed Procedure

### Solution for Fixed Effects

| | | | Solution f | or Fixed Effect | ts | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-D | iabetic tre | atment | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtan | | | | | 1 | <.0001<br><.0001 | 0.05<br>0.05 |
| trtan<br>PREAD<br>PREAD | BASAL INS | | | ONE OTHER OAD | 2 | 0.0012 | 0.05 |
| BASE | BASE | | | | | <.0001 | 0.05 |
| | | | Solution | for Fixed Effec | cts | | |
| | | | | | Actual<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtan<br>trtan | | | | | 1<br>2 | 4.3335<br>-1.0790 | 5.6061<br>-0.7341 |
| PREAD<br>PREAD | BASAL INS | | | ONE OTHER OAD | | -0.4322 | -0.1075 |
| BASE | | | | | | -0.7233 | -0.5855 |
| Ту | rpe 3 Tests | of Fix | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| DIICCC | | | | | | | |
| trtan<br>PREAD<br>BASE | 1<br>1<br>1 | 427<br>427<br>427 | 106.78<br>10.67 | 0.0012 | | | |

| Effect | DF | DF | F Value | Pr > F |
|--------|----|-----|---------|--------|
| trtan | 1 | 427 | 106.78 | <.0001 |
| PREAD | 1 | 427 | 10.67 | 0.0012 |
| BASE | 1 | 427 | 348.31 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.05035<br>0.07183 | 427<br>427 | -38.23<br>-14.18 | <.0001<br><.0001 |
| | Least Squares Mean | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg | | -2.0241<br>-1.1598 | -1.8262<br>-0.8774 | | | |


HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtan 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 431

Number of Observations

Number of Observations Read 431
Number of Observations Used 431
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 87.5168

Fit Statistics

-2 Res Log Likelihood 3147.7 AIC (Smaller is Better) 3149.7 AICC (Smaller is Better) 3149.7 BIC (Smaller is Better) 3153.8

Solution for Fixed Effects

Actual Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 38.9418 2.7492 427 14.16 Intercept -9.9084 0.9589 427 -10.33 trtan trtan BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -2.9498 0.9029 427 -3.27 PREAD -0.6544 BASE 0.03506 427 -18.66

# NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=HBA1CONV

The Mixed Procedure

### Solution for Fixed Effects

| | | | Solution I | or Fixed Effec | ts | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-D | iabetic tre | atment | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtan<br>trtan | | | | | 1 | <.0001<br><.0001 | 0.05<br>0.05 |
| PREAD | BASAL INSU | | | | _ | 0.0012 | 0.05 |
| PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD BASE | | | | <.0001 | 0.05 | | |
| | | | Solution | for Fixed Effe | cts | | |
| | | | | | Actual<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtan<br>trtan | | | | | 1 | 33.5380<br>-11.7931 | 44.3455<br>-8.0237 |
| PREAD<br>PREAD | BASAL INSU | | | ONE OTHER OAD | _ | -4.7244 | -1.1752 |
| BASE | BASAL INS | JLIN + 1 | MEIFORMIN + | ONE OTHER OAD | | -0.7233 | -0.5855 |
| Ту | rpe 3 Tests | of Fix | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtan<br>PREAD<br>BASE | 1<br>1<br>1 | 427<br>427<br>427 | 106.78<br>10.67<br>348.31 | <.0001<br>0.0012<br><.0001 | | | |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.5503<br>0.7851 | 427<br>427 | -38.23<br>-14.18 | <.0001<br><.0001 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg | | 22.1233 | -19.9599<br>-9.5900 | | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 27 of 334 | |

## 4: HbA1c after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – completer analysis set - appendix

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 429

Number of Observations

Number of Observations Read 429 Number of Observations Used 429 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.7214

Fit Statistics

-2 Res Log Likelihood 1089.0 AIC (Smaller is Better) 1091.0 AICC (Smaller is Better) 1091.0 BIC (Smaller is Better) 1095.0

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept 4.9165 0.3212 425 trtpn -0.8833 0.08766 -10.08 trtpn 2 Ω BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD -0.2517 PREAD 0.08217 425 -3.06 PREAD 0.3478 0.03473 425 10.01 BASE

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 28 of 334 | |

 $\label{thm:hbalc} \mbox{HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set - appendix$ 

Parameter Code=C64849B

The Mixed Procedure

### Solution for Fixed Effects

| | | Solution fo | r Fixed Effec | ts | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial a | nti-Diabetic trea | tment | 01 (N) | Pr > t | Alph | ıa | |
| Interce<br>trtpn<br>trtpn | pt | | | 1<br>2 | <.0001<br><.0001 | | | |
| PREAD<br>PREAD | | IN + METFORMIN IN + METFORMIN + | OME OTHER OAD | | 0.0023 | 0.0 | )5 | |
| BASE | DASAL INSUL | IN PERCONTIN | ONE OTHER OAD | | <.0001 | 0.0 | )5 | |
| | | Solution f | or Fixed Effe | cts | | | | |
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| | | nti-Diabetic trea | tment | 01 (N) | Lower | - | pper | |
| Interce<br>trtpn | pt | | | 1 | 4.2851<br>-1.0556 | | 3479<br>7110 | |
| trtpn<br>PREAD | | IN + METFORMIN | | 2 | -0.4132 | -0.09 | 016 | |
| PREAD<br>BASE | BASAL INSUL | IN + METFORMIN + | ONE OTHER OAD | ) | 0.2795 | 5 0.4 | 1160 | |
| | Type 3 Tests o | f Fixed Effects | | | | | | |
| Effect | | Den<br>DF F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 | 425 101.54<br>425 9.38<br>425 100.29 | <.0001<br>0.0023<br><.0001 | | | | | |
| | | Leas | t Squares Mea | ns Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDeg | | | 0.04988<br>0.07206 | 425<br>425 | 140.90<br>109.79 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least | Squares Means | Estimates | | | | |
| Effect | Label | Lower | Upper E | xponentiated | | entiated<br>Lower | | ted<br>per |
| trtpn<br>trtpn | LSMeans, IDeg<br>LSMeans, IDeg | | 7.1265<br>8.0534 | 1128.32<br>2729.27 | | 1022.95<br>2368.82 | 1244<br>3144 | |
| | | Least | Squares Mean | s Estimate | | | | |
| Effect | Label | | Margins | Estim | | andard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -0.8833 0.08766 425 -10.08

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set - appendix

Parameter Code=C64849B

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg <.0001 0.05 -1.0556 -0.7110 0.4134

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.3480 0.4912

# NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set - appendix

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 429

Number of Observations

Number of Observations Read 429
Number of Observations Used 429
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate Residual 86.1783

Fit Statistics

-2 Res Log Likelihood 3126.5 AIC (Smaller is Better) 3128.5 AICC (Smaller is Better) 3128.5 BIC (Smaller is Better) 3132.6

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 38.4099 425 14.07 2.7306 Intercept -9.6545 0.9581 -10.08 1 425 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -2.7507 0.8981 425 -3.06 PREAD 0.3478 BASE 0.03473 425 10.01

| NN9068 | | Date: | 22 January 2020 Novo Nordisk |
|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final |
| Statistical document | | Page: | 31 of 334 |

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set - appendix

Parameter Code=HBA1CONV

The Mixed Procedure

| | | Solution for | Fixed Effe | cts | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial anti-D | iabetic treatme | ent | 01 (N) | Pr > t | Alph | ha | |
| Intercep<br>trtpn<br>trtpn | t | | | 1 2 | <.0001<br><.0001 | | | |
| PREAD<br>PREAD | BASAL INSULIN +<br>BASAL INSULIN + | | E OTHER OA | _ | 0.0023 | 3 0.0 | 05 | |
| BASE | BRIGHT TROUBLY | | D OTHER OH | 5 | <.0001 | 1 0.0 | 05 | |
| | | Solution for | Fixed Eff | ects | | | | |
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial anti-D | iabetic treatme | ent | 01 (N) | Lower | r Ug | pper | |
| Intercep<br>trtpn<br>trtpn | t | | | 1 2 | 33.0428<br>-11.5377 | | | |
| PREAD<br>PREAD | BASAL INSULIN + | | E OTHED OX | _ | -4.5160 | -0.9 | 9855 | |
| PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD<br>BASE | | | | D | 0.2795 | 5 0.4 | 4160 | |
| | Type 3 Tests of Fix | ed Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value P | r > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 425<br>1 425<br>1 425 | 9.38 0 | .0001<br>.0023<br>.0001 | | | | | |
| | | Least | Squares Me | ans Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 53.3214<br>62.9758 | | 425<br>425 | 97.80<br>79.96 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least Sq | uares Mean | s Estimates | | | | |
| Effect | Label | Lower | Upper | Exponentiated | | entiated<br>Lower | Exponentia<br>Up | ted |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | | 54.3930<br>64.5240 | 1.436E23<br>2.239E27 | | 4.918E22<br>4.761E26 | 4.194<br>1.053 | |
| | | Least So | quares Mea | ns Estimate | | | | |
| Effect | Label | | Margin | s Estim | | andard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -9.6545 0.9581 425 -10.08

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set - appendix

Parameter Code=HBA1CONV

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg < .0001 0.05 -11.5377 -7.7713 0.000064

Least Squares Means Estimate

Effect Label Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 9.756E-6 0.000422

# NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set - appendix

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 429

Number of Observations

Number of Observations Read 429
Number of Observations Used 429
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.7214

Fit Statistics

-2 Res Log Likelihood 1089.0
AIC (Smaller is Better) 1091.0
BIC (Smaller is Better) 1095.0

Solution for Fixed Effects

Planned

Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 0.3212 4.9165 425 15.31 Intercept 0.08766 -10.08 1 -0.8833 425 trtpn trtpn BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.2517 0.08217 425 -3.06 PREAD -0.6522 BASE 0.03473 425 -18.78

#### NN9068 Date: 22 January 2020 | Novo Nordisk NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 34 of 334 Statistical document Page:

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set - appendix

Parameter Code=C64849B

The Mixed Procedure

| | | | Solution f | or Fixed Effect | ES | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-Di | abetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn | | | | | 1 2 | <.0001<br><.0001 | 0.05<br>0.05 |
| trtpn<br>PREAD<br>PREAD | BASAL INSU | | | ONE OTHER OAD | 2 | 0.0023 | 0.05 |
| BASE | | | | | | <.0001 | 0.05 |
| | | | Solution | for Fixed Effec | cts | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-Di | abetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn<br>PREAD | BASAL INSU | IT TN 4 N | TETEODMIN | | 1 2 | 4.2851<br>-1.0556<br>-0.4132 | 5.5479<br>-0.7110<br>-0.09016 |
| PREAD | | | | ONE OTHER OAD | | | |
| BASE | | | | | | -0.7205 | -0.5840 |
| Ту | rpe 3 Tests | of Fixe | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 425<br>425<br>425 | 101.54<br>9.38<br>352.70 | <.0001<br>0.0023<br><.0001 | | | |

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| trtpn | 1 | 425 | 101.54 | <.0001 |
| PREAD | 1 | 425 | 9.38 | 0.0023 |
| BASE | 1 | 425 | 352.70 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.04988<br>0.07206 | 425<br>425 | -38.65<br>-14.50 | <.0001<br><.0001 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | | -2.0262<br>-1.1865 | -1.8301<br>-0.9032 | | | |

# NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set - appendix

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 429

Number of Observations

Number of Observations Read 429
Number of Observations Used 429
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate Residual 86.1783

Fit Statistics

-2 Res Log Likelihood 3126.5 AIC (Smaller is Better) 3128.5 AICC (Smaller is Better) 3128.5 BIC (Smaller is Better) 3132.6

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 38.4099 14.07 2.7306 425 Intercept -9.6545 0.9581 1 425 -10.08 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -2.7507 0.8981 425 -3.06 PREAD -0.6522 BASE 0.03473 425 -18.78

#### NN9068 Date: 22 January 2020 | Novo Nordisk NN9068-4166 Version: 1.0 CONFIDENTIAL Final Clinical Trial Report Status: 36 of 334 Statistical document Page:

 $\label{thm:hbalc} \mbox{HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set - appendix$ 

Parameter Code=HBA1CONV

The Mixed Procedure

| | | | Solution f | or Fixed Effect | ts | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | . anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn | | | | | 1 2 | <.0001<br><.0001 | 0.05<br>0.05 |
| trtpn<br>PREAD<br>PREAD | BASAL INS | | | ONE OTHER OAD | _ | 0.0023 | 0.05 |
| BASE | D1101112 1110 | 0221 | | 0112 0111211 0112 | | <.0001 | 0.05 |
| | | | Solution | for Fixed Effe | cts | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | 33.0428<br>-11.5377 | 43.7771<br>-7.7713 |
| PREAD<br>PREAD | BASAL INS | | | ONE OTHER OAD | | -4.5160 | -0.9855 |
| BASE | DIIOIIE IIVO | OBIN I | IIIII OIUIII | ONE OTHER ONE | | -0.7205 | -0.5840 |
| Ту | pe 3 Tests | of Fix | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 425<br>425<br>425 | 101.54<br>9.38<br>352.70 | <.0001<br>0.0023<br><.0001 | | | |

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| trtpn | 1 | 425 | 101.54 | <.0001 |
| PREAD | 1 | 425 | 9.38 | 0.0023 |
| BASE | 1 | 425 | 352.70 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.5452<br>0.7876 | 425<br>425 | -38.65<br>-14.50 | <.0001<br><.0001 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | | 22.1464 | -20.0031<br>-9.8722 | | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 37 of 334 | |

## 5: HbA1c after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – MMRM – full analysis set - appendix

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

### Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method

WORK.ANA\_DATA
AVAL
Unstructured
SUBJID
REML
None
Model-Based
Satterthwaite

### Class Level Information

| Class | Levels | Values |
|---|---|---|
| TRT01PN<br>AVISITN<br>PREAD | 2<br>6<br>2 | 1 2<br>100 150 190 230 270 330<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN +<br>ONE OTHER OAD |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 38 of 334 | |

 $\label{thm:main_model} \begin{tabular}{ll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \\ \end{tabular}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

Class Level Information

Class Levels Values
SUBJID 453



| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 39 of 334 | |

 $\label{thm:main_model} \begin{tabular}{lll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \end{tabular}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure



### Dimensions

| Covariance | Parameters | 21 |
|-------------|------------|-----|
| Columns in | | 31 |
| Columns in | Z | 0 |
| Subjects | | 453 |
| Max Obs per | r Subject | 6 |

### Number of Observations

| Number | of | Observations | Read | 2718 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2595 |
| Number | of | Observations | Not Used | 123 |

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5tatus: Final 

 $\label{thm:main_model} \begin{tabular}{lll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \end{tabular}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

### Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|---|---|---|---|
| 0<br>1<br>2<br>3<br>4 | 1<br>2<br>1<br>1 | 6180.47425772<br>2415.05948115<br>2411.88149460<br>2411.76403647<br>2411.76380269 | 0.00247120<br>0.00009868<br>0.00000020<br>0.00000000 |

Convergence criteria met.

### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|---|---|---|
| UN (1,1)<br>UN (2,1)<br>UN (2,2)<br>UN (3,1)<br>UN (3,2)<br>UN (4,1)<br>UN (4,2)<br>UN (4,3)<br>UN (4,4)<br>UN (5,1)<br>UN (5,1)<br>UN (5,2)<br>UN (5,3)<br>UN (5,5)<br>UN (6,1)<br>UN (6,2) | Subject SUBJID | 0.3328<br>0.3392<br>0.5343<br>0.2998<br>0.5436<br>0.6809<br>0.2578<br>0.4980<br>0.6498<br>0.7191<br>0.2311<br>0.4455<br>0.5985<br>0.6761<br>0.7336<br>0.2068<br>0.4124<br>0.5440 |
| UN (6,4)<br>UN (6,5)<br>UN (6,6) | SUBJID<br>SUBJID<br>SUBJID | 0.6102<br>0.6641<br>0.7317 |

### Fit Statistics

| -2 Res Log Likelihood | 2411.8 |
|--------------------------|--------|
| AIC (Smaller is Better) | 2453.8 |
| AICC (Smaller is Better) | 2454.1 |
| BIC (Smaller is Better) | 2540.2 |

### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 20 | 3768.71 | <.0001 |

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|-------------------|-----------|-----------|---------|--------|
| TRT01PN (AVISITN) | 6 | 435 | 35.96 | <.0001 |
| PREAD(AVISITN) | 6 | 432 | 2.36 | 0.0293 |
| BASE (AVISITN) | 6 | 433 | 213.91 | <.0001 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 41 of 334 | |

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| TRT01PN (AVISITN) TRT01PN (AVISITN) | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ANA_DATA | | 0.05012<br>0.07142 | 427.4<br>437.4 | 140.29<br>111.28 | <.0001<br><.0001 |
| | Least Squares Mea | ns Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| TRT01PN (AVISITN) TRT01PN (AVISITN) | LSMeans, IDegLira<br>LSMeans, IDeg | | | 7.1294<br>8.0883 | | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 42 of 334 | |

 $\label{thm:main_model} \begin{tabular}{ll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \\ \end{tabular}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

### Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method

NORK.ANA\_DATA
AVAL
Unstructured
SUBJID
REML
None
Model-Based
Satterthwaite

#### Class Level Information

| Class Levels | Values |
|---|---|
| AVISITN 6 PREAD 2 1 | 1 2<br>100 150 190 230 270 330<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN +<br>ONE OTHER OAD |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 43 of 334 | |

 $\label{thm:main_model} \begin{tabular}{ll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \\ \end{tabular}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

Class Level Information

Levels Values Class SUBJID 453

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 44 of 334 | |

 $\label{thm:main_model} \begin{tabular}{lll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \end{tabular}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure



### Dimensions

| Covariance | Parameters | 21 |
|-------------|------------|-----|
| Columns in | X | 31 |
| Columns in | Z | 0 |
| Subjects | | 453 |
| Max Obs per | Subject | 6 |

### Number of Observations

| Number | of | Observations | Read | 2718 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2595 |
| Number | of | Observations | Not Used | 123 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 45 of 334 | |

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

### Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 18506.32350920 | |
| 1 | 2 | 14740.90873263 | 0.00056998 |
| 2 | 1 | 14737.73074608 | 0.00002280 |
| 3 | 1 | 14737.61328795 | 0.0000005 |
| 4 | 1 | 14737.61305417 | 0.00000000 |

Convergence criteria met.

### Covariance Parameter Estimates

### Fit Statistics

| -2 Res Log Likelihood | 14737.6 |
|--------------------------|---------|
| AIC (Smaller is Better) | 14779.6 |
| AICC (Smaller is Better) | 14780.0 |
| BIC (Smaller is Better) | 14866.0 |

### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 20 | 3768.71 | <.0001 |

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---|---|---|---|---|
| TRT01PN(AVISITN) PREAD(AVISITN) | 6 | 435<br>432 | 35.96<br>2.36 | <.0001<br>0.0293 |
| BASE (AVISITN) | 6 | 432 | 213.91 | <.0001 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 46 of 334 | |

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| TRT01PN (AVISITN) TRT01PN (AVISITN) | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ANA_DATA<br>WORK.ANA_DATA | 53.3477<br>63.3707 | 0.5478<br>0.7806 | 427.4<br>437.4 | 97.39<br>81.18 | <.0001<br><.0001 |
| | Least Squares Mea | ans Estimates | | | | | |
| Effect | Label | Alpha I | Lower | Upper | | | |
| TRT01PN (AVISITN)<br>TRT01PN (AVISITN) | LSMeans, IDegLira<br>LSMeans, IDeg | | | 4.4243 | | | |

| NN9068 | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|
| Clinical Trial Report | Status: | Final | |
| Statistical document | Page: | 47 of 334 | |

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

### Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Subject Effect
Subject Effect
Subject Effect
Subject Effect
Subject
Stimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Satterthwaite

#### Class Level Information

| Class | Levels | Values |
|---|---|---|
| TRT01PN<br>AVISITN<br>PREAD | 2<br>6<br>2 | 1 2<br>100 150 190 230 270 330<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN +<br>ONE OTHER OAD |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 48 of 334 | |

 $\label{thm:main_model} \begin{tabular}{ll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \\ \end{tabular}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

Class Level Information

Levels Values Class SUBJID 453

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 49 of 334 | |

 $\label{thm:main_model} \begin{tabular}{lll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \end{tabular}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure



### Dimensions

| Covariance | Parameters | 21 |
|------------|------------|-----|
| Columns in | | 31 |
| Columns in | Z | 0 |
| Subjects | | 453 |
| Max Obs pe | r Subject | 6 |

### Number of Observations

| Number | of | Observations | Read | 2718 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2595 |
| Number | of | Observations | Not Used | 123 |

# NN9068 | Date: 22 January 2020 | Novo Nordisk NN9068-4166 | CONFIDENTIAL | Status: Final |  |

 $\label{thm:main_model} \begin{tabular}{lll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \end{tabular}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

### Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|---|---|---|---|
| 0<br>1<br>2<br>3<br>4 | 1<br>2<br>1<br>1 | 6180.47425772<br>2415.05948115<br>2411.88149460<br>2411.76403647<br>2411.76380269 | 0.00247120<br>0.00009868<br>0.00000020<br>0.00000000 |

Convergence criteria met.

### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|---|---|---|
| UN (1,1)<br>UN (2,1)<br>UN (2,2)<br>UN (3,1)<br>UN (3,2)<br>UN (3,3)<br>UN (4,1)<br>UN (4,2)<br>UN (4,3)<br>UN (5,1)<br>UN (5,5)<br>UN (5,5) | Subject SUBJID | 0.3328<br>0.3392<br>0.5343<br>0.2998<br>0.5436<br>0.6809<br>0.2578<br>0.4980<br>0.6498<br>0.7191<br>0.2311<br>0.4455<br>0.5985<br>0.6761<br>0.7336<br>0.2068 |
| | SUBJID<br>SUBJID<br>SUBJID<br>SUBJID | 0.5440<br>0.6102<br>0.6641<br>0.7317 |

### Fit Statistics

| -2 Res Log Likelihood | 2411.8 |
|--------------------------|--------|
| AIC (Smaller is Better) | 2453.8 |
| AICC (Smaller is Better) | 2454.1 |
| BIC (Smaller is Better) | 2540.2 |

### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 20 | 3768.71 | <.0001 |

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|-----------|---------|--------|
| TRT01PN(AVISITN) | 6 | 435 | 35.96 | <.0001 |
| PREAD (AVISITN) | 6 | 432 | 2.36 | 0.0293 |
| BASE (AVISITN) | 6 | 433 | 65.36 | <.0001 |

| NN9068 | | Date: | 22 January 2020 <b>No</b> | vo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 51 of 334 | |

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

| Effect | Label | Margins | Estimate | Standard<br>Error | | t Value |
|---|---|---|---|---|---|---|
| TRT01PN (AVISITN) TRT01PN (AVISITN) | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ANA_DATA<br>WORK.ANA_DATA | | | 2 427.4<br>2 437.4 | -38.59<br>-14.24 |
| Least Squares Means Estimates | | | | | | |
| Effect | Label | Pr > t A | Alpha | Lower | Upper | |
| TRT01PN (AVISITN)<br>TRT01PN (AVISITN) | Change from baseline, IDegLira Change from baseline, IDeg | | | 2.0326 | -1.8356<br>-0.8767 | |
| Least Squares Means Estimate | | | | | | |
| Effect | Label | Margins | Est | imate | Standard<br>Error | DF |
| TRT01PN (AVISITN) | Treatment contrast, IDegLira - | IDeg WORK.ANA_ | _DATA -0 | .9170 | 0.08726 | 434.1 |
| Least Squares Means Estimate | | | | | | |
| Effect | Label | t Value | Pr > t | Alpha | Lower | Upper |
| TRT01PN (AVISITN) | Treatment contrast, IDegLira - | IDeg -10.51 | <.0001 | 0.05 | -1.0885 | -0.7455 |
| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 52 of 334 | |

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

## Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Subject Effect
Stimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Satterthwaite

Class Level Information

| Class | Levels | Values |
|---|---|---|
| TRT01PN<br>AVISITN<br>PREAD | 2<br>6<br>2 | 1 2<br>100 150 190 230 270 330<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN +<br>ONE OTHER OAD |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 53 of 334 | |

 $\label{thm:main_model} \begin{tabular}{ll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \\ \end{tabular}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

Class Level Information

Levels Values Class SUBJID 453

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 54 of 334 | |

 $\label{thm:main_model} \begin{tabular}{lll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \end{tabular}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure



## Dimensions

| Covariance | Parameters | 2.1 |
|-------------|------------|-----|
| Columns in | | 31 |
| Columns in | Z | 0 |
| Subjects | | 453 |
| Max Obs per | r Subject | 6 |

## Number of Observations

| Number | of | Observations | Read | 2718 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2595 |
| Number | of | Observations | Not Used | 123 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 55 of 334 | |

 $\label{thm:main_model} \begin{tabular}{ll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \\ \end{tabular}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

## Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|---|---|---|---|
| 0<br>1<br>2<br>3<br>4 | 1<br>2<br>1<br>1 | 18506.32350920<br>14740.90873263<br>14737.73074608<br>14737.61328795<br>14737.61305417 | 0.00056998<br>0.00002280<br>0.00000005<br>0.00000000 |

Convergence criteria met.

## Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|---|---|---|
| UN (1,1)<br>UN (2,1)<br>UN (2,2)<br>UN (3,1)<br>UN (3,2)<br>UN (3,3)<br>UN (4,1)<br>UN (4,2)<br>UN (4,3)<br>UN (4,4) | Subject SUBJID | 39.7612<br>40.5209<br>63.8318<br>35.8164<br>64.9397<br>81.3416<br>30.8032<br>59.4989<br>77.6293<br>85.9110<br>27.6057<br>53.2163<br>71.5019<br>80.7653<br>87.6338<br>24.7005<br>49.2619<br>64.9837 |
| UN (6, 4)<br>UN (6, 5)<br>UN (6, 6) | SUBJID<br>SUBJID<br>SUBJID | 72.8959<br>79.3406<br>87.4072 |

## Fit Statistics

| -2 Res Log Likelihood | 14737.6 |
|--------------------------|---------|
| AIC (Smaller is Better) | 14779.6 |
| AICC (Smaller is Better) | 14780.0 |
| BIC (Smaller is Better) | 14866.0 |

## Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 20 | 3768.71 | <.0001 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|-------------------|-----------|-----------|---------|--------|
| TRT01PN (AVISITN) | 6 | 435 | 35.96 | <.0001 |
| PREAD (AVISITN) | 6 | 432 | 2.36 | 0.0293 |
| BASE (AVISITN) | 6 | 433 | 65.36 | <.0001 |

| NN9068 | | Date: | 22 January 2020 <b>No</b> | ovo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 56 of 334 | |

 $\label{thm:main_model} \begin{tabular}{lll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix \end{tabular}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

## Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standar<br>Erro | | t Value |
|---|---|---|---|---|---|---|
| TRT01PN (AVISITN) TRT01PN (AVISITN) | | WORK.ANA_DATA<br>WORK.ANA_DATA | | | 8 427.4<br>6 437.4 | |
| | Least Squares Mear | ns Estimates | | | | |
| Effect | Label | Pr > t | Alpha | Lower | Upper | |
| TRT01PN (AVISITN)<br>TRT01PN (AVISITN) | | | | 2.2161 | -20.0628<br>-9.5822 | |
| | Least Squares | Means Estimate | | | | |
| Effect | Label | Margins | Est | imate | Standard<br>Error | DF |
| TRT01PN (AVISITN) | Treatment contrast, IDegLira - | IDeg WORK.ANA_ | _DATA -10 | .0231 | 0.9538 | 434.1 |
| Least Squares Means Estimate | | | | | | |
| Effect | Label | t Value | Pr > t | Alpha | Lower | Upper |
| TRT01PN (AVISITN) | Treatment contrast, IDegLira - | IDeg -10.51 | <.0001 | 0.05 | -11.8977 | -8.1485 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 57 of 334 | |

PARAMSORT=1 Parameter Code=C64849B Label=LSMeans, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME ABS MI

Number of Imputations

Variance Information (1000 Imputations)

-----Variance-----

Parameter Between Within Total

0.004942 0.005254 283778 Estimate 0.000311

Variance Information (1000 Imputations)

Relative Fraction Increase Missing Relative in Variance Information Efficiency Parameter

0.059339 Estimate 0.063075 0.999941

Parameter Estimates (1000 Imputations)

95% Confidence Std Error Limits DF Estimate Minimum Maximum Parameter

Estimate 7.934431 0.072481 7.792370 8.076492 283778 7.884262 7.988346

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter

109.47 <.0001 Estimate

#### 22 January 2020 | Novo Nordisk NN9068 Date: NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

 $\label{thm:hbalc} \mbox{HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set - appendix$ 

PARAMSORT=1 Parameter Code=C64849B Label=LSMeans, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

WORK.LSME\_ABS\_MI Data Set

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.002470 0.002580 550770 Estimate 0.000110

Variance Information (1000 Imputations)

Relative Fraction

Relative Missing Information Increase in Variance Efficiency 0.042592 0.999957 Estimate 0.044484

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits

Minimum Maximum 0.050797 6.951557 7.150676 550770 7.011871 7.088745 7.051117 Estimate

Parameter Estimates (1000 Imputations)

t for H0:

Theta0 Parameter=Theta0 Parameter Pr > |t|0 138.81 <.0001 Estimate

# NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

 $\label{thm:hbalc} \mbox{HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set - appendix$ 

PARAMSORT=2 Parameter Code=HBA1CONV Label=LSMeans, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME ABS MI

Number of Imputations 1000

Variance Information (1000 Imputations)

Parameter Between Within Total DF Estimate 0.037201 0.590373 0.627611 283778

Variance Information (1000 Imputations)

Relative Fraction

Increase Missing Relative Parameter in Variance Information Efficiency
Estimate 0.063075 0.059339 0.999941

Parameter Estimates (1000 Imputations)

95% Confidence

 Parameter
 Estimate
 Std Error
 Limits
 DF
 Minimum
 Maximum

 Estimate
 63.223331
 0.792219
 61.67060
 64.77606
 283778
 62.674980
 63.812625

Parameter Estimates (1000 Imputations)

t for HO:

Parameter Theta0 Parameter=Theta0 Pr > |t|Estimate 0 79.81 <.0001

#### 22 January 2020 | Novo Nordisk NN9068 Date: NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

 $\label{thm:hbalc} \mbox{HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set - appendix$ 

PARAMSORT=2 Parameter Code=HBA1CONV Label=LSMeans, IDeqLira Statement Number=1

The MIANALYZE Procedure

Estimate

Estimate

Model Information

Data Set WORK.LSME ABS MI

0.044484

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.295126 0.308254 550770

0.042592

Estimate 0.013115

Variance Information (1000 Imputations)

Relative Fraction Relative Missing Information Increase in Variance Efficiency

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum 0.555206 52.48052 54.65689 550770 53.139750 53.979986 53.568705

0.999957

Parameter Estimates (1000 Imputations)

t for H0: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 96.48 <.0001 Estimate

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 61 of 334 | |

PARAMSORT=1 Parameter Code=C64849B Label=Change from baseline, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter 0.004942 0.005254 283778 0.000311 Estimate

Variance Information (1000 Imputations)

Relative Fraction

Relative Increase Missing Parameter in Variance Information Efficiency 0.063075 0.059339 0.999941 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits

e DF Minimum Estimate Std Error Parameter Maximum Estimate -1.008395 0.072481 -1.15046 -0.86633 283778 -1.058564 -0.954479

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter Estimate 0 -13.91 <.0001

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 62 of 334 | |

PARAMSORT=1 Parameter Code=C64849B Label=Change from baseline, IDeqLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter 0.002470 0.002580 550770 0.000110 Estimate

Variance Information (1000 Imputations)

Relative Fraction

Relative  $\begin{array}{ccc} & & & & & & \\ & & & & & \\ \text{Parameter} & & \text{in Variance} & & \\ \text{Information} & & & \\ \end{array}$ Efficiency 0.044484 0.042592 0.999957 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits DF Minimum Estimate Std Error Parameter Maximum Estimate -1.891709 0.050797 -1.99127 -1.79215 550770 -1.930955 -1.854080

Parameter Estimates (1000 Imputations)

t for HO:

Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -37.24 <.0001 Estimate

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 63 of 334 | |

PARAMSORT=1 Parameter Code=C64849B Label=Treatment contrast, IDegLira - IDeg Statement Number=2

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.007414 0.007801 406826 Estimate 0.000386

Variance Information (1000 Imputations)

Relative Fraction Relative Increase Missing Parameter in Variance Information Efficiency

0.052138 0.049559 0.999950 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits e DF Minimum Estimate Std Error Parameter Maximum Estimate -0.883314 0.088322 -1.05642 -0.71021 406826 -0.940071 -0.823341

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -10.00 <.0001 Estimate

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 64 of 334 | |

PARAMSORT=2 Parameter Code=HBA1CONV Label=Change from baseline, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter 0.037201 Estimate

Variance Information (1000 Imputations)

Relative Fraction

Relative  $\begin{array}{ccc} & & & & & & \\ & & & & & \\ \text{Parameter} & & \text{in Variance} & & \\ \text{Information} & & & \\ \end{array}$ Efficiency 0.063075 0.059339 0.999941 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits

ce DF Minimum Maximum Estimate Std Error Parameter Estimate -11.021753 0.792219 -12.5745 -9.46903 283778 -11.570104 -10.432458

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -13.91 <.0001 Estimate

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 65 of 334 | |

PARAMSORT=2 Parameter Code=HBA1CONV Label=Change from baseline, IDeqLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter 0.013115 0.295126 0.308254 550770 Estimate

Variance Information (1000 Imputations)

Relative Fraction

Relative Increase Missing Parameter in Variance Information Efficiency 0.044484 0.042592 0.999957 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits

ce DF Minimum Maximum Parameter Estimate Std Error Estimate -20.676379 0.555206 -21.7646 -19.5882 550770 -21.105334 -20.265098

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter Estimate 0 -37.24 <.0001

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 66 of 334 | |

PARAMSORT=2 Parameter Code=HBA1CONV Label=Treatment contrast, IDegLira - IDeg Statement Number=2

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter 0.885743 0.931923 406826 0.046134 Estimate

Variance Information (1000 Imputations)

Relative Fraction

Relative Increase Missing Parameter in Variance Information Efficiency 0.052138 0.049559 0.999950 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits

.e DF Minimum Estimate Std Error Parameter Maximum Estimate -9.654626 0.965362 -11.5467 -7.76255 406826 -10.274981 -8.999121

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -10.00 <.0001 Estimate

NN9068 22 January 2020 Novo Nordisk Date: NN9068-4166 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

## 7: Responder for HbA1c treatment target – supportive statistical analysis – full analysis set

Parameter Code=HBA BL65

The GENMOD Procedure

Model Information

Data Set WORK.ADATA2 Distribution Binomial Link Function Logit

Dependent Variable AVÁLC Analysis Value (C)

Number of Observations Read Number of Observations Used Number of Events Number of Trials 453 453 106

Class Level Information

Class Levels Values TRTPN 1 2

BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 2

Response Profile

| Ordered | | Total |
|---------|-------|-----------|
| Value | AVALC | Frequency |
| 1 | Y | 106 |
| 2 | N | 347 |

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

Parameter Effect TRTPN PREAD Prm1 Intercept Prm2 TRTPN 2 Prm3 TRTPN BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD Prm4 PREAD Prm5 PREAD HBA1CBL Prm6

Criteria For Assessing Goodness Of Fit

Criterion DF Value Value/DF Log Likelihood -218.6220 Full Log Likelihood -218.6220 AIC (smaller is better) AICC (smaller is better) BIC (smaller is better) 445.2439 445.3332 461.7075

Algorithm converged.

| Parameter | | DF | Es | stimate | Standard<br>Error | Wald 95<br>Confidence | |
|---|---|---|---|---|---|---|---|
| Intercept | | 1 | | 0.5081 | 1.0333 | -1.5171 | 2.5332 |
| TRTPN | 1 | 1 | | 1.9218 | 0.3530 | 1.2299 | 2.6138 |
| TRTPN | 2 | 0 | | 0.0000 | 0.0000 | 0.0000 | 0.0000 |

#### NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 Final Clinical Trial Report Status: Statistical document 

Responder for HbAlc treatment target - supportive statistical analysis - full analysis set

Parameter Code=HBA\_BL65 The GENMOD Procedure

| Analysis Of Maximum Likelihood Parameter Estimates | | | | | | | |
|---|---|---|---|---|---|---|---|
| Paramet | er | | DF | Estimate | Standard<br>Error | | l 95%<br>ce Limits |
| PREAD<br>PREAD<br>HBA1CBL<br>Scale | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHE | ER OAD | 1<br>0<br>1<br>0 | 0.3170<br>0.0000<br>-0.3789<br>1.0000 | 0.2359<br>0.0000<br>0.1138<br>0.0000 | -0.1454<br>0.0000<br>-0.6019<br>1.0000 | 0.7795<br>0.0000<br>-0.1559<br>1.0000 |
| | Analysis Of Maximum Likelihood Pa | aramete: | r Est | timates | | | |
| Paramet | er | | Chi- | Wald<br>-Square | Pr > ChiSq | | |
| Interce<br>TRTPN<br>TRTPN | pt | | | 0.24 29.63 | 0.6229<br><.0001 | | |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHE | 7D 07D | | 1.81 | 0.1791 | | |
| HBA1CBL<br>Scale | | IK UAD | | 11.09 | 0.0009 | | |
| NOTE: T | he scale parameter was held fixed. | | | | | | |
| | Least Squares Mea | ans Est | imate | es | | | |
| Effect | Label Estimate | Stan<br>E: | | z Value | Pr > | z Al | pha |
| TRTPN<br>TRTPN | LSMeans frequency, IDegLira -0.7999<br>LSMeans frequency, IDeg -2.7218 | | 1284<br>3318 | | | | .05 |
| | Least Square | es Mean | s Est | timates | | | |
| Effect | Label Lower | Uppe | er I | Exponentiat | | ntiated<br>Lower | Exponentiated Upper |
| TRTPN<br>TRTPN | LSMeans frequency, IDegLira -1.0517<br>LSMeans frequency, IDeg -3.3721 | -0.548<br>-2.07 | | 0.44<br>0.065 | | 0.3494<br>0.03432 | 0.5780<br>0.1260 |
| | Least Square | es Mean | s Est | timate | | | |
| Effect | Label | Estin | mate | Standard<br>Error | z Value | Pr > | z Alpha |
| TRTPN | Treatment odds ratio, IDegLira / IDeg | 1. | 9218 | 0.3530 | 5.44 | <.00 | 01 0.05 |
| | Least Squares Mean | ns Estin | mate | | | | |
| Effect | Label | L | ower | Uppe | r Expon | entiated | |
| TRTPN | Treatment odds ratio, IDegLira / IDeg | 1.3 | 2299 | 2.613 | 8 | 6.8335 | |
| Least Squares Means Estimate | | | | | | | |
| Effect | Label | Expo | | iated Ex<br>Lower | ponentiate<br>Uppe | | |

TRTPN Treatment odds ratio, IDegLira / IDeg 3.4209 13.6505

#### NN9068 22 January 2020 Novo Nordisk Date: NN9068-4166 Version: 1.0 CONFIDENTIAL

Final Clinical Trial Report Status: Statistical document 

Responder for HbA1c treatment target - supportive statistical analysis - full analysis set

Parameter Code=HBA\_BL7

The GENMOD Procedure

Model Information

WORK.ADATA2 Data Set Distribution Binomial Link Function Logit

Dependent Variable AVALC Analysis Value (C)

Number of Observations Read Number of Observations Used Number of Events Number of Trials 453 453 177 453

Class Level Information

Class Levels Values TRTPN 1 2

BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD

Response Profile

Ordered Total Value AVALC Frequency 276 2 Ν

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

Effect TRTPN PREAD Parameter Prm1 Intercept Prm2 TRTPN Prm3 TRTPN 2 BASAL INSULIN + METFORMIN + ONE OTHER OAD Prm4 PREAD PREAD Prm5 HBA1CBL Prm6

Criteria For Assessing Goodness Of Fit

Criterion DF Value Value/DF -260.6635 Log Likelihood

Full Log Likelihood -260.6635 AIC (smaller is better) AICC (smaller is better) 529.3269 529.4162 545.7905 BIC (smaller is better)

Algorithm converged.

| Parameter | | DF | Estimate | Standard<br>Error | Wald 9<br>Confidence | |
|---|---|---|---|---|---|---|
| Intercept | | 1 | 2.0446 | 0.8816 | 0.3168 | 3.7724 |
| TRTPN | 1 | 1 | 1.8428 | 0.2613 | 1.3307 | 2.3550 |
| TRTPN | 2 | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 |

## NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Responder for HbAlc treatment target - supportive statistical analysis - full analysis set

Parameter Code=HBA\_BL7

The GENMOD Procedure

## Analysis Of Maximum Likelihood Parameter Estimates

| | Analysis Of Ma | aximum Likeli | lhood Pa | rameter Est | imates | | |
|---|---|---|---|---|---|---|---|
| Paramete | er | | DF | Estimate | Standard<br>Error | | l 95%<br>ice Limits |
| PREAD<br>PREAD<br>HBA1CBL<br>Scale | BASAL INSULIN + METFORMIN | + ONE OTHER | OAD 0<br>1<br>0 | 0.0000<br>-0.4514 | 0.0000<br>0.0989 | -0.0397<br>0.0000<br>-0.6452<br>1.0000 | 0.7944<br>0.0000<br>-0.2576<br>1.0000 |
| | Analysis Of Maximum Lil | kelihood Para | ameter E | stimates | | | |
| Paramete | er | | Ch | Wald<br>i-Square | Pr > ChiSq | | |
| Intercep<br>TRTPN | pt 1 2 | | | 5.38<br>49.74 | 0.0204<br><.0001 | | |
| TRTPN<br>PREAD<br>PREAD | BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN | T ONE OTHER | OVD | 3.14 | 0.0762 | | |
| HBA1CBL<br>Scale | | TONE OTHER | OAD | 20.83 | <.0001 | | |
| NOTE: Th | he scale parameter was held f | ixed. | | | | | |
| | Least Squares Means Estimates | | | | | | |
| Effect | Label | Estimate | Standar<br>Erro | | ie Pr > : | z Al | pha |
| TRTPN<br>TRTPN | LSMeans frequency, IDegLira<br>LSMeans frequency, IDeg | | 0.119 | | | | 0.05 |
| | Le | east Squares | Means E | stimates | | | |
| Effect | Label | Lower | Upper | Exponentia | | ntiated<br>Lower | Exponentiated Upper |
| TRTPN<br>TRTPN | LSMeans frequency, IDegLira LSMeans frequency, IDeg | | 0.2737<br>-1.3473 | | 400 | 0.8225<br>0.1043 | 1.3149<br>0.2600 |
| | Le | east Squares | Means E | stimate | | | |
| Effect | Label | | Estimat | Standar<br>e Erro | d<br>or z Value | Pr > | z Alpha |
| TRTPN | Treatment odds ratio, IDegLi | ira / IDeg | 1.842 | 8 0.261 | .3 7.05 | <.00 | 0.05 |
| | Least So | quares Means | Estimat | е | | | |
| Effect | Label | | Lowe | r Upp | er Expon | entiated | |
| TRTPN | Treatment odds ratio, IDegLi | ira / IDeg | 1.330 | 7 2.35 | 50 | 6.3145 | |
| | Least Square | es Means Esti | imate | | | | |
| Effect | Label | | Exponen | tiated E<br>Lower | Exponentiate<br>Uppe: | | |

3.7837

10.5380

Treatment odds ratio, IDegLira / IDeg

TRTPN

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 71 of 334 | |

## 8: Responder for HbA1c treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes – supportive statistical analysis – full analysis set

Parameter Code=HB65CHY

The GENMOD Procedure

Model Information

Data Set WORK.ADATA2 Distribution Binomial Link Function Logit

Dependent Variable AVALC Analysis Value (C)

Number of Observations Read Number of Observations Used Number of Events Number of Trials 453 102 453

Class Level Information

Class Levels Values

trtpn BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD 2 PREAD

Response Profile

Ordered Total AVALC Frequency Value

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

Parameter Effect trtpn PREAD

Prm1 Intercept Prm2 trtpn 2 Prm3 trtpn

PREAD BASAL INSULIN + METFORMIN Prm4

Prm5 PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD Prm6 HBA1CBL

Criteria For Assessing Goodness Of Fit

Criterion Value Value/DF Log Likelihood -213.6936 Full Log Likelihood AIC (smaller is better) AICC (smaller is better) -213.6936 435.3871 435.4764 BIC (smaller is better) 451.8507

Algorithm converged.

| Parameter | | DF | Estimate | Confidence |
|--------------------|---|----|----------|-------------------|
| Intercept<br>trtpn | 1 | | | -1.7691<br>1.2673 |

## NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes – supportive statistical analysis – full analysis set

Parameter Code=HB65CHY

The GENMOD Procedure

| | imarjoro or namimam principilo | | u | | | |
|---|---|---|---|---|---|---|
| Paramet | er | DF | Estimate S | tandard<br>Error | Wald 99<br>Confidence | |
| trtpn<br>PREAD<br>PREAD<br>HBA1CBL<br>Scale | 2<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 0.3750<br>0.0000<br>-0.3703 | 0.0000 | -0.0939<br>0.0000<br>-0.5960 | 0.0000 |
| | Analysis Of Maximum Likelihood Paramet | er Es | timates | | | |
| Paramet | er | Chi | Wald<br>-Square P | r > ChiSq | | |
| Interce,<br>trtpn | pt<br>1 | | 0.08<br>29.11 | 0.7836<br><.0001 | | |
| trtpn<br>PREAD<br>PREAD | 2<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 2.46 | 0.1170 | | |
| HBA1CBL<br>Scale | 2.0 2.0022 | | 10.34 | 0.0013 | | |
| NOTE: T | he scale parameter was held fixed. | | | | | |
| | Least Squares Means Es | timat | es | | | |
| | - | | | | | |
| Effect | | ndard<br>Error | z Value | Pr > : | z Alpha | a |
| | | .1296 | | <.000 | | |
| | Least Squares Mea | ns Es | timates | | | |
| | | | | Eurono | ntiated Ex | |
| Effect | Label Lower Up | per | Exponentiate | | Lower | Upper |
| | LSMeans frequency, IDegLira -1.0998 -0.5<br>LSMeans frequency, IDeg -3.5188 -2.1 | | 0.429<br>0.0586 | | 0.3329<br>0.02964 | 0.5533<br>0.1161 |
| | Least Squares Mea | ns Es | timate | | | |
| | | | Standard | | | |
| Effect | Label Est | imate | Error | z Value | Pr > z | Alpha |
| trtpn | Treatment odds ratio, IDegLira / IDeg 1 | .9903 | 0.3689 | 5.40 | <.0001 | 0.05 |
| | Least Squares Means Est | imate | | | | |
| Effect | Label | Lower | Upper | Expone | entiated | |
| trtpn | Treatment odds ratio, IDegLira / IDeg 1 | .2673 | 2.7132 | | 7.3176 | |
| | Least Squares Means Estimat | е | | | | |
| Effect | | | iated Exp<br>Lower | onentiated<br>Upper | | |
| trtpn | Treatment odds ratio, IDegLira / IDeg | 3 | .5513 | 15.0783 | l | |

#### NN9068 22 January 2020 Novo Nordisk Date: NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Final Status: Statistical document 

Responder for HbA1c treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes - supportive statistical analysis - full analysis set

Parameter Code=HB7CHY

The GENMOD Procedure

Model Information

WORK.ADATA2 Data Set Distribution Binomial Link Function Logit

Dependent Variable AVALC Analysis Value (C)

Number of Observations Read Number of Observations Used 453 453 Number of Events Number of Trials 453

Class Level Information

Class Levels Values trtpn

BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 2

Response Profile

Ordered Total Value AVALC Frequency 170 Υ 283 2 Ν

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

Parameter Effect PREAD trtpn

Prm1 Intercept Prm2 trtpn Prm3 trtpn 2

BASAL INSULIN + METFORMIN PREAD Prm4

BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD Prm5

Prm6 HBA1CBL

Criteria For Assessing Goodness Of Fit

Criterion DF Value Value/DF Log Likelihood -260.9980 Full Log Likelihood -260.9980 AIC (smaller is better)
AICC (smaller is better) 529.9960 530.0853 BIC (smaller is better) 546.4596

Algorithm converged.

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidenc | |
|---|---|---|---|---|---|---|
| Intercept<br>trtpn | 1 | _ | | 0.8770<br>0.2638 | -0.1235<br>1.2836 | 3.3144<br>2.3179 |


Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes – supportive statistical analysis – full analysis set

Parameter Code=HB7CHY

The GENMOD Procedure

| | Analysis Of Maximum Likeliho | od Par | ameter Estima | ites | | |
|---|---|---|---|---|---|---|
| Paramete | er | DF | St<br>Estimate | andard<br>Error | Wald 95<br>Confidence | |
| trtpn<br>PREAD<br>PREAD<br>HBA1CBL<br>Scale | 2<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OA | 0<br>1<br>0<br>1<br>0 | | 0.2125<br>0.0000 | -0.0293<br>0.0000<br>-0.5980 - | 0.0000<br>0.8035<br>0.0000<br>0.2142<br>1.0000 |
| | Analysis Of Maximum Likelihood Parame | ter Es | timates | | | |
| Paramete | er | Chi | Wald<br>-Square Pr | c > ChiSq | | |
| Interceptrtpn<br>trtpn<br>trtpn | pt | | 3.31<br>46.58 | 0.0689<br><.0001 | | |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OA | . D | 3.32 | 0.0685 | | |
| HBA1CBL<br>Scale | | .D | 17.21 | <.0001 | | |
| NOTE: Th | he scale parameter was held fixed. | | | | | |
| | Least Squares Means E | Sstimat | es | | | |
| Effect | | andard<br>Error | | Pr > z | Alpha | |
| trtpn<br>trtpn | | 0.1190<br>0.2361 | | 0.724<br><.000 | | |
| | Least Squares Me | ans Es | timates | | | |
| Effect | Label Lower U | ipper | Exponentiated | | tiated Exp<br>Lower | onentiated<br>Upper |
| trtpn<br>trtpn | | 1913<br>3799 | 0.9589<br>0.1584 | | 0.7594<br>.09971 | 1.2108<br>0.2516 |
| | Least Squares Me | ans Es | timate | | | |
| Effect | Label Es | timate | Standard<br>Error | z Value | Pr > z | Alpha |
| trtpn | Treatment odds ratio, IDegLira / IDeg | 1.8007 | 0.2638 | 6.82 | <.0001 | 0.05 |
| | Least Squares Means Es | timate | | | | |
| Effect | Label | Lower | Upper | Expone | ntiated | |
| trtpn | Treatment odds ratio, IDegLira / IDeg | 1.2836 | 2.3179 | | 6.0541 | |
| | Least Squares Means Estima | ite | | | | |
| Effect | Label | ponent | iated Expo | nentiated<br>Upper | | |
| trtpn | Treatment odds ratio, IDegLira / IDeg | 3 | .6096 | 10.1540 | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 75 of 334 | |

## 9: Responder for HbA1c treatment target without weight gain – supportive statistical analysis – full analysis set

Parameter Code=HB65WOWG

The GENMOD Procedure

Model Information

Data Set WORK.ADATA2 Distribution Binomial Link Function Logit

Dependent Variable AVALC Analysis Value (C)

Number of Observations Read Number of Observations Used Number of Events Number of Trials 453 453

Class Level Information

Class Levels Values trtpn

BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD 2 PREAD

Response Profile

Ordered Total AVALC Frequency Value 391

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

Parameter Effect trtpn PREAD

Prm1 Intercept Prm2 trtpn Prm3 trtpn

PREAD BASAL INSULIN + METFORMIN Prm4

Prm5 PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD Prm6 HBA1CBL

Prm7 WGTBL

Criteria For Assessing Goodness Of Fit

Value Criterion Value/DF

-159.3887 -159.3887 328.7775 Log Likelihood Full Log Likelihood
AIC (smaller is better)
AICC (smaller is better)
BIC (smaller is better) 328.9117

Algorithm converged.

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 76 of 334 | |

Responder for HbAlc treatment target without weight gain – supportive statistical analysis – full analysis set

Parameter Code=HB65WOWG

| rarameter code=HB05WOWG | |
|---|---|
| The GENMOD Procedure | |
| Analysis Of Maximum Likelihood Parameter Estimates | |
| Parameter | Standard Wald 95%<br>DF Estimate Error Confidence Limits |
| Intercept trtpn 1 trtpn 2 PREAD BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAL HBA1CBL WGTBL Scale | 1 -0.3826 0.1438 -0.6645 -0.1007<br>1 0.0107 0.0108 -0.0104 0.0318<br>0 1.0000 0.0000 1.0000 1.0000 |
| Analysis Of Maximum Likelihood Paramet | er Estimates |
| Parameter | Wald<br>Chi-Square Pr > ChiSq |
| Intercept trtpn 1 trtpn 2 | 0.78 0.3780<br>16.77 <.0001 |
| PREAD BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAL | 0.03 0.8535 |
| HBAICBL WGTBL Scale | 7.08 0.0078<br>0.99 0.3188 |
| NOTE: The scale parameter was held fixed. | |
| Least Squares Means Es | timates |
| | ndard<br>Error z Value Pr > z Alpha |
| | .1553 -9.61 <.0001 0.05<br>.5867 -6.75 <.0001 0.05 |
| Least Squares Mea | ns Estimates |
| Effect Label Lower Up | Exponentiated Exponentiated oper Exponentiated Lower Upper |
| trtpn LSMeans frequency, IDegLira -1.7965 -1.1<br>trtpn LSMeans frequency, IDeg -5.1113 -2.8 | |
| Least Squares Means Estimate | |
| Effect Label Est | Standard<br>Simate Error z Value Pr > z Alpha |
| trtpn Treatment odds ratio, IDegLira / IDeg | .4694 0.6029 4.10 <.0001 0.05 |
| Least Squares Means Est | imate |
| Effect Label | Lower Upper Exponentiated |

trtpn Treatment odds ratio, IDegLira / IDeg 1.2877

3.6512 11.8157

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 77 of 334 | |

Responder for HbAlc treatment target without weight gain - supportive statistical analysis - full analysis set

Parameter Code=HB65WOWG

The GENMOD Procedure

Least Squares Means Estimate

| Effect | Label | | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|
| trtpn | Treatment or | dds ratio, | IDegLira / IDeg | 3.6243 | 38.5206 |

#### NN9068 22 January 2020 Novo Nordisk Date: NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Responder for HbAlc treatment target without weight gain - supportive statistical analysis - full analysis set

Parameter Code=HBA7WOWG

The GENMOD Procedure

Model Information

Data Set WORK.ADATA2 Distribution Binomial Link Function Logit

Dependent Variable AVALC Analysis Value (C)

Number of Observations Read Number of Observations Used 453 453 Number of Events 105 Number of Trials 453

Class Level Information

Class Levels Values trtpn

BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD

Response Profile

Ordered Total Value AVALC Frequency 105 Υ 2 348

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

Parameter Effect PREAD trtpn Prm1 Intercept Prm2 trtpn Prm3 trtpn 2 BASAL INSULIN + METFORMIN PREAD Prm4 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD Prm5 Prm6 HBA1CBL WGTBL Prm7

Criteria For Assessing Goodness Of Fit

Criterion Value Value/DF Log Likelihood -211.2368 Full Log Likelihood AIC (smaller is better) -211.2368 432.4737 AICC (smaller is better) BIC (smaller is better) 432.6079 453.0531

Algorithm converged.

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 79 of 334 | |

Responder for HbAlc treatment target without weight gain - supportive statistical analysis - full analysis set

Parameter Code=HBA7WOWG

| Parameter Code=HBA7WOWG | | | | | | |
|---|---|---|---|---|---|---|
| The GENI | The GENMOD Procedure | | | | | |
| | Analysis Of Maximum Likelih | ood Para | ameter Est | imates | | |
| Paramet | er | DF | Estimate | Standard<br>Error | Wald 95<br>Confidence | |
| Interceptrtpn trtpn PREAD PREAD HBA1CBL WGTBL Scale | 1<br>2<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER O | 1<br>1<br>0<br>1<br>1<br>0<br>1<br>1<br>1<br>0 | 0.0000<br>-0.4075 | 1.2695<br>0.4097<br>0.0000<br>0.2407<br>0.0000<br>0.1165<br>0.0094<br>0.0000 | 1.5354<br>0.0000<br>-0.2304<br>0.0000<br>-0.6359<br>-0.0200 | 3.0251<br>3.1416<br>0.0000<br>0.7132<br>0.0000<br>0.1791<br>0.0167<br>1.0000 |
| | Analysis Of Maximum Likelihood Param | eter Es | timates | | | |
| Paramete | er | Chi | Wald<br>-Square | Pr > ChiSq | | |
| Intercept trtpn 1 trtpn 2 | | | 0.18<br>32.57 | 0.6724<br><.0001 | | |
| trtpn<br>PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER O | A D | 1.01 | 0.3160 | | |
| HBA1CBL<br>WGTBL<br>Scale | | AD | 12.23 | 0.0005<br>0.8596 | | |
| NOTE: T | he scale parameter was held fixed. | | | | | |
| | Least Squares Means | Estimate | es | | | |
| | S | tandard | | | | |
| Effect | Label Estimate | Error | z Value | e Pr > | z Alpha | |
| trtpn<br>trtpn | LSMeans frequency, IDegLira -0.7744<br>LSMeans frequency, IDeg -3.1129 | 0.1286<br>0.3918 | -6.02<br>-7.99 | | | |
| | Least Squares M | leans Es | timates | | | |
| Effect | Label Lower | Upper 1 | Exponentia | | ntiated Exp<br>Lower | onentiated<br>Upper |
| trtpn<br>trtpn | | .5224 | 0.40 | | 0.3583<br>0.02064 | 0.5931<br>0.09584 |

| Effect | Label | | | Lower | Upper | Exponentiated | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|---|---|---|---|
| _ | | frequency, frequency, | _ | -1.0264<br>-3.8807 | -0.5224<br>-2.3450 | 0.4610<br>0.04447 | 0.3583<br>0.02064 | 0.5931<br>0.09584 |

## Least Squares Means Estimate

| Effect | Label | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|
| trtpn | Treatment odds ratio, IDegLira / IDeg | 2.3385 | 0.4097 | 5.71 | <.0001 | 0.05 |
| Least Squares Means Estimate | | | | | | |
| Effect | Label | Lower | Upper | Exponer | ntiated | |
| trtpn | Treatment odds ratio, IDegLira / IDeg | 1.5354 | 3.1416 | - | 10.3655 | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 80 of 334 | |

Responder for HbAlc treatment target without weight gain - supportive statistical analysis - full analysis set

Parameter Code=HBA7WOWG

The GENMOD Procedure

Least Squares Means Estimate

| | | | | Exponentiated | Exponentiated |
|---|---|---|---|---|---|
| Effect | Label | | | Lower | Upper |
| trtpn | Treatment od | lds ratio. | IDegLira / IDeg | 4.6432 | 23.1402 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 81 of 334 | |

## 10: Responder for HbA1c treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes and weight gain – supportive statistical analysis – full analysis set

Parameter Code=H65WOCHY

The GENMOD Procedure

Model Information

Data Set WORK.ADATA2 Distribution Binomial Link Function Logit

Dependent Variable AVALC Analysis Value (C)

Number of Observations Read Number of Observations Used 453 Number of Events Number of Trials 61 453

Class Level Information

Class Levels Values trtpn

BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD 2 PREAD

Response Profile

Ordered Total AVALC Frequency Value 392

WGTBL

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

Parameter Effect trtpn PREAD Prm1 Intercept Prm2 trtpn Prm3 trtpn PREAD BASAL INSULIN + METFORMIN Prm4 Prm5 PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD Prm6 HBA1CBL

Criteria For Assessing Goodness Of Fit

Value Criterion Value/DF -157.5765 Log Likelihood Full Log Likelihood
AIC (smaller is better) -157.5765 325.1529 AICC (smaller is better)
BIC (smaller is better) 325.2871

Algorithm converged.

Prm7

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 82 of 334 | |

Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes and weight gain – supportive statistical analysis – full analysis set

Parameter Code=H65WOCHY

| The GEN | MOD Procedure | | | | | |
|---|---|---|---|---|---|---|
| | Analysis Of Maximum Likel | ihood Par | rameter Estima | ites | | |
| Paramet | er | DF | | andard<br>Error ( | Wald 95<br>Confidence | |
| Interce<br>trtpn<br>trtpn<br>PREAD<br>PREAD<br>HBA1CBL<br>WGTBL<br>Scale | 1<br>2<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER | 1<br>1<br>0<br>1<br>0 0<br>1<br>1<br>1<br>0 | -1.2594<br>2.4496<br>0.0000<br>0.0944<br>0.0000<br>-0.4041<br>0.0113<br>1.0000 | 0.6033<br>0.0000<br>0.2894<br>0.0000<br>0.1466<br>0.0108 | 1.2671<br>0.0000<br>-0.4728<br>0.0000<br>-0.6915<br>-0.0099 | 1.8454<br>3.6321<br>0.0000<br>0.6615<br>0.0000<br>0.1167<br>0.0325<br>1.0000 |
| | Analysis Of Maximum Likelihood Par | ameter Es | stimates | | | |
| Paramet | er | Chi | Wald<br>Square Pr | > ChiSq | | |
| Interce<br>trtpn<br>trtpn | pt | | 0.63<br>16.48 | 0.4266<br><.0001 | | |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER | COAD | 0.11 | 0.7443 | | |
| HBA1CBL<br>WGTBL<br>Scale | | | 7.59<br>1.09 | 0.0059<br>0.2975 | | |
| NOTE: T | he scale parameter was held fixed. | | | | | |
| | Least Squares Mean | ıs Estimat | es | | | |
| Effect | Label Estimate | Standard<br>Error | | Pr > z | Alpha | |
| trtpn<br>trtpn | LSMeans frequency, IDegLira -1.5204<br>LSMeans frequency, IDeg -3.9700 | 0.1574<br>0.5871 | | <.000 | | |
| | Least Squares | Means Es | stimates | | | |
| Effect | Label Lower | Upper | Exponentiated | | tiated Exp<br>Lower | onentiated<br>Upper |
| trtpn<br>trtpn | | -1.2120<br>-2.8192 | 0.2186<br>0.01887 | | 0.1606<br>005972 | 0.2976<br>0.05965 |
| | Least Squares | Means Es | stimate | | | |
| | | | Standard | | | |
| | Label | Estimate | | | Pr > z | Alpha |
| trtpn | Treatment odds ratio, IDegLira / IDeg | | | 4.06 | <.0001 | 0.05 |
| Effect | Least Squares Means | Lower | | Expone | ntiated | |

trtpn Treatment odds ratio, IDegLira / IDeg 1.2671 3.6321 11.5836

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 83 of 334 | |

Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes and weight gain – supportive statistical analysis – full analysis set

Parameter Code=H65WOCHY

The GENMOD Procedure

Least Squares Means Estimate

| Effect | ffect Label | | Exponentiated<br>Lower | Exponentiated<br>Upper | |
|---|---|---|---|---|---|
| trtpn | Treatment o | odds ratio, | IDegLira / IDeg | 3.5504 | 37.7934 |

#### NN9068 22 January 2020 Novo Nordisk Date: NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Final Status: Statistical document 

Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes and weight gain - supportive statistical analysis - full analysis set

Parameter Code=HB7WOCHY

The GENMOD Procedure

Model Information

WORK.ADATA2 Data Set Distribution Binomial Link Function Logit

Dependent Variable AVALC Analysis Value (C)

Number of Observations Read Number of Observations Used 453 453 Number of Events 101 Number of Trials 453

Class Level Information

Class Levels Values trtpn

BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD

Response Profile

Ordered Total Value AVALC Frequency 101 Υ 352 2

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

Parameter Effect PREAD trtpn Prm1 Intercept Prm2 trtpn Prm3 trtpn 2 BASAL INSULIN + METFORMIN PREAD Prm4 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD Prm5 Prm6 HBA1CBL WGTBL Prm7

Criteria For Assessing Goodness Of Fit

DF Criterion Value Value/DF Log Likelihood -209.2402 Full Log Likelihood AIC (smaller is better) -209.2402 428.4804 AICC (smaller is better) BIC (smaller is better) 428.6146 449.0598

Algorithm converged.

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 85 of 334 | |

Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes and weight gain – supportive statistical analysis – full analysis set

Parameter Code=HB7WOCHY

Effect Label

trtpn Treatment odds ratio, IDegLira / IDeg 1.4609

| The GENMOD Procedure | | | | | | |
|---|---|---|---|---|---|---|
| Analysis Of Maximum Likelihood Parameter Estimates | | | | | | |
| Paramet | er | DF | Sta<br>Estimate | andard<br>Error | Wald !<br>Confidence | |
| Interce<br>trtpn<br>trtpn<br>PREAD<br>PREAD<br>HBA1CBL<br>WGTBL<br>Scale | 1<br>2<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | 1<br>0<br>1<br>0<br>1<br>1<br>0 | 2.2639<br>0.0000<br>0.2414<br>0.0000<br>-0.3788<br>0.0008 | 1.2722<br>0.4097<br>0.0000<br>0.2424<br>0.0000<br>0.1165<br>0.0094<br>0.0000 | -2.3869<br>1.4609<br>0.0000<br>-0.2338<br>0.0000<br>-0.6072<br>-0.0176<br>1.0000 | 2.5998<br>3.0669<br>0.0000<br>0.7166<br>0.0000<br>-0.1505<br>0.0193<br>1.0000 |
| Analysis Of Maximum Likelihood Parameter Estimates | | | | | | |
| Paramet | er | Chi | Wald<br>L-Square Pr | > ChiSq | | |
| Interce<br>trtpn<br>trtpn<br>PREAD<br>PREAD<br>HBA1CBL<br>WGTBL<br>Scale | 1<br>2<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 0.01<br>30.53<br>0.99<br>10.57<br>0.01 | 0.9333<br><.0001<br>0.3194<br>0.0011<br>0.9292 | | |
| NOTE: The scale parameter was held fixed. | | | | | | |
| Least Squares Means Estimates | | | | | | |
| Effect | | ndaro<br>Error | | Pr > | z Alph | na |
| trtpn<br>trtpn | | .1295<br>.3912 | | <.00<br><.00 | | |
| | Least Squares Mean | ns Es | stimates | | | |
| Effect | Label Lower Upp | per | Exponentiated | | ntiated Ex<br>Lower | xponentiated<br>Upper |
| trtpn<br>trtpn | LSMeans frequency, IDegLira -1.0873 -0.57<br>LSMeans frequency, IDeg -3.8640 -2.33 | | 0.4346<br>0.04517 | | 0.3371<br>0.02098 | 0.5601<br>0.09724 |
| Least Squares Means Estimate | | | | | | |
| Effect | Label Est. | imate | Standard<br>Error | z Value | Pr > z | Alpha |
| trtpn | Treatment odds ratio, IDegLira / IDeg 2 | .2639 | 0.4097 | 5.53 | <.0000 | 0.05 |
| Least Squares Means Estimate | | | | | | |

Lower

Upper

3.0669

Exponentiated

9.6205

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 86 of 334 | |

Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes and weight gain – supportive statistical analysis – full analysis set

Parameter Code=HB7WOCHY

The GENMOD Procedure

Least Squares Means Estimate

| Effect | Label | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|
| trtpn | Treatment odds ratio, IDegLira / | IDeg 4.3097 | 21.4759 |

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

## 11: Body weight after 26 weeks of treatment – change from baseline – confirmatory statistical analysis – full analysis set - appendix

Parameter Code=C25208X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 8.0164

Fit Statistics

-2 Res Log Likelihood 2235.4
AIC (Smaller is Better) 2237.4
AICC (Smaller is Better) 2237.4
BIC (Smaller is Better) 2241.5

Solution for Fixed Effects

Planned
Treatment
for
Period Standard
O1 (N) Estimate Error

Intercept
trtpn 1 -1.0762 0.2835

449 trtpn 1 -1.0762 0.2835 -3.80 trtpn 2 Ω BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD 0.3488 PREAD 0.2675 449 1.30 PREAD 1.0227 0.01074 BASE 449 95.25

DF t Value
| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 88 of 334 | |

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=C25208X

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial ant | i-Diabetic treatm | nent | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | a | |
|---|---|---|---|---|---|---|---|---|
| Interce | pt | | | | 0.0811 | | | |
| trtpn<br>trtpn | | | | 1<br>2 | 0.0002 | | | |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | 0.1930 | | | | |
| BASE | | | | | <.0001 | 0.0 | 5 | |
| | | Solution for | Fixed Effec | cts | | | | |
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial ant | i-Diabetic treatm | nent | 01 (N) | Lower | T Up | per | |
| Interce<br>trtpn<br>trtpn | pt | | | 1<br>2 | -3.1625<br>-1.6334 | | 847<br>189 | |
| PREAD<br>PREAD | | | | | -0.1770 | 0.8 | 746 | |
| BASE | | | | | 1.0016 | 1.0 | 438 | |
| | Type 3 Tests of | Fixed Effects | | | | | | |
| Effect | Num De<br>DF D | | r > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 44<br>1 44<br>1 44 | 9 1.70 0 | 0.0002<br>0.1930<br>0.0001 | | | | | |
| | | Least | Squares Mean | ns Estimates | | | | |
| | | | | Standard | | | | |
| Effect | Label | Margins | Estimate | Error | | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLi<br>LSMeans, IDeg | ra WORK.ADATA2<br>WORK.ADATA2 | 75.3159<br>76.3920 | 0.1632<br>0.2311 | 449<br>449 | 461.54<br>330.49 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least So | quares Means | Estimates | | | | |
| Effect | Label | Lower | Upper Ex | xponentiated | | entiated<br>Lower | Exponentia<br>Up | nted |
| trtpn<br>trtpn | LSMeans, IDegLi<br>LSMeans, IDeg | | 75.6366<br>76.8463 | 5.12E32<br>1.502E33 | | 3.715E32<br>9.536E32 | 7.056<br>2.366 | |
| | | Least S | Squares Means | s Estimate | | | | |
| | | | | | Sta | ındard | | |
| Effect | Label | | Margins | Estim | | Error | DF t Vâ | alue |
| trtpn | Treatment contra | st, IDegLira - II | Deg WORK.ADA | ATA2 -1.0 | 762 0 | .2835 | 449 -3 | 3.80 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 89 of 334 | |

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=C25208X

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.0002 0.05 -1.6334 -0.5189 0.3409

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.1953 0.5952


Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=WEIGHTU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453
Number of Observations Used 453
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate Residual 38.9624

Fit Statistics

-2 Res Log Likelihood 2946.9
AIC (Smaller is Better) 2948.9
AICC (Smaller is Better) 2948.9
BIC (Smaller is Better) 2953.0

Solution for Fixed Effects

Planned

Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value -3.2825 1.8774 449 -1.75 Intercept -2.3725 -3.80 1 0.6251 449 trtpn trtpn PREAD BASAL INSULIN + METFORMIN 0.7689 0.5898 449 1.30 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 1.0227 BASE 0.01074 449 95.25

| NN9068 | | Date: | 22 January 2020 Novo Nordisk |
|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final |
| Statistical document | | Page: | 91 of 334 |

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=WEIGHTU

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial an | ti-Diabetic treat | tment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | ıa | |
|---|---|---|---|---|---|---|---|---|
| Intercept<br>trtpn | | | | 1 | 0.081 | | | |
| trtpn<br>PREAD | n<br>D BASAL INSULIN + METFORMIN | | | | 0.193 | 0.0 | 05 | |
| PREAD<br>BASE | BASAL INSULI | N + METFORMIN + ( | ONE OTHER OAD | | <.000 | 1 0.0 | )5 | |
| | | Solution fo | or Fixed Effe | cts | | | | |
| Effect | Pre Trial an | ti-Diabetic treat | tment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lowe | r Ug | pper | |
| Intercept<br>trtpn | | | | 1 | -6.972<br>-3.601 | | 4072<br>1440 | |
| trtpn<br>PREAD BASAL INSULIN + METFORMIN | | | 2 | -0.390 | 2 1.9 | 9281 | | |
| BASE | PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD<br>BASE | | | | 1.001 | 6 1.0 | 0438 | |
| I | ype 3 Tests of | Fixed Effects | | | | | | |
| Effect | | en<br>DF F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 4 | 49 14.40<br>49 1.70<br>49 9072.25 | 0.0002<br>0.1930<br><.0001 | | | | | |
| | | Least | Squares Mea | ns Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| | LSMeans, IDegL<br>LSMeans, IDeg | ira WORK.ADATA2<br>WORK.ADATA2 | | 0.3598<br>0.5096 | 449<br>449 | 461.54<br>330.49 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least S | Squares Means | Estimates | | | | |
| Effect | Label | Lower | Upper E | xponentiated | | entiated<br>Lower | Exponentia<br>Up | ted<br>per |
| | LSMeans, IDegL<br>LSMeans, IDeg | ira 165.34<br>167.41 | 166.75<br>169.42 | 1.293E72<br>1.387E73 | | 6.376E71<br>5.094E72 | 2.622<br>3.775 | |
| | | Least | Squares Mean | s Estimate | | | | |
| Effect L | abel | | Margins | Estim | | andard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -2.3725 0.6251 449 -3.80

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 92 of 334 | |

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=WEIGHTU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.0002 0.05 -3.6010 -1.1440 0.09325

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.02730 0.3185

## NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=C25208X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453
Number of Observations Used 453
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 8.0164

Fit Statistics

-2 Res Log Likelihood 2235.4
AIC (Smaller is Better) 2237.4
AICC (Smaller is Better) 2237.4
BIC (Smaller is Better) 2241.5

Solution for Fixed Effects

Planned

Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value -1.75 -1.4889 0.8516 449 Intercept -3.80 -1.0762 0.2835 449 trtpn trtpn PREAD BASAL INSULIN + METFORMIN 0.3488 0.2675 449 1.30 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.02267 BASE 0.01074 449 2.11

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 94 of 334 | |

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=C25208X

The Mixed Procedure

| | | | Solution fo | or Fixed Effec | ts | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-Di | abetic trea | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | 0.0811<br>0.0002 | 0.05<br>0.05 |
| PREAD | BASAL INSU | | | | _ | 0.1930 | 0.05 |
| PREAD<br>BASE | BASAL INSU | JLIN + M. | ETFORMIN + | ONE OTHER OAD | | 0.0353 | 0.05 |
| | | | Solution : | for Fixed Effe | cts | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-Di | abetic trea | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | -3.1625<br>-1.6334 | 0.1847<br>-0.5189 |
| PREAD<br>PREAD | BASAL INSU | | | ONE OTHER OAD | _ | -0.1770 | 0.8746 |
| BASE | BASAL INSC | JLIN + M. | EIFORMIN + | ONE OTHER OAL | | 0.001572 | 0.04377 |
| Ту | rpe 3 Tests | of Fixe | d Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 449<br>449<br>449 | 14.40<br>1.70<br>4.46 | 0.0002<br>0.1930<br>0.0353 | | | |

### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | -0.6766<br>0.3996 | 0.1632<br>0.2311 | 449<br>449 | -4.15<br>1.73 | <.0001<br>0.0846 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | | -0.9973<br>).05471 | -0.3559<br>0.8538 | | | |


Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=WEIGHTU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453
Number of Observations Used 453
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 38.9624

Fit Statistics

-2 Res Log Likelihood 2946.9
AIC (Smaller is Better) 2948.9
AICC (Smaller is Better) 2948.9
BIC (Smaller is Better) 2953.0

Solution for Fixed Effects

Planned

Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value -1.75 -3.2825 1.8774 449 Intercept -2.3725 -3.80 1 0.6251 449 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.7689 0.5898 449 1.30 PREAD 0.02267 BASE 0.01074 449 2.11

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 96 of 334 | |

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set - appendix

Parameter Code=WEIGHTU

The Mixed Procedure

### Solution for Fixed Effects

| | | | SOTUCTOR I | or rixed Effect | 23 | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-Di | abetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | 0.0811<br>0.0002 | 0.05<br>0.05 |
| PREAD<br>PREAD | BASAL INSU | | | ONE OTHER OAD | 0.1930 | 0.05 | |
| BASE | DASAL INSC | TIN T M | EIFORMIN + | ONE OTHER OAD | | 0.0353 | 0.05 |
| | | | Solution | for Fixed Effe | cts | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-Di | abetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | -6.9722<br>-3.6010 | 0.4072<br>-1.1440 |
| PREAD<br>PREAD | BASAL INSU | | | ONE OTHER OAD | 2 | -0.3902 | 1.9281 |
| BASE | 2110112 1110 | , | | 0112 0111211 0112 | | 0.001572 | 0.04377 |
| Ту | pe 3 Tests | of Fixe | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 449<br>449<br>449 | 14.40<br>1.70<br>4.46 | 0.0002<br>0.1930<br>0.0353 | | | |

### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.3598<br>0.5096 | 449<br>449 | -4.15<br>1.73 | <.0001<br>0.0846 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | | -2.1987<br>-0.1206 | -0.7846<br>1.8823 | | | |

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

### 12: Body weight after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – PP analysis set - appendix

Parameter Code=C25208X

Levels

The Mixed Procedure

Class

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

trtan 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Values

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 431

Number of Observations

Number of Observations Read 431 Number of Observations Used 431 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 8.3053

Fit Statistics

-2 Res Log Likelihood 2142.1 AIC (Smaller is Better) 2144.1 AICC (Smaller is Better) 2144.1 BIC (Smaller is Better) 2148.1

Solution for Fixed Effects

Actual Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error -1.5403 Intercept 0.8925 427 trtan 1 -1.0802 0.2968 427 trtan 2 Λ BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD 0.3398 PREAD 0.2793 427 1.22 PREAD 1.0236 BASE 0.01127 427 90.86

# NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=C25208X

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial anti- | Diabetic treat | ment | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpl | na | |
|---|---|---|---|---|---|---|---|---|
| Intercep | t | | | 1 | 0.085 | | | |
| trtan<br>trtan<br>PREAD | BASAL INSULIN + | METFORMIN | | 2 | 0.000 | | | |
| PREAD<br>BASE | BASAL INSULIN + | METFORMIN + C | NE OTHER OAD | ) | <.000 | 1 0.0 | 05 | |
| | | Solution fo | r Fixed Effe | ects | | | | |
| Effect | Pre Trial anti- | Diabetic treat | ment | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lowe | r Ul | pper | |
| Intercep<br>trtan | t | | | 1 | -3.294<br>-1.663 | | 2140<br>4967 | |
| trtan<br>PREAD | BASAL INSULIN + | | ME OHIED OAR | 2 | -0.209 | 2 0. | 8887 | |
| PREAD<br>BASE | BASAL INSULIN + | METFORMIN + C | INE OTHER OAL | ) | 1.001 | 4 1.0 | 0457 | |
| | Type 3 Tests of Fi | xed Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value | Pr > F | | | | | |
| trtan<br>PREAD<br>BASE | 1 427<br>1 427<br>1 427 | 1.48 | 0.0003<br>0.2244<br><.0001 | | | | | |
| | | Least | Squares Mea | ıns Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtan<br>trtan | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.1698<br>0.2427 | 427<br>427 | | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least S | quares Means | Estimates | | | | |
| Effect | Label | Lower | Upper E | Exponentiated | | entiated<br>Lower | | ted |
| trtan<br>trtan | LSMeans, IDegLira<br>LSMeans, IDeg | 74.9628<br>75.8998 | 75.6303<br>76.8537 | 5.022E32<br>1.479E33 | | 3.597E32<br>9.18E32 | 7.012<br>2.383 | |
| | | Least | Squares Mean | ıs Estimate | | | | |
| Effect | Label | | Margins | : Estim | | andard<br>Error | DF t Va | lue |

trtan Treatment contrast, IDegLira - IDeg WORK.ADATA2 -1.0802 0.2968 427

-3.64

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 99 of 334 | |

Parameter Code=C25208X

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtan Treatment contrast, IDegLira - IDeg 0.0003 0.05 -1.6637 -0.4967 0.3395

Least Squares Means Estimate

Exponentiated Lower Upper trtan Treatment contrast, IDegLira - IDeg 0.1894 Exponentiated 0.6085

### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=WEIGHTU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtan 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 431

Number of Observations

Number of Observations Read 431
Number of Observations Used 431
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 40.3667

Fit Statistics

-2 Res Log Likelihood 2818.8
AIC (Smaller is Better) 2820.8
AICC (Smaller is Better) 2820.8
BIC (Smaller is Better) 2824.8

Solution for Fixed Effects

Actual Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value -3.3957 1.9676 -1.73 427 Intercept -2.3814 -3.64 1 0.6544 427 trtan trtan BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.7491 0.6157 427 1.22 PREAD 1.0236 BASE 0.01127 427 90.86

# NN9068 | Date: 22 January 2020 | Novo Nordisk NN9068-4166 | CONFIDENTIAL | Version: 1.0 | Clinical Trial Report | Status: Final |  |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=WEIGHTU

| The Mixe | ed Procedure | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Solution for | Fixed Effect | ts | | | | |
| Effect | Pre Trial anti-D | iabetic treatr | nent | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpl | na | |
| Intercep<br>trtan | pt | | | 1 | 0.0851 | | | |
| trtan<br>PREAD | BASAL INSULIN + | | | 2 | 0.2244 | | | |
| PREAD<br>BASE | BASAL INSULIN + | METFORMIN + ON | NE OTHER OAD | | <.0001 | 0.0 | 05 | |
| | | Solution for | r Fixed Effe | cts | | | | |
| Effect Interceptrtan trtan PREAD PREAD BASE | Pre Trial anti-D<br>ot<br>BASAL INSULIN +<br>BASAL INSULIN + | METFORMIN | | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lower -7.2631 -3.6677 -0.4611 1.0014 | 0.4 | pper<br>4717<br>9951<br>9593 | |
| | Type 3 Tests of Fix | ed Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value | ?r > F | | | | | |
| trtan<br>PREAD<br>BASE | 1 427<br>1 427<br>1 427 | 1.48 | 0.0003<br>0.2244<br><.0001 | | | | | |
| | | Least | Squares Mean | ns Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.3744<br>0.5350 | | 443.42<br>314.74 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least So | quares Means | Estimates | | | | |
| Effect | Label | Lower | Upper Ex | xponentiated | | ntiated<br>Lower | | ted |
| trtan<br>trtan | LSMeans, IDegLira<br>LSMeans, IDeg | 165.26<br>167.33 | 166.74<br>169.43 | 1.239E72<br>1.341E73 | | .936E71<br>.684E72 | 2.586<br>3.837 | |
| | | Least S | Squares Means | s Estimate | | | | |
| Effect | Label | | Margins | Estim | | ndard<br>Error | DF t Va | lue |

-2.3814

0.6544

427

-3.64

trtan Treatment contrast, IDegLira - IDeg WORK.ADATA2

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 102 of 334 | |

Parameter Code=WEIGHTU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtan Treatment contrast, IDegLira - IDeg 0.0003 0.05 -3.6677 -1.0951 0.09242

Least Squares Means Estimate

Exponentiated Lower Upper trtan Treatment contrast, IDegLira - IDeg 0.02553 0.3345

### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=C25208X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtan 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 431

Number of Observations

Number of Observations Read 431
Number of Observations Used 431
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 8.3053

Fit Statistics

-2 Res Log Likelihood 2142.1
AIC (Smaller is Better) 2144.1
BIC (Smaller is Better) 2148.1

Solution for Fixed Effects

Actual

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value -1.5403 0.8925 -1.73 427 Intercept -1.0802 427 -3.64 1 0.2968 trtan trtan BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.3398 0.2793 427 1.22 PREAD 0.02356 BASE 0.01127 427 2.09

# NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=C25208X

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial anti-Diabetic treatment | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
|---|---|---|---|---|
| Intercept<br>trtan | | 1 | 0.0851<br>0.0003 | 0.05<br>0.05 |
| trtan<br>PREAD<br>PREAD | BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD | 2 | 0.2244 | 0.05 |
| BASE | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 0.0371 | 0.05 |
| | Solution for Fixed Effect | ts | | |
| Effect | Pre Trial anti-Diabetic treatment | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
| Intercept | | | -3.2945 | 0.2140 |
| trtan<br>trtan | | 1 | -1.6637 | -0.4967 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | -0.2092 | 0.8887 |
| BASE | | | 0.001415 | 0.04570 |
| Ту | pe 3 Tests of Fixed Effects | | | |
| Effect | Num Den<br>DF DF F Value Pr > F | | | |

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| trtan | 1 | 427 | 13.24 | 0.0003 |
| PREAD | 1 | 427 | 1.48 | 0.2244 |
| BASE | 1 | 427 | 4.37 | 0.0371 |

### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.1698<br>0.2427 | 427<br>427 | -3.95<br>1.69 | <.0001<br>0.0917 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg | | -1.0038<br>0.06682 | -0.3363<br>0.8871 | | | |

### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=WEIGHTU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtan 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 431

Number of Observations

Number of Observations Read 431
Number of Observations Used 431
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 40.3667

Fit Statistics

-2 Res Log Likelihood 2818.8
AIC (Smaller is Better) 2820.8
AICC (Smaller is Better) 2820.8
BIC (Smaller is Better) 2824.8

Solution for Fixed Effects

Actual

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value -3.3957 1.9676 -1.73 427 Intercept -2.3814 -3.64 1 0.6544 427 trtan trtan BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.7491 0.6157 427 1.22 PREAD 0.02356 BASE 0.01127 427 2.09

#### NN9068 Date: 22 January 2020 | Novo Nordisk NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 106 of 334 Statistical document Page:

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - PP analysis set - appendix

Parameter Code=WEIGHTU

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial anti-Diabetic treatment | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
|---|---|---|---|---|
| Intercept<br>trtan<br>trtan | | 1 | 0.0851<br>0.0003 | |
| PREAD | BASAL INSULIN + METFORMIN | 2 | 0.2244 | 0.05 |
| PREAD<br>BASE | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 0.0371 | 0.05 |
| | Solution for Fixed Effec | ts | | |
| Effect | Pre Trial anti-Diabetic treatment | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
| | The first and blabette electioners | 01 (11) | | 0.4717 |
| Intercept<br>trtan | | 1 2 | -3.6677 | |
| trtan<br>PREAD | BASAL INSULIN + METFORMIN | 2 | -0.4611 | 1.9593 |
| PREAD<br>BASE | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 0.001415 | 0.04570 |
| Ту | pe 3 Tests of Fixed Effects | | | |
| Effect | Num Den<br>DF DF F Value Pr > F | | | |
| + | 1 427 12.24 0.0003 | | | |

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| trtan | 1 | 427 | 13.24 | 0.0003 |
| PREAD | 1 | 427 | 1.48 | 0.2244 |
| BASE | 1 | 427 | 4.37 | 0.0371 |

### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.3744<br>0.5350 | 427<br>427 | -3.95<br>1.69 | <.0001<br>0.0917 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg | | -2.2130<br>-0.1473 | -0.7414<br>1.9558 | | | |

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

### 13: Body weight after 26 weeks of treatment – change from baseline – statistical sensitivity analysis – completer analysis set - appendix

Parameter Code=C25208X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 429

Number of Observations

Number of Observations Read 429 Number of Observations Used 429 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 8.3003

Fit Statistics

-2 Res Log Likelihood 2131.9
AIC (Smaller is Better) 2133.9
AICC (Smaller is Better) 2133.9
BIC (Smaller is Better) 2137.9

Solution for Fixed Effects

Planned Treatment for Period

| Effect | Pre Trial anti-Diabetic treatment | Period<br>01 (N) | Estimate | Standard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn | | 1 2 | -1.3952<br>-1.1604<br>0 | 0.8950<br>0.2986 | 425<br>425 | -1.56<br>-3.89 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 0.3621 | 0.2799 | 425 | 1.29 |
| BASE | | | 1.0225 | 0.01126 | 425 | 90.79 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 108 of 334 | |

Parameter Code=C25208X

The Mixed Procedure

| | | Solution fo | r Fixed Effec | ets | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | Planned<br>Treatment<br>for | | | | | |
| Effect | Pre Trial ar | nti-Diabetic trea | tment | Period<br>01 (N) | Pr > t | alp Alp | ha | |
| Intercep<br>trtpn | t | | | 1<br>2 | 0.119 | | | |
| trtpn<br>PREAD<br>PREAD | | N + METFORMIN | ONE OBJED OAD | | 0.196 | 54 0. | 05 | |
| BASE | BASAL INSULI | N + METFORMIN + | ONE OTHER OAD | , | <.000 | 0. | 05 | |
| | | Solution f | or Fixed Effe | ects | | | | |
| | | | | Planned<br>Treatment<br>for | | | | |
| Effect | Pre Trial an | nti-Diabetic trea | tment | Period<br>01 (N) | Lowe | er U | pper | |
| Intercep<br>trtpn | t | | | 1 2 | -3.154<br>-1.747 | | 3639<br>5735 | |
| trtpn PREAD BASAL INSULIN + METFORMIN | | | -0.188 | 30 0. | 9123 | | | |
| PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD<br>BASE | | | , | 1.000 | 1. | 0446 | | |
| | Type 3 Tests of | Fixed Effects | | | | | | |
| Effect | | Den<br>DF F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 4 | 125 15.10<br>125 1.67<br>125 8243.01 | 0.0001<br>0.1964<br><.0001 | | | | | |
| | | Leas | t Squares Mea | ns Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegI<br>LSMeans, IDeg | ira WORK.ADATA<br>WORK.ADATA | | 0.1694<br>0.2451 | 425<br>425 | 444.45<br>311.93 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least | Squares Means | Estimates | | | | |
| Effect | Label | Lower | Upper E | xponentiated | | nentiated<br>Lower | Exponentia<br>Up | ted<br>per |
| trtpn<br>trtpn | LSMeans, IDegI<br>LSMeans, IDeg | 74.9726<br>75.9842 | 75.6386<br>76.9478 | 5.068E32<br>1.617E33 | | 3.632E32<br>9.989E32 | 7.07<br>2.618 | |
| | | Least | Squares Mean | s Estimate | | | | |
| Effect | Label | | Margins | Estim | | andard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -1.1604 0.2986 425 -3.89

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 109 of 334 | |

Parameter Code=C25208X

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.0001 0.05 -1.7473 -0.5735 0.3134

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.1742 Exponentiated 0.5635

## NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set - appendix

Parameter Code=WEIGHTU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 429

Number of Observations

Number of Observations Read 429
Number of Observations Used 429
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 40.3426

Fit Statistics

-2 Res Log Likelihood 2805.4
AIC (Smaller is Better) 2807.4
AICC (Smaller is Better) 2807.5
BIC (Smaller is Better) 2811.5

Solution for Fixed Effects

Planned

Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value -3.0759 1.9731 425 -1.56Intercept -2.5583 425 -3.89 1 0.6583 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.7984 0.6171 425 1.29 PREAD 1.0225 BASE 0.01126 425 90.79

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 111 of 334 | |

Parameter Code=WEIGHTU

The Mixed Procedure

| THE MIX | ed Procedu | re | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Solution for | Fixed Effe | cts | | | | |
| Effect | Pre Tr | ial anti-D | iabetic treat | ment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > | t Alp | ha | |
| Interce | pt. | | | | | 0.11 | 98 0. | 0.5 | |
| trtpn<br>trtpn | 1 | | | | 1 2 | 0.00 | | | |
| PREAD | | INSULIN + 1 | | | | 0.19 | 64 0. | 05 | |
| PREAD<br>BASE | BASAL | INSULIN + 1 | METFORMIN + O | NE OTHER OA | D | <.00 | 01 0. | 05 | |
| | | | Solution fo | r Fixed Effe | ects | | | | |
| Effect | Pre Tr | ial anti-D | iabetic treat | ment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Low | er U | pper | |
| | | | | | V = (31) | | | | |
| Interce<br>trtpn | pt | | | | 1 | -6.95<br>-3.85 | | 8023<br>2644 | |
| trtpn PREAD BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD BASE | | | 2 | -0.41 | 45 2. | 0113 | | | |
| | | | D | 1.00 | 03 1. | 0446 | | | |
| | Type 3 Te | sts of Fix | ed Effects | | | | | | |
| Effect | Num<br>DF | | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 425 | 1.67 | 0.0001<br>0.1964<br><.0001 | | | | | |
| | | | Least | Squares Mea | ans Estimates | : | | | |
| | | | | | Standard | | | | |
| Effect | Label | | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADATA2<br>WORK.ADATA2 | | | 425<br>425 | 444.45<br>311.93 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least S | quares Mean | s Estimates | | | | |
| Effect | Label | | Lower | Upper 1 | Exponentiated | | nentiated<br>Lower | Exponentia<br>Up | ted |
| trtpn | | IDegLira | 165.29 | 166.75 | 1.264E72 | | 6.066E71 | 2.634 | |
| trtpn | LSMeans, | IDeg | 167.52 | 169.64 | 1.632E73 | i | 5.642E72 | 4.722 | E/3 |
| | | | Least | Squares Mean | ns Estimate | | | | |
| Effect | Label | | | Margin | s Estim | | tandard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -2.5583 0.6583 425 -3.89

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 112 of 334 | |

Parameter Code=WEIGHTU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.0001 0.05 -3.8522 -1.2644 0.07744

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.02123 0.2824

## NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set - appendix

Parameter Code=C25208X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 429

Number of Observations

Number of Observations Read 429
Number of Observations Used 429
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 8.3003

Fit Statistics

-2 Res Log Likelihood 2131.9
AICC (Smaller is Better) 2133.9
AICC (Smaller is Better) 2133.9
BIC (Smaller is Better) 2137.9

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value -1.3952 -1.56 0.8950 425 Intercept 425 -3.89 1 -1.1604 0.2986 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.3621 0.2799 425 1.29 PREAD 0.02247 BASE 0.01126 425 2.00

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 114 of 334 | |

Parameter Code=C25208X

The Mixed Procedure

### Solution for Fixed Effects

| | 001401011 101 111104 211000 | | | |
|---|---|---|---|---|
| Effect | Pre Trial anti-Diabetic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| | | (/ | | |
| Intercept<br>trtpn<br>trtpn | | 1 | 0.1198<br>0.0001 | 0.05<br>0.05 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | _ | 0.1964 | 0.05 |
| BASE | BASAL INSULIN + MELFORMIN + ONE OTHER OAD | | 0.0466 | 0.05 |
| | Solution for Fixed Effec | ts | | |
| Effect | Pre Trial anti-Diabetic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
| Intercept<br>trtpn | | 1 | -3.1543<br>-1.7473 | 0.3639<br>-0.5735 |
| trtpn<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | 2 | -0.1880 | 0.9123 |
| PREAD<br>BASE | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 0.000336 | 0.04461 |
| Ту | pe 3 Tests of Fixed Effects | | | |
| Effect | Num Den<br>DF DF F Value Pr > F | | | |

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| trtpn | 1 | 425 | 15.10 | 0.0001 |
| PREAD | 1 | 425 | 1.67 | 0.1964 |
| BASE | 1 | 425 | 3.98 | 0.0466 |

### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | -0.6760<br>0.4844 | 0.1694<br>0.2451 | 425<br>425 | -3.99<br>1.98 | <.0001<br>0.0488 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | | -1.0090<br>.002600 | -0.3429<br>0.9663 | | | |

### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set - appendix

Parameter Code=WEIGHTU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 429

Number of Observations

Number of Observations Read 429
Number of Observations Used 429
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 40.3426

Fit Statistics

-2 Res Log Likelihood 2805.4
AIC (Smaller is Better) 2807.4
AICC (Smaller is Better) 2807.5
BIC (Smaller is Better) 2811.5

Solution for Fixed Effects

Planned

Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value -3.0759 -1.56 1.9731 425 Intercept -2.5583 425 -3.89 0.6583 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.7984 0.6171 425 1.29 PREAD 0.02247 BASE 0.01126 425 2.00

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 116 of 334 | |

Parameter Code=WEIGHTU

The Mixed Procedure

### Solution for Fixed Effects

| | | | DOIGCION I | or rined brice | | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | l anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn | | | | | 1 | 0.1198<br>0.0001 | 0.05<br>0.05 |
| trtpn<br>PREAD | | | METFORMIN | | _ | 0.1964 | 0.05 |
| PREAD<br>BASE | BASAL INS | SULIN + | METFORMIN + | ONE OTHER OAD | | 0.0466 | 0.05 |
| | | | Solution | for Fixed Effe | cts | | |
| Fffect | Pro Trial | anti-D | iabetic tre | atmont | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
| | rie iliai | anci-D | iabetic tie | acment | OI (N) | | |
| Intercept<br>trtpn<br>trtpn | | | | | 1 | -6.9541<br>-3.8522 | 0.8023<br>-1.2644 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | _ | -0.4145 | 2.0113 |
| BASE | DASAL INC | OUTIN T | METFORMIN T | ONE OTHER OAD | | 0.000336 | 0.04461 |
| Ту | rpe 3 Tests | of Fix | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn | 1 | 425 | 15.10 | 0.0001 | | | |

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| trtpn | 1 | 425 | 15.10 | 0.0001 |
| PREAD | 1 | 425 | 1.67 | 0.1964 |
| BASE | 1 | 425 | 3.98 | 0.0466 |

### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | -1.4903<br>1.0680 | 0.3735<br>0.5404 | 425<br>425 | -3.99<br>1.98 | <.0001<br>0.0488 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | | -2.2245<br>.005731 | -0.7561<br>2.1302 | | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 117 of 334 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

#### Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Subjint
Estimation Method
Residual Variance Method
Prixed Effects SE Method
Degrees of Freedom Method
Satterthwaite

### Class Level Information

| Class | Levels | Values |
|---|---|---|
| TRT01PN<br>avisitn<br>PREAD | 2<br>6<br>2 | 1 2<br>100 150 190 230 270 330<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN +<br>ONE OTHER OAD |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 118 of 334 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

Class Level Information

Levels Class Values SUBJID 453

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 119 of 334 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure



### Dimensions

| Covariance | Parameters | 21 |
|-------------|------------|-----|
| Columns in | X | 31 |
| Columns in | Z | 0 |
| Subjects | | 453 |
| Max Obs per | Subject | 6 |

### Number of Observations

| Number | of | Observations | Read | 2718 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2597 |
| Number | of | Observations | Not Used | 121 |

## NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5tatus: Final 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

### Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 11799.74282062 | |
| 1 | 2 | 8867.20333115 | 0.00000625 |
| 2 | 1 | 8867.19027918 | 0.00000000 |

Convergence criteria met.

#### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|---|---|---|
| UN (1,1)<br>UN (2,1)<br>UN (2,2)<br>UN (3,1)<br>UN (3,2)<br>UN (4,1)<br>UN (4,2)<br>UN (4,3)<br>UN (4,4)<br>UN (5,1)<br>UN (5,2)<br>UN (5,3)<br>UN (5,4)<br>UN (5,5)<br>UN (6,1) | Subject SUBJID | 2.0140<br>1.9791<br>3.9752<br>2.1981<br>3.6319<br>5.2127<br>2.1194<br>3.6227<br>4.9685<br>6.0757<br>2.1682<br>3.7181<br>5.0852<br>5.7532<br>6.9717<br>2.3366<br>3.7858 |
| - ( - / - / | SUBJID<br>SUBJID<br>SUBJID<br>SUBJID | 5.2013<br>5.7740<br>6.5474<br>8.3028 |

### Fit Statistics

| -2 Res Log Likelihood | 8867.2 |
|--------------------------|--------|
| AIC (Smaller is Better) | 8909.2 |
| AICC (Smaller is Better) | 8909.6 |
| BIC (Smaller is Better) | 8995.6 |

### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 20 | 2932.55 | <.0001 |

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|-----------|---------|--------|
| TRT01PN(avisitn) | 6 | 436 | 2.83 | 0.0103 |
| PREAD(avisitn) | 6 | 433 | 1.45 | 0.1950 |
| BASE(avisitn) | 6 | 433 | 5778.27 | <.0001 |

| NN9068 | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|
| Clinical Trial Report | Status: | Final | |
| Statistical document | Page: | 121 of 334 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| TRT01PN(avisitn) TRT01PN(avisitn) | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ANA_DATA<br>WORK.ANA_DATA | 75.2925<br>76.4274 | 0.1691<br>0.2411 | 431.5<br>440.4 | 445.17<br>316.99 | <.0001<br><.0001 |
| Least Squares Means Estimates | | | | | | | |
| Effect | Label | Alpha I | Lower | Upper | | | |
| TRT01PN(avisitn) TRT01PN(avisitn) | LSMeans, IDegLira<br>LSMeans, IDeg | | | 5.6249<br>6.9013 | | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 122 of 334 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

### Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Subject Effect
Stimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Satterthwaite

#### Class Level Information

| Class | Levels | Values |
|---|---|---|
| TRT01PN<br>avisitn<br>PREAD | 2<br>6<br>2 | 1 2<br>100 150 190 230 270 330<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN +<br>ONE OTHER OAD |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 123 of 334 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

Class Level Information

| | 01000 | 20,01 1111011110111 |
|--------|--------|---------------------|
| Class | Levels | Values |
| SUBJID | 453 | |
| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 124 of 334 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure



#### Dimensions

| Covariance | Parameters | 21 |
|-------------|------------|-----|
| Columns in | X | 31 |
| Columns in | Z | 0 |
| Subjects | | 453 |
| Max Obs per | Subject | 6 |

### Number of Observations

| Number | of | Observations | Read | 2718 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2597 |
| Number | of | Observations | Not Used | 121 |

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5tatus: Final 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

#### Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 15877.43246205 | |
| 1 | 2 | 12944.89297256 | 0.00000315 |
| 2 | 1 | 12944.87992061 | 0.00000000 |

Convergence criteria met.

#### Covariance Parameter Estimates

| Subject | Estimate |
|---|---|
| SUBJID<br>SU | 9.7886<br>9.6190<br>19.3211<br>10.6836<br>17.6521<br>25.3355<br>10.3012<br>17.6076<br>24.1485<br>29.5302<br>10.5383<br>18.0715<br>24.7161<br>27.9627<br>33.8849<br>11.3569 |
| SUBJID<br>SUBJID<br>SUBJID<br>SUBJID<br>SUBJID | 18.4005<br>25.2801<br>28.0636<br>31.8228<br>40.3546 |
| | SUBJID<br>SU |

#### Fit Statistics

| -2 Res Log Likelihood | 12944.9 |
|--------------------------|---------|
| AIC (Smaller is Better) | 12986.9 |
| AICC (Smaller is Better) | 12987.2 |
| BIC (Smaller is Better) | 13073.3 |

#### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 20 | 2932.55 | <.0001 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|-----------|---------|--------|
| TRT01PN(avisitn) | 6 | 436 | 2.83 | 0.0103 |
| PREAD(avisitn) | 6 | 433 | 1.45 | 0.1950 |
| BASE(avisitn) | 6 | 433 | 5778.27 | <.0001 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 126 of 334 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| TRT01PN(avisitn) TRT01PN(avisitn) | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ANA_DATA<br>WORK.ANA_DATA | 165.99<br>168.49 | 0.3729<br>0.5315 | 431.5<br>440.4 | 445.17<br>316.99 | <.0001<br><.0001 |
| | Least Squares Mea | ns Estimates | | | | | |
| Effect | Label | Alpha 1 | Lower | Upper | | | |
| TRT01PN(avisitn) TRT01PN(avisitn) | LSMeans, IDegLira<br>LSMeans, IDeg | | 65.26<br>67.45 | 166.72<br>169.54 | | | |

| NN9068 | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|
| Clinical Trial Report | Status: | Final | |
| Statistical document | Page: | 127 of 334 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

#### Model Information

Data Set
Dependent Variable
CHG
Covariance Structure
Subject Effect
Subject Effect
Stimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Satterthwaite

#### Class Level Information

| Class | Levels | Values |
|---|---|---|
| TRT01PN<br>avisitn<br>PREAD | 2<br>6<br>2 | 1 2<br>100 150 190 230 270 330<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN +<br>ONE OTHER OAD |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 128 of 334 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

Class Level Information

Class Levels Values
SUBJID 453



| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 129 of 334 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure



#### Dimensions

| Covariance | Parameters | 2.1 |
|-------------|------------|-----|
| Columns in | | 31 |
| Columns in | Z | 0 |
| Subjects | | 453 |
| Max Obs per | r Subject | 6 |

### Number of Observations

| Number | of | Observations | Read | 2718 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2597 |
| Number | of | Observations | Not Used | 121 |


Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

#### Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 11799.74282062 | |
| 1 | 2 | 8867.20333114 | 0.00000625 |
| 2 | 1 | 8867.19027918 | 0.00000000 |

Convergence criteria met.

#### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|---|---|---|
| UN (1,1)<br>UN (2,1)<br>UN (2,2)<br>UN (3,1)<br>UN (3,2)<br>UN (3,3)<br>UN (4,1)<br>UN (4,2)<br>UN (4,3)<br>UN (4,4)<br>UN (5,1)<br>UN (5,2)<br>UN (5,3)<br>UN (5,4)<br>UN (5,5) | SUBJID | 2.0140<br>1.9791<br>3.9752<br>2.1981<br>3.6319<br>5.2127<br>2.1194<br>3.6227<br>4.9685<br>6.0757<br>2.1682<br>3.7181<br>5.0852<br>5.7532<br>6.9717 |
| UN(6,2) | SUBJID<br>SUBJID<br>SUBJID<br>SUBJID<br>SUBJID<br>SUBJID | 2.3366<br>3.7858<br>5.2013<br>5.7740<br>6.5474<br>8.3028 |
| . , - , | | |

#### Fit Statistics

| -2 Res Log Likelihood | 8867.2 |
|--------------------------|--------|
| AIC (Smaller is Better) | 8909.2 |
| AICC (Smaller is Better) | 8909.6 |
| BIC (Smaller is Better) | 8995.6 |

#### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 20 | 2932.55 | <.0001 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|-----------|---------|--------|
| TRT01PN(avisitn) | 6 | 436 | 2.83 | 0.0103 |
| PREAD(avisitn) | 6 | 433 | 1.45 | 0.1950 |
| BASE(avisitn) | 6 | 433 | 2.12 | 0.0498 |

| NN9068 | | Date: | 22 January 2020 Novo Nord | isk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 131 of 334 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

#### Least Squares Means Estimates

| Effect | Label | Margins Es | Standa<br>Estimate Err | |
|---|---|---|---|---|
| TRT01PN(avisitn) TRT01PN(avisitn) | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ANA_DATA WORK.ANA_DATA | -0.6806 0.16<br>0.4543 0.24 | |
| | Least Squares Mean | s Estimates | | |
| Effect | Label | Pr > t Alph | oha Lower | Upper |
| TRT01PN(avisitn) TRT01PN(avisitn) | | | 05 -1.0131<br>05 -0.01953 | |
| | Least Squares | Means Estimate | | |
| Effect | Label | Margins | Estimate | Standard<br>Error DF |
| TRT01PN(avisitn) | Treatment contrast, IDegLira - | IDeg WORK.ANA_DA | TA -1.1350 | 0.2951 437.4 |
| Least Squares Means Estimate | | | | |
| Effect | Label | t Value Pr | > t Alpha | Lower Upper |
| TRT01PN(avisitn) | Treatment contrast, IDegLira - | IDeg -3.85 | 0.0001 0.05 | -1.7150 -0.5549 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 132 of 334 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

#### Model Information

Data Set
Dependent Variable
CHG
Covariance Structure
Subject Effect
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Satterthwaite

Class Level Information

| Class | Levels | Values |
|---|---|---|
| TRT01PN<br>avisitn<br>PREAD | 2<br>6<br>2 | 1 2<br>100 150 190 230 270 330<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN +<br>ONE OTHER OAD |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 133 of 334 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

Class Level Information

Levels Class Values SUBJID 453

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 134 of 334 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure



### Dimensions

| Covariance | Parameters | 21 |
|-------------|------------|-----|
| Columns in | X | 31 |
| Columns in | Z | 0 |
| Subjects | | 453 |
| Max Obs per | Subject | 6 |

### Number of Observations

| Number | of | Observations | Read | 2718 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2597 |
| Number | of | Observations | Not Used | 121 |

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5tatus: Final 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set - appendix

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

#### Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 15877.43246205 | |
| 1 | 2 | 12944.89297256 | 0.00000315 |
| 2 | 1 | 12944.87992060 | 0.00000000 |

Convergence criteria met.

#### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|---|---|---|
| UN(1,1)<br>UN(2,1)<br>UN(2,2) | Subject SUBJID | 9.7886<br>9.6190<br>19.3211<br>10.6836<br>17.6521<br>25.3355<br>10.3012<br>17.6076<br>24.1485<br>29.5302<br>10.5383<br>18.0715<br>24.7161<br>27.9627<br>33.8849<br>11.3569 |
| UN (6, 2)<br>UN (6, 3)<br>UN (6, 4)<br>UN (6, 5)<br>UN (6, 6) | SUBJID<br>SUBJID<br>SUBJID<br>SUBJID<br>SUBJID | 18.4005<br>25.2801<br>28.0636<br>31.8228<br>40.3546 |

#### Fit Statistics

| -2 Res Log Likelihood | 12944.9 |
|--------------------------|---------|
| AIC (Smaller is Better) | 12986.9 |
| AICC (Smaller is Better) | 12987.2 |
| BIC (Smaller is Better) | 13073.3 |

#### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 20 | 2932.55 | <.0001 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|-----------|---------|--------|
| TRT01PN(avisitn) | 6 | 436 | 2.83 | 0.0103 |
| PREAD(avisitn) | 6 | 433 | 1.45 | 0.1950 |
| BASE(avisitn) | 6 | 433 | 2.12 | 0.0498 |

| NN9068 | | Date: | 22 January 2020 <b>Novo No</b> | ordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 136 of 334 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

#### Least Squares Means Estimates

| Effect | Label | Margins | Standa<br>Estimate Err | |
|---|---|---|---|---|
| TRT01PN(avisitn) TRT01PN(avisitn) | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ANA_DATA<br>WORK.ANA_DATA | -1.5006 0.37<br>1.0016 0.53 | |
| | Least Squares Mear | ns Estimates | | |
| Effect | Label | Pr > t Al | pha Lower | Upper |
| TRT01PN(avisitn) TRT01PN(avisitn) | Change from baseline, IDegLira Change from baseline, IDeg | | -2.2334<br>-0.04305 | -0.7677<br>2.0463 |
| | Least Squares | Means Estimate | | |
| Effect | Label | Margins | Estimate | Standard<br>Error DF |
| TRT01PN(avisitn) | Treatment contrast, IDegLira - | IDeg WORK.ANA_D | DATA -2.5022 | 0.6506 437.4 |
| Least Squares Means Estimate | | | | |
| Effect | Label | t Value P | Pr > t Alpha | Lower Upper |
| TRT01PN(avisitn) | Treatment contrast, IDegLira - | IDeg -3.85 | 0.0001 0.05 | -3.7810 -1.2234 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 137 of 334 | |

### 15: Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis conditional multiple imputation - full analysis set - appendix

paramsort=1 Parameter Code=C25208X Label=LSMeans, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME ABS MI

Number of Imputations

Variance Information (1000 Imputations)

-----Variance-----

Parameter Between Within Total 0.055557 0.058633 362883 Estimate 0.003073

Variance Information (1000 Imputations)

Relative Fraction Increase Missing Relative in Variance Information Efficiency Parameter 0.052474 Estimate 0.055374 0.999948

Parameter Estimates (1000 Imputations)

95% Confidence Std Error Limits DF Estimate Minimum Maximum Parameter Estimate 76.457794 0.242143 75.98320 76.93239 362883 76.282848 76.635672

Parameter Estimates (1000 Imputations)

t for HO:

Theta0 Parameter=Theta0 Pr > |t| Parameter 315.75 <.0001 Estimate

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set - appendix

paramsort=1 Parameter Code=C25208X Label=LSMeans, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME ABS MI

Number of Imputations 1000

Variance Information (1000 Imputations)

Parameter Between Within Total DF

Estimate 0.001029 0.027690 0.028721 776179

Variance Information (1000 Imputations)

Relative Fraction

Increase Missing Relative Parameter in Variance Information Efficiency
Estimate 0.037211 0.035878 0.999964

Parameter Estimates (1000 Imputations)

95% Confidence

 Parameter
 Estimate
 Std Error
 Limits
 DF
 Minimum
 Maximum

 Estimate
 75.358828
 0.169471
 75.02667
 75.69099
 776179
 75.271846
 75.482403

Parameter Estimates (1000 Imputations)

## NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set - appendix

paramsort=2 Parameter Code=WEIGHTU Label=LSMeans, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME ABS MI

Number of Imputations 1000

Variance Information (1000 Imputations)

Parameter Between Within Total DF Estimate 0.014938 0.270027 0.284980 362883

Variance Information (1000 Imputations)

Relative Fraction

Increase Missing Relative Parameter in Variance Information Efficiency
Estimate 0.055374 0.052474 0.999948

Parameter Estimates (1000 Imputations)

0.533835 167.5143 169.6069 362883 168.174892 168.952737

95% Confidence
Parameter Estimate Std Error Limits DF Minimum Maximum

Parameter Estimates (1000 Imputations)

168.560582

Estimate

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set - appendix

paramsort=2 Parameter Code=WEIGHTU Label=LSMeans, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME ABS MI

Number of Imputations 1000

Variance Information (1000 Imputations)

Parameter Between Within Total DF

Estimate 0.005003 0.134584 0.139592 776179

Variance Information (1000 Imputations)

Relative Fraction

Increase Missing Relative Parameter in Variance Information Efficiency
Estimate 0.037211 0.035878 0.999964

Parameter Estimates (1000 Imputations)

95% Confidence

 Parameter
 Estimate
 Std Error
 Limits
 DF
 Minimum
 Maximum

 Estimate
 166.137776
 0.373621
 165.4055
 166.8701
 776179
 165.946014
 166.410213

Parameter Estimates (1000 Imputations)


Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set - appendix

paramsort=1 Parameter Code=C25208X Label=Change from baseline, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME CHG MI

Number of Imputations 1000

Variance Information (1000 Imputations)

Parameter Between Within Total DF Estimate 0.003073 0.055557 0.058633 362883

Variance Information (1000 Imputations)

Relative Fraction

Increase Missing Relative Parameter in Variance Information Efficiency
Estimate 0.055374 0.052474 0.999948

Parameter Estimates (1000 Imputations)

 
 Parameter
 Estimate
 Std Error
 95% Confidence Limits
 DF
 Minimum
 Maximum

 Estimate
 0.465300
 0.242143
 -0.00929
 0.939894
 362883
 0.290354
 0.643178

Parameter Estimates (1000 Imputations)

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 142 of 334 | |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set - appendix

paramsort=1 Parameter Code=C25208X Label=Change from baseline, IDeqLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI Data Set WORK. Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Within Total DF Parameter Between 0.027690 0.028721 776179 Estimate 0.001029

Variance Information (1000 Imputations)

Relative Fraction

Relative Increase Missing in Variance Information Efficiency 0.037211 0.035878 0.999964 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence

DF Minimum Std Error Parameter Estimate Limits Maximum -0.633667 0.169471 -0.96583 -0.30151 776179 -0.720649 -0.510092 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -3.74 0.0002 Estimate

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 143 of 334 | |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set - appendix

paramsort=1 Parameter Code=C25208X Label=Treatment contrast, IDeqLira - IDeq Statement Number=2

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME CHG MI Data Set WORK. Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.083600 0.087324 549385 Estimate 0.003720

Variance Information (1000 Imputations)

Fraction Relative

Relative Increase Missing in Variance Information Efficiency 0.044542 0.042646 0.999957 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Std Error Parameter Estimate Limits

DF Minimum Maximum -1.098966 0.295507 -1.67815 -0.51978 549385 -1.284088 -0.904160 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -3.72 0.0002 Estimate

#### 22 January 2020 | Novo Nordisk NN9068 Date: NN9068-4166 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Final Status: Statistical document 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set - appendix

paramsort=2 Parameter Code=WEIGHTU Label=Change from baseline, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME CHG MI

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total

0.270027 0.284980 362883 Estimate 0.014938

Variance Information (1000 Imputations)

Relative Fraction

1.025810

Estimate

Relative Missing Information Increase in Variance Efficiency 0.055374 0.052474 0.999948 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum 0.533835 -0.02049 2.072111 362883 0.640120

1.417965

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter

0 1.92 0.0547 Estimate

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 145 of 334 | |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set - appendix

paramsort=2 Parameter Code=WEIGHTU Label=Change from baseline, IDeqLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI Data Set WORK. Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.134584 0.139592 776179 Estimate 0.005003

Variance Information (1000 Imputations)

Fraction Relative

Relative Increase Missing in Variance Information Efficiency 0.037211 0.035878 0.999964 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence

DF Minimum Std Error Parameter Estimate Limits Maximum -1.396996 0.373621 -2.12928 -0.66471 776179 -1.588758 -1.124560 Estimate

Parameter Estimates (1000 Imputations)

t for HO:

Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -3.74 0.0002 Estimate

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 146 of 334 | |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set - appendix

paramsort=2 Parameter Code=WEIGHTU Label=Treatment contrast, IDegLira - IDeg Statement Number=2

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME CHG MI Data Set WORK. Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.406328 0.424427 549385 Estimate 0.018081

Variance Information (1000 Imputations)

Fraction Relative

Relative Increase Missing in Variance Information Efficiency 0.044542 0.042646 0.999957 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence

e DF Minimum Std Error Parameter Estimate Limits Maximum -2.422806 0.651481 -3.69969 -1.14592 549385 -2.830930 -1.993332 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter

0 -3.72 0.0002 Estimate

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

### 16: Waist circumference after 26 weeks of treatment – change from baseline – supportive statistical analysis – full analysis set - appendix

Parameter Code=MEANWAIC

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 15.5557

Fit Statistics

-2 Res Log Likelihood 2532.4
AIC (Smaller is Better) 2534.4
AICC (Smaller is Better) 2534.4
BIC (Smaller is Better) 2538.5

Solution for Fixed Effects

Planned Treatment for

| Effect | Pre Trial anti-Diabetic treatment | Period<br>01 (N) | Estimate | Standard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn | | 1 2 | 6.1773<br>-0.8684<br>0 | 2.0732<br>0.3938 | 449<br>449 | 2.98<br>-2.21 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 0.3609 | 0.3724 | 449 | 0.97 |
| BASE | Zidiiz Tilouzii ( izzidiati ( onz diizi diz | | 0.9397 | 0.02113 | 449 | 44.48 |

#### NN9068 22 January 2020 | Novo Nordisk Date: NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Waist circumference after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=MEANWAIC

The Mixed Procedure

| | | Solution for | Fixed Effect | s | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | Planned<br>Treatment<br>for | | | | |
| Effect | Pre Trial anti-D | iabetic treat | ment | Period<br>01 (N) | Pr > t | Alph | a | |
| Interceptrtpn trtpn | pt | | | 1 2 | 0.0030<br>0.0279 | | | |
| PREAD<br>PREAD | BASAL INSULIN +<br>BASAL INSULIN + | | NE OTHER OAD | 2 | 0.3330 | 0.0 | 5 | |
| BASE | DAGAL INSCLIN | HEITOITHIN I C | NUL OTHER OAD | | <.0001 | 0.0 | 5 | |
| | | Solution fo | or Fixed Effec | ets | | | | |
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| | Pre Trial anti-D | iabetic treat | ment | 01 (N) | Lower | - | per | |
| Intercept trtpn | pt | | | 1 2 | 2.1029<br>-1.6422 | | | |
| trtpn<br>PREAD<br>PREAD | BASAL INSULIN +<br>BASAL INSULIN + | | ME OHIED OAD | ۷ | -0.3710 | 1.0 | 928 | |
| BASE | DASAL INSULIN 1 | MEIPONMIN I C | NE OTHER OAD | | 0.8982 | 0.9 | 812 | |
| | Type 3 Tests of Fix | ed Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 449<br>1 449<br>1 449 | | 0.0279<br>0.3330<br><.0001 | | | | | |
| | | Least | : Squares Mear | ns Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.2271<br>0.3213 | 449<br>449 | 423.69<br>302.13 | <.0001<br><.0001 | 0.05 |
| | | Least S | Gquares Means | Estimates | | | | |
| Effect | Label | Lower | Upper Ex | xponentiated | | ntiated<br>Lower | | ted<br>per |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | 95.7661<br>96.4493 | 96.6586<br>97.7123 | 6.088E41<br>1.451E42 | | .897E41<br>.716E41 | 9.513<br>2.728 | |
| | | Least | Squares Means | s Estimate | | | | |
| Effect | Label | | Margins | Estim | | ndard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -0.8684 0.3938 449

-2.21

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 149 of 334 | |

Waist circumference after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=MEANWAIC

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.0279 0.05 -1.6422 -0.09459 0.4196

Least Squares Means Estimate

Exponentiated Label Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.1935 0.9097

# NN9068 NN9068-4166 Clinical Trial Report Statistical document CONFIDENTIAL Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

Waist circumference after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=MEANWAIC

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453
Number of Observations Used 453
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 15.5557

Fit Statistics

-2 Res Log Likelihood 2532.4
AIC (Smaller is Better) 2534.4
AICC (Smaller is Better) 2534.4
BIC (Smaller is Better) 2538.5

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 6.1773 2.0732 449 2.98 Intercept 1 -0.8684 0.3938 -2.21 449 trtpn trtpn PREAD BASAL INSULIN + METFORMIN 0.3609 449 0.97 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.06029 BASE 0.02113 449 -2.85

#### NN9068 Date: 22 January 2020 | Novo Nordisk NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 151 of 334 Statistical document Page:

Waist circumference after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=MEANWAIC

The Mixed Procedure

| Solution for Fixed Effects | | | | | | |
|---|---|---|---|---|---|---|
| Effect | Pre Trial anti-Dia | abetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept | | | | 1 | 0.0030<br>0.0279 | 0.05<br>0.05 |
| trtpn<br>PREAD<br>PREAD | BASAL INSULIN + MI<br>BASAL INSULIN + MI | | ONE OTHER OAD | 2 | 0.3330 | 0.05 |
| BASE | | | | | 0.0045 | 0.05 |
| | | Solution | for Fixed Effec | ts | | |
| | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial anti-Dia | abetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn<br>PREAD<br>PREAD | BASAL INSULIN + MI<br>BASAL INSULIN + MI | | ONE OTHER OAD | 1 2 | 2.1029<br>-1.6422<br>-0.3710 | 10.2517<br>-0.09459<br>1.0928 |
| BASE | BASAL INSULIN + MI | SIFORMIN + | ONE OTHER OAD | | -0.1018 | -0.01877 |
| Ту | pe 3 Tests of Fixed | d Effects | | | | |
| Effect | Num Den<br>DF DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1 449<br>1 449<br>1 449 | 4.86<br>0.94<br>8.15 | 0.0279<br>0.3330<br>0.0045 | | | |

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| trtpn | 1 | 449 | 4.86 | 0.0279 |
| PREAD | 1 | 449 | 0.94 | 0.3330 |
| BASE | 1 | 449 | 8.15 | 0.0045 |

### Least Squares Means Estimates

Standard

| Effect | Label | Margins | Estimate | Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.2271<br>0.3213 | 449<br>449 | -1.50<br>1.64 | 0.1335<br>0.1016 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | | -0.7876<br>-0.1044 | 0.1049<br>1.1585 | | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 152 of 334 | |

### 17: Fasting plasma glucose after 26 weeks of treatment – change from baseline – supportive statistical analysis – full analysis set - appendix

Parameter Code=C105585P

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REMI Residual Variance Method Fixed Effects SE Method Profile Model-Based Degrees of Freedom Method Residual

Class Level Information

Levels Values Class

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters Columns in X Columns in Z 6 Ω Subjects Max Obs per Subject

Number of Observations

Number of Observations Read Number of Observations Used 453 453 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 2.9791

Fit Statistics

-2 Res Log Likelihood AIC (Smaller is Better) 1790.0 AICC (Smaller is Better) 1790.0 BIC (Smaller is Better) 1794.1

Solution for Fixed Effects

DF t Value

18.16

-0.75

3.64

449

449

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate 01 (N) Error Intercept 5.8339 0.3212 trtpn -0.4165 0.1722 2 Ω

trtpn BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD -0.1213 PREAD 0.1624 449 PREAD 0.1052 0.02893 BASE

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 153 of 334 | |

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=C105585P

The Mixed Procedure

| The Mixe | ed Procedure | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Solution for F: | ixed Effec | cts | | | | |
| Effect | Pre Trial anti- | Diabetic treatmen | nt | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | ıa | |
| | | pragocio creatmer | | 01 (11) | | - | | |
| Intercep<br>trtpn<br>trtpn | ot | | | 1 2 | <.0001<br>0.0160 | 0.0 | | |
| PREAD<br>PREAD | BASAL INSULIN + | METFORMIN<br>METFORMIN + ONE | OTHER ONE | | 0.4557 | 0.0 | )5 | |
| BASE | BASAL INSULIN T | METFORMIN + ONE | OIRER OAL | ) | 0.0003 | 0.0 | )5 | |
| | | Solution for I | Fixed Effe | ects | | | | |
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial anti- | Diabetic treatmen | nt | 01 (N) | Lower | Uŗ | oper | |
| Interceptrtpn<br>trtpn<br>trtpn | ot | | | 1 2 | 5.2026<br>-0.7550 | | 1651<br>7803 | |
| PREAD | BASAL INSULIN + | | -0.4405 | 0.1980 | | | | |
| PREAD<br>BASE | BASAL INSULIN + | ) | 0.04833 | 0.1 | L621 | | | |
| | Type 3 Tests of Fi | xed Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value Pr | > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 449<br>1 449<br>1 449 | 0.56 0.4 | 0160<br>4557<br>0003 | | | | | |
| | | Least So | quares Mea | ans Estimates | | | | |
| | | | | Standard | | | | |
| Effect | Label | Margins | Estimate | Error | DF t | : Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 6.3857<br>6.8022 | 0.09936<br>0.1406 | 449<br>449 | 64.27<br>48.39 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least Squa | ares Means | s Estimates | | | | |
| Effect | Label | Lower | Upper E | Exponentiated | | ntiated<br>Lower | Exponentia<br>Up | ted<br>per |
| trtpn<br>trtpn | LSMeans, IDegLira | | 6.5809<br>7.0784 | 593.28<br>899.79 | | 488.05<br>682.61 | 721<br>1186 | |
| | | T | | - Batimat | | | | |
| | | Least Sqi | uares Mean | ns Estimate | | | | |
| Effect | Label | | Margins | s Estim | | ndard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -0.4165 0.1722 449 -2.42

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 154 of 334 | |

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=C105585P

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.0160 0.05 -0.7550 -0.07803 0.6594

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.4700 0.9249

# NN9068 NN9068-4166 Clinical Trial Report Statistical document CONFIDENTIAL Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=FPGU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 967.38

Fit Statistics

-2 Res Log Likelihood 4390.3
AIC (Smaller is Better) 4392.3
AICC (Smaller is Better) 4392.3
BIC (Smaller is Better) 4396.4

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 105.13 5.7880 449 18.16 Intercept -7.5052 1 -2.42 3.1034 449 trtpn 0 trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -2.1852 -0.75 PREAD 0.1052 BASE 0.02893 449 3.64

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 156 of 334 | |

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=FPGU

The Mixed Procedure

### Solution for Fixed Effects

| Solution for Fixed Effects | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | Planned<br>Treatment<br>for | | | | |
| Effect | Pre Tr | ial anti-D | iabetic treat | ment | Period<br>01 (N) | Pr > t | alp Alp | ha | |
| Intercept | | | | | 1<br>2 | <.000<br>0.016 | | 05<br>05 | |
| trtpn<br>PREAD<br>PREAD | | INSULIN + I | METFORMIN<br>METFORMIN + C | NE OTHER ON | | 0.455 | 0. | 05 | |
| BASE | DASAL . | INSOLIN | ABIFORMIN I C | ONE OTHER OA | ND | 0.000 | 0. | 05 | |
| | | | Solution fo | or Fixed Eff | ects | | | | |
| Effort | Dro Tr | ial anti-D | iabetic treat | rmont | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lovo | | 222 | |
| | | iai anti-D. | iabetic treat | lileirc | OI (N) | Lowe<br>93.751 | | pper<br>6.50 | |
| Intercept trtpn trtpn | , i | | | | 1 2 | -13.604 | | 4062 | |
| PREAD<br>PREAD | | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | -7.937 | 78 3. | 3.5675 | |
| BASE | DAGAE . | INSOLIN | ALII OIGIIN T | NE OTHER OF | LD | 0.0483 | 33 0. | 1621 | |
| | Type 3 Te | sts of Fixe | ed Effects | | | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | | 5.85<br>0.56<br>13.22 | 0.0160<br>0.4557<br>0.0003 | | | | | |
| | | | Least | : Squares Me | ans Estimates | | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADATA2 | | | 449<br>449 | 64.27<br>48.39 | <.0001<br><.0001 | 0.05 |
| - | | 3 | Least S | Squares Mean | s Estimates | | | | |
| Effect | Label | | Lower | Upper | Exponentiated | | nentiated<br>Lower | Exponentia<br>Up | ited<br>oper |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | 111.55<br>117.60 | 118.59<br>127.55 | 9.423E49<br>1.713E53 | | 2.793E48<br>1.18E51 | 3.179<br>2.486 | |
| | | | Least | Squares Mea | ıns Estimate | | | | |
| Effect | Label | | | Margin | s Estim | | andard<br>Error | DF t Va | ılue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -7.5052 3.1034 449 -2.42

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 157 of 334 | |

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=FPGU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.0160 0.05 -13.6042 -1.4062 0.000550

Least Squares Means Estimate

Effect Label Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 1.235E-6 0.2451


Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=C105585P

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 2.9791

Fit Statistics

-2 Res Log Likelihood 1788.0 AIC (Smaller is Better) 1790.0 AICC (Smaller is Better) 1790.0 BIC (Smaller is Better) 1794.1

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 5.8339 449 0.3212 18.16 Intercept -0.4165 0.1722 1 -2.42 449 trtpn 0 trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.1213 0.1624 449 -0.75 PREAD -0.8948 BASE 0.02893 449 -30.93

#### NN9068 Date: 22 January 2020 | Novo Nordisk NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 159 of 334 Statistical document Page:

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=C105585P

The Mixed Procedure

| Solution for Fixed Effects | | | | | | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-D | labetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn | | | | | 1 2 | <.0001<br>0.0160 | 0.05<br>0.05 |
| trtpn<br>PREAD | BASAL INSULIN + METFORMIN | | | | Ζ | 0.4557 | 0.05 |
| PREAD<br>BASE | BASAL INS | JLIN + 1 | 4ETFORMIN + | ONE OTHER OAD | | <.0001 | 0.05 |
| | | | Solution | for Fixed Effe | cts | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | labetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | 5.2026<br>-0.7550 | 6.4651<br>-0.07803 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | 2 | -0.4405 | 0.1980 |
| BASE | DAGAE INS | ADIN 1 I | IBIT ORTIN | ONE OTHER OAD | | -0.9517 | -0.8379 |
| Ту | rpe 3 Tests | of Fixe | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 449<br>449<br>449 | 5.85<br>0.56<br>956.44 | 0.0160<br>0.4557<br><.0001 | | | |

### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.09936<br>0.1406 | 449<br>449 | -33.88<br>-20.98 | <.0001<br><.0001 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | | -3.5615<br>-3.2260 | -3.1709<br>-2.6735 | | | |

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=FPGU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 967.38

Fit Statistics

-2 Res Log Likelihood 4390.3
AIC (Smaller is Better) 4392.3
AICC (Smaller is Better) 4392.3
BIC (Smaller is Better) 4396.4

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 105.13 5.7880 449 18.16 Intercept -7.5052 -2.42 3.1034 449 trtpn 0 trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -2.1852 449 -0.75 PREAD -0.8948 BASE 0.02893 449 -30.93


Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=FPGU

The Mixed Procedure

#### Solution for Fixed Effects

| Solution for Fixed Effects | | | | | | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn | | | | | 1 2 | <.0001<br>0.0160 | 0.05<br>0.05 |
| trtpn<br>PREAD | BASAL INS | | | | ۷ | 0.4557 | 0.05 |
| PREAD<br>BASE | BASAL INS | JLIN + I | METFORMIN + | ONE OTHER OAD | | <.0001 | 0.05 |
| | | | Solution | for Fixed Effe | cts | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | labetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | 93.7515<br>-13.6042 | 116.50<br>-1.4062 |
| PREAD<br>PREAD | BASAL INS | | | ONE OTHER OAD | _ | -7.9378 | 3.5675 |
| BASE | DASAL INS | JLIN T I | TEIFORMIN T | ONE OTHER OAD | | -0.9517 | -0.8379 |
| Ту | pe 3 Tests | of Fixe | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 449<br>449<br>449 | 5.85<br>0.56<br>956.44 | 0.0160<br>0.4557<br><.0001 | | | |

# Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 1.7904<br>2.5330 | 449<br>449 | -33.88<br>-20.98 | <.0001<br><.0001 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | | 54.1776<br>58.1318 | -57.1403<br>-48.1758 | | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 162 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure

Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method

WORK.ANA\_DATA
AVAL
Compound Symmetry
USUBJID
REML
REML
Profile
Kenward-Roger
Kenward-Roger

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 163 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure

Class Level Information

| Class | Levels | Values |
|---------|--------|--------|
| USUBJID | 453 | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 164 of 334 | |

Parameter Code=C105585Y



| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 165 of 334 | |

Parameter Code=C105585Y



| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 166 of 334 | |

Parameter Code=C105585Y



| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 167 of 334 | |

Parameter Code=C105585Y



| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 168 of 334 | |

Parameter Code=C105585Y



| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 169 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure



TRTPN 2 1 2 3 4 5 6 7 8 9
PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

# Dimensions

| Covarian | ce | Parameters | 2 |
|----------|----|------------|----|
| Columns | in | X | 39 |
| Columns | in | Z | 0 |


9-point self-measured plasma glucose profile after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C105585Y

The Mixed Procedure

Dimensions

Subjects 453 Max Obs per Subject 9

Number of Observations

Number of Observations Read 4077 Number of Observations Used 3987 Number of Observations Not Used 90

Iteration History

 Iteration
 Evaluations
 -2 Res Log Like
 Criterion

 0
 1
 17980.86879431
 0.00000000

 1
 2
 16986.47007207
 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate | Standard<br>Error | Z<br>Value | Pr Z | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| CS | USUBJID | 1.9446 | 0.1557 | 12.49 | <.0001 | 0.05 | 1.6394 | 2.2499 |
| Residual | | 3.3601 | 0.08020 | 41.90 | <.0001 | 0.05 | 3.2083 | 3.5230 |

Asymptotic Covariance Matrix of Estimates

Row Cov Parm CovP1 CovP2

1 CS 0.02425 -0.00074
2 Residual -0.00074 0.006432

Fit Statistics

-2 Res Log Likelihood 16986.5 AIC (Smaller is Better) 16990.5 AICC (Smaller is Better) 16990.5 BIC (Smaller is Better) 16998.7

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1 994.40 <.0001

Solution for Fixed Effects

Planned Treatment Analysis for Period Standard Timepoint Effect Pre Trial anti-Diabetic treatment Estimate 01 (N) (N) Error 0.2158 5.9802 Intercept TRTPN -0.3993 0.2304 TRTPN 2 0

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 171 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Tr | rial ant: | i.— I | Diabetic tr | cea | atmer | nt | | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Estimate | Standard<br>Error |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | | | | | | | | | 1 | 1 | 0.03903 | 0.1878 |
| TRTPN (ATPTN) | | | | | | | | | 2 | 1 | 0.1496 | 0.2428 |
| TRTPN (ATPTN) | | | | | | | | | 1 | 2 | 3.9868 | 0.1890 |
| TRTPN (ATPTN) | | | | | | | | | 2 | 2 | 4.8504 | 0.2441 |
| TRTPN (ATPTN) | | | | | | | | | 1 | 3 | 1.2229 | 0.1887 |
| TRTPN (ATPTN) | | | | | | | | | 2 | 3 | 2.1036 | 0.2445 |
| TRTPN (ATPTN) | | | | | | | | | 1 | 4 | 4.0424 | 0.1883 |
| TRTPN (ATPTN) | | | | | | | | | 2 | 4 | 5.1013 | 0.2434 |
| TRTPN (ATPTN) | | | | | | | | | 1 | 5 | 1.8419 | 0.1886 |
| TRTPN (ATPTN) | | | | | | | | | 2 | 5 | 2.1763 | 0.2442 |
| TRTPN (ATPTN) | | | | | | | | | 1 | 6 | 4.4428 | 0.1885 |
| TRTPN (ATPTN) | | | | | | | | | 2 | 6 | 5.0832 | 0.2451 |
| TRTPN (ATPTN) | | | | | | | | | 1 | 7 | 3.0157 | 0.1906 |
| TRTPN (ATPTN) | | | | | | | | | 2 | 7 | 3.6866 | 0.2462 |
| TRTPN (ATPTN) | | | | | | | | | 1 | 8 | 0.4344 | 0.1905 |
| TRTPN (ATPTN) | | | | | | | | | 2 | 8 | 0.7451 | 0.2450 |
| TRTPN (ATPTN) | | | | | | | | | 1 | 9 | 0 | |
| TRTPN (ATPTN) | | | | | | | | | 2 | 9 | 0 | |
| PREAD (ATPTN) | BASAL | INSULIN | + | METFORMIN | | | | | | 1 | -0.1512 | 0.2168 |
| PREAD (ATPTN) | BASAL | INSULIN | + | METFORMIN | + | ONE | OTHER | OAD | | 1 | 0 | |
| PREAD (ATPTN) | BASAL | INSULIN | + | METFORMIN | | | | | | 2 | -0.03748 | 0.2188 |
| PREAD (ATPTN) | BASAL | INSULIN | + | METFORMIN | + | ONE | OTHER | OAD | | 2 | 0 | |
| ( , | | | | METFORMIN | | | | | | 3 | 0.3374 | 0.2187 |
| PREAD (ATPTN) | | | | METFORMIN | + | ONE | OTHER | OAD | | 3 | 0 | |
| PREAD (ATPTN) | | | | | | | | | | 4 | 0.2126 | 0.2180 |
| , | | | | METFORMIN | + | ONE | OTHER | OAD | | 4 | 0 | |
| | | | | METFORMIN | | | | | | 5 | -0.1693 | 0.2183 |
| PREAD (ATPTN) | | | | METFORMIN | + | ONE | OTHER | OAD | | 5 | 0 | |
| , | | | | METFORMIN | | | | | | 6 | -0.09171 | 0.2191 |
| , | | | | METFORMIN | + | ONE | OTHER | OAD | | 6 | 0 | |
| PREAD (ATPTN) | | | | METFORMIN | | 0115 | 0.000 | 07.5 | | 7 | 0.05532 | 0.2205 |
| PREAD (ATPTN) | | | | METFORMIN | + | ONE | OTHER | OAD | | 7 | 0 | 0 0001 |
| , | | | | METFORMIN | | 0115 | 0.000 | 07.5 | | 8 | -0.05872 | 0.2204 |
| | | | | METFORMIN | + | ONE | OTHER | OAD | | | 0 | 0 0170 |
| PREAD (ATPTN) | | | | METFORMIN | | ONTE | OMILED | 07.0 | | 9 | -0.02011 | 0.2172 |
| PREAD (ATPTN) | BASAL | INSOTIN | + | METFORMIN | + | ONE | OTHER | UAD | | 9 | 0 | |

| Pre Trial anti-Diabetic treatment | Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | DF | t Value |
|---|---|---|---|---|
| | | | 1934 | 27.71 |
| | 1 | | 1940 | -1.73 |
| | 2 | | | |
| | 1 | 1 | 3512 | 0.21 |
| | 2 | 1 | 3513 | 0.62 |
| | 1 | | 3516 | 21.09 |
| | 2 | | 3514 | 19.87 |
| | 1 | | | 6.48 |
| | 2 | | | 8.60 |
| | 1 | | | 21.47 |
| | 2 | | | 20.96 |
| | 1 | | | 9.77 |
| | 2 | | | 8.91 |
| | 1 | 6 | 3515 | 23.57 |
| | Pre Trial anti-Diabetic treatment | Pre Trial anti-Diabetic treatment 1 2 1 | Treatment for Analysis Period Timepoint (N) 1 2 1 1 1 1 1 1 2 1 1 1 2 2 1 1 1 2 2 2 2 2 2 2 2 1 3 3 1 4 4 4 4 1 5 5 | Treatment for Analysis Period Timepoint 01 (N) |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 172 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure

| Pre Trial anti-Diabetic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | DF t Value |
|---|---|---|---|
| | 2<br>1<br>2<br>1<br>2 | 6<br>7<br>7<br>8<br>8 | 3516 20.74<br>3518 15.82<br>3517 14.98<br>3518 2.28<br>3516 3.04 |
| BASAL INSULIN + METFORMIN | 2 | 1 | 1927 -0.70 |
| BASAL INSULIN + METFORMIN | | 2 | 1970 -0.17 |
| BASAL INSULIN + METFORMIN | | 3 | 1965 1.54 |
| BASAL INSULIN + METFORMIN | | 4 | 1949 0.98 |
| BASAL INSULIN + METFORMIN | | 5 | 1956 -0.78 |
| BASAL INSULIN + METFORMIN | | 6 | 1975 -0.42 |
| BASAL INSULIN + METFORMIN | | 7 | 2009 0.25 |
| BASAL INSULIN + METFORMIN | | 8 | 2006 -0.27 |
| BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 9 | 1934 -0.09 |
| Solution for Fixed Effects | 5 | | |
| Pre Trial anti-Diabetic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Pr > t |
| | | | <.0001 |
| BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD | 1<br>2<br>1<br>2 | 1<br>1<br>2<br>2<br>3<br>3<br>4<br>4<br>5<br>5<br>6<br>6<br>7<br>7<br>8<br>8<br>9<br>9<br>1<br>1<br>2<br>2<br>2 | 0.0833<br>0.8354<br>0.5380<br><.0001<br><.00027<br>0.0024 |
| | BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD BASAL INSULIN + METFORMIN + ONE OTHER OAD BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD SOLUTION FOR FIXED EFFECTS Pre Trial anti-Diabetic treatment BASAL INSULIN + METFORMIN + ONE OTHER OAD SOLUTION FOR FIXED EFFECTS BASAL INSULIN + METFORMIN + ONE OTHER OAD | Pre Trial anti-Diabetic treatment Pre Trial anti-Diabetic treatment | Pre Trial anti-Diabetic treatment |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 173 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure

#### Solution for Fixed Effects

| | | Planned<br>Treatment<br>for<br>Period | Analysis<br>Timepoint | |
|---|---|---|---|---|
| Effect | Pre Trial anti-Diabetic treatment | 01 (N) | (N) | Pr > t |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 3 | 0.1230 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 3 | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 4 | 0.3295 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 4 | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 5 | 0.4381 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 5 | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 6 | 0.6755 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 6 | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 7 | 0.8020 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 7 | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 8 | 0.7900 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 8 | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 9 | 0.9262 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 9 | |

Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------------|-----------|-----------|---------|--------|
| TRTPN | 1 | 451 | 38.01 | <.0001 |
| TRTPN (ATPTN) | 8 | 3517 | 3.99 | 0.0001 |
| PREAD (ATPTN) | 9 | 3357 | 0.83 | 0.5889 |

# Least Squares Means

| | Planned<br>Treatment<br>for<br>Period | Analysis<br>Timepoint | | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | 01 (N) | (N) | Margins | Estimate | Error | DF | t Value | Pr > t |
| TRTPN (ATPTN) | 1 | 1 | WORK.ANA DATA | 5.5482 | 0.1325 | 1927 | 41.86 | <.0001 |
| TRTPN (ATPTN) | 2 | 1 | WORK.ANA DATA | 6.0580 | 0.1875 | 1927 | 32.32 | <.0001 |
| TRTPN (ATPTN) | 1 | 2 | WORK.ANA DATA | 9.5499 | 0.1332 | 1950 | 71.70 | <.0001 |
| TRTPN (ATPTN) | 2 | 2 | WORK.ANA DATA | 10.8128 | 0.1909 | 2006 | 56.65 | <.0001 |
| TRTPN (ATPTN) | 1 | 3 | WORK.ANA DATA | 6.9640 | 0.1330 | 1943 | 52.34 | <.0001 |
| TRTPN (ATPTN) | 2 | 3 | WORK.ANA DATA | 8.2440 | 0.1909 | 2006 | 43.20 | <.0001 |
| TRTPN (ATPTN) | 1 | 4 | WORK.ANA DATA | 9.7242 | 0.1331 | 1944 | 73.08 | <.0001 |

#### Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Alpha | Lower | Upper |
|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | 0.05 | 5.2882 | 5.8081 |
| TRTPN (ATPTN) | 2 | 1 | 0.05 | 5.6903 | 6.4256 |
| TRTPN (ATPTN) | 1 | 2 | 0.05 | 9.2887 | 9.8111 |
| TRTPN (ATPTN) | 2 | 2 | 0.05 | 10.4385 | 11.1871 |
| TRTPN (ATPTN) | 1 | 3 | 0.05 | 6.7030 | 7.2249 |
| TRTPN (ATPTN) | 2 | 3 | 0.05 | 7.8697 | 8.6182 |
| TRTPN (ATPTN) | 1 | 4 | 0.05 | 9.4632 | 9.9851 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 174 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure

#### Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 2 | 4 | WORK.ANA DATA | 11.1823 | 0.1890 | 1957 | 59.18 | <.0001 |
| TRTPN (ATPTN) | 1 | 5 | WORK.ANA DATA | 7.3424 | 0.1330 | 1943 | 55.19 | <.0001 |
| TRTPN (ATPTN) | 2 | 5 | WORK.ANA DATA | 8.0761 | 0.1899 | 1981 | 42.52 | <.0001 |
| TRTPN (ATPTN) | 1 | 6 | WORK.ANA DATA | 9.9802 | 0.1332 | 1950 | 74.92 | <.0001 |
| TRTPN (ATPTN) | 2 | 6 | WORK.ANA DATA | 11.0199 | 0.1913 | 2018 | 57.60 | <.0001 |
| TRTPN (ATPTN) | 1 | 7 | WORK.ANA DATA | 8.6229 | 0.1343 | 1992 | 64.20 | <.0001 |
| TRTPN (ATPTN) | 2 | 7 | WORK.ANA_DATA | 9.6930 | 0.1923 | 2044 | 50.41 | <.0001 |
| TRTPN (ATPTN) | 1 | 8 | WORK.ANA DATA | 5.9875 | 0.1345 | 1998 | 44.52 | <.0001 |
| TRTPN (ATPTN) | 2 | 8 | WORK.ANA_DATA | 6.6974 | 0.1914 | 2018 | 35.00 | <.0001 |
| TRTPN (ATPTN) | 1 | 9 | WORK.ANA_DATA | 5.5714 | 0.1325 | 1927 | 42.03 | <.0001 |
| TRTPN (ATPTN) | 2 | 9 | WORK.ANA_DATA | 5.9706 | 0.1884 | 1947 | 31.69 | <.0001 |

#### Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Alpha | Lower | Upper |
|---|---|---|---|---|---|
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 2<br>1<br>2<br>1 | 4<br>5<br>5<br>6 | 0.05<br>0.05<br>0.05<br>0.05 | 10.8118<br>7.0815<br>7.7036<br>9.7190 | 11.5529<br>7.6034<br>8.4486<br>10.2415 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 6<br>7 | 0.05 | 10.6446 | 11.3951 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2<br>1 | 7 | 0.05 | 9.3159<br>5.7237 | 10.0701 6.2512 |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 2<br>1<br>2 | 8<br>9<br>9 | 0.05<br>0.05<br>0.05 | 6.3221<br>5.3114<br>5.6011 | 7.0727<br>5.8313<br>6.3402 |

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | 2 | 1 | WORK.ANA DATA | -0.5098 | 0.2296 | 1927 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 2 | WORK.ANA DATA | -4.0018 | 0.1498 | 3513 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 2 | WORK.ANA DATA | -5.2646 | 0.2324 | 1979 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 3 | WORK.ANA DATA | -1.4158 | 0.1496 | 3514 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 3 | WORK.ANA_DATA | -2.6958 | 0.2324 | 1979 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 4 | WORK.ANA DATA | -4.1760 | 0.1496 | 3514 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 4 | WORK.ANA_DATA | -5.6342 | 0.2308 | 1947 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 5 | WORK.ANA_DATA | -1.7943 | 0.1496 | 3514 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 5 | WORK.ANA_DATA | -2.5279 | 0.2316 | 1963 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 6 | WORK.ANA_DATA | -4.4321 | 0.1498 | 3514 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 6 | WORK.ANA_DATA | -5.4717 | 0.2328 | 1988 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 7 | WORK.ANA_DATA | -3.0747 | 0.1508 | 3516 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 7 | WORK.ANA_DATA | -4.1448 | 0.2336 | 2005 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 8 | WORK.ANA_DATA | -0.4393 | 0.1509 | 3516 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 8 | WORK.ANA_DATA | -1.1492 | 0.2328 | 1988 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 9 | WORK.ANA_DATA | -0.02320 | 0.1492 | 3511 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 9 | WORK.ANA_DATA | -0.4225 | 0.2304 | 1940 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 2 | WORK.ANA_DATA | -3.4920 | 0.2300 | 1934 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 175 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 2 | 1 | 2 | 2 | WORK.ANA DATA | -4.7548 | 0.2140 | 3526 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 3 | WORK.ANA DATA | -0.9060 | 0.2299 | 1932 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 3 | WORK.ANA DATA | -2.1860 | 0.2140 | 3526 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 4 | WORK.ANA DATA | -3.6662 | 0.2299 | 1932 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 4 | WORK.ANA DATA | -5.1244 | 0.2123 | 3522 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 5 | WORK.ANA DATA | -1.2845 | 0.2299 | 1932 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 5 | WORK.ANA DATA | -2.0181 | 0.2132 | 3525 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 6 | WORK.ANA DATA | -3.9223 | 0.2300 | 1934 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 6 | WORK.ANA_DATA | -4.9619 | 0.2144 | 3527 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 7 | WORK.ANA_DATA | -2.5649 | 0.2306 | 1948 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 7 | WORK.ANA_DATA | -3.6350 | 0.2153 | 3528 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 8 | WORK.ANA_DATA | 0.07050 | 0.2307 | 1950 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 8 | WORK.ANA_DATA | -0.6394 | 0.2145 | 3527 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 9 | WORK.ANA_DATA | 0.4866 | 0.2296 | 1926 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 9 | WORK.ANA_DATA | 0.08734 | 0.2119 | 3517 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 2 | WORK.ANA_DATA | -1.2629 | 0.2327 | 1987 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 3 | WORK.ANA_DATA | 2.5860 | 0.1501 | 3513 |
| TRTPN (ATPTN) | 1 | 2 2 | 2 | 3 | WORK.ANA_DATA | 1.3060 | 0.2327 | 1987 |
| TRTPN (ATPTN) | 1 | 2 | 1 2 | 4 | WORK.ANA_DATA | -0.1742 | 0.1501<br>0.2312 | 3513<br>1954 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 2 | 1 | 5 | WORK.ANA_DATA<br>WORK.ANA DATA | -1.6324<br>2.2075 | 0.2312 | 3513 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 5 | WORK.ANA DATA | 1.4738 | 0.2320 | 1970 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 6 | WORK.ANA DATA | -0.4303 | 0.1503 | 3513 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 6 | WORK.ANA DATA | -1.4699 | 0.2331 | 1995 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 7 | WORK.ANA DATA | 0.9271 | 0.1513 | 3515 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 7 | WORK.ANA DATA | -0.1431 | 0.2339 | 2013 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 8 | WORK.ANA DATA | 3.5625 | 0.1514 | 3515 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 8 | WORK.ANA DATA | 2.8525 | 0.2331 | 1995 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 9 | WORK.ANA DATA | 3.9786 | 0.1498 | 3513 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 9 | WORK.ANA DATA | 3.5793 | 0.2308 | 1947 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 3 | WORK.ANA DATA | 3.8488 | 0.2327 | 1985 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 3 | WORK.ANA DATA | 2.5689 | 0.2163 | 3516 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 4 | WORK.ANA_DATA | 1.0886 | 0.2327 | 1985 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 4 | WORK.ANA_DATA | -0.3695 | 0.2148 | 3515 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 5 | WORK.ANA_DATA | 3.4704 | 0.2327 | 1985 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 5 | WORK.ANA_DATA | 2.7367 | 0.2156 | 3516 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 6 | WORK.ANA_DATA | 0.8326 | 0.2328 | 1987 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 6 | WORK.ANA_DATA | -0.2071 | 0.2166 | 3514 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 7 | WORK.ANA_DATA | 2.1900 | 0.2334 | 2001 |
| TRTPN (ATPTN) | 2 | 2 2 | 2 | 7<br>8 | WORK.ANA_DATA | 1.1198 | 0.2175 | 3515 |
| TRTPN (ATPTN) | 2 | 2 | 1 2 | 8 | WORK.ANA_DATA<br>WORK.ANA DATA | 4.8253<br>4.1154 | 0.2335<br>0.2167 | 2003<br>3516 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 2 | 1 | 9 | WORK.ANA DATA | 5.2414 | 0.2324 | 1979 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 9 | WORK.ANA DATA | 4.8422 | 0.2146 | 3520 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 3 | WORK.ANA DATA | -1.2800 | 0.2327 | 1985 |
| TRTPN (ATPTN) | i | 3 | 1 | 4 | WORK.ANA DATA | -2.7602 | 0.1500 | 3511 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 4 | WORK.ANA DATA | -4.2184 | 0.2311 | 1952 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 5 | WORK.ANA DATA | -0.3785 | 0.1500 | 3511 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 5 | WORK.ANA DATA | -1.1121 | 0.2319 | 1968 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 6 | WORK.ANA DATA | -3.0163 | 0.1501 | 3512 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 6 | WORK.ANA DATA | -4.0559 | 0.2330 | 1993 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 7 | WORK.ANA DATA | -1.6589 | 0.1511 | 3513 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 7 | WORK.ANA_DATA | -2.7290 | 0.2338 | 2011 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 8 | WORK.ANA_DATA | 0.9765 | 0.1512 | 3514 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 8 | WORK.ANA_DATA | 0.2666 | 0.2331 | 1993 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 9 | WORK.ANA_DATA | 1.3926 | 0.1496 | 3514 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 9 | WORK.ANA_DATA | 0.9933 | 0.2307 | 1945 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 4 | WORK.ANA_DATA | -1.4802 | 0.2327 | 1985 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 4 | WORK.ANA_DATA | -2.9384 | 0.2149 | 3518 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 176 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure

| | | DILL | erences or | neast squar | es means | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
| TRTPN (ATPTN) | 2 | 3 | 1 | 5 | WORK, ANA DATA | 0.9015 | 0.2327 | 1985 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 5 | WORK.ANA DATA | 0.1679 | 0.2154 | 3512 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 6 | WORK.ANA DATA | -1.7363 | 0.2328 | 1987 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 6 | WORK.ANA DATA | -2.7759 | 0.2167 | 3516 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 7 | WORK.ANA DATA | -0.3789 | 0.2334 | 2001 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 7 | WORK.ANA DATA | -1.4490 | 0.2176 | 3518 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 8 | WORK.ANA DATA | 2.2565 | 0.2335 | 2003 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 8 | WORK.ANA DATA | 1.5466 | 0.2166 | 3513 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 9 | WORK.ANA DATA | 2.6726 | 0.2324 | 1979 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 9 | WORK.ANA DATA | 2.2733 | 0.2146 | 3520 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 4 | WORK.ANA DATA | -1.4582 | 0.2311 | 1952 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 5 | WORK.ANA DATA | 2.3817 | 0.1500 | 3511 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 5 | WORK.ANA_DATA | 1.6481 | 0.2319 | 1968 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 6 | WORK.ANA_DATA | -0.2561 | 0.1501 | 3511 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 6 | WORK.ANA_DATA | -1.2957 | 0.2331 | 1993 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 7 | WORK.ANA_DATA | 1.1013 | 0.1511 | 3514 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 7 | WORK.ANA_DATA | 0.03118 | 0.2338 | 2011 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 8 | WORK.ANA_DATA | 3.7367 | 0.1512 | 3514 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 8 | WORK.ANA_DATA | 3.0268 | 0.2331 | 1993 |
| TRTPN (ATPTN) | 1 | 4 | 1 2 | 9 | WORK.ANA_DATA | 4.1528 | 0.1496 | 3514 |
| TRTPN (ATPTN) | 1 2 | 4 | 1 | 5 | WORK.ANA_DATA<br>WORK.ANA DATA | 3.7535<br>3.8399 | 0.2307<br>0.2311 | 1945<br>1952 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 4 | 2 | 5 | _ | 3.1062 | 0.2141 | 3517 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 6 | WORK.ANA_DATA<br>WORK.ANA DATA | 1.2021 | 0.2312 | 1954 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 6 | WORK.ANA DATA | 0.1625 | 0.2152 | 3516 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 7 | WORK.ANA DATA | 2.5595 | 0.2318 | 1968 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 7 | WORK.ANA DATA | 1.4894 | 0.2160 | 3517 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 8 | WORK.ANA DATA | 5.1949 | 0.2319 | 1970 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 8 | WORK.ANA DATA | 4.4850 | 0.2152 | 3516 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 9 | WORK.ANA DATA | 5.6110 | 0.2308 | 1947 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 9 | WORK.ANA DATA | 5.2117 | 0.2129 | 3516 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 5 | WORK.ANA DATA | -0.7336 | 0.2319 | 1968 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 6 | WORK.ANA DATA | -2.6378 | 0.1501 | 3512 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 6 | WORK.ANA_DATA | -3.6774 | 0.2330 | 1993 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 7 | WORK.ANA_DATA | -1.2804 | 0.1511 | 3513 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 7 | WORK.ANA_DATA | -2.3505 | 0.2338 | 2011 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 8 | WORK.ANA_DATA | 1.3550 | 0.1512 | 3513 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 8 | WORK.ANA_DATA | 0.6451 | 0.2331 | 1993 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 9 | WORK.ANA_DATA | 1.7711 | 0.1496 | 3514 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 9 | WORK.ANA_DATA | 1.3718 | 0.2307 | 1945<br>1970 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 5<br>5 | 2 | 6<br>6 | WORK.ANA_DATA<br>WORK.ANA DATA | -1.9041<br>-2.9438 | 0.2320<br>0.2159 | 3515 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 7 | WORK.ANA DATA | -0.5468 | 0.2326 | 1984 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 7 | WORK.ANA DATA | -1.6169 | 0.2168 | 3516 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 8 | WORK.ANA DATA | 2.0886 | 0.2327 | 1986 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 8 | WORK.ANA DATA | 1.3787 | 0.2158 | 3513 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 9 | WORK.ANA DATA | 2.5047 | 0.2316 | 1963 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 9 | WORK.ANA DATA | 2.1055 | 0.2138 | 3519 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 6 | WORK.ANA DATA | -1.0396 | 0.2331 | 1995 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 7 | WORK.ANA DATA | 1.3574 | 0.1512 | 3514 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 7 | WORK.ANA DATA | 0.2872 | 0.2339 | 2013 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 8 | WORK.ANA DATA | 3.9928 | 0.1514 | 3514 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 8 | WORK.ANA_DATA | 3.2828 | 0.2332 | 1995 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 9 | WORK.ANA_DATA | 4.4089 | 0.1498 | 3514 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 9 | WORK.ANA_DATA | 4.0096 | 0.2308 | 1947 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 7 | WORK.ANA_DATA | 2.3970 | 0.2338 | 2009 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 7 | WORK.ANA_DATA | 1.3269 | 0.2180 | 3518 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 8 | WORK.ANA_DATA | 5.0324 | 0.2339 | 2011 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 8 | WORK.ANA_DATA | 4.3225 | 0.2170 | 3515 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 177 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure

#### Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 2 | 6 | 1 | 9 | WORK.ANA DATA | 5.4485 | 0.2328 | 1988 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 9 | WORK.ANA DATA | 5.0492 | 0.2150 | 3521 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 7 | WORK.ANA DATA | -1.0701 | 0.2346 | 2026 |
| TRTPN (ATPTN) | 1 | 7 | 1 | 8 | WORK.ANA DATA | 2.6354 | 0.1523 | 3514 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 8 | WORK.ANA DATA | 1.9255 | 0.2338 | 2009 |
| TRTPN (ATPTN) | 1 | 7 | 1 | 9 | WORK.ANA_DATA | 3.0515 | 0.1508 | 3516 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 9 | WORK.ANA DATA | 2.6522 | 0.2314 | 1961 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 8 | WORK.ANA DATA | 3.7055 | 0.2347 | 2029 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 8 | WORK.ANA DATA | 2.9956 | 0.2179 | 3516 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 9 | WORK.ANA_DATA | 4.1216 | 0.2336 | 2005 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 9 | WORK.ANA DATA | 3.7224 | 0.2159 | 3522 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 8 | WORK.ANA DATA | -0.7099 | 0.2339 | 2011 |
| TRTPN (ATPTN) | 1 | 8 | 1 | 9 | WORK.ANA_DATA | 0.4161 | 0.1509 | 3516 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 9 | WORK.ANA DATA | 0.01684 | 0.2315 | 1964 |
| TRTPN (ATPTN) | 2 | 8 | 1 | 9 | WORK.ANA_DATA | 1.1260 | 0.2328 | 1988 |
| TRTPN (ATPTN) | 2 | 8 | 2 | 9 | WORK.ANA_DATA | 0.7268 | 0.2151 | 3522 |
| TRTPN (ATPTN) | 1 | 9 | 2 | 9 | WORK.ANA_DATA | -0.3993 | 0.2304 | 1940 |

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | 1<br>1 | 2<br>1<br>2<br>1 | 1<br>2<br>2<br>3<br>3<br>4<br>4<br>5<br>5<br>6<br>6<br>6<br>7<br>7<br>8<br>8<br>9<br>9<br>2<br>2<br>3<br>3<br>4<br>4<br>4<br>5<br>5<br>6<br>6<br>6<br>6<br>7<br>7<br>8<br>8<br>8<br>8<br>9 | -2.22 -26.72 -22.66 -9.46 -11.60 -27.91 -24.41 -11.99 -10.91 -29.59 -23.51 -20.39 -17.75 -2.91 -4.94 -0.16 -1.83 -15.18 -22.22 -3.94 -10.21 -15.95 -24.13 -5.59 -9.47 -17.05 -23.14 | 0.0265 <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 1 | 2 | 7 | -11.12<br>-16.88 | <.0001<br><.0001 | 0.05<br>0.05 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 8 | 0.31 | 0.7600 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 8 | -2.98 | 0.0029 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 9 | 2.12 | 0.0342 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 9 | 0.41 | 0.6802 | 0.05 |
| ILILIN (AILIN) | ∠ | 1 | ∠ | <b>フ</b> | U.41 | 0.0002 | 0.05 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 178 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure

| | | DITTELEUC | es or heast | squares Me | allo | | |
|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
| TRTPN (ATPTN) | 1<br>1 | 2<br>2 | 2<br>1<br>2<br>1 | 2 3 3 4 4 4 5 5 6 6 6 7 7 8 8 9 9 3 3 4 4 4 5 5 6 6 6 7 | -5.43<br>17.22<br>5.61<br>-1.16<br>-7.06<br>14.70<br>6.35<br>-2.86<br>-6.31<br>6.13<br>-0.61<br>23.53<br>12.24<br>26.57<br>15.51<br>16.54<br>11.87<br>4.68<br>-1.72<br>14.92<br>12.69<br>3.58<br>-0.96 | <.0001 <.0001 <.0001 0.2459 <.0001 0.0042 <.0001 0.5409 <.0001 0.5409 <.0001 0.03392 | 0.05 |
| TRTPN (ATPTN) | 2<br>2<br>2<br>2<br>2<br>2<br>1 | 2<br>3<br>3 | 1<br>2<br>1<br>2<br>1<br>2<br>2<br>1<br>2<br>1<br>2<br>1<br>2<br>1<br>2<br>1<br>2<br>1<br>2<br>1 | 7<br>7<br>8<br>8<br>9<br>9<br>3<br>4<br>4<br>5<br>5<br>6<br>6<br>7<br>7<br>8<br>8 | 9.38<br>5.15<br>20.67<br>18.99<br>22.56<br>22.56<br>-5.50<br>-18.41<br>-18.25<br>-2.52<br>-4.80<br>-20.09<br>-17.40<br>-10.98<br>-11.67<br>6.46<br>1.14 | <.0001 <. | 0.05 |
| TRTPN (ATPTN) | 1<br>1<br>2 | 3<br>4<br>4<br>4<br>4 | 1<br>2<br>1<br>2 | 9<br>9<br>4<br>4<br>5<br>5<br>6<br>6<br>7<br>7<br>8<br>8<br>9<br>9<br>4<br>5<br>5<br>6 | 9.31<br>4.31<br>-6.36<br>-13.67<br>3.87<br>0.78<br>-7.46<br>-12.81<br>-1.62<br>-6.66<br>9.66<br>7.14<br>11.50<br>10.59<br>-6.31<br>15.88<br>7.11<br>-1.71<br>-5.56 | <.0001<br><.0001<br><.0001<br><.0001<br>0.0001<br>0.4358<br><.0001 | 0.05 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 179 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure

| | | DILIELEUC | es or heast | oquares Me | allo | | |
|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
| TRTPN (ATPTN) | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 | 1 2 | 778899556677888995667788899667788899667788899667788899667788899667788899667788899667788899667788899967 | 7.29 0.13 24.71 12.99 27.75 16.27 16.62 14.51 5.20 0.75 11.04 6.89 22.40 20.84 24.31 24.48 -3.16 -17.57 -15.78 -8.48 -10.05 8.96 2.77 11.84 5.95 -8.21 -13.63 -2.35 -7.46 8.97 6.39 10.81 9.85 -4.46 8.98 | <pre></pre> | 0.05 |
| TRTPN (ATPTN) | 1<br>1<br>1<br>1<br>1<br>1<br>2<br>1<br>1<br>1<br>1<br>2<br>1<br>1<br>1<br>1<br>1<br>1<br>1<br>2 | 6<br>7<br>7<br>7<br>7<br>7 | 1<br>2<br>1<br>2 | 7<br>7<br>8<br>8<br>9<br>9<br>7<br>7<br>8<br>8<br>9<br>9<br>7<br>7<br>8<br>8<br>9<br>9<br>9<br>9<br>8<br>8<br>9 | 8.98<br>1.23<br>26.38<br>14.08<br>29.44<br>17.38<br>10.25<br>6.09<br>21.52<br>19.91<br>23.41<br>23.48<br>-4.56<br>17.31<br>8.24<br>20.24<br>11.46<br>15.79<br>13.75<br>17.65<br>17.24<br>-3.04<br>2.76<br>0.07<br>4.84 | <.0001 0.2196 <.0001 | 0.05 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 180 of 334 | |

Parameter Code=C105585Y

The Mixed Procedure

#### Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 2 | 8 | 2 2 | 9 | 3.38 | 0.0007 | 0.05 |
| TRTPN (ATPTN) | 1 | 9 | | 9 | -1.73 | 0.0833 | 0.05 |

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
|---|---|---|---|---|---|---|
| TRTPN (ATPTN) TRTPN (ATPTN) | 1<br>1<br>1 | 1<br>1<br>1 | 2<br>1<br>2 | 1<br>2<br>2 | -0.9601<br>-4.2954<br>-5.7204 | -0.05948<br>-3.7081<br>-4.8089 |
| TRTPN (ATPTN) | | | 1 | 3 | | |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 1 | 2 | 3 | -1.7092<br>-3.1515 | -1.1224<br>-2.2401 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 4 | -4.4694 | -3.8826 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 4 | -6.0869 | -5.1815 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 5 | -2.0876 | -1.5009 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 5 | -2.9821 | -2.0737 |
| TRTPN (ATPTN) | 1 | ī | 1 | 6 | -4.7257 | -4.1384 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 6 | -5.9282 | -5.0152 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 7 | -3.3703 | -2.7791 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 7 | -4.6028 | -3.6868 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 8 | -0.7352 | -0.1434 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 8 | -1.6057 | -0.6927 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 9 | -0.3157 | 0.2693 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 9 | -0.8743 | 0.02937 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 2 | -3.9430 | -3.0410 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 2 | -5.1744 | -4.3352 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 3 | -1.3569 | -0.4552 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 3 | -2.6056<br>-4.1171 | -1.7664<br>-3.2153 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 4 | -5.5407 | -3.2153<br>-4.7081 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 1 | 1 | 5 | -1.7353 | -0.8336 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 5 | -2.4361 | -1.6002 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 6 | -4.3733 | -3.4712 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 6 | -5.3823 | -4.5415 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 7 | -3.0172 | -2.1126 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 7 | -4.0571 | -3.2129 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 8 | -0.3820 | 0.5230 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 8 | -1.0599 | -0.2189 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 9 | 0.03632 | 0.9369 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 9 | -0.3280 | 0.5027 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 2 | -1.7193 | -0.8065 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 3 | 2.2916 | 2.8803 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 3 | 0.8495 | 1.7624 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 4 | -0.4686 | 0.1201 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 4 | -2.0858 | -1.1790 |
| TRTPN (ATPTN) | 1 | 2 | 1 2 | 5<br>5 | 1.9131 | 2.5018 |
| TRTPN (ATPTN) | | 2 | 1 | 6 | 1.0189 | 1.9288<br>-0.1357 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 2 | 2 | 6 | -0.7250<br>-1.9271 | -1.0127 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 7 | 0.6305 | 1.2237 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 7 | -0.6018 | 0.3157 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 8 | 3.2656 | 3.8593 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 8 | 2.3953 | 3.3098 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 9 | 3.6849 | 4.2722 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 9 | 3.1268 | 4.0318 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 181 of 334 | |

Parameter Code=C105585Y

Differences of Least Squares Means

| | | | I Deade byu | arco neano | | |
|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
| TRTPN (ATPTN) | 2<br>2 | 2<br>2 | 1<br>2<br>1<br>2 | 3<br>3<br>4<br>4<br>5<br>5<br>6<br>6<br>7<br>7<br>7<br>8<br>8<br>9 | 3.3925<br>2.1447<br>0.6323<br>-0.7906<br>3.0141<br>2.3140<br>0.3761<br>-0.6318<br>1.7322<br>0.6934<br>4.3674<br>3.6905<br>4.7857 | 4.3051<br>2.9930<br>1.5449<br>0.05156<br>3.9266<br>3.1594<br>1.2890<br>0.2177<br>2.6477<br>1.5462<br>5.2832<br>4.5404<br>5.6972 |
| TRTPN (ATPTN) | 2<br>1<br>1<br>1<br>1<br>1<br>1<br>1 | 2<br>3 | 2<br>2<br>1<br>2<br>1<br>2<br>1<br>2<br>1<br>2 | 9<br>4<br>4<br>5<br>5<br>6<br>6<br>7 | 4.4214<br>-1.7362<br>-3.0542<br>-4.6716<br>-0.6725<br>-1.5669<br>-3.3106<br>-4.5129<br>-1.9551 | 5.2630<br>-0.8237<br>-2.4662<br>-3.7651<br>-0.08446<br>-0.6573<br>-2.7220<br>-3.5989<br>-1.3627 |
| TRTPN (ATPTN) | 1<br>1<br>1<br>1<br>2<br>2<br>2<br>2 | 3<br>3 | 2<br>1<br>2<br>1<br>2<br>1<br>2<br>1<br>2 | 7<br>8<br>9<br>9<br>4<br>4<br>5<br>5 | -3.1876<br>0.6800<br>-0.1905<br>1.0992<br>0.5410<br>-1.9365<br>-3.3597<br>0.4452<br>-0.2544 | -2.2704<br>1.2730<br>0.7237<br>1.6860<br>1.4457<br>-1.0239<br>-2.5170<br>1.3578<br>0.5901 |
| TRTPN (ATPTN) | 2<br>2 | 3<br>4 | 1<br>2<br>1<br>2<br>1<br>2<br>1<br>2<br>2 | 6<br>6<br>7<br>7<br>8<br>8<br>9<br>9 | -2.1927<br>-3.2009<br>-0.8366<br>-1.8756<br>1.7986<br>1.1220<br>2.2169<br>1.8525<br>-1.9114 | -1.2798<br>-2.3510<br>0.07881<br>-1.0224<br>2.7144<br>1.9712<br>3.1283<br>2.6941<br>-1.0049 |
| TRTPN (ATPTN) | 1<br>1<br>1<br>1<br>1<br>1<br>1 | 4<br>4<br>4<br>4<br>4<br>4<br>4<br>4 | 1<br>2<br>1<br>2<br>1<br>2<br>1<br>2 | 5<br>5<br>6<br>6<br>7<br>7<br>8 | 2.0877<br>1.1933<br>-0.5503<br>-1.7527<br>0.8051<br>-0.4274<br>3.4402<br>2.5697 | 2.6757<br>2.1029<br>0.03819<br>-0.8386<br>1.3976<br>0.4898<br>4.0332<br>3.4839 |
| TRTPN (ATPTN) | 1<br>1<br>2 | 4<br>4 | 1<br>2<br>1<br>2<br>1<br>2<br>1<br>2<br>1<br>2<br>1<br>2<br>1<br>2 | 9<br>9<br>5<br>5<br>6<br>6<br>7<br>7<br>8<br>8<br>8<br>9 | 3.8594<br>3.3011<br>3.3866<br>2.6865<br>0.7487<br>-0.2594<br>2.1048<br>1.0658<br>4.7400<br>4.0630<br>5.1583 | 4.4462<br>4.2059<br>4.2931<br>3.5260<br>1.6555<br>0.5844<br>3.0142<br>1.9129<br>5.6497<br>4.9069<br>6.0637 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 182 of 334 | |

Parameter Code=C105585Y

Differences of Least Squares Means

| | Planned<br>Treatment<br>for<br>Period | Analysis<br>Timepoint | Planned<br>Treatment<br>for<br>Period | Analysis<br>Timepoint | | |
|---|---|---|---|---|---|---|
| Effect | 01 (N) | (N) | 01 (N) | (N) | Lower | Upper |
| TRTPN (ATPTN) | 2 | 4 | 2 | 9 | 4.7942 | 5.6292 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 5 | -1.1884 | -0.2789 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 6 | -2.9321 | -2.3435 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 6 | -4.1345 | -3.2204 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 7 | -1.5766 | -0.9842 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 7 | -2.8091 | -1.8920 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 8 | 1.0585 | 1.6514 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 8 | 0.1880 | 1.1021 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 9 | 1.4777 | 2.0645 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 9 | 0.9194 | 1.8242 |
| TRTPN (ATPTN) | 2 | 5<br>5 | 1 2 | 6<br>6 | -2.3591 | -1.4492 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 7 | -3.3671<br>-1.0030 | -2.5205<br>-0.09055 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 5 | 2 | 7 | -2.0419 | -1.1919 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 8 | 1.6322 | 2.5450 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 8 | 0.9556 | 1.8018 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 9 | 2.0505 | 2.9589 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 9 | 1.6863 | 2.5246 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 6 | -1.4969 | -0.5824 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 7 | 1.0609 | 1.6539 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 7 | -0.1715 | 0.7460 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 8 | 3.6960 | 4.2896 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 8 | 2.8256 | 3.7401 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 9 | 4.1152 | 4.7025 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 9 | 3.5570 | 4.4622 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 7 | 1.9385 | 2.8555 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 7 | 0.8995 | 1.7543 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 8 | 4.5737 | 5.4911 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 8 | 3.8969 | 4.7480 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 9 | 4.9920 | 5.9050 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 9 | 4.6276 | 5.4709 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 7 | -1.5301 | -0.6101 |
| TRTPN (ATPTN) | 1 | 7<br>7 | 1 2 | 8 | 2.3368 | 2.9339 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 7 | 1 | 8<br>9 | 1.4670<br>2.7559 | 2.3840<br>3.3471 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 9 | 2.1984 | 3.1061 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 8 | 3.2453 | 4.1657 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 8 | 2.5684 | 3.4228 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 9 | 3.6636 | 4.5796 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 9 | 3.2991 | 4.1457 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 8 | -1.1686 | -0.2512 |
| TRTPN (ATPTN) | 1 | 8 | 1 | 9 | 0.1202 | 0.7120 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 9 | -0.4372 | 0.4709 |
| TRTPN (ATPTN) | 2 | 8 | 1 | 9 | 0.6695 | 1.5825 |
| TRTPN (ATPTN) | 2 | 8 | 2 | 9 | 0.3051 | 1.1484 |
| TRTPN (ATPTN) | 1 | 9 | 2 | 9 | -0.8511 | 0.05258 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 183 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Setimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
WORK.ANA\_DATA
AVAL
Compound Symmetry
USUBJID
REML
REML
Profile
Kenward-Roger
Kenward-Roger

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 184 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

Class Level Information

| | CIASS | Level Informacion |
|---------|--------|-------------------|
| Class | Levels | Values |
| USUBJID | 453 | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 185 of 334 | |

Parameter Code=SMPGCOL



| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 186 of 334 | |

Parameter Code=SMPGCOL



| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 187 of 334 | |

Parameter Code=SMPGCOL



| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 188 of 334 | |

Parameter Code=SMPGCOL



| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 189 of 334 | |

Parameter Code=SMPGCOL



| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 190 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure



TRTPN 2 1 2 3 4 5 6 7 8 9
PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

# Dimensions

| Covarian | ce | Parameters | 2 |
|----------|----|------------|----|
| Columns | in | X | 39 |
| Columns | in | Z | 0 |


9-point self-measured plasma glucose profile after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=SMPGCOL

The Mixed Procedure

Dimensions

Subjects 453 Max Obs per Subject 9

Number of Observations

Number of Observations Read 4077 Number of Observations Used 3987 Number of Observations Not Used 90

Iteration History

 Iteration
 Evaluations
 -2 Res Log Like
 Criterion

 0
 1
 40881.40823158
 0.00000000

 1
 2
 39887.00950934
 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate | Standard<br>Error | Value | Pr Z | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| CS | USUBJID | 631.46 | 50.5711 | 12.49 | <.0001 | 0.05 | 532.34 | 730.57 |
| Residual | | 1091.10 | 26.0426 | 41.90 | <.0001 | 0.05 | 1041.80 | 1143.99 |

Asymptotic Covariance Matrix of Estimates

| Row | Cov Parm | CovP1 | CovP2 |
|-----|----------|----------|----------|
| 1 2 | CS | 2557.44 | -77.8457 |
| | Residual | -77.8457 | 678.22 |

Fit Statistics

-2 Res Log Likelihood 39887.0 AIC (Smaller is Better) 39891.0 AICC (Smaller is Better) 39891.0 BIC (Smaller is Better) 39899.2

Null Model Likelihood Ratio Test

| Effect | Pre Trial anti-Diabetic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Estimate | Standard<br>Error |
|---|---|---|---|---|---|
| Intercept<br>TRTPN | | 1 | | 107.76<br>-7.1946 | 3.8891<br>4.1516 |
| TRTPN | | 2 | | 0 | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 192 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial anti-Diabetic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Estimate | Standard<br>Error |
|---|---|---|---|---|---|
| TRTPN (ATPTN) | | 1<br>2<br>1<br>2<br>1<br>2<br>1<br>2<br>1<br>2 | 1<br>1<br>2<br>2<br>3<br>3<br>4<br>4<br>5<br>5 | 0.7033<br>2.6952<br>71.8421<br>87.4046<br>22.0372<br>37.9077<br>72.8432<br>91.9248<br>33.1905<br>39.2162 | 4.3979<br>3.4006<br>4.4057<br>3.3924<br>4.3856<br>3.3989<br>4.3997 |
| TRTPN (ATPTN) | | 1<br>2<br>1<br>2<br>1<br>2<br>1 | 6<br>7<br>7<br>8<br>8<br>9 | 80.0601<br>91.5997<br>54.3426<br>66.4318<br>7.8283<br>13.4264 | 3.3967<br>4.4173<br>3.4347<br>4.4361<br>3.4334<br>4.4143 |
| PREAD (ATPTN) PREAD (ATPTN) PREAD (ATPTN) PREAD (ATPTN) PREAD (ATPTN) | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OF<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OF<br>BASAL INSULIN + METFORMIN | DAD<br>DAD | 1<br>1<br>2<br>2<br>3 | -2.7250<br>0<br>-0.6754<br>0<br>6.0799 | 3.9060<br>3.9435<br>3.9403 |
| PREAD (ATPTN) PREAD (ATPTN) PREAD (ATPTN) PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER C<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER C<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER C | DAD | 3<br>4<br>4<br>5<br>5 | 3.8311<br>0<br>-3.0503 | 3.9276<br>3.9334 |
| PREAD (ATPTN) PREAD (ATPTN) | BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER C BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER C BASAL INSULIN + METFORMIN | | 6<br>6<br>7<br>7<br>8 | -1.6527<br>0<br>0.9968<br>0<br>-1.0581 | 3.9476<br>3.9739<br>3.9719 |
| | BASAL INSULIN + METFORMIN + ONE OTHER C<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER C | | 8<br>9<br>9 | -0.3624<br>0 | 3.9131 |

| Effect | Pre Trial anti-Diabetic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | DF | t Value |
|---|---|---|---|---|---|
| Intercept | | | | 1934 | 27.71 |
| TRTPN | | 1 | | 1940 | -1.73 |
| TRTPN | | 2 | | | |
| TRTPN (ATPTN) | | 1 | 1 | 3512 | 0.21 |
| TRTPN (ATPTN) | | 2 | 1 | 3513 | 0.62 |
| TRTPN (ATPTN) | | 1 | 2 | 3516 | 21.09 |
| TRTPN (ATPTN) | | 2 | 2 | 3514 | 19.87 |
| TRTPN (ATPTN) | | 1 | 3 | 3515 | 6.48 |
| TRTPN (ATPTN) | | 2 | 3 | 3516 | 8.60 |
| TRTPN (ATPTN) | | 1 | 4 | 3514 | 21.47 |
| TRTPN (ATPTN) | | 2 | 4 | 3513 | 20.96 |
| TRTPN (ATPTN) | | 1 | 5 | 3515 | 9.77 |
| TRTPN (ATPTN) | | 2 | 5 | 3515 | 8.91 |
| TRTPN (ATPTN) | | 1 | 6 | 3515 | 23.57 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 193 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| | Solution for Fixed Effe | cts | | | |
|---|---|---|---|---|---|
| Effect | Pre Trial anti-Diabetic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | DF | t Value |
| | | 2 | 6 | 3516 | 20.74 |
| TRTPN (ATPTN) TRTPN (ATPTN) | | 1 | 7 | 3518 | |
| | | 2 | 7 | 3310 | 14.98 |
| TRTPN (ATPTN) | | 1 | 8 | 3517<br>3518 | 2.28 |
| TRTPN (ATPTN) | | 2 | 8 | 3516 | 3.04 |
| TRTPN (ATPTN) TRTPN (ATPTN) | | 1 | 9 | 3310 | 3.04 |
| TRTPN (ATPTN) | | 2 | 9 | | |
| , , | BASAL INSULIN + METFORMIN | 2 | 1 | 1927 | -0.70 |
| | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 1 | 1321 | -0.70 |
| | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 2 | 1970 | -0.17 |
| | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 2 | 1370 | 0.17 |
| | BASAL INSULIN + METFORMIN | | 3 | 1965 | 1.54 |
| | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 3 | 1000 | 1.04 |
| , , | BASAL INSULIN + METFORMIN | | 4 | 1949 | 0.98 |
| , , | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 4 | 1010 | 0.30 |
| | BASAL INSULIN + METFORMIN | | 5 | 1956 | -0.78 |
| | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 5 | | |
| | BASAL INSULIN + METFORMIN | | 6 | 1975 | -0.42 |
| | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 6 | | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 7 | 2009 | 0.25 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 7 | | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 8 | 2006 | -0.27 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 8 | | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 9 | 1934 | -0.09 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 9 | | |
| | Solution for Fixed Effects | | | | |
| | | Planned | | | |
| | | Treatment | Analysis | | |

| Effect | Pre Trial anti-Diabetic treatment | Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Pr > t |
|---|---|---|---|---|
| Intercept TRTPN TRTPN TRTPN TRTPN (ATPTN) PREAD (ATPTN) PREAD (ATPTN) | BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD BASAL INSULIN + METFORMIN | 1<br>2<br>1<br>2 | 1<br>1<br>2<br>2<br>3<br>3<br>4<br>4<br>4<br>5<br>5<br>6<br>6<br>6<br>7<br>7<br>7<br>8<br>8<br>8<br>9<br>9<br>1<br>1<br>1<br>2<br>1<br>2 | <.0001 0.0833 0.8354 0.5380 <.0001 <.0002 0.0001 <.0001 0.0002 0.0001 0.0227 0.0024 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 2 | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 194 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial anti-Diabetic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Pr > t |
|---|---|---|---|---|
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 3 | 0.1230 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 3 | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 4 | 0.3295 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 4 | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 5 | 0.4381 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 5 | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 6 | 0.6755 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 6 | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 7 | 0.8020 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 7 | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 8 | 0.7900 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 8 | |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN | | 9 | 0.9262 |
| PREAD (ATPTN) | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 9 | |

Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------------|-----------|-----------|---------|--------|
| TRTPN | 1 | 451 | 38.01 | <.0001 |
| TRTPN (ATPTN) | 8 | 3517 | 3.99 | 0.0001 |
| PREAD (ATPTN) | 9 | 3357 | 0.83 | 0.5889 |

# Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | WORK.ANA DATA | 99.9780 | 2.3885 | 1927 | 41.86 | <.0001 |
| TRTPN (ATPTN) | 2 | 1 | WORK.ANA DATA | 109.16 | 3.3781 | 1927 | 32.32 | <.0001 |
| TRTPN (ATPTN) | 1 | 2 | WORK.ANA DATA | 172.09 | 2.4000 | 1950 | 71.70 | <.0001 |
| TRTPN (ATPTN) | 2 | 2 | WORK.ANA DATA | 194.85 | 3.4392 | 2006 | 56.65 | <.0001 |
| TRTPN (ATPTN) | 1 | 3 | WORK.ANA DATA | 125.49 | 2.3975 | 1943 | 52.34 | <.0001 |
| TRTPN (ATPTN) | 2 | 3 | WORK.ANA DATA | 148.56 | 3.4392 | 2006 | 43.20 | <.0001 |
| TRTPN (ATPTN) | 1 | 4 | WORK.ANA_DATA | 175.23 | 2.3976 | 1944 | 73.08 | <.0001 |

#### Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Alpha | Lower | Upper |
|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | 0.05 | 95.2938 | 104.66 |
| TRTPN (ATPTN) | 2 | 1 | 0.05 | 102.54 | 115.79 |
| TRTPN (ATPTN) | 1 | 2 | 0.05 | 167.38 | 176.80 |
| TRTPN (ATPTN) | 2 | 2 | 0.05 | 188.10 | 201.59 |
| TRTPN (ATPTN) | 1 | 3 | 0.05 | 120.79 | 130.19 |
| TRTPN (ATPTN) | 2 | 3 | 0.05 | 141.81 | 155.30 |
| TRTPN (ATPTN) | 1 | 4 | 0.05 | 170.53 | 179.93 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 195 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

#### Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 2 | 4 | WORK.ANA DATA | 201.51 | 3.4051 | 1957 | 59.18 | <.0001 |
| TRTPN (ATPTN) | 1 | 5 | WORK.ANA DATA | 132.31 | 2.3975 | 1943 | 55.19 | <.0001 |
| TRTPN (ATPTN) | 2 | 5 | WORK.ANA DATA | 145.53 | 3.4223 | 1981 | 42.52 | <.0001 |
| TRTPN (ATPTN) | 1 | 6 | WORK.ANA DATA | 179.84 | 2.4005 | 1950 | 74.92 | < .0001 |
| TRTPN (ATPTN) | 2 | 6 | WORK.ANA DATA | 198.58 | 3.4477 | 2018 | 57.60 | <.0001 |
| TRTPN (ATPTN) | 1 | 7 | WORK.ANA DATA | 155.38 | 2.4205 | 1992 | 64.20 | <.0001 |
| TRTPN (ATPTN) | 2 | 7 | WORK.ANA_DATA | 174.67 | 3.4650 | 2044 | 50.41 | <.0001 |
| TRTPN (ATPTN) | 1 | 8 | WORK.ANA DATA | 107.89 | 2.4234 | 1998 | 44.52 | <.0001 |
| TRTPN (ATPTN) | 2 | 8 | WORK.ANA DATA | 120.69 | 3.4481 | 2018 | 35.00 | <.0001 |
| TRTPN (ATPTN) | 1 | 9 | WORK.ANA_DATA | 100.40 | 2.3885 | 1927 | 42.03 | <.0001 |
| TRTPN (ATPTN) | 2 | 9 | WORK.ANA_DATA | 107.59 | 3.3954 | 1947 | 31.69 | <.0001 |

#### Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Alpha | Lower | Upper |
|---|---|---|---|---|---|
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 2<br>1<br>2<br>1<br>2 | 4<br>5<br>5<br>6<br>6 | 0.05<br>0.05<br>0.05<br>0.05<br>0.05 | 194.83<br>127.61<br>138.82<br>175.14<br>191.82 | 208.18<br>137.01<br>152.24<br>184.55<br>205.34 |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 1<br>2<br>1<br>2<br>1<br>2 | 7<br>7<br>8<br>8<br>9<br>9 | 0.05<br>0.05<br>0.05<br>0.05<br>0.05 | 150.64<br>167.87<br>103.14<br>113.92<br>95.7118<br>100.93 | 160.13<br>181.46<br>112.65<br>127.45<br>105.08<br>114.25 |

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | 2 | 1 | WORK.ANA DATA | -9.1865 | 4.1376 | 1927 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 2 | WORK.ANA DATA | -72.1116 | 2.6986 | 3513 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 2 | WORK.ANA DATA | -94.8687 | 4.1874 | 1979 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 3 | WORK.ANA DATA | -25.5128 | 2.6963 | 3514 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 3 | WORK.ANA_DATA | -48.5780 | 4.1874 | 1979 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 4 | WORK.ANA_DATA | -75.2515 | 2.6964 | 3514 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 4 | WORK.ANA_DATA | -101.53 | 4.1594 | 1947 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 5 | WORK.ANA_DATA | -32.3329 | 2.6964 | 3514 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 5 | WORK.ANA_DATA | -45.5531 | 4.1735 | 1963 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 6 | WORK.ANA_DATA | -79.8657 | 2.6990 | 3514 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 6 | WORK.ANA_DATA | -98.6000 | 4.1944 | 1988 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 7 | WORK.ANA_DATA | -55.4058 | 2.7168 | 3516 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 7 | WORK.ANA_DATA | -74.6896 | 4.2086 | 2005 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 8 | WORK.ANA_DATA | -7.9162 | 2.7194 | 3516 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 8 | WORK.ANA_DATA | -20.7089 | 4.1947 | 1988 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 9 | WORK.ANA_DATA | -0.4180 | 2.6883 | 3511 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 9 | WORK.ANA_DATA | -7.6126 | 4.1515 | 1940 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 2 | WORK.ANA_DATA | -62.9251 | 4.1440 | 1934 |
| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 196 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| Differences of Beast Squares Means | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
| TRTPN (ATPTN) | 2 | 1 | 2 | 2 | WORK.ANA DATA | -85.6821 | 3.8566 | 3526 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 3 | WORK.ANA DATA | -16.3263 | 4.1425 | 1932 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 3 | WORK.ANA DATA | -39.3915 | 3.8565 | 3526 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 4 | WORK.ANA DATA | -66.0650 | 4.1426 | 1932 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 4 | WORK.ANA DATA | -92.3412 | 3.8262 | 3522 |
| TRTPN (ATPTN) | 2 | ī | 1 | 5 | WORK.ANA DATA | -23.1463 | 4.1426 | 1932 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 5 | WORK.ANA DATA | -36.3666 | 3.8415 | 3525 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 6 | WORK.ANA DATA | -70.6792 | 4.1443 | 1934 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 6 | WORK.ANA DATA | -89.4134 | 3.8642 | 3527 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 7 | WORK.ANA DATA | -46.2192 | 4.1559 | 1948 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 7 | WORK.ANA DATA | -65.5031 | 3.8796 | 3528 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 8 | WORK.ANA DATA | 1.2704 | 4.1576 | 1950 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 8 | WORK.ANA DATA | -11.5224 | 3.8645 | 3527 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 9 | WORK.ANA DATA | 8.7685 | 4.1373 | 1926 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 9 | WORK.ANA_DATA | 1.5739 | 3.8176 | 3517 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 2 | WORK.ANA_DATA | -22.7570 | 4.1938 | 1987 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 3 | WORK.ANA_DATA | 46.5988 | 2.7054 | 3513 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 3 | WORK.ANA_DATA | 23.5336 | 4.1939 | 1987 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 4 | WORK.ANA_DATA | -3.1399 | 2.7055 | 3513 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 4 | WORK.ANA_DATA | -29.4161 | 4.1660 | 1954 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 5 | WORK.ANA_DATA | 39.7788 | 2.7054 | 3513 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 5 | WORK.ANA_DATA | 26.5585 | 4.1801 | 1970 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 6 | WORK.ANA_DATA | -7.7541 | 2.7081 | 3513 |
| TRTPN (ATPTN) | 1 | 2 2 | 2 | 6<br>7 | WORK.ANA_DATA | -26.4884 | 4.2009 | 1995 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 7 | WORK.ANA_DATA | 16.7059<br>-2.5780 | 2.7258<br>4.2151 | 3515<br>2013 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 2 | 1 | 8 | WORK.ANA_DATA<br>WORK.ANA DATA | 64.1955 | 2.7279 | 3515 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 8 | WORK.ANA DATA | 51.4027 | 4.2012 | 1995 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 9 | WORK.ANA DATA | 71.6936 | 2.6986 | 3513 |
| TRTPN (ATPTN) | 1 | 2 2 | 2 | 9 | WORK.ANA DATA | 64.4990 | 4.1581 | 1947 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 3 | WORK.ANA DATA | 69.3559 | 4.1925 | 1985 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 3 | WORK.ANA DATA | 46.2907 | 3.8985 | 3516 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 4 | WORK.ANA DATA | 19.6172 | 4.1926 | 1985 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 4 | WORK.ANA DATA | -6.6591 | 3.8703 | 3515 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 5 | WORK.ANA DATA | 62.5358 | 4.1925 | 1985 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 5 | WORK.ANA_DATA | 49.3156 | 3.8851 | 3516 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 6 | WORK.ANA_DATA | 15.0029 | 4.1943 | 1987 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 6 | WORK.ANA_DATA | -3.7313 | 3.9037 | 3514 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 7 | WORK.ANA_DATA | 39.4629 | 4.2057 | 2001 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 7 | WORK.ANA_DATA | 20.1791 | 3.9190 | 3515 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 8 | WORK.ANA_DATA | 86.9525 | 4.2074 | 2003 |
| TRTPN (ATPTN) | 2 | 2 2 | 2 | 8 | WORK.ANA_DATA | 74.1598 | 3.9057 | 3516 |
| TRTPN (ATPTN) | 2 | 2 | 1 2 | 9 | WORK.ANA_DATA | 94.4506 | 4.1874 | 1979 |
| TRTPN (ATPTN) | 2 | 2 3 | 2 | 3 | WORK.ANA_DATA | 87.2560 | 3.8675 | 3520<br>1985 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 3 | 1 | 4 | WORK.ANA_DATA<br>WORK.ANA DATA | -23.0652<br>-49.7387 | 4.1924<br>2.7023 | 3511 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 4 | WORK.ANA DATA | -76.0149 | 4.1646 | 1952 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 5 | WORK.ANA DATA | -6.8201 | 2.7022 | 3511 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 5 | WORK.ANA DATA | -20.0403 | 4.1787 | 1968 |
| TRTPN (ATPTN) | ī | 3 | 1 | 6 | WORK.ANA DATA | -54.3530 | 2.7049 | 3512 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 6 | WORK.ANA DATA | -73.0872 | 4.1995 | 1993 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 7 | WORK.ANA DATA | -29.8930 | 2.7221 | 3513 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 7 | WORK.ANA DATA | -49.1768 | 4.2137 | 2011 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 8 | WORK.ANA DATA | 17.5966 | 2.7253 | 3514 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 8 | WORK.ANA DATA | 4.8039 | 4.1998 | 1993 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 9 | WORK.ANA_DATA | 25.0948 | 2.6963 | 3514 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 9 | WORK.ANA_DATA | 17.9001 | 4.1567 | 1945 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 4 | WORK.ANA_DATA | -26.6735 | 4.1926 | 1985 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 4 | WORK.ANA_DATA | -52.9497 | 3.8725 | 3518 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 197 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 2 | 3 | 1 | 5 | WORK.ANA DATA | 16.2451 | 4.1925 | 1985 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 5 | WORK.ANA DATA | 3.0249 | 3.8810 | 3512 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 6 | WORK.ANA_DATA | -31.2878 | 4.1942 | 1987 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 6 | WORK.ANA_DATA | -50.0220 | 3.9056 | 3516 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 7 | WORK.ANA_DATA | -6.8278 | 4.2056 | 2001 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 7 | WORK.ANA_DATA | -26.1116 | 3.9209 | 3518 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 8 | WORK.ANA_DATA | 40.6618 | 4.2074 | 2003 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 8 | WORK.ANA_DATA | 27.8691 | 3.9024<br>4.1873 | 3513<br>1979 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 3 | 2 | 9 | WORK.ANA_DATA<br>WORK.ANA DATA | 48.1600<br>40.9653 | 3.8674 | 3520 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 4 | WORK.ANA DATA | -26.2762 | 4.1647 | 1952 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 5 | WORK.ANA DATA | 42.9186 | 2.7023 | 3511 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 5 | WORK.ANA DATA | 29.6984 | 4.1788 | 1968 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 6 | WORK.ANA DATA | -4.6142 | 2.7045 | 3511 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 6 | WORK.ANA_DATA | -23.3485 | 4.1996 | 1993 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 7 | WORK.ANA_DATA | 19.8457 | 2.7227 | 3514 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 7 | WORK.ANA_DATA | 0.5619 | 4.2138 | 2011 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 8 | WORK.ANA_DATA | 67.3353 | 2.7254 | 3514 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 8<br>9 | WORK.ANA_DATA | 54.5426<br>74.8335 | 4.1999<br>2.6964 | 1993<br>3514 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 4 | 2 | 9 | WORK.ANA_DATA<br>WORK.ANA DATA | 67.6388 | 4.1568 | 1945 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 5 | WORK.ANA DATA | 69.1949 | 4.1646 | 1952 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 5 | WORK.ANA DATA | 55.9746 | 3.8575 | 3517 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 6 | WORK.ANA DATA | 21.6620 | 4.1663 | 1954 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 6 | WORK.ANA_DATA | 2.9278 | 3.8778 | 3516 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 7 | WORK.ANA_DATA | 46.1220 | 4.1778 | 1968 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 7 | WORK.ANA_DATA | 26.8381 | 3.8932 | 3517 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 8 | WORK.ANA_DATA | 93.6116 | 4.1796 | 1970 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 8<br>9 | WORK.ANA_DATA<br>WORK.ANA DATA | 80.8188<br>101.11 | 3.8782<br>4.1594 | 3516<br>1947 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 4 | 2 | 9 | WORK.ANA DATA | 93.9151 | 3.8371 | 3516 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 5 | WORK.ANA DATA | -13.2203 | 4.1788 | 1968 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 6 | WORK.ANA DATA | -47.5329 | 2.7049 | 3512 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 6 | WORK.ANA DATA | -66.2671 | 4.1995 | 1993 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 7 | WORK.ANA_DATA | -23.0729 | 2.7221 | 3513 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 7 | WORK.ANA_DATA | -42.3568 | 4.2137 | 2011 |
| TRTPN (ATPTN) | 1 | 5<br>5 | 1 2 | 8 | WORK.ANA_DATA | 24.4167 | 2.7247<br>4.1998 | 3513 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 5 | 1 | 9 | WORK.ANA_DATA<br>WORK.ANA DATA | 11.6240<br>31.9148 | 2.6964 | 1993<br>3514 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 9 | WORK.ANA DATA | 24.7202 | 4.1567 | 1945 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 6 | WORK.ANA DATA | -34.3126 | 4.1804 | 1970 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 6 | WORK.ANA DATA | -53.0469 | 3.8907 | 3515 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 7 | WORK.ANA_DATA | -9.8526 | 4.1919 | 1984 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 7 | WORK.ANA_DATA | -29.1365 | 3.9060 | 3516 |
| TRTPN (ATPTN) | 2 | 5<br>5 | 1 | 8 | WORK.ANA_DATA | 37.6369 | 4.1936 | 1986 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 8<br>9 | WORK.ANA_DATA | 24.8442 | 3.8890<br>4.1735 | 3513 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 5 | 2 | 9 | WORK.ANA_DATA<br>WORK.ANA DATA | 45.1351<br>37.9405 | 3.8524 | 1963<br>3519 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 6 | WORK.ANA DATA | -18.7342 | 4.2012 | 1995 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 7 | WORK.ANA DATA | 24.4600 | 2.7253 | 3514 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 7 | WORK.ANA DATA | 5.1761 | 4.2154 | 2013 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 8 | WORK.ANA_DATA | 71.9496 | 2.7279 | 3514 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 8 | WORK.ANA_DATA | 59.1568 | 4.2015 | 1995 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 9 | WORK.ANA_DATA | 79.4477 | 2.6990 | 3514 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 9 | WORK.ANA_DATA | 72.2531 | 4.1584 | 1947 |
| TRTPN (ATPTN) | 2 | 6<br>6 | 1 2 | 7<br>7 | WORK.ANA_DATA | 43.1942 | 4.2127 | 2009 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 6 | 1 | 8 | WORK.ANA_DATA<br>WORK.ANA DATA | 23.9104<br>90.6838 | 3.9282<br>4.2144 | 3518<br>2011 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 8 | WORK.ANA DATA | 77.8911 | 3.9112 | 3515 |
| ,, | | | | | | | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 198 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

### Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 2<br>2<br>1<br>1<br>1 | 6<br>7<br>7<br>7 | 1<br>2<br>2<br>1<br>2 | 9<br>9<br>7<br>8<br>8 | WORK.ANA_DATA WORK.ANA_DATA WORK.ANA_DATA WORK.ANA_DATA WORK.ANA_DATA WORK.ANA_DATA | 98.1819<br>90.9873<br>-19.2838<br>47.4896<br>34.6969<br>54.9877 | 4.1944<br>3.8750<br>4.2268<br>2.7440<br>4.2130<br>2.7168 | 1988<br>3521<br>2026<br>3514<br>2009<br>3516 |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 1<br>2<br>2<br>2 | 7<br>7<br>7<br>7 | 2<br>1<br>2<br>1 | 9<br>8<br>8<br>9 | WORK.ANA_DATA<br>WORK.ANA_DATA<br>WORK.ANA_DATA<br>WORK.ANA_DATA | 47.7931<br>66.7734<br>53.9807<br>74.2716 | 4.1700<br>4.2285<br>3.9265<br>4.2086 | 1961<br>2029<br>3516<br>2005 |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 2<br>1<br>1<br>2<br>2 | 7<br>8<br>8<br>8<br>8 | 2<br>2<br>1<br>2<br>1<br>2 | 9<br>8<br>9<br>9<br>9 | WORK.ANA_DATA WORK.ANA_DATA WORK.ANA_DATA WORK.ANA_DATA WORK.ANA_DATA WORK.ANA_DATA | 67.0770<br>-12.7927<br>7.4981<br>0.3035<br>20.2909<br>13.0962 | 3.8904<br>4.2147<br>2.7194<br>4.1717<br>4.1947<br>3.8754 | 3522<br>2011<br>3516<br>1964<br>1988<br>3522 |
| TRTPN (ATPTN) | Τ | 9 | 2 | 9 | WORK.ANA_DATA | -7.1946 | 4.1516 | 1940 |

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1<br>1 | | 2<br>1<br>2<br>1 | 1<br>2<br>2<br>3<br>3<br>4<br>4<br>4<br>5<br>5<br>6<br>6<br>7<br>7<br>8<br>8<br>9<br>9<br>2<br>2<br>2<br>3<br>3<br>4<br>4<br>4<br>5<br>5<br>6<br>6<br>7<br>7<br>8<br>8<br>9<br>9<br>9<br>2<br>9<br>2<br>3<br>3<br>4<br>4<br>5<br>5<br>6<br>6<br>6<br>7<br>8<br>9<br>9<br>2<br>9<br>2<br>3<br>3<br>4<br>4<br>5<br>5<br>6<br>6<br>7<br>7<br>8<br>7 | -2.22<br>-26.72<br>-22.66<br>-9.46<br>-11.60<br>-27.91<br>-24.41<br>-11.99<br>-10.91<br>-29.59<br>-23.51<br>-20.39<br>-17.75<br>-2.91<br>-4.94<br>-0.16<br>-1.83<br>-15.18<br>-2.22<br>-2.32<br>-15.95<br>-24.13<br>-15.95<br>-24.13<br>-15.59<br>-9.47<br>-17.05<br>-23.14<br>-11.12 | 0.0265 <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 2<br>2<br>2<br>2<br>2 | 1<br>1<br>1<br>1 | 2<br>1<br>2<br>1<br>2 | 7<br>8<br>8<br>9<br>9 | -16.88<br>0.31<br>-2.98<br>2.12<br>0.41 | <.0001<br>0.7600<br>0.0029<br>0.0342<br>0.6802 | 0.05<br>0.05<br>0.05<br>0.05<br>0.05 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 199 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 2 | 2 | 2 | -5.43 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 3 | 17.22 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 3 | 5.61 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 4 | -1.16 | 0.2459 | 0.05 |
| TRTPN (ATPTN) | 1 | 2 2 | 2 | 4<br>5 | -7.06<br>14.70 | <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 2 | 2 | 5 | 6.35 | <.0001<br><.0001 | 0.05<br>0.05 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 6 | -2.86 | 0.0042 | 0.05 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 6 | -6.31 | <.0001 | 0.05 |
| TRTPN (ATPTN) | ī | 2 | ī | 7 | 6.13 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 7 | -0.61 | 0.5409 | 0.05 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 8 | 23.53 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 8 | 12.24 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 9 | 26.57 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 9 | 15.51 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 2 2 | 1 2 | 3 | 16.54 | <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 2 | 1 | 4 | 11.87<br>4.68 | <.0001<br><.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 4 | -1.72 | 0.0854 | 0.05 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 5 | 14.92 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 5 | 12.69 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 6 | 3.58 | 0.0004 | 0.05 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 6 | -0.96 | 0.3392 | 0.05 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 7 | 9.38 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 7 | 5.15 | <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 2 | 2 2 | 1 2 | 8 | 20.67<br>18.99 | <.0001<br><.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 9 | 22.56 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 9 | 22.56 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 3 | -5.50 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 4 | -18.41 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 4 | -18.25 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 5 | -2.52 | 0.0117 | 0.05 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 5 | -4.80 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 3 | 1 2 | 6<br>6 | -20.09<br>-17.40 | <.0001<br><.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 3 | 1 | 7 | -10.98 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 7 | -11.67 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 8 | 6.46 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 8 | 1.14 | 0.2528 | 0.05 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 9 | 9.31 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 9 | 4.31 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 4 | -6.36 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 4 | -13.67 | <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 2 | 3 | 2 | 5<br>5 | 3.87<br>0.78 | 0.0001<br>0.4358 | 0.05 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 6 | -7.46 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 6 | -12.81 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 7 | -1.62 | 0.1046 | 0.05 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 7 | -6.66 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 8 | 9.66 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 8 | 7.14 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 9 | 11.50 | <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2<br>1 | 3 4 | 2 2 | 9<br>4 | 10.59<br>-6.31 | <.0001<br><.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 5 | 15.88 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 5 | 7.11 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 6 | -1.71 | 0.0881 | 0.05 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 6 | -5.56 | <.0001 | 0.05 |
| • | | | | | | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 200 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 4 | 1 | 7 | 7.29 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 7 | 0.13 | 0.8939 | 0.05 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 8 | 24.71 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 8 | 12.99 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 9 | 27.75 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 9 | 16.27 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 5 | 16.62 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 5 | 14.51 | <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 2 | 4 | 1 2 | 6<br>6 | 5.20<br>0.75 | <.0001<br>0.4503 | 0.05 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 7 | 11.04 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 7 | 6.89 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 8 | 22.40 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 8 | 20.84 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 9 | 24.31 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 9 | 24.48 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 5 | -3.16 | 0.0016 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 6 | -17.57 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 6 | -15.78 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1<br>1 | 5<br>5 | 1 2 | 7<br>7 | -8.48<br>-10.05 | <.0001<br><.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 5 | 1 | 8 | 8.96 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 8 | 2.77 | 0.0057 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 9 | 11.84 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 9 | 5.95 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 6 | -8.21 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 6 | -13.63 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 7 | -2.35 | 0.0189 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 7<br>8 | -7.46 | <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 2 | 5<br>5 | 2 | 8 | 8.97<br>6.39 | <.0001<br><.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 9 | 10.81 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 9 | 9.85 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 6 | -4.46 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 7 | 8.98 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 7 | 1.23 | 0.2196 | 0.05 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 8 | 26.38 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1<br>1 | 6<br>6 | 2 | 8<br>9 | 14.08<br>29.44 | <.0001<br><.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 6 | 2 | 9 | 17.38 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 7 | 10.25 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 7 | 6.09 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 8 | 21.52 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 8 | 19.91 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 9 | 23.41 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 9 | 23.48 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 7 | -4.56 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 7<br>7 | 1 2 | 8 | 17.31<br>8.24 | <.0001 | 0.05<br>0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 7 | 1 | 9 | 20.24 | <.0001<br><.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 9 | 11.46 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 8 | 15.79 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 8 | 13.75 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 9 | 17.65 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 9 | 17.24 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 8 | -3.04 | 0.0024 | 0.05 |
| TRTPN (ATPTN) | 1 | 8 | 1 | 9 | 2.76 | 0.0059 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 2 | 8 | 2 | 9 | 0.07<br>4.84 | 0.9420<br><.0001 | 0.05 |
| TIVIEN (WILIN) | ۷ | J | ± | J | 4.04 | <.000± | 0.00 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 201 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

### Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN)<br>TRTPN (ATPTN) | 2 | 8<br>9 | 2 2 | 9<br>9 | 3.38<br>-1.73 | 0.0007<br>0.0833 | 0.05<br>0.05 |

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | 2 | 1 | -17.3012 | -1.0719 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 2 | -77.4025 | -66.8207 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 2 | -103.08 | -86.6565 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 3 | -30.7993 | -20.2263 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 3 | -56.7901 | -40.3659 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 4 | -80.5382 | -69.9648 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 4 | -109.69 | -93.3704 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 5 | -37.6195 | -27.0463 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 5 | -53.7382 | -37.3681 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 6 | -85.1576 | -74.5739 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 6 | -106.83 | -90.3741 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 7 | -60.7324 | -50.0791 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 7 | -82.9433 | -66.4359 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 8 | -13.2480 | -2.5843 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 8 | -28.9354 | -12.4824 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 9 | -5.6888 | 4.8528 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 9 | -15.7546 | 0.5293 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 2 | -71.0522 | -54.7980 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 2 | -93.2435 | -78.1208 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 3 | -24.4506 | -8.2020 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 3 | -46.9527 | -31.8302 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 4 | -74.1894 | -57.9405 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 4 | -99.8429 | -84.8395 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 5 | -31.2707 | -15.0220 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 5 | -43.8984 | -28.8347 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 6 | -78.8069 | -62.5515 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 6 | -96.9897 | -81.8372 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 7 | -54.3697 | -38.0688 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 7 | -73.1096 | -57.8966 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 8 | -6.8835 | 9.4242 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 8 | -19.0993 | -3.9454 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 9 | 0.6544 | 16.8826 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 9 | -5.9110 | 9.0588 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 2 | -30.9818 | -14.5323 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 3 | 41.2945 | 51.9031 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 3 | 15.3088 | 31.7585 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 4 | -8.4444 | 2.1646 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 4 | -37.5863 | -21.2459 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 5 | 34.4744 | 45.0831 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 5 | 18.3606 | 34.7564 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 6 | -13.0637 | -2.4445 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 6 | -34.7270 | -18.2497 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 7 | 11.3615 | 22.0503 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 7 | -10.8444 | 5.6884 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 8 | 58.8470 | 69.5440 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 8 | 43.1635 | 59.6420 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 9 | 66.4027 | 76.9845 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 9 | 56.3441 | 72.6538 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 202 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| Differences of Least Squares fleating | | | | | | |
|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
| TRTPN (ATPTN) | 2 | 2 | 1 | 3 | 61.1337 | 77.5781 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 3 | 38.6471 | 53.9343 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 4 | 11.3948 | 27.8396 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 4 | -14.2472 | 0.9291 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 5 | 54.3136 | 70.7581 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 5 | 41.6983 | 56.9329 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 6 | 6.7773 | 23.2285 |
| TRTPN (ATPTN) | 2 | 2<br>2<br>2 | 2 | 6<br>7 | -11.3851<br>31.2149 | 3.9225<br>47.7109 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 2 | 1 2 | 7 | 12.4953 | 27.8629 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 8 | 78.7012 | 95.2038 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 8 | 66.5021 | 81.8174 |
| TRTPN (ATPTN) | 2 | 2 2 | 1 | 9 | 86.2385 | 102.66 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 9 | 79.6733 | 94.8387 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 3 | -31.2872 | -14.8432 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 4 | -55.0370 | -44.4405 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 4 | -84.1824 | -67.8475 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 5 | -12.1182 | -1.5220 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 5 | -28.2354 | -11.8452 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 6 | -59.6563 | -49.0497 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 6 | -81.3230 | -64.8513 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 7 | -35.2301 | -24.5559 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 3 | 2 | 7<br>8 | -57.4405<br>12.2533 | -40.9131<br>22.9399 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 8 | -3.4326 | 13.0404 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 9 | 19.8082 | 30.3813 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 9 | 9.7481 | 26.0522 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 4 | -34.8958 | -18.4512 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 4 | -60.5424 | -45.3571 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 5 | 8.0230 | 24.4673 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 5 | -4.5845 | 10.6342 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 6 | -39.5132 | -23.0623 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 6 | -57.6795 | -42.3645 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 7<br>7 | -15.0757 | 1.4201 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 8 | -33.7992 | -18.4241 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 3 | 2 | 8 | 32.4106<br>20.2179 | 48.9131<br>35.5202 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 9 | 39.9479 | 56.3720 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 9 | 33.3828 | 48.5479 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 4 | -34.4440 | -18.1084 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 5 | 37.6203 | 48.2170 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 5 | 21.5031 | 37.8936 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 6 | -9.9167 | 0.6882 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 6 | -31.5845 | -15.1125 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 7 | 14.5074 | 25.1841 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 7 | -7.7019 | 8.8257 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 8 | 61.9919 | 72.6788 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 8<br>9 | 46.3059<br>69.5467 | 62.7793<br>80.1202 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 4 | 2 | 9 | 59.4867 | 75.7910 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 5 | 61.0274 | 77.3624 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 5 | 48.4114 | 63.5379 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 6 | 13.4911 | 29.8328 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 6 | -4.6753 | 10.5308 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 7 | 37.9285 | 54.3154 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 7 | 19.2050 | 34.4713 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 8 | 85.4148 | 101.81 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 8 | 73.2151 | 88.4226 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 9 | 92.9524 | 109.27 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 203 of 334 | |

Parameter Code=SMPGCOL

The Mixed Procedure

Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint | Lower | Upper |
|---|---|---|---|---|---|---|
| | , , | , | . , | , | | -11 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 9 | 86.3920 | 101.44 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 5 | -21.4155 | -5.0250 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 6 | -52.8363 | -42.2295 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 6 | -74.5030 | -58.0312 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 7 | -28.4099 | -17.7359 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 7 | -50.6205 | -34.0930 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 8 | 19.0745 | 29.7589 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 8 | 3.3874 | 19.8605 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 9 | 26.6282 | 37.2014 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 9 | 16.5681 | 32.8723 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 6 | -42.5111 | -26.1142 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 6 | -60.6751 | -45.4187 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 7 | -18.0737 | -1.6316 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 7 | -36.7948 | -21.4782 |
| TRTPN (ATPTN) | 2 | 5<br>5 | 1 2 | 8 | 29.4126 | 45.8613 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 9 | 17.2193<br>36.9501 | 32.4692<br>53.3201 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 5 | 2 | 9 | 30.3873 | 45.4936 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 6 | -26.9735 | -10.4950 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 7 | 19.1166 | 29.8033 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 7 | -3.0909 | 13.4432 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 8 | 66.6011 | 77.2981 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 8 | 50.9170 | 67.3967 |
| TRTPN (ATPTN) | i | 6 | 1 | 9 | 74.1559 | 84.7395 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 9 | 64.0976 | 80.4086 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 7 | 34.9326 | 51.4559 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 7 | 16.2086 | 31.6121 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 8 | 82.4188 | 98.9488 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 8 | 70.2227 | 85.5595 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 9 | 89.9561 | 106.41 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 9 | 83.3898 | 98.5849 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 7 | -27.5732 | -10.9945 |
| TRTPN (ATPTN) | 1 | 7 | 1 | 8 | 42.1096 | 52.8696 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 8 | 26.4346 | 42.9591 |
| TRTPN (ATPTN) | 1 | 7 | 1 | 9 | 49.6611 | 60.3144 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 9 | 39.6150 | 55.9712 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 8 | 58.4808 | 75.0661 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 8 | 46.2823 | 61.6792 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 9 | 66.0179 | 82.5252 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 9 | 59.4492 | 74.7047 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 8 | -21.0583 | -4.5272 |
| TRTPN (ATPTN) | 1 | 8 | 1 | 9 | 2.1663 | 12.8300 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 9 | -7.8779 | 8.4850 |
| TRTPN (ATPTN) | 2 | 8 | 1 | 9 | 12.0644 | 28.5173 |
| TRTPN (ATPTN) | 2 | 8 | 2 | 9 | 5.4980 | 20.6945 |
| TRTPN (ATPTN) | 1 | 9 | 2 | 9 | -15.3368 | 0.9475 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 204 of 334 | |

# 19: Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment – change from baseline – supportive statistical analysis – full analysis set - appendix

Parameter Code=P9PSMPGM

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 443

Number of Observations

Number of Observations Read 453 Number of Observations Used 443 Number of Observations Not Used 10

Covariance Parameter Estimates

Cov Parm Estimate
Residual 2.4827

Fit Statistics

-2 Res Log Likelihood 1668.3 AIC (Smaller is Better) 1670.3 AICC (Smaller is Better) 1670.3 BIC (Smaller is Better) 1674.4

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept 7.2884 0.3649 439 19.97 trtpn -0.9761 0.1585 -6.16 trtpn 2 Ω BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD -0.02534 PREAD 0.1500 439 -0.17 PREAD 0.1399 0.03066 439 4.56 BASE

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 tatus: Final 

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PSMPGM

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial | l anti-Di | abetic treat | ment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | ıa | |
|---|---|---|---|---|---|---|---|---|---|
| Intercept | t | | | | | <.0001 | | | |
| trtpn<br>trtpn<br>PREAD | DACAT INC | SIIT TN I N | IEMEODMIN | | 1<br>2 | <.0001<br>0.8659 | | | |
| PREAD<br>PREAD<br>BASE | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | | <.0001 | | | |
| BIIOE | | | Solution fo | or Fixed Effe | cts | 1.0001 | 0.0 | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial anti-Diabetic treatment | | | | 01 (N) | Lower | Up | per | |
| Intercept<br>trtpn<br>trtpn | ept | | | | 1 2 | 6.5712<br>-1.2877 | | | |
| PREAD<br>PREAD | READ BASAL INSULIN + METFORMIN | | | ۷ | -0.3201 | 0.2 | 695 | | |
| BASE | | | | | | 0.07968 | 0.2 | 002 | |
| | Type 3 Tests | s of Fixe | d Effects | | | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 439<br>439<br>439 | 37.90<br>0.03<br>20.83 | <.0001<br>0.8659<br><.0001 | | | | | |
| | | | Least | Squares Mear | ns Estimates | | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, II<br>LSMeans, II | | WORK.ADATA2 | | 0.09191<br>0.1291 | 439<br>439 | 85.40<br>68.34 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least S | Squares Means | Estimates | | | | |
| Effect | Label | | Lower | Upper Ex | kponentiated | | ntiated<br>Lower | Exponentia<br>Up | ted<br>per |
| | LSMeans, II | | 7.6685<br>8.5714 | 8.0298<br>9.0790 | 2563.52<br>6803.49 | | 2139.86<br>5278.49 | 3071<br>8769 | |
| | | | Least | Squares Means | s Estimate | | | | |
| | | | | | | | ndard | | |
| Effect 1 | Label | | | Margins | Estim | ate | Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -0.9761 0.1585 439

-6.16

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PSMPGM

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg <.0001 0.05 -1.2877 -0.6645 0.3768

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.2759 0.5146


Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9SMPGMU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 443

Number of Observations

Number of Observations Read 453 Number of Observations Used 443 Number of Observations Not Used 10

Covariance Parameter Estimates

Cov Parm Estimate
Residual 806.17

Fit Statistics

-2 Res Log Likelihood 4212.8
AIC (Smaller is Better) 4214.8
AICC (Smaller is Better) 4214.8
BIC (Smaller is Better) 4218.9

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 6.5753 131.34 439 19.97 Intercept -17.5886 2.8570 1 439 -6.16 trtpn trtpn PREAD BASAL INSULIN + METFORMIN -0.4567 2.7030 -0.17 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD BASE 0.1399 0.03066 439 4.56

#### NN9068 22 January 2020 | Novo Nordisk Date: NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9SMPGMU

The Mixed Procedure

| | Solution for Fixed Effects | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | Planned<br>Treatment<br>for | | | | |
| Effect | Pre Trial anti-D | iabetic treatm | nent | Period<br>01 (N) | Pr > t | Alph | ıa | |
| Interceptrtpn<br>trtpn<br>trtpn | pt | | 1 2 | <.0001<br><.0001 | | | | |
| PREAD<br>PREAD | BASAL INSULIN +<br>BASAL INSULIN + | | IE OTHER OAD | 2 | 0.8659 | 0.0 | 5 | |
| BASE | BROTH INCOLIN | IIIII OITIIN , OI | d official official | | <.0001 | 0.0 | 15 | |
| | | Solution for | Fixed Effec | cts | | | | |
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| | Pre Trial anti-D | iabetic treatm | nent | 01 (N) | Lower | _ | pper | |
| Intercept trtpn | pt | | | 1 | 118.41<br>-23.2036 | | .26<br>9735 | |
| trtpn<br>PREAD | BASAL INSULIN + | | | 2 | -5.7691 | 4.8 | 557 | |
| PREAD<br>BASE | BASAL INSULIN + | | 0.07968 | 0.2 | 2002 | | | |
| Type 3 Tests of Fixed Effects | | | | | | | | |
| Effect | Num Den<br>DF DF | F Value F | r > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 439<br>1 439<br>1 439 | 0.03 | (.0001<br>(.8659<br>(.0001 | | | | | |
| | | Least | Squares Mean | ns Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF 1 | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 141.44<br>159.03 | 1.6563<br>2.3270 | 439<br>439 | 85.40<br>68.34 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least So | quares Means | Estimates | | | | |
| Effect | Label | Lower | Upper Ex | xponentiated | | ntiated<br>Lower | Exponentia<br>Up | ted<br>per |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | 138.19<br>154.46 | 144.70<br>163.60 | 2.674E61<br>1.164E69 | | .032E60<br>.201E67 | 6.933<br>1.127 | |
| | | Least S | Squares Means | s Estimate | | | | |
| Effect | Label | | Margins | Estim | | ndard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -17.5886 2.8570 439

-6.16

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9SMPGMU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg <.0001 0.05 -23.2036 -11.9735 2.298E-8

Least Squares Means Estimate

Effect Label Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 8.37E-11 6.309E-6

# NN9068 NN9068-4166 Clinical Trial Report Statistical document CONFIDENTIAL Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PSMPGM

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 443

Number of Observations

Number of Observations Read 453 Number of Observations Used 443 Number of Observations Not Used 10

Covariance Parameter Estimates

Cov Parm Estimate
Residual 2.4827

Fit Statistics

-2 Res Log Likelihood 1668.3 AIC (Smaller is Better) 1670.3 AICC (Smaller is Better) 1670.3 BIC (Smaller is Better) 1674.4

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 7.2884 0.3649 439 19.97 Intercept -0.9761 439 -6.16 0.1585 trtpn 0 trtpn PREAD BASAL INSULIN + METFORMIN -0.02534 439 -0.17 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.8601 BASE 0.03066 439 -28.05

# NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PSMPGM

The Mixed Procedure

# Solution for Fixed Effects

| Solution for Fixed Effects | | | | |
|---|---|---|---|---|
| Effect | Pre Trial anti-Diabetic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn<br>trtpn | | 1 2 | <.0001<br><.0001 | 0.05<br>0.05 |
| PREAD | BASAL INSULIN + METFORMIN | _ | 0.8659 | 0.05 |
| PREAD<br>BASE | BASAL INSULIN + METFORMIN + ONE OTHER C | DAD | <.0001 | 0.05 |
| Solution for Fixed Effects | | | | |
| | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial anti-Diabetic treatment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | 1 2 | 6.5712<br>-1.2877 | 8.0055<br>-0.6645 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER C | 2 | -0.3201 | 0.2695 |
| BASE | DAGAE INSUER - FEITOREIN - ONE CIMEN C | )AD | -0.9203 | -0.7998 |
| Ту | pe 3 Tests of Fixed Effects | | | |
| Effect | Num Den<br>DF DF F Value Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1 439 37.90 <.0001<br>1 439 0.03 0.8659<br>1 439 786.85 <.0001 | | | |

# Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.09191<br>0.1291 | 439<br>439 | -35.03<br>-17.38 | <.0001<br><.0001 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | | -3.4004<br>-2.4975 | -3.0391<br>-1.9899 | | | |


Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9SMPGMU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 443

Number of Observations

Number of Observations Read 453 Number of Observations Used 443 Number of Observations Not Used 10

Covariance Parameter Estimates

Cov Parm Estimate
Residual 806.17

Fit Statistics

-2 Res Log Likelihood 4212.8
AIC (Smaller is Better) 4214.8
AICC (Smaller is Better) 4214.8
BIC (Smaller is Better) 4218.9

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 131.34 6.5753 439 19.97 Intercept -17.5886 2.8570 439 -6.16 trtpn 0 trtpn PREAD BASAL INSULIN + METFORMIN -0.4567 2.7030 439 -0.17 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.8601 BASE 0.03066 439 -28.05

#### NN9068 22 January 2020 | Novo Nordisk Date: NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9SMPGMU

The Mixed Procedure

| Solution for Fixed Effects | | | | | | |
|---|---|---|---|---|---|---|
| Effect | Pre Trial ant | i-Diabetic trea | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn | | | | 1 | <.0001<br><.0001 | 0.05<br>0.05 |
| trtpn<br>PREAD | BASAL INSULIN | | 2 | 0.8659 | 0.05 | |
| PREAD<br>BASE | BASAL INSULIN | 1 + METFORMIN + | ONE OTHER OAD | | <.0001 | 0.05 |
| Solution for Fixed Effects | | | | | | |
| 755 | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial ant | i-Diabetic trea | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | 1 2 | 118.41<br>-23.2036 | 144.26<br>-11.9735 |
| PREAD<br>PREAD | BASAL INSULIN | | _ | -5.7691 | 4.8557 | |
| BASE | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | -0.9203 | -0.7998 |
| Т | rpe 3 Tests of | Fixed Effects | | | | |
| Effect | Num De<br>DF I | | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1 43<br>1 43<br>1 43 | 0.03 | <.0001<br>0.8659<br><.0001 | | | |

# Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 1.6563<br>2.3270 | 439<br>439 | -35.03<br>-17.38 | <.0001<br><.0001 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | | 51.2758<br>15.0054 | -54.7654<br>-35.8586 | | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 214 of 334 | |

Parameter Code=P9PGIBU

The Mixed Procedure

Class

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

trtpn 2 1 2 PREAD 2 BASAL INSULIN +

Levels

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Values

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 449

Number of Observations

Number of Observations Read 453 Number of Observations Used 449 Number of Observations Not Used 4

Covariance Parameter Estimates

Cov Parm Estimate
Residual 2154.91

Fit Statistics

-2 Res Log Likelihood 4708.0
AIC (Smaller is Better) 4710.0
AICC (Smaller is Better) 4710.0
BIC (Smaller is Better) 4714.1

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept 62.1279 5.6099 11.07 trtpn -13.8531 4.6458 -2.98 trtpn 2 Ω BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD 3.8477 PREAD 4.3900 445 0.88 PREAD 0.2690 0.03980 6.76 BASE 445

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 215 of 334 | |

Parameter Code=P9PGIBU

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial anti-D. | iabetic treatme | ent | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | a | |
|---|---|---|---|---|---|---|---|---|
| Intercep | | | | , | <.0001 | 0.0 | | |
| trtpn<br>trtpn | | | | 1 2 | 0.0030 | 0.0 | 5 | |
| PREAD<br>PREAD | BASAL INSULIN + I<br>BASAL INSULIN + I | | E OTHER OAD | | 0.3813 | 0.0 | | |
| BASE | | | | | <.0001 | 0.0 | 5 | |
| | | Solution for | Fixed Effec | | | | | |
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial anti-D | iabetic treatme | ent | 01 (N) | Lower | Up | per | |
| Intercep<br>trtpn<br>trtpn | t | | | 1 2 | 51.1026<br>-22.9835 | 73.1<br>-4.7 | | |
| PREAD<br>PREAD | | | | -4.7801 | 12.4 | 754 | | |
| BASE | | | | | 0.1908 | 0.3 | 472 | |
| | Type 3 Tests of Fixe | ed Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value Pr | r > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 445<br>1 445<br>1 445 | 0.77 0. | .0030<br>.3813<br>.0001 | | | | | |
| | | Least S | Squares Mear | ns Estimates | | | | |
| | | | - | Standard | | | | |
| Effect | Label | Margins | Estimate | Error | DF t | Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 73.0519<br>86.9050 | 2.6908<br>3.7824 | 445<br>445 | 27.15<br>22.98 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least Squ | uares Means | Estimates | | | | |
| Effect | Label | Lower | Upper Ex | xponentiated | | tiated<br>Lower | Exponentia<br>Up | ted<br>per |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | | 78.3402<br>94.3386 | 5.322E31<br>5.525E37 | | 688E29<br>266E34 | 1.054<br>9.348 | |
| | | Least So | quares Means | s Estimate | | | | |
| Effect | Label | | Margins | Estima | | dard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -13.8531 4.6458 445 -2.98

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
5 tatus:
Final
Page:

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGIBU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.0030 0.05 -22.9835 -4.7226 9.632E-7

Least Squares Means Estimate

Effect Label Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 1.04E-10 0.008892

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGIEU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 446

Number of Observations

Number of Observations Read 453 Number of Observations Used 446 Number of Observations Not Used 7

Covariance Parameter Estimates

Cov Parm Estimate
Residual 1879.19

Fit Statistics

-2 Res Log Likelihood 4616.1
AIC (Smaller is Better) 4618.1
AICC (Smaller is Better) 4618.1
BIC (Smaller is Better) 4622.2

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 45.9181 4.3240 442 10.62 Intercept -4.3682 -1.00 4.3513 442 trtpn 0 trtpn PREAD BASAL INSULIN + METFORMIN -0.5936 4.1296 -0.14 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.1500 BASE 0.03431 442 4.37

| NN9068 | | Date: | 22 January 2020 Novo Nordis |
|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final |
| Statistical document | | Page: | 218 of 334 |

Parameter Code=P9PGIEU

The Mixed Procedure

| The Mix | ed Procedu | re | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Solution for | Fixed Effe | ects | | | | |
| Effect | Pro Tr | ial anti-D | iabetic treat | mant | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | n a | |
| FILECC | rie ii. | iai anci-b. | iabetic tieat | menc | 01 (N) | | _ | | |
| Interce<br>trtpn<br>trtpn | pt | | | | 1 2 | <.0001<br>0.3160 | | | |
| PREAD | | INSULIN + I | | | | 0.8858 | 0.0 | )5 | |
| PREAD<br>BASE | BASAL | INSULIN + I | METFORMIN + O | NE OTHER OF | AD | <.0001 | 0.0 | )5 | |
| | | | Solution fo | r Fixed Ef | fects | | | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Tr | ial anti-D | iabetic treat | ment | 01 (N) | Lower | Up | pper | |
| Interce<br>trtpn<br>trtpn | pt | | | | 1 2 | 37.4199<br>-12.9200 | | 1163<br>1836 | |
| PREAD | | INSULIN + I | | | _ | -8.7098 | 7.5 | 5226 | |
| PREAD<br>BASE | BASAL | INSULIN + I | METFORMIN + O | NE OTHER OA | AD | 0.08253 | 0.2 | 2174 | |
| | Туре 3 Те | sts of Fixe | ed Effects | | | | | | |
| Effect | Num<br>DF | | F Value | Pr > F | | | | | |
| trtpn | 1 | | | 0.3160 | | | | | |
| PREAD<br>BASE | 1<br>1 | | | 0.8858<br><.0001 | | | | | |
| | | | Least | Squares Me | eans Estimates | 3 | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADATA2<br>WORK.ADATA2 | | | 442<br>442 | 18.93<br>14.70 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least S | quares Mean | ns Estimates | | | | |
| | | | _ | | _ | | ntiated | Exponentia | |
| Effect | Label | | Lower | Upper | Exponentiated | | Lower | Up | per |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | 42.7758<br>45.1352 | 52.6848<br>59.0618 | 5.358E20<br>4.228E22 | | .778E18 | 7.598<br>4.469 | |
| | | | Least | Squares Mea | ans Estimate | | | | |
| Effect | Label | | | Margin | ns Estim | | ndard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -4.3682 4.3513 442 -1.00

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 219 of 334 | |

Parameter Code=P9PGIEU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.3160 0.05 -12.9200 4.1836 0.01267

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 2.449E-6 65.6022

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 1.0 Status: Final Page: 22 January 2020 Avov Nordisk Post 22 January 2020 22 January 2020 Status: 1.0 Status: Final Page: 22 January 2020

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGILU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 449

Number of Observations

Number of Observations Read 453 Number of Observations Used 449 Number of Observations Not Used 4

Covariance Parameter Estimates

Cov Parm Estimate
Residual 2310.04

Fit Statistics

-2 Res Log Likelihood 4739.1 AIC (Smaller is Better) 4741.1 AICC (Smaller is Better) 4741.1 BIC (Smaller is Better) 4745.2

Solution for Fixed Effects

Planned Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 44.9769 9.45 4.7616 445 Intercept -1.2247 -0.25 1 445 4.8065 trtpn trtpn PREAD BASAL INSULIN + METFORMIN -4.4637 4.5624 -0.98 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.2018 BASE 0.03834 445 5.26

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 221 of 334 | |

Parameter Code=P9PGILU

The Mixed Procedure

| IIIC IIIAC | ou iloccuu | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Solution for | Fixed Effe | ects | | | | |
| Effect | Pre Tr | ial anti-D: | iabetic treatm | ment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | ıa | |
| Intercer | ot | | | | | <.0001 | 0.0 | )5 | |
| trtpn<br>trtpn | | | | | 1<br>2 | 0.7990 | 0.0 | )5 | |
| PREAD<br>PREAD | | INSULIN + N | METFORMIN<br>METFORMIN + OI | NE OTHER OF | A D | 0.3284 | 0.0 | )5 | |
| BASE | 2110112 | 111002211 | | 0111211 01 | | <.0001 | 0.0 | )5 | |
| | | | Solution for | r Fixed Eff | fects | | | | |
| Effect | Pre Tr | ial anti-Di | iabetic treatm | ment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Uŗ | pper | |
| Intercep | ot | | | | | 35.6189 | | | |
| trtpn<br>trtpn | | | | | 1<br>2 | -10.6710 | | 2215 | |
| PREAD<br>PREAD | | INSULIN + 1<br>INSULIN + 1 | METFORMIN<br>METFORMIN + OI | NE OTHER OF | AD | -13.4301 | | 5028 | |
| BASE | | | | | | 0.1264 | 0.2 | 2771 | |
| | Туре 3 Те | sts of Fixe | ed Effects | | | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | | | |
| trtpn<br>PREAD | 1 | | | 0.7990<br>0.3284 | | | | | |
| BASE | 1 | | | <.0001 | | | | | |
| | | | Least | Squares Me | eans Estimates | | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF t | . Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADATA2<br>WORK.ADATA2 | | | 445<br>445 | 18.01<br>13.13 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least So | quares Mear | ns Estimates | | | | |
| Effect | Label | | Lower | Upper | Exponentiated | | ntiated<br>Lower | | ted<br>per |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | 44.6786<br>43.6845 | 55.6264<br>59.0699 | 6.039E21<br>2.055E22 | | .533E19<br>.374E18 | 1.44<br>4.505 | |
| | | | Least : | Squares Mea | ans Estimate | | | | |
| | | | | | | Star | ndard | | |
| Effect | Label | | | Margir | ns Estim | ate I | Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -1.2247 4.8065 445 -0.25

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
5 tatus:
Final
Page:
22 January 2020
Pove Nordisk
Pove Nordisk

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGILU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.7990 0.05 -10.6710 8.2215 0.2938

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.000023 3720.21

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final Page: 22 January 2020 Power Nordisk Power Nordisk Power Status: Final Page: 22 January 2020 Power Nordisk Power Status: Final Page: Page: Page: Page: Power Nordisk

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGINC

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 452

Number of Observations

Number of Observations Read 453 Number of Observations Used 452 Number of Observations Not Used 1

Covariance Parameter Estimates

Cov Parm Estimate
Residual 2.9392

Fit Statistics

-2 Res Log Likelihood 1777.4
AICC (Smaller is Better) 1779.4
AICC (Smaller is Better) 1779.4
BIC (Smaller is Better) 1783.5

Solution for Fixed Effects

Planned Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 2.7808 0.2026 448 13.73 Intercept 1 -0.4039 0.1715 -2.36 448 trtpn 0 trtpn PREAD BASAL INSULIN + METFORMIN -0.09210 0.1624 -0.57 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.2575 BASE 0.03900 448 6.60

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 224 of 334 | |

Parameter Code=P9PGINC

The Mixed Procedure

| | | | Solution for | Fixed Eff | ects | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial | anti-Di | abetic treatm | ment | 01 (N) | Pr > t | Alp | ha | |
| Intercept | | | | | 1 2 | <.0001<br>0.018 | | | |
| trtpn<br>PREAD | BASAL INS | | | IE OMIJED O | _ | 0.5709 | 9 0.0 | 05 | |
| PREAD<br>BASE | BASAL INS | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | AD | <.0000 | 1 0.0 | 05 | | |
| Solution for Fixed Effects | | | | | | | | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial | anti-Di | abetic treatm | ment | 01 (N) | Lowe | r Ul | pper | |
| Intercep<br>trtpn<br>trtpn | ot | | | | 1 2 | 2.382 | | 1789<br>6690 | |
| PREAD<br>PREAD | BASAL INS | | ETFORMIN<br>ETFORMIN + ON | IE OTUED O | _ | -0.4112 | 2 0.3 | 2271 | |
| BASE | DAGAL INS | OLIN I P. | ETTORMIN OF | VE OTHER O. | AD | 0.1808 | 8 0.3 | 3341 | |
| | Type 3 Tests | of Fixe | d Effects | | | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value F | ?r > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 448<br>448<br>448 | 0.32 | 0.0189<br>0.5709<br><.0001 | | | | | |
| | | | Least | Squares M | eans Estimates | 3 | | | |
| Effect | Label | | Margins | Estimat | Standard<br>e Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, ID<br>LSMeans, ID | | WORK.ADATA2<br>WORK.ADATA2 | 3.146<br>3.550 | | 448<br>448 | 31.80<br>25.39 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least So | quares Mea | ns Estimates | | | | |
| Effect | Label | | Lower | Upper | Exponentiated | | entiated<br>Lower | Exponentia<br>Up | ted<br>per |
| trtpn<br>trtpn | LSMeans, ID<br>LSMeans, ID | | 2.9516<br>3.2752 | 3.3404<br>3.8247 | 23.2435<br>34.8123 | | 19.1370<br>26.4488 | 28.2<br>45.8 | |
| | | | Least S | Squares Me | ans Estimate | | | | |
| Effect | Label | | | Margi | ns Estin | | andard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -0.4039 0.1715 448 -2.36

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 225 of 334 | |

Parameter Code=P9PGINC

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.0189 0.05 -0.7410 -0.06690 0.6677

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.4766 Exponentiated 0.9353

#### 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGINCB

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 449

Number of Observations

Number of Observations Read 453 Number of Observations Used 449 Number of Observations Not Used 4

Covariance Parameter Estimates

Cov Parm Estimate
Residual 6.6362

Fit Statistics

-2 Res Log Likelihood 2128.8
AIC (Smaller is Better) 2130.8
AICC (Smaller is Better) 2130.8
BIC (Smaller is Better) 2134.9

Solution for Fixed Effects

Planned Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 3.4477 445 11.07 0.3113 Intercept -0.7688 -2.98 1 0.2578 445 trtpn 0 trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.2135 0.2436 0.88 PREAD 0.2690 BASE 0.03980 445 6.76

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 227 of 334 | |

Parameter Code=P9PGINCB

The Mixed Procedure

| Solution for Fixed Effects | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial anti | -Diabetic treat | ment | 01 (N) | Pr > t | Alph | na | |
| Intercep<br>trtpn | t | | | 1 2 | <.0001<br>0.0030 | | | |
| trtpn PREAD BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | | 0.3813 | 0.0 | )5 | |
| PREAD<br>BASE | DAGAL INSULIN | METFORMIN 1 0 | NE OTHER OA | D | <.0001 | 0.0 | )5 | |
| | | Solution fo | r Fixed Effe | ects | | | | |
| | | | | Planned<br>Treatment<br>for | | | | |
| Effect | Pre Trial anti | -Diabetic treat | ment | Period<br>01 (N) | Lower | . Ur | pper | |
| Intercep | pt | | | 1 2 | 2.8359<br>-1.2754 | | )596<br>2621 | |
| trtpn<br>PREAD | | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | 3 0.6 | 5923 | |
| PREAD<br>BASE | BASAL INSULIN | | | | | 0.3 | 3472 | |
| | Type 3 Tests of F | ixed Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 445<br>1 445<br>1 445 | 0.77 | 0.0030<br>0.3813<br><.0001 | | | | | |
| | | Least | Squares Mea | ans Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLir<br>LSMeans, IDeg | a WORK.ADATA2<br>WORK.ADATA2 | | | 445<br>445 | 27.15<br>22.98 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least S | quares Mean: | s Estimates | | | | |
| Effect | Label | Lower | Upper 1 | Exponentiated | Expone | entiated<br>Lower | Exponentia<br>Up | ted<br>per |
| trtpn<br>trtpn | LSMeans, IDegLir<br>LSMeans, IDeg | 3.7605<br>4.4102 | 4.3474<br>5.2352 | 57.6238<br>124.30 | | 42.9686<br>82.2838 | 77.2<br>187 | |
| Least Squares Means Estimate | | | | | | | | |
| Effect | Label | | Margin | s Estima | | andard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -0.7688 0.2578 445 -2.98

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 228 of 334 | |

Parameter Code=P9PGINCB

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.0030 0.05 -1.2754 -0.2621 0.4636

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.2793 0.7695

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 1.0 Status: Final Page: 22 January 2020 Version: 22 January 2020 Version: 1.0 Status: Final 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGINCE

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 446

Number of Observations

Number of Observations Read 453 Number of Observations Used 446 Number of Observations Not Used 7

Covariance Parameter Estimates

Cov Parm Estimate
Residual 5.7871

Fit Statistics

-2 Res Log Likelihood 2054.2
AIC (Smaller is Better) 2056.2
AICC (Smaller is Better) 2056.3
BIC (Smaller is Better) 2060.3

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 2.5482 442 0.2400 10.62 Intercept -0.2424 0.2415 442 -1.00 trtpn trtpn PREAD BASAL INSULIN + METFORMIN -0.03294 -0.14 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.1500 BASE 0.03431 442 4.37

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 230 of 334 | |

Parameter Code=P9PGINCE

The Mixed Procedure

| IIIC IIIAC | d IIOCCau. | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Solution for | Fixed Effe | cts | | | | |
| Effect | Pre Tr | ial anti-D | iabetic treatm | nent | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alp | ha | |
| Intercer | o.t | | | | | <.000 | | | |
| trtpn | | | | | 1<br>2 | 0.316 | | | |
| trtpn<br>PREAD | | INSULIN + 1 | | | | 0.885 | 8 0. | 05 | |
| PREAD<br>BASE | BASAL . | INSULIN + 1 | METFORMIN + ON | NE OTHER OA | .D | <.000 | 1 0. | 05 | |
| | | | Solution for | Fixed Eff | ects | | | | |
| Effect | Pre Tr | ial anti-D | iabetic treatm | nent. | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lowe | r U | pper | |
| Intercep | | | | | , | 2.076 | | 0198 | |
| trtpn<br>trtpn | | | | | 1 2 | -0.717 | | 2322 | |
| PREAD | | INSULIN + 1 | | IE OBUIED OZ | | -0.483 | 3 0. | 4175 | |
| PREAD<br>BASE | BASAL . | BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | 0.0825 | 3 0. | 2174 | |
| | Type 3 Te: | sts of Fix | ed Effects | | | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value F | ?r > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 442 | 0.02 | 0.3160<br>0.8858<br><.0001 | | | | | |
| | | | Least | Squares Me | ans Estimates | | | | |
| | | | | | Standard | | | | |
| Effect | Label | | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADATA2<br>WORK.ADATA2 | | | 442<br>442 | 18.93<br>14.70 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least So | quares Mean | s Estimates | | | | |
| Effect | Label | | Lower | Upper | Exponentiated | | entiated<br>Lower | | ted<br>per |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | 2.3738<br>2.5047 | 2.9237<br>3.2776 | 14.1362<br>18.0140 | | 10.7381<br>12.2402 | 18.6<br>26.5 | |
| | | | Least S | Squares Mea | ns Estimate | | | | |
| | | | | | _ : | | andard | | _ |
| Effect | Label | | | Margin | s Estim | ate | Error | DF t Va | Lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -0.2424 0.2415 442 -1.00

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 231 of 334 | |

Parameter Code=P9PGINCE

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.3160 0.05 -0.7170 0.2322 0.7847

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.4882 Exponentiated T.2613
### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGINCL

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 449

Number of Observations

Number of Observations Read 453 Number of Observations Used 449 Number of Observations Not Used 4

Covariance Parameter Estimates

Cov Parm Estimate
Residual 7.1139

Fit Statistics

-2 Res Log Likelihood 2159.9
AIC (Smaller is Better) 2161.9
AICC (Smaller is Better) 2161.9
BIC (Smaller is Better) 2166.0

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 2.4959 9.45 0.2642 445 Intercept -0.06796 -0.25 0.2667 445 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.98 PREAD 0.2018 BASE 0.03834 445 5.26

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 233 of 334 | |

Parameter Code=P9PGINCL

The Mixed Procedure

| | | | Solution for | Fixed Effe | ects | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Tri | ial anti-Di | labetic treatm | nent | 01 (N) | Pr > t | Alph | na | |
| Intercept<br>trtpn | | | | | 1<br>2 | <.0001<br>0.7990 | | | |
| trtpn<br>PREAD | | INSULIN + N | | | | 0.3284 | 4 0.0 | )5 | |
| PREAD<br>BASE | BASAL . | INSULIN + N | METFORMIN + ON | NE OTHER OF | AD | <.0000 | 1 0.0 | )5 | |
| | | | Solution for | Fixed Eff | fects | | | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Tri | ial anti-Di | labetic treatm | nent | 01 (N) | Lower | _ | oper | |
| Intercept<br>trtpn<br>trtpn | | | | | 1<br>2 | 1.9766<br>-0.5922 | | 0153<br>4562 | |
| PREAD BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAL | | | | | -0.7453 | 3 0.2 | 2499 | | |
| BASE | DITOTIE | INCOLIN , I | | VE OTHER OF | 15 | 0.1264 | 4 0.2 | 2771 | |
| Ту | ype 3 Tes | sts of Fixe | ed Effects | | | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value F | ?r > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 445<br>445<br>445 | 0.96 | 0.7990<br>0.3284<br><.0001 | | | | | |
| | | | Least | Squares Me | eans Estimates | | | | |
| Effect I | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADATA2<br>WORK.ADATA2 | 2.7832<br>2.8511 | | 445<br>445 | 18.01<br>13.13 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least So | quares Mear | ns Estimates | | | | |
| Effect I | Label | | Lower | Upper | Exponentiated | | entiated<br>Lower | Exponentia<br>Up | ted<br>per |
| | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | 2.4794<br>2.4242 | 3.0869<br>3.2780 | 16.1700<br>17.3072 | | 11.9340<br>11.2935 | 21.9<br>26.5 | |
| | | | Least S | Squares Mea | ans Estimate | | | | |
| Effect La | abel | | | Margin | ns Estim | | andard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -0.06796 0.2667 445 -0.25

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 234 of 334 | |

Parameter Code=P9PGINCL

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.7990 0.05 -0.5922 0.4562 0.9343

Least Squares Means Estimate

Effect Label Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.5531 Exponentiated T.5781

### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGIU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 452

Number of Observations

Number of Observations Read 453 Number of Observations Used 452 Number of Observations Not Used 1

Covariance Parameter Estimates

Cov Parm Estimate
Residual 954.43

Fit Statistics

-2 Res Log Likelihood 4373.9
AIC (Smaller is Better) 4375.9
AICC (Smaller is Better) 4376.0
BIC (Smaller is Better) 4380.1

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 50.1099 448 3.6507 13.73 Intercept -7.2791 3.0904 -2.36 448 trtpn 0 trtpn PREAD BASAL INSULIN + METFORMIN -1.6597 -0.57 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.2575 BASE 0.03900 448 6.60

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 236 of 334 | |

Parameter Code=P9PGIU

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial anti-D: | labetic treatment | | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | ıa | |
|---|---|---|---|---|---|---|---|---|
| Intercept | | | | | <.0001 | | | |
| trtpn<br>trtpn | | | | 1 2 | 0.0189 | 0.0 | | |
| PREAD<br>PREAD | BASAL INSULIN + 1<br>BASAL INSULIN + 1 | | THER OAD | | 0.5709 | 0.0 | | |
| BASE | | Columbia for Di | DEE | <b>.</b> . | <.0001 | 0.0 | 15 | |
| | | Solution for Fi: | xea Ellec | Planned | | | | |
| | | | | Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial anti-D | labetic treatment | | 01 (N) | Lower | - | per | |
| Intercept<br>trtpn<br>trtpn | | | | 1 | 42.9353<br>-13.3526 | | | |
| PREAD<br>PREAD | BASAL INSULIN + 1<br>BASAL INSULIN + 1 | | _ | -7.4108 | 4.0 | 914 | | |
| BASE | 5110112 11100211 | ETT OTHER COME O | 111211 0112 | | 0.1808 | 0.3 | 341 | |
| Т | Type 3 Tests of Fixe | ed Effects | | | | | | |
| | Num Den | | | | | | | |
| Effect | | F Value Pr > | F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 448<br>1 448<br>1 448 | 5.55 0.01:<br>0.32 0.57:<br>43.59 <.00 | 09 | | | | | |
| | | Least Squ | ares Mean | s Estimates | | | | |
| | | | | Standard | | | | |
| Effect | Label | Margins E | stimate | Error | DF t | . Value | Pr > t | Alpha |
| | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 56.6914<br>63.9705 | 1.7825<br>2.5193 | 448<br>448 | 31.80<br>25.39 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least Square | es Means | Estimates | | | | |
| Effect | Label | Lower U | pper Ex | ponentiated | | ntiated<br>Lower | | ted<br>per |
| | LSMeans, IDegLira<br>LSMeans, IDeg | 53.1882 60.<br>59.0193 68. | 1946<br>9216 | 4.176E24<br>6.054E27 | | .257E23<br>.283E25 | 1.3871<br>8.5561 | |
| | | Least Squa | res Means | Estimate | | | | |
| | | - | | | Star | ndard | | |
| Effect L | abel | | Margins | Estim | ate E | Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -7.2791 3.0904 448 -2.36

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
5 tatus:
Final
Page:

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGIU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.0189 0.05 -13.3526 -1.2055 0.000690

Least Squares Means Estimate

Effect Label Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 1.589E-6 0.2995

### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5tatus: Final 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGIBU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 449

Number of Observations

Number of Observations Read 453 Number of Observations Used 449 Number of Observations Not Used 4

Covariance Parameter Estimates

Cov Parm Estimate
Residual 2154.91

Fit Statistics

-2 Res Log Likelihood 4708.0 AIC (Smaller is Better) 4710.0 AICC (Smaller is Better) 4710.0 BIC (Smaller is Better) 4714.1

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 62.1279 11.07 5.6099 445 Intercept -13.8531 -2.98 4.6458 445 trtpn trtpn PREAD BASAL INSULIN + METFORMIN 3.8477 4.3900 445 0.88 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.7310 BASE 0.03980 445 -18.37


Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGIBU

The Mixed Procedure

#### Solution for Fixed Effects

| | | | Solution f | or Fixed Effect | S | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | L anti-D: | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn | | | | | 1 2 | <.0001<br>0.0030 | 0.05<br>0.05 |
| trtpn<br>PREAD | BASAL INS | | | | 2 | 0.3813 | 0.05 |
| PREAD<br>BASE | | | | | | <.0001 | 0.05 |
| | | | Solution | for Fixed Effec | cts | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | 1<br>2 | 51.1026<br>-22.9835 | 73.1532<br>-4.7226 |
| PREAD<br>PREAD | BASAL INS | | | ONE OTHER OAD | | -4.7801 | 12.4754 |
| BASE | | | | | | -0.8092 | -0.6528 |
| Ту | pe 3 Tests | s of Fixe | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 445<br>445<br>445 | 8.89<br>0.77<br>337.31 | 0.0030<br>0.3813<br><.0001 | | | |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | -12.3083<br>1.5448 | 2.6908<br>3.7824 | 445<br>445 | -4.57<br>0.41 | <.0001<br>0.6832 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | | 7.5966<br>-5.8889 | -7.0200<br>8.9784 | | | |

### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGIEU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 446

Number of Observations

Number of Observations Read 453 Number of Observations Used 446 Number of Observations Not Used 7

Covariance Parameter Estimates

Cov Parm Estimate
Residual 1879.19

Fit Statistics

-2 Res Log Likelihood 4616.1
AIC (Smaller is Better) 4618.1
AICC (Smaller is Better) 4618.1
BIC (Smaller is Better) 4622.2

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 45.9181 442 4.3240 10.62 Intercept -4.3682 -1.00 4.3513 442 trtpn trtpn PREAD BASAL INSULIN + METFORMIN -0.5936 4.1296 -0.14 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.8500 BASE 0.03431 442 -24.78

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 241 of 334 | |

Parameter Code=P9PGIEU

The Mixed Procedure

#### Solution for Fixed Effects

| | | Solution f | or Fixed Effec | ts | | |
|---|---|---|---|---|---|---|
| Pre Trial | anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| | | | | 1 | <.0001<br>0.3160 | 0.05<br>0.05 |
| tpn<br>EAD BASAL INSULIN + METFORMIN<br>EAD BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | _ | 0.8858 | 0.05 | |
| BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | | <.0001 | 0.05 |
| | | Solution | for Fixed Effe | cts | | |
| | | | | Planned<br>Treatment<br>for<br>Period | | |
| Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Upper |
| | | | | 1 2 | 37.4199<br>-12.9200 | 54.4163<br>4.1836 |
| | | | ONE OTHER OAD | _ | -8.7098 | 7.5226 |
| | | | | | -0.9175 | -0.7826 |
| pe 3 Tests | of Fix | ed Effects | | | | |
| Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| 1<br>1<br>1 | 442<br>442<br>442 | 1.01<br>0.02<br>613.81 | 0.3160<br>0.8858<br><.0001 | | | |
| | BASAL INSUBASAL INSUBASA | BASAL INSULIN + I BASAL INSULIN + I Pre Trial anti-D BASAL INSULIN + I BASAL INSULIN + I Pe 3 Tests of Fixe Num Den DF DF 1 442 1 442 | Pre Trial anti-Diabetic tre BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + Solution Pre Trial anti-Diabetic tre BASAL INSULIN + METFORMIN + BASAL INSULIN + METFORMIN + pe 3 Tests of Fixed Effects Num Den DF DF F Value 1 442 1.01 1 442 0.02 | Pre Trial anti-Diabetic treatment BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD Solution for Fixed Effe Pre Trial anti-Diabetic treatment BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD pe 3 Tests of Fixed Effects Num Den DF DF F Value Pr > F 1 442 1.01 0.3160 1 442 0.02 0.8858 | Planned Treatment for Period O1 (N) BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD Solution for Fixed Effects Planned Treatment for Period O1 (N) 1 2 BASAL INSULIN + METFORMIN + ONE OTHER OAD Planned Treatment for Period O1 (N) 1 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD Pe 3 Tests of Fixed Effects Num Den DF DF F Value Pr > F 1 442 1.01 0.3160 1 442 0.02 0.8858 | Pre Trial anti-Diabetic treatment for Period (01 (N)) Pr > t BASAL INSULIN + METFORMIN |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 2.5209<br>3.5430 | 442<br>442 | 1.84<br>2.54 | 0.0671<br>0.0115 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | 0.05<br>0.05 | -0.3267<br>2.0327 | 9.5823<br>15.9593 | | | |

### NN9068 NN9068-4166 Clinical Trial Report Statistical document CONFIDENTIAL Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGILU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 449

Number of Observations

Number of Observations Read 453 Number of Observations Used 449 Number of Observations Not Used 4

Covariance Parameter Estimates

Cov Parm Estimate
Residual 2310.04

Fit Statistics

-2 Res Log Likelihood 4739.1
AIC (Smaller is Better) 4741.1
AICC (Smaller is Better) 4741.1
BIC (Smaller is Better) 4745.2

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 44.9769 9.45 445 4.7616 Intercept -0.25 -1.2247 445 4.8065 trtpn trtpn PREAD BASAL INSULIN + METFORMIN -4.4637 4.5624 -0.98 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.7982 BASE 0.03834 445 -20.82

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 243 of 334 | |

Parameter Code=P9PGILU

The Mixed Procedure

#### Solution for Fixed Effects

| | | | SOTULTON I | or rixed Filect | .5 | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | <.0001<br>0.7990 | 0.05<br>0.05 |
| PREAD | BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | ۷ | 0.3284 | 0.05 |
| PREAD<br>BASE | BASAL INS | ULIN + I | 4ETFORMIN + | ONE OTHER OAD | | <.0001 | 0.05 |
| | | | Solution | for Fixed Effec | cts | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | 35.6189<br>-10.6710 | 54.3350<br>8.2215 |
| PREAD<br>PREAD | BASAL INS | | | ONE OTHER OAD | ۷ | -13.4301 | 4.5028 |
| BASE | DASAL INS | OTILI | TETFORMIN I | ONE OTHER OAD | | -0.8736 | -0.7229 |
| DASE | | | | | | 0.0700 | 0.7223 |
| | pe 3 Tests | of Fixe | ed Effects | | | 0.0700 | 0.7223 |
| | pe 3 Tests<br>Num<br>DF | of Fixe | | Pr > F | | | 0.7223 |
| Ту | Num | Den | | Pr > F<br>0.7990<br>0.3284<br><.0001 | | 313733 | 0.7223 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 7.8878<br>9.1125 | 2.7853<br>3.9142 | 445<br>445 | 2.83 | 0.0048<br>0.0204 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | 0.05<br>0.05 | 2.4138<br>1.4198 | 13.3617<br>16.8052 | | | |

### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGINC

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 452

Number of Observations

Number of Observations Read 453 Number of Observations Used 452 Number of Observations Not Used 1

Covariance Parameter Estimates

Cov Parm Estimate
Residual 2.9392

Fit Statistics

-2 Res Log Likelihood 1777.4
AICC (Smaller is Better) 1779.4
AICC (Smaller is Better) 1779.4
BIC (Smaller is Better) 1783.5

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 2.7808 0.2026 448 13.73 Intercept -0.4039 0.1715 -2.36 448 trtpn 0 trtpn PREAD BASAL INSULIN + METFORMIN -0.09210 0.1624 448 -0.57 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.7425 BASE 0.03900 448 -19.04

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 245 of 334 | |

Parameter Code=P9PGINC

The Mixed Procedure

#### Solution for Fixed Effects

| | | | Solution I | or Fixed Effect | S | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn | | | | | 1 2 | <.0001<br>0.0189 | 0.05<br>0.05 |
| trtpn<br>PREAD | BASAL INSU | | | | ۷ | 0.5709 | 0.05 |
| PREAD<br>BASE | BASAL INSU | JLIN + 1 | METFORMIN + | ONE OTHER OAD | | <.0001 | 0.05 |
| | | | Solution | for Fixed Effec | cts | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | 2.3826<br>-0.7410 | 3.1789<br>-0.06690 |
| PREAD | BASAL INSU | | | ONE OFFICE OAD | ۷ | -0.4112 | 0.2271 |
| PREAD<br>BASE | RASAL INSC | JLIN + I | METFORMIN + | ONE OTHER OAD | | -0.8192 | -0.6659 |
| Ту | pe 3 Tests | of Fix | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 448<br>448<br>448 | 5.55<br>0.32<br>362.57 | 0.0189<br>0.5709<br><.0001 | | | |

| trtpn | 1 | 448 | 5.55 | 0.0189 |
|-------|---|-----|--------|--------|
| PREAD | 1 | 448 | 0.32 | 0.5709 |
| BASE | 1 | 448 | 362.57 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.09892<br>0.1398 | 448<br>448 | -0.12<br>2.81 | 0.9061<br>0.0052 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | 0.05<br>0.05 | -0.2061<br>0.1175 | 0.1827<br>0.6670 | | | |

### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGINCB

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 449

Number of Observations

Number of Observations Read 453 Number of Observations Used 449 Number of Observations Not Used 4

Covariance Parameter Estimates

Cov Parm Estimate
Residual 6.6362

Fit Statistics

-2 Res Log Likelihood 2128.8 AIC (Smaller is Better) 2130.8 AICC (Smaller is Better) 2130.8 BIC (Smaller is Better) 2134.9

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 3.4477 0.3113 445 11.07 Intercept -0.7688 0.2578 -2.98 445 trtpn trtpn PREAD BASAL INSULIN + METFORMIN 0.2135 0.2436 445 0.88 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.7310 BASE 0.03980 445 -18.37

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 247 of 334 | |

Parameter Code=P9PGINCB

The Mixed Procedure

#### Solution for Fixed Effects

| | | | Solution f | or Fixed Effec | ts | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn | | | | | 1 2 | <.0001<br>0.0030 | 0.05<br>0.05 |
| trtpn<br>PREAD | BASAL INS | | | | _ | 0.3813 | 0.05 |
| PREAD<br>BASE | BASAL INS | JLIN + I | METFORMIN + | ONE OTHER OAD | | <.0001 | 0.05 |
| | | | Solution | for Fixed Effe | cts | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | 2.8359<br>-1.2754 | 4.0596<br>-0.2621 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | _ | -0.2653 | 0.6923 | |
| BASE | DADAE IND | OHIN , 1 | ALII ORUIIN | ONE OTHER OAD | | -0.8092 | -0.6528 |
| Ту | rpe 3 Tests | of Fixe | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 445<br>445<br>445 | 8.89<br>0.77<br>337.31 | 0.0030<br>0.3813<br><.0001 | | | |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.1493<br>0.2099 | 445<br>445 | -4.57<br>0.41 | <.0001<br>0.6832 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | | -0.9765<br>-0.3268 | -0.3896<br>0.4982 | | | |


Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGINCE

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 446

Number of Observations

Number of Observations Read 453 Number of Observations Used 446 Number of Observations Not Used 7

Covariance Parameter Estimates

Cov Parm Estimate
Residual 5.7871

Fit Statistics

-2 Res Log Likelihood 2054.2
AIC (Smaller is Better) 2056.2
AICC (Smaller is Better) 2056.3
BIC (Smaller is Better) 2060.3

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 2.5482 0.2400 442 10.62 Intercept -0.2424 0.2415 -1.00 442 trtpn 0 trtpn PREAD BASAL INSULIN + METFORMIN -0.03294 -0.14 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.8500 BASE 0.03431 442 -24.78

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 249 of 334 | |

Parameter Code=P9PGINCE

The Mixed Procedure

#### Solution for Fixed Effects

| Alpha |
|------------------|
| Aipiia |
| 0.05<br>0.05 |
| 0.05 |
| 0.05 |
| Upper |
| 3.0198<br>0.2322 |
| 0.4175 |
| -0.7826 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 0.2568<br>0.4992 | 0.1399<br>0.1966 | 442<br>442 | 1.84<br>2.54 | 0.0671<br>0.0115 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | | 0.01813<br>0.1128 | 0.5318<br>0.8856 | | | |

## NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 tatus: Final 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGINCL

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 449

Number of Observations

Number of Observations Read 453 Number of Observations Used 449 Number of Observations Not Used 4

Covariance Parameter Estimates

Cov Parm Estimate
Residual 7.1139

Fit Statistics

-2 Res Log Likelihood 2159.9
AIC (Smaller is Better) 2161.9
BIC (Smaller is Better) 2166.0

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 2.4959 9.45 0.2642 445 Intercept -0.06796 0.2667 -0.25 1 445 trtpn trtpn PREAD BASAL INSULIN + METFORMIN -0.98 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.7982 BASE 0.03834 445 -20.82

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 251 of 334 | |

Parameter Code=P9PGINCL

The Mixed Procedure

#### Solution for Fixed Effects

| | | | Solution I | or Fixed Effec | ts | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-D: | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn | | | | | 1 | <.0001<br>0.7990 | 0.05<br>0.05 |
| trtpn<br>PREAD | BASAL INS | | | | _ | 0.3284 | 0.05 |
| PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD BASE | | | | Planned Treatment for Period 01 (N) Pr > t Alph | 0.05 | | |
| | | | Solution | for Fixed Effe | cts | | |
| | | | | | Treatment for | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | | | 3.0153<br>0.4562 |
| PREAD<br>PREAD | BASAL INS | | | ONE OTHER OAD | | -0.7453 | 0.2499 |
| BASE | DASAL INS | OLIN I | ALIFORMIN ( | ONE OTHER OAL | , | -0.8736 | -0.7229 |
| Ту | pe 3 Tests | of Fixe | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 445<br>445<br>445 | 0.06<br>0.96<br>433.46 | 0.7990<br>0.3284<br><.0001 | | | |

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| trtpn | 1 | 445 | 0.06 | 0.7990 |
| PREAD | 1 | 445 | 0.96 | 0.3284 |
| BASE | 1 | 445 | 433.46 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.1546<br>0.2172 | 445<br>445 | 2.83 | 0.0048<br>0.0204 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | 0.05<br>0.05 | 0.1340<br>0.07879 | 0.7415<br>0.9326 | | | |

### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=P9PGIU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 452

Number of Observations

Number of Observations Read 453 Number of Observations Used 452 Number of Observations Not Used 1

Covariance Parameter Estimates

Cov Parm Estimate
Residual 954.43

Fit Statistics

-2 Res Log Likelihood 4373.9
AIC (Smaller is Better) 4375.9
AICC (Smaller is Better) 4376.0
BIC (Smaller is Better) 4380.1

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 50.1099 3.6507 448 13.73 Intercept -7.2791 3.0904 -2.36 448 trtpn 0 trtpn PREAD BASAL INSULIN + METFORMIN -1.6597 2.9264 448 -0.57 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.7425 BASE 0.03900 448 -19.04

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 253 of 334 | |

Parameter Code=P9PGIU

The Mixed Procedure

#### Solution for Fixed Effects

| Solution for Fixed Effects | | | | | | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn | | | | | 1 2 | <.0001<br>0.0189 | 0.05<br>0.05 |
| trtpn<br>PREAD | BASAL INSU | | | | ۷ | 0.5709 | 0.05 |
| PREAD<br>BASE | BASAL INSU | JLIN + 1 | METFORMIN + | ONE OTHER OAD | | <.0001 | 0.05 |
| | Solution for Fixed Effects | | | | | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | 42.9353<br>-13.3526 | 57.2845<br>-1.2055 |
| PREAD<br>PREAD | BASAL INSU | | | ONE OTHER OAD | _ | -7.4108 | 4.0914 |
| BASE | DASAL INSC | )TIN T I | MEIFORMIN T | ONE OTHER OAD | | -0.8192 | -0.6659 |
| Ту | Type 3 Tests of Fixed Effects | | | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 448<br>448<br>448 | 5.55<br>0.32<br>362.56 | 0.0189<br>0.5709<br><.0001 | | | |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 1.7825<br>2.5193 | 448<br>448 | -0.12<br>2.81 | 0.9061<br>0.0052 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | 0.05<br>0.05 | -3.7136<br>2.1174 | 3.2927<br>12.0198 | | | |

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

### 21: Fasting insulin after 26 weeks of treatment – supportive statistical analysis – full analysis set – appendix

Parameter Code=INS\_TO\_S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN

BASAL INSULIN + METFORMIN + ONE OTHER OAD

0112 0111211 0

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 452

max obs per subject

Number of Observations

Number of Observations Read 453 Number of Observations Used 452 Number of Observations Not Used 1

Covariance Parameter Estimates

Cov Parm Estimate

Residual 0.5659

Fit Statistics

-2 Res Log Likelihood 1037.6
AIC (Smaller is Better) 1039.6
AICC (Smaller is Better) 1039.6
BIC (Smaller is Better) 1043.7

Solution for Fixed Effects

Planned Treatment for

| Effect | Pre Trial anti-Diabetic treatment | for<br>Period<br>01 (N) | Estimate | Standard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn | | 1 2 | 1.4173<br>0.2632<br>0 | 0.1666<br>0.07509 | 448<br>448 | 8.50<br>3.50 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | -0.01274<br>0 | 0.07095 | 448 | -0.18 |
| base_log | | | 0.4230 | 0.04125 | 448 | 10.26 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 255 of 334 | |

Fasting insulin after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

| appendix | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Paramete | er Code=INS_TO_S | | | | | | | |
| The Mixe | ed Procedure | | | | | | | |
| | | Solution for | Fixed Effect | ts | | | | |
| Effect Interceptrtpn trtpn PREAD PREAD base loc | BASAL INSULIN +<br>BASAL INSULIN + | METFORMIN | | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t <.0001 0.0005 0.8576 <.0001 | Alpl<br>0.0<br>0.0 | 05<br>05<br>05 | |
| | , | Solution for | Fixed Effe | cts | | | | |
| Effect Interceptrtpn trtpn PREAD PREAD base_log | BASAL INSULIN +<br>BASAL INSULIN + | Diabetic treatm<br>METFORMIN | ent | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower 1.0897 0.1156 -0.1522 0.3419 | 1.7 | pper<br>7448<br>1107<br>1267<br>5041 | |
| | Type 3 Tests of Fi | xed Effects | | | | | | |
| Effect<br>trtpn<br>PREAD | Num Den<br>DF DF<br>1 448<br>1 448 | 12.28 0 | r > F<br>.0005<br>.8576 | | | | | |
| base_log | | | .0001 | | | | | |
| | | Least | Squares Mean | ns Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF t | Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 3.2281<br>2.9649 | 0.04337<br>0.06126 | 448<br>448 | 74.42<br>48.40 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least Sq | uares Means | Estimates | | | | |
| Effect | Label | Lower | Upper E | xponentiated | Exponen | tiated<br>Lower | Exponentia<br>Up | ted |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | 3.1428<br>2.8445 | 3.3133<br>3.0853 | 25.2310<br>19.3931 | | 3.1694<br>7.1935 | 27.4<br>21.8 | |
| | | Least | Squares Mean | ns Estimate | | | | |

| Effect | Label | | Margins | Estimate | Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | 0.2632 | 0.07509 | 448 | 3.50 | 0.0005 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 256 of 334 | |

Fasting insulin after 26 weeks of treatment – supportive statistical analysis – full analysis set – appendix

Parameter Code=INS\_TO\_S

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 0.1156 0.4107 1.3010

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 1.1225 1.5079

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 257 of 334 | |

### 22: Fasting C-peptide after 26 weeks of treatment – supportive statistical analysis – full analysis set – appendix

Parameter Code=C74736S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 449

Number of Observations

Number of Observations Read 453 Number of Observations Used 449 Number of Observations Not Used 4

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.3774

Fit Statistics

-2 Res Log Likelihood 849.9
AIC (Smaller is Better) 851.9
AICC (Smaller is Better) 851.9
BIC (Smaller is Better) 856.0

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept -0.9362 0.06948 -13.47 trtpn 0.2201 0.06149 3.58 trtpn 2 Ω BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD 0.04696 0.05821 PREAD 445 0.81 PREAD base\_log 0.7072 0.04482 445 15.78


Fasting C-peptide after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

| Paramete | er Code=C7 | 4736S | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| The Mixe | d Procedu | re | | | | | | | |
| | | | Solution fo | r Fixed Effect | S | | | | |
| Effect | Pre Tr | ial anti-D | iabetic trea | tment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alp | ha | |
| Intercep | t | | | | | <.000 | 1 0. | 05 | |
| trtpn<br>trtpn | | | | | 1 2 | 0.000 | 4 0. | 05 | |
| PREAD<br>PREAD | BASAL<br>BASAL | INSULIN + N<br>INSULIN + N | | ONE OTHER OAD | | 0.420 | 3 0. | 05 | |
| base_log | | | | | | <.000 | 1 0. | 05 | |
| | | | Solution f | or Fixed Effec | ets | | | | |
| | | ial anti-Di | iabetic trea | tment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lowe | | pper | |
| Intercep<br>trtpn | t | | | | 1 | -1.072<br>0.0992 | | 7997<br>3410 | |
| trtpn PREAD BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD base log | | 2 | -0.0674 | 5 0. | 1614 | | | | |
| | | | 0.619 | 1 0. | 7953 | | | | |
| _ | | | | | | | | | |
| | Туре 3 Те | sts of Fixe | ed Effects | | | | | | |
| Effect | Num<br>DF | | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>base_log | 1<br>1<br>1 | 445 | 12.82<br>0.65<br>249.02 | 0.0004<br>0.4203<br><.0001 | | | | | |
| | | | Leas | t Squares Mear | ns Estimates | | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| | LSMeans,<br>LSMeans, | | WORK.ADATA<br>WORK.ADATA | | 0.03553<br>0.05017 | 445<br>445 | -37.88<br>-31.21 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least | Squares Means | Estimates | | | | |
| Effect | Label | | Lower | Upper Ex | ponentiated | | entiated<br>Lower | | ted<br>per |
| | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | -1.4158<br>-1.6647 | -1.2761<br>-1.4675 | 0.2603<br>0.2089 | | 0.2427<br>0.1892 | | 791<br>305 |
| | | | Leas | t Squares Mear | ns Estimate | | | | |
| D. 6 | T - 1 1 | | | Manadaa | Datimata | Standar | | + 17-1 D | > 151 |

| Effect | Label | | Margins | Estimate | Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | 0.2201 | 0.06149 | 445 | 3.58 | 0.0004 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 259 of 334 | |

Fasting C-peptide after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

Parameter Code=C74736S

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 0.09929 0.3410 1.2463

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 1.1044 1.4064

### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

Fasting C-peptide after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

Parameter Code=CPEPTI U

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 449

Number of Observations

Number of Observations Read 453
Number of Observations Used 449
Number of Observations Not Used 4

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.3774

Fit Statistics

-2 Res Log Likelihood 849.9
AIC (Smaller is Better) 851.9
BIC (Smaller is Better) 856.0

Solution for Fixed Effects

Planned Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value -10.42 -0.6126 0.05878 445 Intercept 3.58 0.2201 0.06149 445 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.04696 0.05821 0.81 PREAD 0.7072 base log 0.04482 445 15.78

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 261 of 334 | |

Fasting C-peptide after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

| Paramete | r Code=CPEPTI_U | | | | | |
|---|---|---|---|---|---|---|
| The Mixe | d Procedure | | | | | |
| | Solution for Fixed Effects | | | | | |
| Effect | Pre Trial anti-D | iabetic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha | |
| Intercep<br>trtpn | t | | 1 | <.0001<br>0.0004 | 0.05<br>0.05 | |
| trtpn<br>PREAD | trtpn | | | 0.4203 | 0.05 | |
| PREAD<br>base log | BASAL INSULIN + 1 | METFORMIN + ONE OTHER O | AD | <.0001 | 0.05 | |
| base_rog | | Solution for Fixed Ef | foots | ₹.000± | 0.03 | |
| | | Solution for fixed El | | | | |
| Effect | Pre Trial anti-D | iabatic treatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper | |
| | | rapetic treatment | 01 (11) | | | |
| Intercep<br>trtpn<br>trtpn | t | | 1 2 | -0.7282<br>0.09929 | -0.4971<br>0.3410 | |
| PREAD<br>PREAD | BASAL INSULIN + 1<br>BASAL INSULIN + 1 | METFORMIN<br>METFORMIN + ONE OTHER O | AD | -0.06745 | 0.1614 | |
| base_log | | | | 0.6191 | 0.7953 | |
| | Type 3 Tests of Fix | ed Effects | | | | |
| Effect | Num Den<br>DF DF | F Value Pr > F | | | | |
| trtpn<br>PREAD<br>base_log | 1 445<br>1 445<br>1 445 | 12.82 0.0004<br>0.65 0.4203<br>249.02 <.0001 | | | | |
| | | Least Squares M | eans Estimates | | | |
| | | | Standard | | | |
| Effect | Label | Margins Estimat | e Error | DF t | Value Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2 -0.240<br>WORK.ADATA2 -0.460 | | | -6.77 <.0001<br>-9.18 <.0001 | 0.05<br>0.05 |
| | | Least Squares Mea | ns Estimates | | | |
| Effect | Label | Lower Upper | Exponentiated | Exponent | | ated<br>oper |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | -0.3105 -0.1709<br>-0.5595 -0.3622 | 0.7861<br>0.6308 | | | 3429<br>5961 |

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | 0.2201 | 0.06149 | 445 | 3.58 | 0.0004 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 262 of 334 | |

Fasting C-peptide after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

Parameter Code=CPEPTI\_U

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 0.09929 0.3410 1.2463

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 1.1044 Exponentiated 1.4064

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

### 23: Fasting glucagon after 26 weeks of treatment – supportive statistical analysis – full analysis set - appendix

Parameter Code=C74859P

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 451

Number of Observations

Number of Observations Read 453 Number of Observations Used 451 Number of Observations Not Used 2

Covariance Parameter Estimates

Cov Parm Estimate Residual 0.2747

Fit Statistics

-2 Res Log Likelihood 711.8
AIC (Smaller is Better) 713.8
AICC (Smaller is Better) 713.8
BIC (Smaller is Better) 717.9

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept 2.5453 0.1201 447 trtpn 1 -0.03858 0.05240 -0.74 trtpn 2 Λ BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD -0.06470 PREAD 0.04944 447 -1.31 PREAD 0.2213 0.03481 6.36 base\_log 447

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 264 of 334 | |

Fasting glucagon after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

| - append | 11X | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Paramete | er Code=C74859P | | | | | | | |
| The Mixe | ed Procedure | | | | | | | |
| | | Solution for | Fixed Effect | S | | | | |
| Effect | Pre Trial ant | i-Diabetic treat | ment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alp | ha | |
| Intercep<br>trtpn | ot | | | 1 | <.000<br>0.461 | | | |
| trtpn<br>PREAD<br>PREAD | BASAL INSULIN | | NE OTHER OAR | 2 | 0.191 | 3 0. | 05 | |
| base_log | BASAL INSULIN + METFORMIN + ONE OTHER OAD og | | | <.000 | 1 0. | 05 | | |
| | | Solution fo | r Fixed Effec | :ts | | | | |
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial ant | i-Diabetic treat | ment | 01 (N) | Lowe | r U | pper | |
| Intercep<br>trtpn | ot | | | 1 2 | 2.309 | | 7814<br>6440 | |
| trtpn PREAD BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 2 | -0.161 | 9 0.0 | 3246 | | | |
| base_log | | THEIT ORTHIN TO | NE OTHER OAD | | 0.152 | 9 0. | 2898 | |
| | Type 3 Tests of | Fixed Effects | | | | | | |
| Effect | Num De<br>DF D | | Pr > F | | | | | |
| trtpn<br>PREAD<br>base_log | 1 44<br>1 44<br>1 44 | 7 1.71 | 0.4619<br>0.1913<br><.0001 | | | | | |
| | | Least | Squares Mean | s Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLi<br>LSMeans, IDeg | ra WORK.ADATA2<br>WORK.ADATA2 | | 0.03021<br>0.04280 | 447<br>447 | 105.07<br>75.06 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least S | quares Means | Estimates | | | | |
| Effect | Label | Lower | Upper Ex | ponentiated | | entiated<br>Lower | Exponentia<br>Up | ted |
| trtpn<br>trtpn | LSMeans, IDegLi<br>LSMeans, IDeg | 3.1149<br>3.1287 | 3.2336<br>3.2970 | 23.9091<br>24.8495 | | 22.5308<br>22.8447 | 25.3<br>27.0 | |
| | | Least | Squares Mean | ıs Estimate | | | | |
| | | | | | Standar | d | | |

| Effect | Label | | Margins | Estimate | Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | -0.03858 | 0.05240 | 447 | -0.74 | 0.4619 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 265 of 334 | |

Fasting glucagon after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

Parameter Code=C74859P

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.1416 0.06440 0.9622

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.8680 Exponentiated 1.0665

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 266 of 334 | |

#### 24: HOMA-B after 26 weeks of treatment – supportive statistical analysis – full analysis set - appendix

Parameter Code=HOMA BCS

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 aval\_log Diagonal Dependent Variable Covariance Structure Estimation Method Residual Variance Method Profile Fixed Effects SE Method Model-Based Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

1 2 2 trtpn

BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters Columns in X Columns in Z 0 Subjects Max Obs per Subject 452

Number of Observations

Number of Observations Read Number of Observations Used 452 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 0.5070

Fit Statistics

-2 Res Log Likelihood 988.5 AIC (Smaller is Better) AICC (Smaller is Better) BIC (Smaller is Better) 990.5 994.6

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 1.8932 0.1322 448 14.32 Intercept 1 0.3901 0.07103 448 5.49 trtpn trtpn PREAD BASAL INSULIN + METFORMIN -0.01262 0.06714 -0.19 PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD 0.3927 0.03605 448 10.89 base\_log

### NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 1.0 Status: Final 

Planned

HOMA-B after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix Parameter Code=HOMA\_BCS

The Mixed Procedure

#### Solution for Fixed Effects

| | | | | | Treatment<br>for<br>Period | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Pre Tr | ial anti-D | iabetic treat | ment | 01 (N) | Pr > t | Alp | ha | |
| Interce<br>trtpn<br>trtpn | pt | | | | 1 2 | <.0001<br><.0001 | | 05<br>05 | |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | 2 | 0.8510 | 0. | 05 | |
| base_lo | | | | | | <.0001 | 0. | 05 | |
| Solution for Fixed Effects | | | | | | | | | |
| Effect | Pre Tr | ial anti-D | iabetic treat: | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | U | Jpper | | |
| Intercept | | | | | | 1.6334 | | 1530 | |
| trtpn<br>trtpn | 1 - | | | | 1 2 | 0.2505 | | 5297 | |
| PREAD<br>PREAD | | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | -0.1446 | 0. | 0.1193 | |
| base_lo | | | | | | 0.3218 | 0. | 4635 | |
| Type 3 Tests of Fixed Effects | | | | | | | | | |
| Effect | Num<br>DF | | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>base_lo | 1<br>1<br>1 | 448 | 0.04 | <.0001<br>0.8510<br><.0001 | | | | | |
| Least Squares Means Estimates | | | | | | | | | |
| | | | | | Standard | | | | |
| Effect | | | Margins | Estimate | | | | Pr > t | _ |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.04105<br>0.05796 | 448<br>448 | 85.64<br>53.92 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least S | quares Means | Estimates | | | | |
| Effect | Label | Label Lower | | | xponentiated | | | Exponentiated<br>Upper | |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | | 3.4348<br>3.0114 | 3.5961<br>3.2393 | 33.6300<br>22.7680 | | | 36.4553<br>25.5149 | |
| Least Squares Means Estimate | | | | | | | | | |
| nee : | T - 1 3 | | | 26 | B-+ ' | Standard | | + 17-3 | See S. 11.1 |
| Effect | | | | - | Estimate | Error | | t Value I | |
| trtpn | rreatment | ratio, ID | egLira - IDeg | WORK.ADATA2 | 2 0.3901 | 0.07103 | 448 | 5.49 | <.0001 |
| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 268 of 334 | |

HOMA-B after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix Parameter Code=HOMA\_BCS

The Mixed Procedure

Least Squares Means Estimate

Effect Label Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 0.2505 0.5297 1.4771

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 1.2846 1.6984

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

## 25: HDL cholesterol after 26 weeks of treatment – supportive statistical analysis – full analysis set – appendix

Parameter Code=C105587S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.02369

Fit Statistics

-2 Res Log Likelihood -387.4
AIC (Smaller is Better) -385.4
AICC (Smaller is Better) -385.3
BIC (Smaller is Better) -381.2

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept 0.05515 0.01465 449 trtpn 1 -0.02691 0.01535 trtpn 2 Λ BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD -0.01619 PREAD 0.01449 449 -1.12 PREAD 0.7660 0.02813 27.23 base\_log 449

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 270 of 334 | |

HDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set appendix

| appendix | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Paramete | er Code=C1 | 05587S | | | | | | | |
| The Mixe | ed Procedu | re | | | | | | | |
| | | | Solution for | Fixed Effec | ts | | | | |
| Effect. | Pre Tr | ial anti-D | iabetic treat | ment. | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alp | ha | |
| | | iai anci b | idbeere erede | | 01 (14) | | _ | | |
| Intercep<br>trtpn<br>trtpn | )t | | | | 1<br>2 | 0.000 | | 05<br>05 | |
| PREAD<br>PREAD | | INSULIN + : | METFORMIN<br>METFORMIN + O | NE OTHER OAD | ) | 0.264 | 3 0. | 05 | |
| base_log | | INCOLIN | | NE OTHER ONE | | <.000 | 1 0. | 05 | |
| | | | Solution fo | r Fixed Effe | cts | | | | |
| | | ial anti-D | iabetic treat | ment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lowe<br>0.0263 | | pper<br>8395 | |
| Intercep<br>trtpn | , , | | | | 1 | -0.0570 | | | |
| trtpn<br>PREAD BASAL INSULIN + METFORMIN | | | 2 | -0.0446 | 6 0.0 | 1228 | | | |
| PREAD base_log | | INSULIN + 1 | METFORMIN + O | NE OTHER OAD | ) | 0.710 | 7 0. | 8213 | |
| | Type 3 Te | sts of Fix | ed Effects | | | | | | |
| Effect | Num<br>DF | | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>base_log | 1<br>1<br>1 | 449 | 1.25 | 0.0802<br>0.2643<br><.0001 | | | | | |
| | | | Least | Squares Mea | ns Estimates | | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.008859<br>0.01253 | 449<br>449 | 11.10<br>10.00 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least S | quares Means | Estimates | | | | |
| Effect | Label | | Lower | Upper E | xponentiated | | entiated<br>Lower | Exponentia<br>Ug | ated<br>oper |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | 0.08095<br>0.1006 | 0.1158<br>0.1499 | 1.1034<br>1.1335 | | 1.0843<br>1.1059 | | 1227<br>1617 |
| | | | Least | Squares Mea | ns Estimate | | | | |
| Effect | Label | | | Margins | Estimate | Standar<br>Erro | | t Value Pr | c > t |

trtpn Treatment ratio, IDegLira - IDeg WORK.ADATA2 -0.02691 0.01535 449 -1.75 0.0802

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 271 of 334 | |

 ${\tt HDL}\ cholesterol\ after\ 26\ weeks\ of\ treatment\ -\ supportive\ statistical\ analysis\ -\ full\ analysis\ set\ -\ appendix$ 

Parameter Code=C105587S

The Mixed Procedure

Least Squares Means Estimate

Effect Label Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.05708 0.003252 0.9734

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.9445 Exponentiated 1.0033


 $\mathtt{HDL}$  cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set -  $\mathtt{appendix}$ 

Parameter Code=HDL SU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453
Number of Observations Used 453
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.02369

Fit Statistics

-2 Res Log Likelihood -387.4
AIC (Smaller is Better) -385.4
AICC (Smaller is Better) -385.3
BIC (Smaller is Better) -381.2

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 0.9101 0.1065 449 8.55 Intercept 0.01535 1 -0.02691 -1.75 449 trtpn trtpn PREAD BASAL INSULIN + METFORMIN -0.01619 0.01449 449 -1.12 BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.7660 base log 0.02813 449 27.23

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 273 of 334 | |

HDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

Parameter Code=HDL\_SU

| | Paramete: | r Code=HD | L_SU | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | The Mixed | d Procedu | re | | | | | | |
| | | | | Solution fo | or Fixed Effec | ts | | | |
| | Effect | Pre Tr | ial anti-D | iabetic trea | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpi | ha |
| | Intercept | | 141 41101 2 | 1420010 010 | 200110 | 01 (11) | <.000 | _ | |
| | trtpn<br>trtpn | _ | | | | 1 2 | 0.0802 | | |
| | PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | | 0.2643 | 3 0. | 05 |
| | base_log | | INSULIN + I | METFORMIN + | ONE OTHER OAD | | <.0000 | 1 0. | 05 |
| | | | | Solution | for Fixed Effe | cts | | | |
| | | | | | | Planned<br>Treatment<br>for<br>Period | | | |
| | Effect | Pre Tr | ial anti-D | iabetic trea | atment | 01 (N) | Lowe | r Uj | pper |
| Intercept trtpn trtpn | | | | 1 2 | 0.7008 | 8 1.1 | 1194<br>3252 | | |
| | PREAD<br>PREAD | | INSULIN + 1 | | ONE OTHER OAD | _ | -0.0446 | 0.0 | 1228 |
| | base_log | | 111002111 | | one officer one | | 0.710 | 7 0. | 8213 |
| | ŗ | Type 3 Te | sts of Fixe | ed Effects | | | | | |
| | Effect | Num<br>DF | | F Value | Pr > F | | | | |
| | trtpn<br>PREAD<br>base_log | 1<br>1<br>1 | 449 | 1.25 | | | | | |
| | | | | Leas | st Squares Mea | ns Estimates | 5 | | |
| | Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
| | | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | | | 0.008859<br>0.01253 | | 423.51<br>301.57 | <.0001<br><.0001 |
| | | | | Least | Squares Means | Estimates | | | |
| | Effort | Tabal | | Lover | Hnnor E | vnonontiatos | | entiated | Exponentiat |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 3.7519<br>3.7788 | | 449<br>449 | 423.51<br>301.57 | <.0001<br><.0001 | 0.05<br>0.05 |
| Least Squares Means Estimates | | | | | | | | |
| Effect | Label | Lower | Upper | Exponentiated | Expor | nentiated<br>Lower | Exponentia<br>Up | ted<br>per |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | 3.7345<br>3.7542 | 3.7693<br>3.8034 | 42.6008<br>43.7629 | | 41.8655<br>42.6983 | 43.3<br>44.8 | |
| | Least Squares Means Estimate | | | | | | | |

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | -0.02691 | 0.01535 | 449 | -1.75 | 0.0802 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 274 of 334 | |

 ${\tt HDL}\ cholesterol\ after\ 26\ weeks\ of\ treatment\ -\ supportive\ statistical\ analysis\ -\ full\ analysis\ set\ -\ appendix$ 

Parameter Code=HDL\_SU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.05708 0.003252 0.9734

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.9445 Exponentiated 1.0033

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

## 26: LDL cholesterol after 26 weeks of treatment – supportive statistical analysis – full analysis set – appendix

Parameter Code=C105588S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 443

Number of Observations

Number of Observations Read 453 Number of Observations Used 443 Number of Observations Not Used 10

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.09192

Fit Statistics

-2 Res Log Likelihood 217.4
AIC (Smaller is Better) 219.4
AICC (Smaller is Better) 219.4
BIC (Smaller is Better) 223.4

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept 0.2451 0.04507 439 5.44 trtpn 1 -0.05261 0.03067 trtpn 2 0 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD 0.01684 PREAD 0.02889 439 0.58 PREAD 0.6372 0.04110 base\_log 439 15.50

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 276 of 334 | |

LDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set appendix

| Paramete | er Code=C105588S | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| The Mixe | ed Procedure | | | | | | | |
| | | Solution for Fixe | ed Effect | S | | | | |
| Effect | Pre Trial anti- | Diabetic treatment | | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | ıa | |
| Intercep | ot | | | | <.0001 | 0.0 | | |
| trtpn<br>trtpn | | | | 1 2 | 0.0869 | 0.0 | | |
| PREAD<br>PREAD | BASAL INSULIN +<br>BASAL INSULIN + | METFORMIN + ONE OT | THER OAD | | 0.5603 | 0.0 | | |
| base_log | | | | | <.0001 | 0.0 | )5 | |
| | | Solution for Fix | ked Effec | ts | | | | |
| Effect | Pre Trial anti- | Diabetic treatment | | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Up | pper | |
| Intercep | ot | | | | 0.1565 | 0.3 | 3337 | |
| trtpn<br>trtpn | | | | 1 2 | -0.1129 | 0.007 | 7660 | |
| PREAD BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | -0.03995 | 0.07 | 7363 | | | |
| base_log | | | | | 0.5564 | 0.7 | 179 | |
| | Type 3 Tests of Fi | ked Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value Pr > | F | | | | | |
| trtpn<br>PREAD<br>base_log | 1 439<br>1 439<br>1 439 | 2.94 0.086<br>0.34 0.560<br>240.29 <.000 | 03 | | | | | |
| | | Least Squa | ares Mean | s Estimates | | | | |
| Effect | Label | Margins Es | stimate | Standard<br>Error | DF t | . Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | | 0.7561<br>0.8087 | 0.01760<br>0.02510 | 439<br>439 | 42.97<br>32.21 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least Square | es Means | Estimates | | | | |
| Effect | Label | Lower Up | pper Ex | ponentiated | | tiated<br>Lower | Exponentia<br>Up | ted<br>per |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | | 7906<br>3580 | 2.1299<br>2.2449 | | 2.0575<br>2.1369 | 2.2 | |
| | | Least Squa | ares Mean | s Estimate | | | | |
| Effect | Label | Mar | rgins | Estimate | Standard<br>Error | DF | t Value Pr | > t |

trtpn Treatment ratio, IDegLira - IDeg WORK.ADATA2 -0.05261 0.03067 439 -1.72 0.0869

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 277 of 334 | |

 ${\tt LDL}\ cholesterol\ after\ 26\ weeks\ of\ treatment\ -\ supportive\ statistical\ analysis\ -\ full\ analysis\ set\ -\ appendix$ 

Parameter Code=C105588S

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.1129 0.007660 0.9487

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.8933 1.0077


 ${ t LDL}$  cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set -  ${ t appendix}$ 

Parameter Code=LDL SU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 443

Number of Observations

Number of Observations Read 453
Number of Observations Used 443
Number of Observations Not Used 10

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.09192

Fit Statistics

-2 Res Log Likelihood 217.4
AICC (Smaller is Better) 219.4
AICC (Smaller is Better) 219.4
BIC (Smaller is Better) 223.4

Solution for Fixed Effects

Planned

Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 1.5708 0.1870 439 8.40 Intercept -0.05261 0.03067 -1.72 439 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.01684 0.02889 439 0.58 PREAD 0.6372 base log 0.04110 439 15.50

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 279 of 334 | |

LDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

Parameter Code=LDL\_SU

The Mixed Procedure

| | | | Solution for | r Fixed Effe | cts | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Pre Tr | ial anti-D | iabetic trea | tment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpl | ha |
| Interceptrtpn | t | | | | 1 | <.000<br>0.086 | | |
| trtpn<br>PREAD | | INSULIN + I | | ONE OFFIER OF | 2 | 0.560 | 3 0.0 | 05 |
| PREAD<br>base_log | BASAL | INSULIN + I | METFORMIN + ( | ONE OTHER OA | D | <.000 | 1 0.0 | 05 |
| | | | Solution fo | or Fixed Eff | ects | | | |
| Effect | Pre Tr | ial anti-D | iabetic trea | tment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lowe | r U] | pper |
| Intercept<br>trtpn<br>trtpn | | | | | 1<br>2 | 1.203<br>-0.112 | 9 0.00 | |
| PREAD<br>PREAD<br>base_log | | INSULIN + I | METFORMIN<br>METFORMIN + ( | ONE OTHER OA | D | -0.0399 | | 7363<br>7179 |
| | Type 3 Te | sts of Fixe | ed Effects | | | | | |
| Effect | Num<br>DF | | F Value | Pr > F | | | | |
| trtpn<br>PREAD<br>base_log | 1<br>1<br>1 | 439 | | 0.0869<br>0.5603<br><.0001 | | | | |
| | | | Least | t Squares Me | ans Estimates | 3 | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADATA | 2 4.4096<br>2 4.4622 | | 439<br>439 | | <.0001<br><.0001 |
| | | | Least : | Squares Mean | s Estimates | | | |
| Effect | Label | | Lower | Upper | Exponentiated | | entiated<br>Lower | Exponentia<br>Un |

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | LSMeans, I | _ | 4.3750<br>4.4129 | 4.4442<br>4.5115 | 82.2346<br>86.6770 | 79.4392<br>82.5043 | 85.1283<br>91.0608 |

Alpha 0.05 0.05

### Least Squares Means Estimate

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | -0.05261 | 0.03067 | 439 | -1.72 | 0.0869 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 280 of 334 | |

 ${\tt LDL}\ cholesterol\ after\ 26\ weeks\ of\ treatment\ -\ supportive\ statistical\ analysis\ -\ full\ analysis\ set\ -\ appendix$ 

Parameter Code=LDL\_SU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.1129 0.007660 0.9487

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.8933 1.0077

22 January 2020 | Novo Nordisk NN9068 Date: NN9068-4166 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

## 27: VLDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set -

Parameter Code=C105589S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable aval\_log Covariance Structure
Estimation Method
Residual Variance Method
Fixed Effects SE Method Diagonal REMI Profile Model-Based Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn

PREAD 2 BASAL INSULIN + METFORMIN

BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters Columns in X Columns in Z 6 Ω Subjects Max Obs per Subject 453

Number of Observations

Number of Observations Read Number of Observations Used 453 453 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 0.1867

Fit Statistics

-2 Res Log Likelihood AIC (Smaller is Better) 543.2 AICC (Smaller is Better) 543.2 BIC (Smaller is Better)

Solution for Fixed Effects

Planned Treatment for

| Effect | Pre Trial anti-Diabetic treatment | Period<br>01 (N) | Estimate | Standard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn | | 1 2 | -0.1883<br>-0.01158 | 0.04107<br>0.04308 | 449<br>449 | -4.58<br>-0.27 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 0.07290 | 0.04067 | 449 | 1.79 |
| base_log | | | 0.6095 | 0.03509 | 449 | 17.37 |

### NN9068 Date: 22 January 2020 | Novo Nordisk NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

VLDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

Effect Label

| Paramete | r Code=C1 | 05589S | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| The Mixe | d Procedu: | re | | | | | | | |
| | | | Solution fo | r Fixed Effe | cts | | | | |
| Effect | Pre Tr | ial anti-Di | labetic trea | tment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | : Alpl | na | |
| Intercep | t | | | | | <.000 | 1 0.0 | 05 | |
| trtpn<br>trtpn | | | | | 1 2 | 0.788 | 1 0.0 | 05 | |
| PREAD<br>PREAD | | INSULIN + N | | ONE OTHER OA | | 0.073 | 7 0.0 | 05 | |
| base_log | | INSOLIN , I | IDIT ORTIN | ONE OTHER OA | D | <.000 | 1 0.0 | 05 | |
| | | | Solution f | or Fixed Eff | ects | | | | |
| Effect | Pre Tr | ial anti-Di | labetic trea | tment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lowe | er Uj | pper | |
| Intercept trtpn | | | | | 1 | -0.269<br>-0.0962 | | 1076<br>7308 | |
| trtpn<br>PREAD BASAL INSULIN + METFORMIN | | | | 2 | -0.0070 | | 1528 | | |
| PREAD<br>base_log | BASAL : | | | ONE OTHER OA | D | 0.540 | | 6784 | |
| | Type 3 Te: | sts of Fixe | ed Effects | | | | | | |
| | Num | | | | | | | | |
| Effect | DF | DF | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>base_log | 1<br>1<br>1 | | 0.07<br>3.21<br>301.77 | 0.7881<br>0.0737<br><.0001 | | | | | |
| | | | Leas | t Squares Me | ans Estimates | | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADATA<br>WORK.ADATA | | | 449<br>449 | -11.76<br>-7.98 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least | Squares Mean | s Estimates | | | | |
| Effect | Label | | Lower | Upper | Exponentiated | | entiated<br>Lower | | ted |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | -0.3413<br>-0.3500 | -0.2436<br>-0.2117 | 0.7464<br>0.7551 | | 0.7108<br>0.7047 | | 838<br>092 |

Least Squares Means Estimate

trtpn Treatment ratio, IDegLira - IDeg WORK.ADATA2 -0.01158 0.04308 449 -0.27 0.7881

Margins Estimate Error

Standard

DF t Value Pr > |t|

| NN9068 | | Date: | 22 January 2020 Novo Nordis | sk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 283 of 334 | |

 $\hbox{\tt VLDL cholesterol after 26 weeks of treatment-supportive statistical analysis-full analysis set-appendix}$ 

Parameter Code=C105589S

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.09625 0.07308 0.9885

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.9082 1.0758


 ${ t VLDL}$  cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

Parameter Code=VLDL SU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453
Number of Observations Used 453
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.1867

Fit Statistics

-2 Res Log Likelihood 541.2
AIC (Smaller is Better) 543.2
AICC (Smaller is Better) 543.2
BIC (Smaller is Better) 547.3

Solution for Fixed Effects

Planned

Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 1.2385 0.1275 449 9.71 Intercept -0.01158 0.04308 1 -0.27 449 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.07290 0.04067 449 1.79 PREAD 0.6095 base log 0.03509 449 17.37

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 285 of 334 | |

VLDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

| Paramete | r Code=VLDL_SU | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| The Mixe | d Procedure | | | | | | | |
| | | Solution for | Fixed Effe | cts | | | | |
| Effect | Pre Trial anti-I | Diabetic treatm | nent | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alp | na | |
| Intercep | t | | | | <.000 | | | |
| trtpn<br>trtpn | | | | 1<br>2 | 0.788 | | | |
| PREAD<br>PREAD | | | | D | 0.073 | 7 0.0 | 05 | |
| base_log | base_log | | | | <.000 | 1 0.0 | 05 | |
| Solution for Fixed Effects | | | | | | | | |
| Effect | Pre Trial anti-I | Diabetic treatm | nent | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lowe | r U] | pper | |
| Intercep | 1 | 0.987 | | 4890 | | | | |
| trtpn<br>trtpn | 2 | -0.0962 | | 7308 | | | | |
| PREAD<br>PREAD | BASAL INSULIN +<br>BASAL INSULIN + | | NE OTHER OA | D | -0.0070 | | 1528 | |
| base_log | | | | | 0.540 | 5 0.1 | 6784 | |
| | Type 3 Tests of Fix | ked Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value F | ?r > F | | | | | |
| trtpn<br>PREAD<br>base_log | 1 449<br>1 449<br>1 449 | 3.21 | 0.7881<br>0.0737<br><.0001 | | | | | |
| | | Loast | Squares Mo | ans Estimates | | | | |
| | | Least | oquares me | Standard | | | | |
| Effect | Label | Margins | Estimate | | DF | t Value | Pr > t | Alpha |
| | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.02487<br>0.03517 | 449<br>449 | 135.15<br>95.89 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least So | quares Mean | s Estimates | | | | |
| Effect | Label | Lower | Upper | Exponentiated | | entiated<br>Lower | | ted<br>per |
| | LSMeans, IDegLira<br>LSMeans, IDeg | 3.3122<br>3.3035 | 3.4099<br>3.4418 | 28.8201<br>29.1559 | | 27.4455<br>27.2086 | 30.2<br>31.2 | |
| | | Least | Squares Me | ans Estimate | | | | |

### Least Squares Means Estimate

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | -0.01158 | 0.04308 | 449 | -0.27 | 0.7881 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 286 of 334 | |

 $\hbox{\tt VLDL cholesterol after 26 weeks of treatment-supportive statistical analysis-full analysis set-appendix}$ 

Parameter Code=VLDL\_SU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.09625 0.07308 0.9885

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.9082 Exponentiated 1.00758

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

## 28: Triglycerides after 26 weeks of treatment – supportive statistical analysis – full analysis set – appendix

Parameter Code=C64812S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.2371

Fit Statistics

-2 Res Log Likelihood 648.7 AIC (Smaller is Better) 650.7 AICC (Smaller is Better) 650.7 BIC (Smaller is Better) 654.8

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept 0.1298 0.05020 449 2.59 trtpn 1 -0.01325 0.04855 -0.27 trtpn 2 Ω BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD 0.06990 PREAD 0.04585 449 1.52 PREAD 0.6028 0.03500 base\_log 449 17.22

### NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 288 of 334 Statistical document Page:

Triglycerides after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

| Paramete | r Code=C648 | 12S | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| The Mixe | d Procedure | | | | | | | | | |
| | | | Solution fo | or Fixed | Effect | s | | | | |
| Effect | Pre Tria | l anti-D: | iabetic trea | atment | | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpl | na | |
| Intercep<br>trtpn<br>trtpn<br>PREAD<br>PREAD<br>base log | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAL | | | | | 1 2 | 0.0100<br>0.7851<br>0.1281 | L 0.0 | 05 | |
| | | | Solution : | for Fixe | d Effec | ts | | | | |
| Effect Interceptrtpntrtpn | Pre Tria | l anti-D: | | | | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower<br>0.03115<br>-0.1087 | 5 0.2 | pper<br>2285<br>3216 | |
| PREAD<br>PREAD<br>base_log | BASAL IN | | METFORMIN<br>METFORMIN + | ONE OTH | ER OAD | | 0.5340 | | 1600<br>6716 | |
| | Type 3 Test | s of Fixe | ed Effects | | | | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | | | | |
| trtpn<br>PREAD<br>base_log | 1<br>1<br>1 | 449<br>449<br>449 | 0.07<br>2.32<br>296.62 | 0.7851<br>0.1281<br><.0001 | | | | | | |
| | | | Leas | st Squar | es Mear | s Estimates | | | | |
| Effect | Label | | Margins | Est | imate | Standard<br>Error | DF | t Value | Pr > t | Z |
| trtpn<br>trtpn | LSMeans, I | | WORK.ADATA | | .5207<br>.5340 | 0.02802<br>0.03963 | 449<br>449 | 18.58<br>13.47 | <.0001<br><.0001 | |
| | | | Least | Squares | Means | Estimates | | | | |
| Effect | Label | | Lower | Upp | er Ex | ponentiated | | entiated<br>Lower | Exponenti<br>U | ateo<br>Jppe: |

| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADATA2<br>WORK.ADATA2 | 0.520<br>0.534 | | 449<br>449 | 18.58<br>13.47 | <.0001<br><.0001 | 0.05<br>0.05 |
|---|---|---|---|---|---|---|---|---|---|
| Least Squares Means Estimates | | | | | | | | | |
| Effect | Label | | Lower | Upper | Exponentiated | Expone | entiated<br>Lower | Exponentiat<br>Upp | |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | 0.4657<br>0.4561 | 0.5758<br>0.6119 | 1.6833<br>1.7057 | | 1.5931<br>1.5779 | 1.77<br>1.84 | |
| | Least Squares Means Estimate | | | | | | | | |

Alpha

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | -0.01325 | 0.04855 | 449 | -0.27 | 0.7851 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 289 of 334 | |

Triglycerides after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

Parameter Code=C64812S

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.1087 0.08216 0.9868

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.8970 1.0856


 $\hbox{Triglycerides after 26 weeks of treatment - supportive statistical analysis - full analysis set-appendix } \\$ 

Parameter Code=TRIG SU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453
Number of Observations Used 453
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.2371

Fit Statistics

-2 Res Log Likelihood 648.7 AICC (Smaller is Better) 650.7 AICC (Smaller is Better) 650.7 BIC (Smaller is Better) 654.8

Solution for Fixed Effects

Planned

Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 0.1840 1.9126 449 10.40 Intercept -0.01325 0.04855 -0.27 1 449 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.06990 0.04585 449 1.52 PREAD 0.6028 base log 0.03500 449 17.22

| NN9068 | | Date: | 22 January 2020 Novo Nordisi |
|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final |
| Statistical document | | Page: | 291 of 334 |

Triglycerides after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

| Paramete | r Code=TR | IG_SU | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| The Mixe | d Procedu | re | | | | | | | |
| | | | Solution f | or Fixed Effec | :ts | | | | |
| Effect | Pre Tr | ial anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | a | |
| Intercep<br>trtpn | t | | | | 1<br>2 | <.0001<br>0.7851 | | | |
| PREAD<br>PREAD | | | | | | 0.1281 | 0.0 | 5 | |
| base_log | | INSULIN + 1 | MEIFORMIN T | ONE OTHER OAL | , | <.0001 | 0.0 | 5 | |
| | | | Solution | for Fixed Effe | ects | | | | |
| Effect | Pre Tr | ial anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | c UD | per | |
| Intercep | t | | | | | 1.5511 | - | 741 | |
| trtpn<br>trtpn | | | | | 1 2 | -0.1087 | 7 0.08 | 216 | |
| PREAD<br>PREAD<br>base_log | BASAL : | INSULIN + I<br>INSULIN + I | | ONE OTHER OAD | ) | 0.5340 | | 716 | |
| | Type 3 Tes | sts of Fixe | ed Effects | | | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>base_log | 1<br>1<br>1 | | 0.07<br>2.32<br>296.62 | 0.7851<br>0.1281<br><.0001 | | | | | |
| | | | Lea | st Squares Mea | ıns Estimates | | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | 1 |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | IDegLira<br>IDeg | WORK.ADAT<br>WORK.ADAT | | 0.02802<br>0.03963 | 449<br>449 | 178.76<br>126.73 | <.0001<br><.0001 | |
| | | | Least | Squares Means | Estimates | | | | |
| | | | | | | Expone | entiated | Exponenti | ate |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | LSMeans, IDeo | | 5.0094<br>5.022 | | 449<br>449 | 178.76<br>126.73 | <.0001<br><.0001 | |
| | Least Squares Means Estimates | | | | | | | |
| Effect | Label | Lower | Upper | Exponentiated | Expone | entiated<br>Lower | Exponent | iated<br>Upper |
| trtpn<br>trtpn | LSMeans, IDeo | | 5.0645<br>5.1005 | 149.81<br>151.81 | | 141.78<br>140.43 | _ | .58.29<br>.64.11 |
| | | Least | Squares Me | eans Estimate | | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Erron | | t Value | Pr > t |

trtpn Treatment ratio, IDegLira - IDeg WORK.ADATA2 -0.01325 0.04855 449 -0.27 0.7851

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 292 of 334 | |

Triglycerides after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

Parameter Code=TRIG\_SU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.1087 0.08216 0.9868

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.8970 Exponentiated 1.0856

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

## 29: Total cholesterol after 26 weeks of treatment – supportive statistical analysis – full analysis set - appendix

Parameter Code=C105586S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.03056

Fit Statistics

-2 Res Log Likelihood -273.4
AIC (Smaller is Better) -271.4
AICC (Smaller is Better) -271.4
BIC (Smaller is Better) -267.3

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept 0.4374 0.05797 449 7.55 trtpn 1 -0.03841 0.01743 -2.20 trtpn 2 Ω BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD 0.02172 PREAD 0.01647 449 1.32 PREAD 0.6782 0.03724 base\_log 449 18.21

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 294 of 334 | |

Total cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

| Paramete | er Code=C105 | 5586S | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| The Mixe | ed Procedure | è | | | | | | | |
| | | | Solution for | Fixed Effe | ects | | | | |
| Effect | Pre Tria | al anti-D | iabetic treat | ment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | na | |
| Intercep | ot | | | | <.000 | _ | | | |
| trtpn<br>trtpn | trtpn | | | | | 0.028 | 1 0.0 | )5 | |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | 4 D | 0.187 | 9 0.0 | )5 | |
| base_log | | .002111 | | 0111211 01 | 12 | <.000 | 1 0.0 | )5 | |
| | | | Solution fo | r Fixed Eft | fects | | | | |
| Effect | Dro Trio | 1 anti-D | iabetic treat | mont | Planned<br>Treatment<br>for<br>Period | Toyyo | × II | nor. | |
| | | i anti-Di | labetic treat | ment | 01 (N) | Lowe | - | pper | |
| Intercep<br>trtpn | )t | | | | 1 | 0.323<br>-0.0726 | | 5513<br>0415 | |
| PREAD | | | | | 2 | -0.0106 | 4 0.05 | 5409 | |
| PREAD<br>base_log | | ISULIN + 1 | METFORMIN + O | NE OTHER OF | AD | 0.605 | 0 0. | 7513 | |
| | Type 3 Test | | ed Effects | | | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>base_log | 1<br>1<br>1 | 449<br>449<br>449 | 1.74 | 0.0281<br>0.1879<br><.0001 | | | | | |
| | | | Least | Squares Me | eans Estimates | 3 | | | |
| | | | | 1 | Standard | | | | |
| Effect | Label | | Margins | Estimate | | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, I<br>LSMeans, I | | WORK.ADATA2<br>WORK.ADATA2 | | | 449<br>449 | 142.39<br>103.37 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least S | quares Mear | ns Estimates | | | | |
| Effect | Label | | Lower | Upper | Exponentiated | | entiated<br>Lower | | ted |
| trtpn<br>trtpn | LSMeans, I<br>LSMeans, I | | 1.4128<br>1.4430 | 1.4523<br>1.4990 | 4.1895<br>4.3535 | | 4.1075<br>4.2335 | | 731<br>770 |
| | | | Least | Squares Me | eans Estimate | | | | |

### Least Squares Means Estimate

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | -0.03841 | 0.01743 | 449 | -2.20 | 0.0281 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 295 of 334 | |

 $\hbox{Total cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix } \\$ 

Parameter Code=C105586S

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.07267 -0.00415 0.9623

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.9299 0.9959


 $\hbox{Total cholesterol after 26 weeks of treatment-supportive statistical analysis-full analysis set-appendix } \\$ 

Parameter Code=T\_CHOL\_U

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453
Number of Observations Used 453
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.03056

Fit Statistics

-2 Res Log Likelihood -273.4
AIC (Smaller is Better) -271.4
AICC (Smaller is Better) -271.4
BIC (Smaller is Better) -267.3

Solution for Fixed Effects

Planned

Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 1.6132 0.1924 449 8.39 Intercept 0.01743 -2.20 1 -0.03841 449 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 0.02172 0.01647 449 1.32 PREAD 0.6782 base log 0.03724 449 18.21

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 297 of 334 | |

 $\hbox{Total cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix } \\$ 

| - append | ix | zo weeks or tre | acment - supp | JICIVE SCACI | Stical a | nalysis - | ruir anarys | is set |
|---|---|---|---|---|---|---|---|---|
| Paramete | r Code=T_CHOL_U | | | | | | | |
| The Mixe | d Procedure | | | | | | | |
| | | Solution fo | r Fixed Effec | ts | | | | |
| Effect. | Pre Trial ant | i-Diabetic trea | tment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpl | na | |
| Intercep<br>trtpn | | | | 1 | <.000 | 1 0.0 | )5 | |
| trtpn<br>PREAD | BASAL INSULIN | + METFORMIN | | 2 | 0.187 | | | |
| PREAD<br>base log | BASAL INSULIN | + METFORMIN + | ONE OTHER OAD | | <.000 | | | |
| | | Solution f | or Fixed Effe | cts | | | | |
| Effect | Pre Trial ant | | | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lowe | r U) | pper | |
| Intercep<br>trtpn<br>trtpn<br>PREAD<br>PREAD<br>base_log | BASAL INSULIN<br>BASAL INSULIN | + METFORMIN<br>+ METFORMIN + | ONE OTHER OAD | 1 2 | 1.235<br>-0.0726<br>-0.0106<br>0.605 | 7 -0.00<br>4 0.09 | | |
| | Type 3 Tests of | Fixed Effects | | | | | | |
| Effect | Num De:<br>DF D: | | Pr > F | | | | | |
| trtpn<br>PREAD<br>base_log | 1 44<br>1 44<br>1 44 | 9 1.74 | 0.0281<br>0.1879<br><.0001 | | | | | |
| | | Leas | t Squares Mea | ns Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLi | ra WORK.ADATA<br>WORK.ADATA | | 0.01006<br>0.01423 | 449<br>449 | 505.54<br>360.12 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least | Squares Means | Estimates | | | | |
| Effect | Label | Lower | Upper E | xponentiated | | entiated<br>Lower | Exponentia<br>Up | ted |
| trtpn<br>trtpn | LSMeans, IDegLi<br>LSMeans, IDeg | | 5.1059<br>5.1525 | 161.76<br>168.09 | | 158.59<br>163.45 | | .99 |
| | | Leas | t Squares Mea | ns Estimate | | | | |

trtpn Treatment ratio, IDegLira - IDeg WORK.ADATA2 -0.03841 0.01743 449 -2.20 0.0281

Effect Label

Standard
Margins Estimate Error DF t Value Pr > |t|

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 298 of 334 | |

 $\hbox{Total cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix } \\$ 

Parameter Code= $T_CHOL_U$ 

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.07267 -0.00415 0.9623

Least Squares Means Estimate

Exponentiated Label Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.9299 0.9959

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
1.0
Status:
Final
Page:

## 30: Free fatty acid after 26 weeks of treatment – supportive statistical analysis – full analysis set – appendix

Parameter Code=C80200S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 452

Number of Observations

Number of Observations Read 453 Number of Observations Used 452 Number of Observations Not Used 1

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.2601

Fit Statistics

-2 Res Log Likelihood 688.4
AIC (Smaller is Better) 690.4
AICC (Smaller is Better) 690.4
BIC (Smaller is Better) 694.5

Solution for Fixed Effects

Planned Treatment for

| Effect | Pre Trial anti-Diabetic treatment | Period<br>01 (N) | Estimate | Standard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn | | 1 2 | -1.1035<br>-0.01181<br>0 | 0.06468<br>0.05099 | 448<br>448 | -17.06<br>-0.23 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | -0.03834<br>0 | 0.04808 | 448 | -0.80 |
| base_log | | | 0.2370 | 0.04606 | 448 | 5.15 |

| NN9068 | | Date: | 22 January 2020 Novo Nordi | sk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 300 of 334 | |

Free fatty acid after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

| appendix | ty acid after 26 we | eks of treatm | ent - suppor | tive statist | ical ana | lysis - i | ull analysis | set - |
|---|---|---|---|---|---|---|---|---|
| Paramete | r Code=C80200S | | | | | | | |
| The Mixe | d Procedure | | | | | | | |
| | | Solution for | Fixed Effec | ts | | | | |
| Effect | Pre Trial anti-D | iabetic treat | ment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alp | ha | |
| Intercep<br>trtpn | t | | | 1 2 | <.000<br>0.817 | | | |
| trtpn<br>PREAD | BASAL INSULIN + | | NIE OBUED OAD | | 0.425 | 6 0. | 05 | |
| PREAD<br>base_log | BASAL INSULIN + | METFORMIN + C | NE OTHER OAD | | <.000 | 1 0. | 05 | |
| | | Solution fo | r Fixed Effe | cts | | | | |
| Effect | Pre Trial anti-D | iabetic treat | ment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lowe | r Uj | pper | |
| Intercep<br>trtpn<br>trtpn<br>PREAD<br>PREAD<br>base_log | trtpn PREAD BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | -1.230<br>-0.112<br>-0.132 | 0 0.0 | -0.9764<br>0.08841<br>0.05615<br>0.3275 | |
| | Type 3 Tests of Fix | ed Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>base_log | 1 448<br>1 448<br>1 448 | 0.64 | 0.8170<br>0.4256<br><.0001 | | | | | |
| | | Least | Squares Mea | ns Estimates | ; | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.02936<br>0.04167 | 448<br>448 | -46.29<br>-32.33 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least S | quares Means | Estimates | | | | |
| Effect | Label | Lower | Upper E | xponentiated | | entiated<br>Lower | | ted |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | -1.4167<br>-1.4291 | -1.3013<br>-1.2653 | 0.2569<br>0.2600 | | 0.2425<br>0.2395 | | 722<br>822 |

### Least Squares Means Estimate

| Effect | Label | | Margins | Estimate | Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | -0.01181 | 0.05099 | 448 | -0.23 | 0.8170 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 301 of 334 | |

Free fatty acid after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix  $\mathbf{x}$ 

Parameter Code=C80200S

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.1120 0.08841 0.9883

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.8940 Exponentiated 1.0924


Free fatty acid after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix

Parameter Code=FFAU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 452

Number of Observations

Number of Observations Read 453
Number of Observations Used 452
Number of Observations Not Used 1

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.2601

Fit Statistics

-2 Res Log Likelihood 688.4
AIC (Smaller is Better) 690.4
BIC (Smaller is Better) 694.5

Solution for Fixed Effects

Planned Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 1.4444 0.1203 448 12.01 Intercept 0.05099 -0.23 -0.01181 448 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.03834 0.04808 -0.80 PREAD 0.2370 base log 0.04606 448 5.15

| NN9068 | | Date: | 22 January 2020 Novo Nordisi |
|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final |
| Statistical document | | Page: | 303 of 334 |

Free fatty acid after 26 weeks of treatment - supportive statistical analysis - full analysis set appendix

| Paramete | r Code=FFAU | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| The Mixed | d Procedure | | | | | | | |
| Solution for Fixed Effects | | | | | | | | |
| Refort | Pre Trial anti- | Diabetia tuestm | ont | Planned<br>Treatment<br>for<br>Period | Dro N. J. E. J. | 7.1.0.0.0 | | |
| FILECT | Pre Trial anti- | Diabetic treatm | ent | 01 (N) | Pr > t | Alpha | | |
| Intercept<br>trtpn<br>trtpn | t | | | 1<br>2 | <.0001<br>0.8170 | 0.05 | | |
| PREAD<br>PREAD | BASAL INSULIN +<br>BASAL INSULIN + | | E OTHER OAI | ) | 0.4256 | 0.05 | 5 | |
| base_log | | | | | <.0001 | 0.05 | 5 | |
| | | Solution for | Fixed Effe | ects | | | | |
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial anti- | Diabetic treatm | ent | 01 (N) | Lower | Upp | per | |
| Intercept<br>trtpn<br>trtpn | t | | | 1 2 | 1.2080<br>-0.1120 | 1.68<br>0.088 | | |
| PREAD BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | ) | -0.1328 | 0.056 | 515 | | |
| base_log | | | n omner om | , | 0.1465 | 0.32 | 275 | |
| - | Type 3 Tests of Fi | xed Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value P | r > F | | | | | |
| trtpn<br>PREAD<br>base_log | 1 448<br>1 448<br>1 448 | 0.64 0 | .8170<br>.4256<br>.0001 | | | | | |
| | | Least | Squares Mea | ans Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF t | Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 1.9803<br>1.9921 | 0.02936<br>0.04167 | 448<br>448 | 67.45<br>47.81 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least Sq | uares Means | s Estimates | | | | |
| Effect | Label | Lower | Upper I | Exponentiated | | tiated<br>Lower | Exponenti<br>U | ated<br>pper |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | 1.9226<br>1.9102 | 2.0380<br>2.0740 | 7.2452<br>7.3312 | | 6.8390<br>6.7548 | | 6755<br>9568 |
| | | Least | Squares Mea | ans Estimate | | | | |
| Effect 1 | Label | | Margins | Estimate | Standard<br>Error | DF t | . Value P | r > t |

trtpn Treatment ratio, IDegLira - IDeg WORK.ADATA2 -0.01181 0.05099 448 -0.23 0.8170
| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 304 of 334 | |

Free fatty acid after 26 weeks of treatment - supportive statistical analysis - full analysis set - appendix  $\mathbf{x}$ 

Parameter Code=FFAU

The Mixed Procedure

Least Squares Means Estimate

Effect Label Alpha Lower Upper Exponentiated trtpn Treatment ratio, IDegLira - IDeg 0.05 -0.1120 0.08841 0.9883

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment ratio, IDegLira - IDeg 0.8940 Exponentiated 1.0924

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 305 of 334 | |

#### 31: Hypoglycaemic episodes – treatment emergent – confirmatory statistical analysis – full analysis set

Parameter Code=HYCNFSE

The GENMOD Procedure

Model Information

Data Set WORK.ANA\_DATA
Distribution Negative Binomial
Link Function
Dependent Vi

Dependent Variable Offset Variable AVAĹ Analysis Value LOGOFF

Number of Observations Read Number of Observations Used Missing Values 453 452

Class Level Information

Values Class Levels TRTPN

BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 2

Parameter Information

Parameter Effect TRTPN PREAD Prm1 Intercept TRTPN Prm2 TRTPN 2 Prm3 Prm4 PREAD BASAL INSULIN + METFORMIN

Prm5 PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD

Iteration History For Parameter Estimates

| Iter | Ridge | Log<br>Likelihood | Prm1 | Prm2 | Prm4 | Dispersion |
|---|---|---|---|---|---|---|
| 0 | 0 | -272.05183 | 4.8722249 | -0.133255 | 0.0535432 | 0.9030346 |
| 1 | 1 | -210.31256 | 4.3017337 | -0.38207 | -0.019395 | 0.5621385 |
| 2 | 1 | -196.63064 | 4.0111682 | -0.544379 | 0.0204517 | 0.7702072 |
| 3 | 0.06 | -192.79932 | 4.0350243 | -0.558915 | 0.0141844 | 6.3310514 |
| 4 | 0 | -189.55465 | 3.6343238 | -0.650209 | 0.3457195 | 3.2510687 |
| 5 | 0 | -189.37048 | 3.755194 | -0.639949 | 0.2514424 | 3.1348703 |
| 6 | 0 | -189.3701 | 3.7514615 | -0.640906 | 0.2552308 | 3.154036 |
| 7 | 0 | -189.3701 | 3.7514508 | -0.640908 | 0.2552416 | 3.1540135 |

#### Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|--------------------------|-----|-----------|----------|
| Deviance | 449 | 191.5532 | 0.4266 |
| Scaled Deviance | 449 | 191.5532 | 0.4266 |
| Pearson Chi-Square | 449 | 572.5233 | 1.2751 |
| Scaled Pearson X2 | 449 | 572.5233 | 1.2751 |
| Log Likelihood | | -189.3701 | |
| Full Log Likelihood | | -208.8157 | |
| AIC (smaller is better) | | 425.6314 | |
| AICC (smaller is better) | | 425.7209 | |
| BIC (smaller is better) | | 442.0862 | |

# NN9068 | Date: 22 January 2020 | Novo Nordisk NN9068-4166 | Confidential Report | Status: Final  |

 ${\tt Hypoglycaemic\ episodes\ -\ treatment\ emergent\ -\ confirmatory\ statistical\ analysis\ -\ full\ analysis\ set}$ 

Parameter Code=HYCNFSE

The GENMOD Procedure

Last Evaluation Of The Negative Of The Gradient and Hessian

| 4.205977 -0.177<br>3.519355 -0.138<br>4.205977 -0.132 | 861<br>454<br>367 |
|---|---|
| | 4.205977 -0.177<br>3.519355 -0.138 |

Algorithm converged.

#### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidence | 95%<br>ce Limits |
|---|---|---|---|---|---|---|
| Intercept<br>TRTPN<br>TRTPN<br>PREAD<br>PREAD<br>Dispersion | 1<br>2<br>BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | 1<br>0<br>1<br>0 | 3.7515<br>-0.6409<br>0.0000<br>0.2552<br>0.0000<br>3.1540 | 0.2710<br>0.2948<br>0.0000<br>0.2919<br>0.0000<br>1.0834 | 3.2202<br>-1.2187<br>0.0000<br>-0.3170<br>0.0000<br>1.6087 | 4.2827<br>-0.0632<br>0.0000<br>0.8274<br>0.0000<br>6.1837 |

#### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|
| Intercept<br>TRTPN<br>TRTPN | 1 2 | 191.58<br>4.73 | <.0001<br>0.0297 |
| PREAD<br>PREAD<br>Dispersion | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | 0.76 | 0.3820 |

NOTE: The negative binomial dispersion parameter was estimated by maximum likelihood.

#### TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|---|
| 1 2 | 3.2382 | 0.1931 | 16.77 | <.0001 | 0.05 | 2.8596 | 3.6167 | 25.4869 |
| | 3.8791 | 0.2228 | 17.41 | <.0001 | 0.05 | 3.4424 | 4.3157 | 48.3793 |

TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Exponentiated Lower | Exponentiated Upper |
|-----------------------------|---------------------|---------------------|
| 1 2 | 17.4553<br>31.2620 | 37.2140<br>74.8691 |

#### Differences of TRTPN Least Squares Means

| Planned<br>Treatment | Planned<br>Treatment | | Standard | | | | | |
|---|---|---|---|---|---|---|---|---|
| (N) | (N) | Estimate | | z Value | Pr > z | Alpha | Lower | Upper |
| 1 | 2 | -0.6409 | 0.2948 | -2.17 | 0.0297 | 0.05 | -1.2187 | -0.06315 |

#### NN9068 NN9068-4166 Date: 22 January 2020 Novo Nordisk Version: 1.0

Clinical Trial Report Status: Final Statistical document 

Hypoglycaemic episodes - treatment emergent - confirmatory statistical analysis - full analysis set

Parameter Code=HYCNFSE

The GENMOD Procedure

Differences of TRTPN Least Squares Means

Planned Planned

Treatment (N) Exponentiated Lower Upper

1 2 0.5268 0.2956 0.9388

Least Squares Means Estimate

Standard

Least Squares Means Estimate

Exponentiated Exponentiated Lower Upper TRTPN IDegLira / IDeg 0.5268 0.2956 0.9388

### 32: Hypoglycaemic episodes – treatment emergent – statistical sensitivity analysis – multiple imputation – full analysis set

Parameter Code=HYCNFSE Planned Treatment (N)=1 Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSM\_MI

Number of Imputations 1000

Variance Information (1000 Imputations)

Parameter Between Within Total DF Estimate 0.003123 0.035506 0.038632 152521

Variance Information (1000 Imputations)

Relative Fraction
Increase Missing Relative
Parameter in Variance Information Efficiency

Estimate 0.088058 0.080943 0.999919

Parameter Estimates (1000 Imputations)

 
 Parameter
 Estimate
 Std Error
 25% Confidence Limits
 DF
 Minimum
 Maximum

 Estimate
 3.271298
 0.196551
 2.886063
 3.656534
 152521
 3.193123
 3.464076

Parameter Estimates (1000 Imputations)

t for HO:

Parameter Theta0 Parameter=Theta0 Pr > |t|Estimate 0 16.64 <.0001

## NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 tatus: Final 

 $\label{thm:mapping} \mbox{Hypoglycaemic episodes - treatment emergent - statistical sensitivity analysis - multiple imputation - full analysis set$ 

Parameter Code=HYCNFSE Planned Treatment (N)=2 Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSM MI

Number of Imputations 1000

Variance Information (1000 Imputations)

Parameter Between Within Total DF

Estimate 0.002588 0.048444 0.051034 387717

Variance Information (1000 Imputations)

Relative Fraction

Increase Missing Relative Parameter in Variance Information Efficiency
Estimate 0.053475 0.050765 0.999949

Parameter Estimates (1000 Imputations)

95% Confidence

 Parameter
 Estimate
 Std Error
 Limits
 DF
 Minimum
 Maximum

 Estimate
 3.880257
 0.225908
 3.437485
 4.323030
 387717
 3.817666
 4.255104

Parameter Estimates (1000 Imputations)

t for HO:

Parameter Theta0 Parameter=Theta0 Pr > |t|Estimate 0 17.18 <.0001


DF

 $\label{thm:mapping} \mbox{Hypoglycaemic episodes - treatment emergent - statistical sensitivity analysis - multiple imputation - full analysis set$ 

Parameter Code=HYCNFSE Label=IDegLira / IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME MI

Number of Imputations 1000

Variance Information (1000 Imputations)

Parameter Between Within Total

Estimate 0.005649 0.083893 0.089548 250504

Variance Information (1000 Imputations)

Relative Fraction

Increase Missing Relative Parameter in Variance Information Efficiency
Estimate 0.067407 0.063158 0.999937

Parameter Estimates (1000 Imputations)

95% Confidence

 Parameter
 Estimate
 Std Error
 Limits
 DF
 Minimum
 Maximum

 Estimate
 -0.608959
 0.299246
 -1.19547
 -0.02244
 250504
 -1.010738
 -0.360220

Parameter Estimates (1000 Imputations)

t for HO:

Parameter Theta0 Parameter=Theta0 Pr > |t|Estimate 0 -2.03 0.0419

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 310 of 334 | |

#### 33: Hypoglycaemic episodes – treatment emergent – supportive statistical analysis – full analysis set

Parameter Code=HYCNFSES

The GENMOD Procedure

Model Information

WORK.ANA DATA Data Set Distribution Negative Binomial Link Function Log

Dependent Variable Offset Variable AVAĹ Analysis Value logoff

Number of Observations Read Number of Observations Used Missing Values 453 452

Class Level Information

Values Class Levels TRTPN

BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 2

Parameter Information

Parameter Effect TRTPN PREAD Prm1 Intercept

TRTPN Prm2 TRTPN 2 Prm3 Prm4 PREAD

BASAL INSULIN + METFORMIN Prm5 PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD

Iteration History For Parameter Estimates

| | | Log | | | | |
|------|-------|------------|-----------|-----------|-----------|------------|
| Iter | Ridge | Likelihood | Prm1 | Prm2 | Prm4 | Dispersion |
| 0 | 0 | -248.88659 | 4.7823425 | -0.097818 | 0.0546535 | 0.8596882 |
| 1 | 1 | -150.683 | 3.7018963 | -0.473071 | -0.076207 | 0.0626182 |
| 2 | 0.06 | -144.39901 | 3.2524477 | -0.570648 | 0.3099962 | 0.1619065 |
| 3 | 1 | -143.90765 | 3.1384215 | -0.614858 | 0.4166656 | 0.1781804 |
| 4 | 1 | -143.75331 | 3.0873625 | -0.619769 | 0.482044 | 0.1989049 |
| 5 | 1 | -143.6442 | 3.0615369 | -0.615829 | 0.514276 | 0.2241457 |
| 6 | 1 | -143.53327 | 3.0479009 | -0.611319 | 0.5296764 | 0.2550337 |
| 7 | 1 | -143.40811 | 3.040686 | -0.60782 | 0.5369217 | 0.2932181 |
| 8 | 1 | -143.26397 | 3.0369288 | -0.605294 | 0.5401102 | 0.3408479 |
| 9 | 1 | -143.09875 | 3.0350577 | -0.603396 | 0.541174 | 0.400609 |
| 10 | 0.06 | -141.69204 | 3.0387866 | -0.593892 | 0.5282424 | 2.4021374 |
| 11 | 0 | -141.64987 | 3.0413466 | -0.583393 | 0.5170532 | 2.0466411 |
| 12 | 0 | -141.64952 | 3.0412361 | -0.583948 | 0.5177205 | 2.0124952 |
| 13 | 0 | -141.64952 | 3.041235 | -0.583949 | 0.5177226 | 2.0121329 |
| 14 | 0 | -141.64952 | 3.041235 | -0.583949 | 0.5177226 | 2.0121329 |

Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|--------------------------|-----|-----------|----------|
| Deviance | 449 | 161.6466 | 0.3600 |
| Scaled Deviance | 449 | 161.6466 | 0.3600 |
| Pearson Chi-Square | 449 | 487.6689 | 1.0861 |
| Scaled Pearson X2 | 449 | 487.6689 | 1.0861 |
| Log Likelihood | | -141.6495 | |
| Full Log Likelihood | | -146.6193 | |
| AIC (smaller is better) | | 301.2387 | |
| AICC (smaller is better) | | 301.3281 | |

### NN9068 Date: 22 January 2020 Novo Nordisk NN9068-4166 Version: 1.0 Clinical Trial Report Status: Final

Page:


Hypoglycaemic episodes - treatment emergent - supportive statistical analysis - full analysis set

Parameter Code=HYCNFSES

The GENMOD Procedure

Statistical document

Criteria For Assessing Goodness Of Fit

Criterion DF Value Value/DF

BIC (smaller is better) 317.6934

Last Evaluation Of The Negative Of The Gradient and Hessian

| | Prm1 | Prm2 | Prm4 | Dispersion |
|---|---|---|---|---|
| Gradient<br>Prm1 | -2.874E-9<br>35.798234 | -2.428E-9<br>19.712382 | -2.36E-10<br>21.111393 | 2.4602E-8<br>-0.077305 |
| Prm2 | 19.712382 | 19.712382 | 11.018598 | -0.12625 |
| Prm4 | 21.111393 | 11.018598 | 21.111393 | 0.0691198 |
| Dispersion | -0.077305 | -0.12625 | 0.0691198 | 0.5954467 |

Algorithm converged.

#### Analysis Of Maximum Likelihood Parameter Estimates

| | | | | | | | | | Standard | Wald 9 | 5% |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | | | | | | DF | Estimate | Error | Confidence | Limits |
| Intercept | | | | | | | 1 | 3.0412 | 0.3284 | 2.3975 | 3.6850 |
| TRTPN | 1 | | | | | | 1 | -0.5839 | 0.3370 | -1.2444 | 0.0765 |
| TRTPN | 2 | | | | | | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 |
| PREAD | BASAL | INSULIN | + METFORMIN | | | | 1 | 0.5177 | 0.3410 | -0.1506 | 1.1861 |
| PREAD | BASAL | INSULIN | + METFORMIN | + ONE | OTHER | OAD | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 |
| Dispersion | | | | | | | 1 | 2.0121 | 1.2985 | 0.5680 | 7.1278 |

#### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|
| Intercept<br>TRTPN<br>TRTPN | 1 2 | 85.74<br>3.00 | <.0001<br>0.0831 |
| PREAD<br>PREAD<br>Dispersion | BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAL | 2.31 | 0.1290 |

NOTE: The negative binomial dispersion parameter was estimated by maximum likelihood.

#### TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|---|
| 1 | 2.7161 | 0.2263 | 12.00 | <.0001 | 0.05 | 2.2726 | 3.1597 | 15.1219 |
| 2 | 3.3001 | 0.2531 | 13.04 | <.0001 | 0.05 | 2.8041 | 3.7961 | 27.1153 |

#### TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Exponentiated Lower | Exponentiated<br>Upper |
|-----------------------------|---------------------|------------------------|
| 1 | 9.7044 | 23.5640 |
| 2 | 16.5114 | 44.5290 |

| NN9068<br>NN9068-4166<br>Clinical Trial Report<br>Statistical document | CONFIDE | | Date:<br>Version:<br>Status:<br>Page: | 22 January 2020<br>1.0<br>Fina<br>312 of 33- | 0 1 |
|---|---|---|---|---|---|
| Hypoglycaemic episodes - | treatment emergent - s | supportive stat | istical analysis | - full analys | is set |
| Parameter Code=HYCNFSES | | | | | |
| The GENMOD Procedure | | | | | |
| | Differences of TRTPN | Least Squares | Means | | |
| Planned Planned<br>Treatment Treatment<br>(N) (N) E | Standard<br>Estimate Error z | : Value Pr > | z Alpha | Lower U | pper |
| 1 2 | -0.5839 0.3370 | -1.73 0.0 | 831 0.05 | -1.2444 0.0 | 7654 |
| Difference | es of TRTPN Least Squar | es Means | | | |
| Planned Planned<br>Treatment Treatment<br>(N) (N) E | Expone<br>Exponentiated | entiated Exp<br>Lower | onentiated<br>Upper | | |
| 1 2 | 0.5577 | 0.2881 | 1.0795 | | |
| Least Squares Means Estimate | | | | | |
| Effect Label | Standard<br>Estimate Error | z Value Pr | > z Alpha | Lower | Upper |
| TRTPN IDegLira / IDeg | -0.5839 0.3370 | -1.73 | 0.0831 0.05 | -1.2444 | 0.07654 |
| Le | Least Squares Means Estimate | | | | |
| Effect Label | Exp<br>Exponentiated | onentiated<br>Lower | Exponentiated<br>Upper | | |

Effect Label Exponentiated Lower Upper TRTPN IDegLira / IDeg 0.5577 0.2881 1.0795

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 313 of 334 | |

### 34: Nocturnal hypoglycaemic episodes – treatment emergent – supportive statistical analysis – full analysis set

Parameter Code=HYNOCSE

The GENMOD Procedure

Model Information

Data Set WORK.ANA DATA Distribution Negative Binomial Log AVAL Link Function Dependent Variable Offset Variable

Analysis Value logoff

Number of Observations Read 453 Number of Observations Used Missing Values

Class Level Information

Values Class Levels TRTPN

1 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD

Parameter Information

Effect TRTPN PREAD Parameter

Intercept Prm1 TRTPN Prm2 Prm3 TRTPN 2

PREAD BASAL INSULIN + METFORMIN Prm4

Prm5 PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD

Iteration History For Parameter Estimates

| Iter | Ridge | Log<br>Likelihood | Prm1 | Prm2 | Prm4 | Dispersion |
|---|---|---|---|---|---|---|
| 0<br>1<br>2<br>3<br>4<br>5<br>6<br>7<br>8<br>9<br>10<br>11<br>12<br>13<br>14<br>15<br>16<br>17<br>18<br>19<br>20<br>21<br>22 | 0<br>16<br>1<br>0.06<br>0.06<br>0.06<br>0.06<br>0.06<br>0.06<br>0.0 | Likelihood -215.96192 -167.98527 -90.768506 -72.013485 -67.946168 -67.192355 -67.124605 -67.121743 -67.121031 -67.121031 -67.120625 -67.12915 -67.118547 -67.11712 -67.11712 -67.11712 -67.115266 -67.112806 -67.112806 | 4.6893282<br>4.4687164<br>3.5294783<br>2.6019258<br>1.9188902<br>1.4811743<br>1.3101504<br>1.2752562<br>1.2704551<br>1.2697436<br>1.2697436<br>1.2697436<br>1.2697247<br>1.2697247<br>1.2697144<br>1.269703<br>1.2696902<br>1.2696902<br>1.2696593<br>1.2696593<br>1.2696404<br>1.2695928<br>1.2695524 | -0.053017 -0.190605 -0.439246 -0.475368 -0.540226 -0.565808 -0.5559066 -0.559966 -0.558894 -0.558812 -0.558878 -0.55878 -0.55878 -0.55878 -0.558656 -0.5586565 -0.558857 -0.558857 | 0.0516002<br>-0.037648<br>-0.082759<br>0.3715303<br>0.9677594<br>1.4152555<br>1.5891586<br>1.6240807<br>1.6287998<br>1.6293805<br>1.6294463<br>1.6294478<br>1.6294408<br>1.6294319<br>1.6294219<br>1.6294107<br>1.6293982<br>1.629384<br>1.629384<br>1.629384<br>1.6293879<br>1.6293879<br>1.6293279<br>1.6293027 | 0.8341748<br>0.8571859<br>0.170072<br>0.0162736<br>0.0165235<br>0.0170752<br>0.0177306<br>0.0184492<br>0.0192286<br>0.0200756<br>0.0220114<br>0.0231238<br>0.0243527<br>0.0257169<br>0.0257169<br>0.0272398<br>0.0289502<br>0.03308844<br>0.0330885<br>0.0356219<br>0.0385624<br>0.0420137<br>0.0461171 |
| 23<br>24<br>25<br>26 | 0.06<br>0.06<br>0.06<br>0.06 | -67.109383<br>-67.107124<br>-67.104336<br>-67.100824 | 1.2695258<br>1.269481<br>1.269425<br>1.2693535 | -0.558262<br>-0.558143<br>-0.557995<br>-0.557805 | 1.629237<br>1.629193<br>1.629138<br>1.6290678 | 0.0510694<br>0.0571518<br>0.0647792<br>0.0745844 |

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5tatus: Final 

 ${\tt Nocturnal\ hypoglycaemic\ episodes\ -\ treatment\ emergent\ -\ supportive\ statistical\ analysis\ -\ full\ analysis\ set}$ 

Parameter Code=HYNOCSE

The GENMOD Procedure

#### Iteration History For Parameter Estimates

| Iter | Ridge | Log<br>Likelihood | Prm1 | Prm2 | Prm4 | Dispersion |
|---|---|---|---|---|---|---|
| 27<br>28 | 0.06 | -67.096295<br>-67.090299 | 1.2692595<br>1.2691315 | -0.557556<br>-0.557218 | 1.6289753<br>1.6288495 | 0.0875714<br>0.1054017 |
| 29 | 0.06 | -67.08214 | 1.2689504 | -0.556738 | 1.6286715 | 0.1309448 |
| 30 | 0.06 | -67.070793 | 1.2686826 | -0.556029 | 1.6284083 | 0.1693051 |
| 31<br>32 | 0.06 | -67.055061<br>-67.034869 | 1.2682702 | -0.554938<br>-0.553245 | 1.6280038 | 0.2293512 |
| 33 | 0.06 | -67.014505 | 1.2667097 | -0.55083 | 1.6264928 | 0.4546296 |
| 34 | 0 | -67.000492 | 1.2637589 | -0.5432 | 1.6237742 | 1.0469637 |
| 35 | 0 | -66.994046 | 1.2635923 | -0.542893 | 1.623724 | 0.8558277 |
| 36 | 0 | -66.993831 | 1.2637759 | -0.543338 | 1.6238771 | 0.8174085 |
| 37 | 0 | -66.99383 | 1.2637833 | -0.543357 | 1.6238838 | 0.8156145 |
| 38 | 0 | -66.99383 | 1.2637833 | -0.543357 | 1.6238838 | 0.8156145 |

#### Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|---|---|---|---|
| Deviance Scaled Deviance Pearson Chi-Square Scaled Pearson X2 Log Likelihood Full Log Likelihood AIC (smaller is better) AICC (smaller is better) BIC (smaller is better) | 449<br>449<br>449<br>449 | 91.8805<br>91.8805<br>471.5693<br>471.5693<br>-66.9938<br>-67.6870<br>143.3740<br>143.4634<br>159.8287 | 0.2046<br>0.2046<br>1.0503<br>1.0503 |

### Last Evaluation Of The Negative Of The Gradient and Hessian

| | Prm1 | Prm2 | Prm4 | Dispersion |
|---|---|---|---|---|
| Gradient | 7.2041E-8 | -9.852E-8 8.6776345 8.6776345 7.0138944 -0.053721 | 8.936E-8 | 1.0772E-6 |
| Prm1 | 16.193152 | | 13.226628 | 0.0434796 |
| Prm2 | 8.6776345 | | 7.0138944 | -0.053721 |
| Prm4 | 13.226628 | | 13.226628 | 0.0530582 |
| Dispersion | 0.0434796 | | 0.0530582 | 0.272279 |

Algorithm converged.

#### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | F | Estimate | Standard<br>Error | Wald 95<br>Confidence | |
|---|---|---|---|---|---|---|---|
| Intercept<br>TRTPN<br>TRTPN | 1 2 | | 1<br>1<br>0 | | 0.4998 | -1.5229 | 2.5271<br>0.4362<br>0.0000 |

### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | Wald<br>Chi-Square | Pr > ChiSq |
|-----------------------------|-----|--------------------|------------------|
| Intercept<br>TRTPN<br>TRTPN | 1 2 | 3.84<br>1.18 | 0.0499<br>0.2769 |

#### NN9068 22 January 2020 | Novo Nordisk Date: NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Nocturnal hypoglycaemic episodes - treatment emergent - supportive statistical analysis - full analysis set

Parameter Code=HYNOCSE

The GENMOD Procedure

#### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | | DF | Estimate | Standard<br>Error | Wald<br>Confidenc | |
|---|---|---|---|---|---|---|---|
| | BASAL INSULIN +<br>BASAL INSULIN + | <br>ONE OTHER | _ | 0.0000 | 0.6427<br>0.0000<br>1.9224 | 0.3642<br>0.0000<br>0.0080 | 2.8836<br>0.0000<br>82.7552 |

Analysis Of Maximum Likelihood Parameter Estimates

Parameter Chi-Square Pr > ChiSq

BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 6.38 0.0115

PREAD

Dispersion

NOTE: The negative binomial dispersion parameter was estimated by maximum likelihood.

#### TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|---|
| 1 | 1.5324 | 0.3934 | 3.90 | <.0001 | 0.05 | 0.7614 | 2.3033 | 4.6291 |
| 2. | 2.0757 | 0.4214 | 4.93 | < .0001 | 0.05 | 1.2499 | 2.9016 | 7.9703 |

#### TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Exponentiated Lower | Exponentiated<br>Upper |
|-----------------------------|---------------------|------------------------|
| 1 2 | 2.1413<br>3.4899 | 10.0075<br>18.2029 |

#### Differences of TRTPN Least Squares Means

| Planned<br>Treatmer | | | Standard | | | | | |
|---|---|---|---|---|---|---|---|---|
| (N) | (N) | Estimate | | z Value | Pr > z | Alpha | Lower | Upper |
| 1 | 2 | -0.5434 | 0.4998 | -1.09 | 0.2769 | 0.05 | -1.5229 | 0.4362 |

#### Differences of TRTPN Least Squares Means

| Treatment (N) | Treatment (N) | Exponentiated | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|
| 1 | 2 | 0.5808 | 0.2181 | 1.5468 |

#### Least Squares Means Estimate

| Effect | Label | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| TRTPN | IDegLira / IDeg | -0.5434 | 0.4998 | -1.09 | 0.2769 | 0.05 | -1.5229 | 0.4362 |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 316 of 334 | |

 ${\tt Nocturnal\ hypoglycaemic\ episodes\ -\ treatment\ emergent\ -\ supportive\ statistical\ analysis\ -\ full\ analysis\ set}$ 

Parameter Code=HYNOCSE

The GENMOD Procedure

Least Squares Means Estimate

| Effect | Label | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| TRTPN | IDegLira / IDeg | 0.5808 | 0.2181 | 1.5468 |

#### NN9068 22 January 2020 | Novo Nordisk Date: NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final  Statistical document

Nocturnal hypoglycaemic episodes - treatment emergent - supportive statistical analysis - full analysis set

Parameter Code=HYNOCSES

The GENMOD Procedure

Model Information

Data Set WORK.ANA DATA Distribution Link Function Negative Binomial Log Dependent Variable AVAL

Analysis Value logoff

Offset Variable

Number of Observations Read Number of Observations Used 453 452 Missing Values

Class Level Information

Class Levels Values TRTPN

BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 2

Parameter Information

Parameter Effect TRTPN PREAD

Prm1 Intercept TRTPN TRTPN Prm2 Prm3 2 Prm4

BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD Prm5 PREAD

Iteration History For Parameter Estimates

| Iter | Ridge | Log<br>Likelihood | Prm1 | Prm2 | Prm4 | Dispersion |
|---|---|---|---|---|---|---|
| 0 | 0 | -212.11027 | 4.6898332 | -0.053761 | 0.038275 | 0.8351092 |
| 1 | 16 | -162.95238 | 4.4666039 | -0.193 | -0.053776 | 0.8590154 |
| 2 | 1 | -81.103474 | 3.4686626 | -0.455285 | -0.129406 | 0.125644 |
| 3 | 0.06 | -63.352907 | 2.6085205 | -0.526344 | 0.230995 | 0.0522172 |
| 4 | 0.06 | -59.275366 | 1.9430772 | -0.623397 | 0.7585306 | 0.0580303 |
| 5 | | -58.55622 | 1.5250015 | -0.677486 | 1.1872585 | 0.073142 |
| 6<br>7 | 0.06 | -58.483218<br>-58.448149 | 1.3669014 | -0.682462<br>-0.67888 | 1.35142 | 0.1028472 |
| 8 | 0.06 | -58.351696 | 1.3337319 | -0.675113 | 1.3819333 | 0.421137 |
| 9 | 0.06 | -58.185224 | 1.3299425 | -0.662876 | 1.3760787 | 1.7256941 |
| 10 | | -58.184617 | 1.3257512 | -0.649048 | 1.3695915 | 1.7974982 |
| 11 | 0 | -58.184617 | 1.3256893 | -0.648998 | 1.3695947 | 1.7956447 |
| 12 | | -58.184617 | 1.3256893 | -0.648998 | 1.3695947 | 1.7956447 |

#### Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|--------------------------|-----|----------|----------|
| Deviance | 449 | 74.9894 | 0.1670 |
| Scaled Deviance | 449 | 74.9894 | 0.1670 |
| Pearson Chi-Square | 449 | 474.3927 | 1.0566 |
| Scaled Pearson X2 | 449 | 474.3927 | 1.0566 |
| Log Likelihood | | -58.1846 | |
| Full Log Likelihood | | -58.8778 | |
| AIC (smaller is better) | | 125.7555 | |
| AICC (smaller is better) | | 125.8450 | |
| BIC (smaller is better) | | 142.2103 | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 318 of 334 | |

 ${\tt Nocturnal\ hypoglycaemic\ episodes\ -\ treatment\ emergent\ -\ supportive\ statistical\ analysis\ -\ full\ analysis\ set}$ 

Parameter Code=HYNOCSES

The GENMOD Procedure

Last Evaluation Of The Negative Of The Gradient and Hessian

| | Prm1 | Prm2 | Prm4 | Dispersion |
|---|---|---|---|---|
| Gradient Prm1 Prm2 Prm4 Dispersion | -9.349E-9<br>12.891925<br>6.6108821<br>9.9666887<br>0.0342268 | -3.309E-8 6.6108821 6.6108821 5.0193772 -0.037243 | 3.9818E-9<br>9.9666887<br>5.0193772<br>9.9666887<br>0.0460269 | 1.6756E-7<br>0.0342268<br>-0.037243<br>0.0460269<br>0.1113227 |

Algorithm converged.

#### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | DF | Estimate | Standard<br>Error | Wald<br>Confidenc | |
|---|---|---|---|---|---|
| Intercept TRTPN 1 TRTPN 2 PREAD BASAL INSULIN + METFORMIN PREAD BASAL INSULIN + METFORMIN + Dispersion | 00 OTHER OAD 0 1 | 1.3257<br>-0.6490<br>0.0000<br>1.3696<br>0.0000<br>1.7956 | 0.6589<br>0.5598<br>0.0000<br>0.6658<br>0.0000<br>3.0130 | 0.0343<br>-1.7462<br>0.0000<br>0.0647<br>0.0000<br>0.0670 | 2.6170<br>0.4482<br>0.0000<br>2.6745<br>0.0000<br>48.1374 |

#### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | | | | | | Wald<br>Chi-Square | Pr | > | ChiSq |
|---|---|---|---|---|---|---|---|---|---|---|
| Intercept<br>TRTPN<br>TRTPN | 1 | | | | | | 4.05<br>1.34 | | - | .0442 |
| PREAD<br>PREAD<br>Dispersion | BASAL | METFORMIN<br>METFORMIN | + | ONE | OTHER | OAD | 4.23 | | 0 | .0397 |

NOTE: The negative binomial dispersion parameter was estimated by maximum likelihood.

### TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|---|
| 1 | 1.3615 | 0.4261 | 3.20 | 0.0014 | 0.05 | 0.5264 | 2.1966 | 3.9020 |
| 2 | 2.0105 | 0.4434 | 4.53 | <.0001 | 0.05 | 1.1415 | 2.8795 | 7.4670 |

TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Exponentiated Lower | Exponentiated<br>Upper |
|-----------------------------|---------------------|------------------------|
| 1 2 | 1.6927<br>3.1314 | 8.9946<br>17.8055 |

| NN9068<br>NN9068-4166<br>Clinical Trial Report<br>Statistical document | | | | CONFIDER | <del>VTIAL</del> | Date:<br>Version<br>Status:<br>Page: | : | 22 January<br>319 o | 1.0<br>Final |
|---|---|---|---|---|---|---|---|---|---|
| | Nocturna<br>analysis | | c episodes - t | reatment eme | ergent - s | supportive | statistica | al analysis | - full |
| | Parameter Code=HYNOCSES | | | | | | | | |
| | The GENM | OD Procedure | | | | | | | |
| | Differences of TRTPN Least Squares Means | | | | | | | | |
| | Planned<br>Treatmen<br>(N) | Planned<br>t Treatment<br>(N) | S<br>Estimate | tandard<br>Error z | Value F | Pr > z | Alpha | Lower | Upper |
| | 1 | 2 | -0.6490 | 0.5598 | -1.16 | 0.2463 | 0.05 | -1.7462 | 0.4482 |
| | Differences of TRTPN Least Squares Means | | | | | | | | |
| | Planned<br>Treatmen<br>(N) | Planned<br>Treatment<br>(N) | Exponentiate | | ntiated<br>Lower | Exponenti<br>U | ated<br>oper | | |
| | 1 | 2 | 0.522 | 6 | 0.1744 | 1. | 5655 | | |
| | | | T, | east Squares | s Means Es | stimate | | | |
| | | | | Standard | | | | | |
| | Effect | Label | Estimate | Error | z Value | Pr > z | Alpha | Lower | Upper |
| | TRTPN | IDegLira / ID | eg -0.6490 | 0.5598 | -1.16 | 0.2463 | 0.05 | -1.7462 | 0.4482 |
| | | | Least Squares | Means Estir | nate | | | | |
| | Effect | Label | Exponenti | | onentiated<br>Lower | | ntiated<br>Upper | | |
| | TRTPN | IDegLira / ID | )eg 0. | 5226 | 0.1744 | l | 1.5655 | | |

Nordisk

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 320 of 334 | |

### 35: Pulse after 26 weeks of treatment – change from baseline – supportive statistical analysis – full analysis set - appendix

Parameter Code=C49676X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Dimensions

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 65.0379

Fit Statistics

-2 Res Log Likelihood 3174.8
AIC (Smaller is Better) 3176.8
AICC (Smaller is Better) 3176.9
BIC (Smaller is Better) 3180.9

Solution for Fixed Effects

Planned Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment Estimate DF t Value 01 (N) Error Intercept 39.2829 3.1653 449 trtpn 4.4149 0.8040 5.49 trtpn 2 Ω BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN + ONE OTHER OAD -0.2566 0.7591 PREAD 449 -0.34 PREAD 0.5115 0.03986 BASE 449 12.83


Pulse after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=C49676X

The Mixed Procedure

| | | | Solution for | r Fixed Effec | ets | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Tri | ial anti-Di | iabetic treat | tment | 01 (N) | Pr > t | Alph | ıa | |
| Interce<br>trtpn<br>trtpn | pt | | | | 1 2 | <.0001 | | | |
| PREAD<br>PREAD | | INSULIN + N | | ONE OTHER OAD | | 0.7355 | 5 0.0 | 15 | |
| BASE | DASAL | INSOLIN 1 I | ABIFORMIN I V | ONE OTHER OAL | , | <.0000 | 1 0.0 | 15 | |
| Solution for Fixed Effects | | | | | | | | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| | | ial anti-Di | iabetic treat | ment | 01 (N) | Lower | _ | per | |
| Interce<br>trtpn<br>trtpn | pt | | | | 1<br>2 | 33.0623<br>2.8348 | | 1950 | |
| PREAD<br>PREAD | | INSULIN + N | | ONE OTHER OAD | | -1.7485 | 5 1.2 | 1352 | |
| BASE | DINOTIE | INDOBIN , I | IBIT OTHIEN T | JNE OTHER ONE | , | 0.4332 | 2 0.5 | 898 | |
| | Type 3 Tes | sts of Fixe | ed Effects | | | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | | 30.15<br>0.11<br>164.70 | <.0001<br>0.7355<br><.0001 | | | | | |
| | | | Least | Squares Mea | ans Estimates | | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | | WORK.ADATA | | 0.4641<br>0.6564 | 449<br>449 | 179.18<br>119.97 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | | Least : | Squares Means | Estimates | | | | |
| Effect | Label | | Lower | Upper E | Exponentiated | | entiated<br>Lower | Exponentia<br>Up | ted<br>per |
| trtpn<br>trtpn | LSMeans,<br>LSMeans, | | 82.2483<br>77.4555 | 84.0725<br>80.0355 | 1.306E36<br>1.58E34 | | 5.248E35<br>4.35E33 | 3.252<br>5.741 | |
| | | | Least | Squares Mean | ns Estimate | | | | |
| Effect | Label | | | Margins | | | andard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 4.4149 0.8040 449

5.49

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 322 of 334 | |

Pulse after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=C49676X

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg <.0001 0.05 2.8348 5.9950 82.6739

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 17.0278 Exponentiated 401.40

## NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Pulse after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=C49676X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453
Number of Observations Used 453
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 65.0379

Fit Statistics

-2 Res Log Likelihood 3174.8
AICC (Smaller is Better) 3176.9
BIC (Smaller is Better) 3180.9

Solution for Fixed Effects

Planned

Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 39.2829 449 3.1653 12.41 Intercept 4.4149 0.8040 5.49 449 trtpn 0 trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD -0.2566 0.7591 449 -0.34 PREAD -0.4885 BASE 0.03986 449 -12.26


Pulse after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=C49676X

The Mixed Procedure

#### Solution for Fixed Effects

| | | | Solution f | or Fixed Effect | S | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | . anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn | | | | | 1 2 | <.0001<br><.0001 | 0.05<br>0.05 |
| trtpn<br>PREAD | BASAL INS | | | | 2 | 0.7355 | 0.05 |
| PREAD<br>BASE | BASAL INS | SULIN + I | METFORMIN + | ONE OTHER OAD | | <.0001 | 0.05 |
| | Solution for Fixed Effects | | | | | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | 33.0623<br>2.8348 | 45.5036<br>5.9950 |
| PREAD<br>PREAD | BASAL INS | | | ONE OTHER OAD | | -1.7485 | 1.2352 |
| BASE | DINOTED TIVE | OBIN . I | ibir Oldiliv T | ONE OTHER ONE | | -0.5668 | -0.4102 |
| Ту | pe 3 Tests | of Fixe | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD<br>BASE | 1<br>1<br>1 | 449<br>449<br>449 | 30.15<br>0.11<br>150.22 | <.0001<br>0.7355<br><.0001 | | | |

### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.4641<br>0.6564 | 449<br>449 | 12.44<br>2.07 | <.0001<br>0.0393 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | 0.05<br>0.05 | 4.8598<br>0.06695 | 6.6839<br>2.6470 | | | |

22 January 2020 | Novo Nordisk NN9068 Date: NN9068-4166 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

### 36: Systolic blood pressure after 26 weeks of treatment – change from baseline – supportive statistical analysis – full analysis set - appendix

Parameter Code=SYSBPMEA

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method Residual Variance Method Fixed Effects SE Method REMI Profile Model-Based Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters Columns in X Columns in Z 6 Ω Subjects Max Obs per Subject 453

Number of Observations

Number of Observations Read Number of Observations Used 453 453 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 125.53

Fit Statistics

-2 Res Log Likelihood AIC (Smaller is Better) 3472.8 AICC (Smaller is Better) 3472.9 BIC (Smaller is Better) 3476.9

Solution for Fixed Effects

Planned Treatment for

| Effect | Pre Trial anti-Diabetic treatment | Period<br>01 (N) | Estimate | Standard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn | | 1 2 | 64.3085<br>-3.1299<br>0 | 4.9405<br>1.1171 | 449<br>449 | 13.02<br>-2.80 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 1.2168 | 1.0553 | 449 | 1.15 |
| BASE | Enough Francisco | | 0.4942 | 0.03775 | 449 | 13.09 |

| NN9068 | | Date: | 22 January 2020 Novo Nor | disk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 326 of 334 | |

Systolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=SYSBPMEA

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial anti-D: | iabetic treatme | nt | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | ıa | |
|---|---|---|---|---|---|---|---|---|
| Intercep | t | | | | <.0001 | - | | |
| trtpn<br>trtpn | | | | 1 2 | 0.0053 | | | |
| PREAD<br>PREAD | BASAL INSULIN + 1<br>BASAL INSULIN + 1 | | 0.2495 | | | | | |
| BASE | | 0-1 | nia nee | | <.0001 | 0.0 | 15 | |
| | | Solution for 1 | rixed Ellec | | | | | |
| | | | | Planned<br>Treatment<br>for<br>Period | | | | |
| Effect | Pre Trial anti-D | labetic treatmen | nt | 01 (N) | Lower | Up | per | |
| Intercep<br>trtpn<br>trtpn | t | | 1 2 | 54.5991<br>-5.3252 | | | | |
| PREAD<br>PREAD | BASAL INSULIN + N<br>BASAL INSULIN + N | | -0.8572 | 3.2 | 909 | | | |
| BASE | | | 0.4200 | 0.5 | 684 | | | |
| Type 3 Tests of Fixed Effects | | | | | | | | |
| Effect | Num Den<br>DF DF | F Value Pr | > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 449<br>1 449<br>1 449 | 1.33 0.3 | 0053<br>2495<br>0001 | | | | | |
| | | Least So | quares Mear | ns Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 125.38<br>128.51 | 0.6448<br>0.9120 | 449<br>449 | 194.45<br>140.92 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least Squa | ares Means | Estimates | | | | |
| Effect | Label | Lower | Upper Ex | kponentiated | Expone | ntiated<br>Lower | | ted<br>per |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | | 126.65<br>130.30 | 2.834E54<br>6.482E55 | | .981E53<br>1.08E55 | 1.006<br>3.891 | |
| | | Least Sq | uares Means | s Estimate | | | | |
| Effect | Label | | Margins | Estima | | ndard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 -3.1299 1.1171 449 -2.80

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 327 of 334 | |

Systolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=SYSBPMEA

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.0053 0.05 -5.3252 -0.9345 0.04372

Least Squares Means Estimate

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.004867 0.3928

# NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Systolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=SYSBPMEA

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 125.53

Fit Statistics

-2 Res Log Likelihood 3470.8
AIC (Smaller is Better) 3472.8
AICC (Smaller is Better) 3472.9
BIC (Smaller is Better) 3476.9

Solution for Fixed Effects

Planned

Treatment for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 64.3085 4.9405 449 13.02 Intercept -3.1299 -2.80 1 1.1171 449 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 1.2168 1.0553 449 1.15 PREAD -0.5058 BASE 0.03775 449 -13.40

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 329 of 334 | |

Systolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=SYSBPMEA

The Mixed Procedure

#### Solution for Fixed Effects

| Solution for Fixed Effects | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-D | iabetic tre | eatment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha | |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | <.0001<br>0.0053 | 0.05<br>0.05 | |
| PREAD | BASAL INS | | | _ | 0.2495 | 0.05 | | |
| PREAD BASAL INSULIN + METFORMIN + ONE OTHER OAD BASE | | | | | D | <.0001 | 0.05 | |
| Solution for Fixed Effects | | | | | | | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Uppe | r |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | 54.5991<br>-5.3252 | 74.0178<br>-0.9345 | |
| PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | | | D _ | -0.8572 | 3.2909 | 9 |
| BASE | DADAH IND | OLLIN I | METI ORMIN I | ONE OTHER OA | D | -0.5800 | -0.431 | 6 |
| Ту | rpe 3 Tests | of Fix | ed Effects | | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | | |
| | | 449 | 7.85 | 0.0053 | | | | |
| PREAD<br>PREAD<br>BASE<br>Ty | BASAL INS | OLIN + : of Fix Den DF | METFORMIN + ed Effects F Value | Pr > F | _ | | | |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.6448<br>0.9120 | 449<br>449 | -5.22<br>-0.26 | <.0001<br>0.7937 |
| | Least Squares Means | Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | | -4.6357<br>-2.0309 | -2.1014<br>1.5536 | | | |

| NN9068 | | Date: | 22 January 2020 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 330 of 334 | |

### 37: Diastolic blood pressure after 26 weeks of treatment – change from baseline – supportive statistical analysis – full analysis set - appendix

Parameter Code=DIABPMEA

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 2 1 2

PREAD 2 BASAL INSULIN + METFORMIN BASAL INSULIN + METFORMIN +

ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 49.8665

Fit Statistics

-2 Res Log Likelihood 3055.4
AIC (Smaller is Better) 3057.4
AICC (Smaller is Better) 3057.4
BIC (Smaller is Better) 3061.5

Solution for Fixed Effects

Planned Treatment for

| Effect | Pre Trial anti-Diabetic treatment | Period<br>01 (N) | Estimate | Standard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn | | 1 2 | 31.4557<br>0.3195<br>0 | 3.1010<br>0.7041 | 449<br>449 | 10.14 |
| PREAD<br>PREAD | BASAL INSULIN + METFORMIN<br>BASAL INSULIN + METFORMIN + ONE OTHER OAD | | 1.0538 | 0.6650 | 449 | 1.58 |
| BASE | | | 0.5940 | 0.03829 | 449 | 15.51 |

# NN9068 | Date: 22 January 2020 | Novo Nordisk NN9068-4166 | CONFIDENTIAL | Status: Final |  |

Diastolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=DIABPMEA

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial anti-D | iabetic treatr | ment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alph | na | |
|---|---|---|---|---|---|---|---|---|
| Intercep<br>trtpn | t | | | 1 | <.0003<br>0.6503 | | | |
| trtpn<br>PREAD | tpn | | 2 | 0.113 | | | | |
| PREAD<br>BASE | BASAL INSULIN + | | <.000 | 1 0.0 | )5 | | | |
| | | Solution for | r Fixed Effe | cts | | | | |
| D55 | Dua Muial auti D | | | Planned<br>Treatment<br>for<br>Period | | | | |
| | Pre Trial anti-D | labetic treati | nent | 01 (N) | Lowe: | _ | pper | |
| Intercep<br>trtpn<br>trtpn | 00 | | | 1 2 | 25.3613<br>-1.0643 | | 7031 | |
| PREAD<br>PREAD | READ BASAL INSULIN + METFORMIN | | | | -0.253 | 0 2.3 | 3606 | |
| BASE | DAGAE INCOLLIN | | 0.518 | 8 0.6 | 5693 | | | |
| | Type 3 Tests of Fix | ed Effects | | | | | | |
| Effect | Num Den<br>DF DF | F Value | Pr > F | | | | | |
| trtpn<br>PREAD<br>BASE | 1 449<br>1 449<br>1 449 | 2.51 | 0.6502<br>0.1137<br><.0001 | | | | | |
| | | Least | Squares Mean | ns Estimates | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | WORK.ADATA2<br>WORK.ADATA2 | | 0.4064<br>0.5748 | 449<br>449 | 195.22<br>137.47 | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least So | quares Means | Estimates | | | | |
| Effect | Label | Lower | Upper E | xponentiated | | entiated<br>Lower | | ted<br>per |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | 78.5374<br>77.8870 | 80.1347<br>80.1462 | 2.852E34<br>2.072E34 | | 1.283E34<br>6.697E33 | 6.34<br>6.413 | |
| | | Least S | Squares Mean: | s Estimate | | | | |
| Effect | Label | | Margins | Estim | | andard<br>Error | DF t Va | lue |

trtpn Treatment contrast, IDegLira - IDeg WORK.ADATA2 0.3195 0.7041 449

0.45

NN9068
NN9068-4166
Clinical Trial Report
Statistical document

Date:
22 January 2020
Version:
5tatus:
Final
Page:

Diastolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=DIABPMEA

The Mixed Procedure

Least Squares Means Estimate

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - IDeg 0.6502 0.05 -1.0642 1.7031 1.3764

Least Squares Means Estimate

Effect Label Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - IDeg 0.3450 5.4912

## NN9068 NN9068-4166 Clinical Trial Report Statistical document Date: 22 January 2020 Version: 5 Status: Final 

Diastolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=DIABPMEA

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2
PREAD 2 BASAL INSULIN + METFORMIN
BASAL INSULIN + METFORMIN +
ONE OTHER OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 453

Number of Observations

Number of Observations Read 453 Number of Observations Used 453 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 49.8665

Fit Statistics

-2 Res Log Likelihood 3055.4
AIC (Smaller is Better) 3057.4
AICC (Smaller is Better) 3057.4
BIC (Smaller is Better) 3061.5

Solution for Fixed Effects

Planned

Treatment. for Period Standard Effect Pre Trial anti-Diabetic treatment 01 (N) Estimate Error DF t Value 31.4557 3.1010 449 10.14 Intercept 0.3195 0.7041 0.45 1 449 trtpn trtpn BASAL INSULIN + METFORMIN + ONE OTHER OAD PREAD 1.0538 0.6650 449 1.58 PREAD -0.4060 BASE 0.03829 449 -10.60

#### NN9068 Date: 22 January 2020 | Novo Nordisk NN9068-4166 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 334 of 334 Statistical document Page:

Diastolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set - appendix

Parameter Code=DIABPMEA

The Mixed Procedure

| | | | Solution f | or Fixed Effect | ts | | |
|---|---|---|---|---|---|---|---|
| Effect | Pre Trial | anti-D | iabetic tre | atment | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Pr > t | Alpha |
| Intercept<br>trtpn<br>trtpn | pt | | | | 1 2 | <.0001<br>0.6502 | 0.05<br>0.05 |
| PREAD<br>PREAD | BASAL INS | | METFORMIN<br>METFORMIN + | _ | 0.1137 | 0.05 | |
| BASE | BASAL INS | OLIN + | MEIFORMIN + | ONE OTHER OAD | | <.0001 | 0.05 |
| Solution for Fixed Effects | | | | | | | |
| | | | | | Planned<br>Treatment<br>for<br>Period | | |
| Effect | Pre Trial | anti-D | iabetic tre | atment | 01 (N) | Lower | Upper |
| Intercept<br>trtpn<br>trtpn | | | | | 1 2 | 25.3613<br>-1.0642 | 37.5500<br>1.7031 |
| PREAD<br>PREAD | BASAL INS | | | ONE OTHER OAD | 2 | -0.2530 | 2.3606 |
| BASE | DASAL INS | OLIN | METRONMIN | ONE OTHER OAD | | -0.4812 | -0.3307 |
| Ту | pe 3 Tests | of Fix | ed Effects | | | | |
| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F | | | |
| trtpn<br>PREAD | 1<br>1<br>1 | 449<br>449 | 0.21<br>2.51 | 0.6502<br>0.1137 | | | |

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| trtpn | 1 | 449 | 0.21 | 0.6502 |
| PREAD | 1 | 449 | 2.51 | 0.1137 |
| BASE | 1 | 449 | 112.39 | <.0001 |

### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | WORK.ADATA2<br>WORK.ADATA2 | 0.1124<br>-0.2071 | 0.4064<br>0.5748 | 449<br>449 | 0.28<br>-0.36 | 0.7823<br>0.7188 |
| | Least Squares Means Estimates | | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg | | -0.6863<br>-1.3367 | 0.9111<br>0.9225 | | | |